CLINICAL TRIAL: NCT02893878
Title: Post-authorisation Passive Enhanced Safety Surveillance of Seasonal Influenza Vaccines: Pilot Study in England
Brief Title: Post-authorisation Passive Enhanced Safety Surveillance of Seasonal Influenza Vaccines
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: 202056
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-09

CONDITIONS: Influenza, Human
Keywords: Seasonal influenza vaccines; Passive Enhanced Safety surveillance; England; Pilot study
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (3):
- Vaccinated_Fluarix Tetra Group: Volunteered subjects who received GlaxoSmithKline's (GSK's) influenza vaccination (Fluarix Tetra) in approximately 10 volunteer practices.
  Interventions: Other: Vaccine safety surveillance
- Vaccinated_Non GSK Group: Volunteered subjects who received Non-GSK influenza vaccination in approximately 10 volunteer practices.
  Interventions: Other: Vaccine safety surveillance
- Vaccinated_Unknown Group: Volunteered subjects who received influenza vaccination (GSK or Non-GSK not known) in approximately 10 volunteer practices.
  Interventions: Other: Vaccine safety surveillance

INTERVENTIONS:
Other: Vaccine safety surveillance — Extraction of routinely collected primary care data from approximately 10 volunteer English general practices by using an improved card-based ADR reporting system to estimate proportions of AEIs among seasonal influenza-vaccinated individuals.

SUMMARY:
The purpose of this 2016/17 pilot study is to improve the combination of a card-based adverse drug reaction (ADR) system and the use of routine data to collect adverse events following vaccination with seasonal influenza vaccines, as per European Medicines Agency (EMA) guidance and Pharmacovigilance Risk Assessment Committee of EMA (PRAC) requirements, and to identify additional data which may need to be collected in order to appropriately address the requirement.

ELIGIBILITY:
Inclusion Criteria:

• Volunteers receiving an influenza vaccine and receiving an ADR card at the beginning of the 2016/17 season.

Exclusion Criteria:

• In the database analysis, registered patients who have explicitly opted out of data sharing will be excluded from the analysis.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Registered patients in up to 10 volunteer English general practices immunized against seasonal influenza at the beginning of 2016/17 season.
Sampling Method: Non-Probability Sample
Enrollment: 19334 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2016-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included vaccinated subjects only.
Groups:
- Vaccinated_Fluarix Tetra Group: Volunteered subjects who received GlaxoSmithKline's (GSK's) influenza vaccination (Fluarix Tetra) in 10 volunteer practices.
- Vaccinated_Non GSK Group: Volunteered subjects who received Non-GSK influenza vaccination in 10 volunteer practices.
- Vaccinated_Unknown Group: Volunteered subjects who received influenza vaccination (GSK or Non-GSK not known) in 10 volunteer practices.
Period: Overall Study
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Started | 13861 | 2295 | 3178
Completed | 13861 | 2295 | 3178
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group | Total
Number analyzed (Participants) | 13861 | 2295 | 3178 | 19334
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66 (16.2) | 24 (29.7) | 57 (24.9) | 60 (24.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7661 | 1159 | 1808 | 10628
  Male | 6200 | 1136 | 1370 | 8706
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 327 | 244 | 123 | 694
  Black | 275 | 334 | 133 | 742
  White | 9581 | 906 | 1506 | 11993
  Mixed | 39 | 64 | 10 | 113
  Other | 36 | 19 | 5 | 60
  Missing | 3603 | 728 | 1401 | 5732

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined Adverse Events of Interest (AEIs) (Any) & Onset Dates of AEIs Using a Card Based-adverse Drug Reaction (ADR) Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis.
Description: AEIs were presented by categories depending of the nature of the event. -Fever or other febrile illness; - Local reaction; - General reaction (fatigue, myalgia,etc); - All other presentations that were reported following vaccination (e .g., Bell's palsy, Guillain-Barre syndrome). The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: The Weekly safety vaccinated cohorts (for each calendar Week 38 to 48) included subjects who were vaccinated the week before the week of interest and were registered during the safety follow-up period (from vaccination up to 7 days post vaccination).
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Week 37: number analyzed (Participants) | 6
  Week 37 | 0
  Week 38: number analyzed (Participants) | 1269
  Week 38 | 67
  Week 39: number analyzed (Participants) | 2626
  Week 39 | 169
  Week 40: number analyzed (Participants) | 2146
  Week 40 | 164
  Week 41: number analyzed (Participants) | 2458
  Week 41 | 112
  Week 42: number analyzed (Participants) | 1362
  Week 42 | 85
  Week 43: number analyzed (Participants) | 738
  Week 43 | 29
  Week 44: number analyzed (Participants) | 769
  Week 44 | 31
  Week 45: number analyzed (Participants) | 704
  Week 45 | 28
  Week 46: number analyzed (Participants) | 945
  Week 46 | 13
  Week 47: number analyzed (Participants) | 474
  Week 47 | 3
  Week 48: number analyzed (Participants) | 364
  Week 48 | 2

2. Primary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Any) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis (Cumulative).
Description: as for outcome 1
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: Cumulative weekly safety vaccinated cohorts (for each calendar Week 38 to 48) included subjects who were vaccinated at any point from study start up to the week before the week of interest (i.e. cumulatively since the beginning of the study) and were registered during the safety follow-up period (from vaccination up to 7 days post vaccination).
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Week 37: number analyzed (Participants) | 6
  Week 37 | 0
  Week 38: number analyzed (Participants) | 1275
  Week 38 | 67
  Week 39: number analyzed (Participants) | 3901
  Week 39 | 236
  Week 40: number analyzed (Participants) | 6047
  Week 40 | 400
  Week 41: number analyzed (Participants) | 8505
  Week 41 | 512
  Week 42: number analyzed (Participants) | 9867
  Week 42 | 597
  Week 43: number analyzed (Participants) | 10605
  Week 43 | 626
  Week 44: number analyzed (Participants) | 11374
  Week 44 | 657
  Week 45: number analyzed (Participants) | 12078
  Week 45 | 685
  Week 46: number analyzed (Participants) | 13023
  Week 46 | 698
  Week 47: number analyzed (Participants) | 13497
  Week 47 | 701
  Week 48 | 703

3. Primary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis.
Description: The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Week 37: number analyzed (Participants) | 6
  Week 37 | 0
  Week 38: number analyzed (Participants) | 1269
  Week 38 | 4
  Week 39: number analyzed (Participants) | 2626
  Week 39 | 15
  Week 40: number analyzed (Participants) | 2146
  Week 40 | 8
  Week 41: number analyzed (Participants) | 2458
  Week 41 | 10
  Week 42: number analyzed (Participants) | 1362
  Week 42 | 9
  Week 43: number analyzed (Participants) | 738
  Week 43 | 3
  Week 44: number analyzed (Participants) | 769
  Week 44 | 2
  Week 45: number analyzed (Participants) | 704
  Week 45 | 3
  Week 46: number analyzed (Participants) | 945
  Week 46 | 4
  Week 47: number analyzed (Participants) | 474
  Week 47 | 0
  Week 48: number analyzed (Participants) | 364
  Week 48 | 0

4. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis in a (Cumulative).
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Week 37: number analyzed (Participants) | 6
  Week 37 | 0
  Week 38: number analyzed (Participants) | 1275
  Week 38 | 4
  Week 39: number analyzed (Participants) | 3901
  Week 39 | 19
  Week 40: number analyzed (Participants) | 6047
  Week 40 | 27
  Week 41: number analyzed (Participants) | 8505
  Week 41 | 37
  Week 42: number analyzed (Participants) | 9867
  Week 42 | 46
  Week 43: number analyzed (Participants) | 10605
  Week 43 | 49
  Week 44: number analyzed (Participants) | 11374
  Week 44 | 51
  Week 45: number analyzed (Participants) | 12078
  Week 45 | 54
  Week 46: number analyzed (Participants) | 13023
  Week 46 | 58
  Week 47: number analyzed (Participants) | 13497
  Week 47 | 58
  Week 48 | 58

5. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis.
Description: Local symptoms include local erythema. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Week 37: number analyzed (Participants) | 6
  Week 37 | 0
  Week 38: number analyzed (Participants) | 1269
  Week 38 | 16
  Week 39: number analyzed (Participants) | 2626
  Week 39 | 20
  Week 40: number analyzed (Participants) | 2146
  Week 40 | 24
  Week 41: number analyzed (Participants) | 2458
  Week 41 | 28
  Week 42: number analyzed (Participants) | 1362
  Week 42 | 15
  Week 43: number analyzed (Participants) | 738
  Week 43 | 6
  Week 44: number analyzed (Participants) | 769
  Week 44 | 7
  Week 45: number analyzed (Participants) | 704
  Week 45 | 8
  Week 46: number analyzed (Participants) | 945
  Week 46 | 3
  Week 47: number analyzed (Participants) | 474
  Week 47 | 0
  Week 48: number analyzed (Participants) | 364
  Week 48 | 0

6. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis in a (Cumulative).
Description: as for outcome 5
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Week 37: number analyzed (Participants) | 6
  Week 37 | 0
  Week 38: number analyzed (Participants) | 1275
  Week 38 | 16
  Week 39: number analyzed (Participants) | 3901
  Week 39 | 36
  Week 40: number analyzed (Participants) | 6047
  Week 40 | 60
  Week 41: number analyzed (Participants) | 8505
  Week 41 | 88
  Week 42: number analyzed (Participants) | 9867
  Week 42 | 103
  Week 43: number analyzed (Participants) | 10605
  Week 43 | 109
  Week 44: number analyzed (Participants) | 11374
  Week 44 | 116
  Week 45: number analyzed (Participants) | 12078
  Week 45 | 124
  Week 46: number analyzed (Participants) | 13023
  Week 46 | 127
  Week 47: number analyzed (Participants) | 13497
  Week 47 | 127
  Week 48 | 127

7. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (General Non-specific Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis.
Description: General non-specific symptoms include any general non-specific symptoms, drowsiness, fatigue, irritability and malaise. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1269
  Any, Week 38 | 20
  Any, Week 39: number analyzed (Participants) | 2626
  Any, Week 39 | 47
  Any, Week 40: number analyzed (Participants) | 2146
  Any, Week 40 | 43
  Any, Week 41: number analyzed (Participants) | 2458
  Any, Week 41 | 25
  Any, Week 42: number analyzed (Participants) | 1362
  Any, Week 42 | 20
  Any, Week 43: number analyzed (Participants) | 738
  Any, Week 43 | 3
  Any, Week 44: number analyzed (Participants) | 769
  Any, Week 44 | 6
  Any, Week 45: number analyzed (Participants) | 704
  Any, Week 45 | 9
  Any, Week 46: number analyzed (Participants) | 945
  Any, Week 46 | 6
  Any, Week 47: number analyzed (Participants) | 474
  Any, Week 47 | 2
  Any, Week 48: number analyzed (Participants) | 364
  Any, Week 48 | 1
  Drowsiness, Week 37: number analyzed (Participants) | 6
  Drowsiness, Week 37 | 0
  Drowsiness, Week 38: number analyzed (Participants) | 1269
  Drowsiness, Week 38 | 8
  Drowsiness, Week 39: number analyzed (Participants) | 2626
  Drowsiness, Week 39 | 20
  Drowsiness, Week 40: number analyzed (Participants) | 2146
  Drowsiness, Week 40 | 18
  Drowsiness, Week 41: number analyzed (Participants) | 2458
  Drowsiness, Week 41 | 10
  Drowsiness, Week 42: number analyzed (Participants) | 1362
  Drowsiness, Week 42 | 9
  Drowsiness, Week 43: number analyzed (Participants) | 738
  Drowsiness, Week 43 | 1
  Drowsiness, Week 44: number analyzed (Participants) | 769
  Drowsiness, Week 44 | 1
  Drowsiness, Week 45: number analyzed (Participants) | 704
  Drowsiness, Week 45 | 2
  Drowsiness, Week 46: number analyzed (Participants) | 945
  Drowsiness, Week 46 | 2
  Drowsiness, Week 47: number analyzed (Participants) | 474
  Drowsiness, Week 47 | 1
  Drowsiness, Week 48: number analyzed (Participants) | 364
  Drowsiness, Week 48 | 0
  Fatigue, Week 37: number analyzed (Participants) | 6
  Fatigue, Week 37 | 0
  Fatigue, Week 38: number analyzed (Participants) | 1269
  Fatigue, Week 38 | 20
  Fatigue, Week 39: number analyzed (Participants) | 2626
  Fatigue, Week 39 | 40
  Fatigue, Week 40: number analyzed (Participants) | 2146
  Fatigue, Week 40 | 35
  Fatigue, Week 41: number analyzed (Participants) | 2458
  Fatigue, Week 41 | 20
  Fatigue, Week 42: number analyzed (Participants) | 1362
  Fatigue, Week 42 | 13
  Fatigue, Week 43: number analyzed (Participants) | 738
  Fatigue, Week 43 | 3
  Fatigue, Week 44: number analyzed (Participants) | 769
  Fatigue, Week 44 | 6
  Fatigue, Week 45: number analyzed (Participants) | 704
  Fatigue, Week 45 | 9
  Fatigue, Week 46: number analyzed (Participants) | 945
  Fatigue, Week 46 | 6
  Fatigue, Week 47: number analyzed (Participants) | 474
  Fatigue, Week 47 | 1
  Fatigue, Week 48: number analyzed (Participants) | 364
  Fatigue, Week 48 | 1
  Irritability, Week 37: number analyzed (Participants) | 6
  Irritability, Week 37 | 0
  Irritability, Week 38: number analyzed (Participants) | 1269
  Irritability, Week 38 | 3
  Irritability, Week 39: number analyzed (Participants) | 2626
  Irritability, Week 39 | 2
  Irritability, Week 40: number analyzed (Participants) | 2146
  Irritability, Week 40 | 6
  Irritability, Week 41: number analyzed (Participants) | 2458
  Irritability, Week 41 | 1
  Irritability, Week 42: number analyzed (Participants) | 1362
  Irritability, Week 42 | 1
  Irritability, Week 43: number analyzed (Participants) | 738
  Irritability, Week 43 | 1
  Irritability, Week 44: number analyzed (Participants) | 769
  Irritability, Week 44 | 1
  Irritability, Week 45: number analyzed (Participants) | 704
  Irritability, Week 45 | 1
  Irritability, Week 46: number analyzed (Participants) | 945
  Irritability, Week 46 | 0
  Irritability, Week 47: number analyzed (Participants) | 474
  Irritability, Week 47 | 0
  Irritability, Week 48: number analyzed (Participants) | 364
  Irritability, Week 48 | 0
  Malaise, Week 37: number analyzed (Participants) | 6
  Malaise, Week 37 | 0
  Malaise, Week 38: number analyzed (Participants) | 1269
  Malaise, Week 38 | 0
  Malaise, Week 39: number analyzed (Participants) | 2626
  Malaise, Week 39 | 0
  Malaise, Week 40: number analyzed (Participants) | 2146
  Malaise, Week 40 | 0
  Malaise, Week 41: number analyzed (Participants) | 2458
  Malaise, Week 41 | 0
  Malaise, Week 42: number analyzed (Participants) | 1362
  Malaise, Week 42 | 0
  Malaise, Week 43: number analyzed (Participants) | 738
  Malaise, Week 43 | 0
  Malaise, Week 44: number analyzed (Participants) | 769
  Malaise, Week 44 | 0
  Malaise, Week 45: number analyzed (Participants) | 704
  Malaise, Week 45 | 0
  Malaise, Week 46: number analyzed (Participants) | 945
  Malaise, Week 46 | 0
  Malaise, Week 47: number analyzed (Participants) | 474
  Malaise, Week 47 | 0
  Malaise, Week 48: number analyzed (Participants) | 364
  Malaise, Week 48 | 0

8. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (General Non-specific Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis (Cumulative).
Description: as for outcome 7
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1275
  Any, Week 38 | 20
  Any, Week 39: number analyzed (Participants) | 3901
  Any, Week 39 | 67
  Any, Week 40: number analyzed (Participants) | 6047
  Any, Week 40 | 110
  Any, Week 41: number analyzed (Participants) | 8505
  Any, Week 41 | 135
  Any, Week 42: number analyzed (Participants) | 9867
  Any, Week 42 | 155
  Any, Week 43: number analyzed (Participants) | 10605
  Any, Week 43 | 158
  Any, Week 44: number analyzed (Participants) | 11374
  Any, Week 44 | 164
  Any, Week 45: number analyzed (Participants) | 12078
  Any, Week 45 | 173
  Any, Week 46: number analyzed (Participants) | 13023
  Any, Week 46 | 179
  Any, Week 47: number analyzed (Participants) | 13497
  Any, Week 47 | 181
  Any, Week 48 | 182
  Drowsiness, Week 37: number analyzed (Participants) | 6
  Drowsiness, Week 37 | 0
  Drowsiness, Week 38: number analyzed (Participants) | 1275
  Drowsiness, Week 38 | 8
  Drowsiness, Week 39: number analyzed (Participants) | 3901
  Drowsiness, Week 39 | 28
  Drowsiness, Week 40: number analyzed (Participants) | 6047
  Drowsiness, Week 40 | 46
  Drowsiness, Week 41: number analyzed (Participants) | 8505
  Drowsiness, Week 41 | 56
  Drowsiness, Week 42: number analyzed (Participants) | 9867
  Drowsiness, Week 42 | 65
  Drowsiness, Week 43: number analyzed (Participants) | 10605
  Drowsiness, Week 43 | 66
  Drowsiness, Week 44: number analyzed (Participants) | 11374
  Drowsiness, Week 44 | 67
  Drowsiness, Week 45: number analyzed (Participants) | 12078
  Drowsiness, Week 45 | 69
  Drowsiness, Week 46: number analyzed (Participants) | 13023
  Drowsiness, Week 46 | 71
  Drowsiness, Week 47: number analyzed (Participants) | 13497
  Drowsiness, Week 47 | 72
  Drowsiness, Week 48 | 72
  Fatigue, Week 37: number analyzed (Participants) | 6
  Fatigue, Week 37 | 0
  Fatigue, Week 38: number analyzed (Participants) | 1275
  Fatigue, Week 38 | 20
  Fatigue, Week 39: number analyzed (Participants) | 3901
  Fatigue, Week 39 | 60
  Fatigue, Week 40: number analyzed (Participants) | 6047
  Fatigue, Week 40 | 95
  Fatigue, Week 41: number analyzed (Participants) | 8505
  Fatigue, Week 41 | 115
  Fatigue, Week 42: number analyzed (Participants) | 9867
  Fatigue, Week 42 | 128
  Fatigue, Week 43: number analyzed (Participants) | 10605
  Fatigue, Week 43 | 131
  Fatigue, Week 44: number analyzed (Participants) | 11374
  Fatigue, Week 44 | 137
  Fatigue, Week 45: number analyzed (Participants) | 12078
  Fatigue, Week 45 | 146
  Fatigue, Week 46: number analyzed (Participants) | 13023
  Fatigue, Week 46 | 152
  Fatigue, Week 47: number analyzed (Participants) | 13497
  Fatigue, Week 47 | 153
  Fatigue, Week 48 | 154
  Irritability, Week 37: number analyzed (Participants) | 6
  Irritability, Week 37 | 0
  Irritability, Week 38: number analyzed (Participants) | 1275
  Irritability, Week 38 | 3
  Irritability, Week 39: number analyzed (Participants) | 3901
  Irritability, Week 39 | 5
  Irritability, Week 40: number analyzed (Participants) | 6047
  Irritability, Week 40 | 11
  Irritability, Week 41: number analyzed (Participants) | 8505
  Irritability, Week 41 | 12
  Irritability, Week 42: number analyzed (Participants) | 9867
  Irritability, Week 42 | 13
  Irritability, Week 43: number analyzed (Participants) | 10605
  Irritability, Week 43 | 14
  Irritability, Week 44: number analyzed (Participants) | 11374
  Irritability, Week 44 | 15
  Irritability, Week 45: number analyzed (Participants) | 12078
  Irritability, Week 45 | 16
  Irritability, Week 46: number analyzed (Participants) | 13023
  Irritability, Week 46 | 16
  Irritability, Week 47: number analyzed (Participants) | 13497
  Irritability, Week 47 | 16
  Irritability, Week 48 | 16
  Malaise, Week 37: number analyzed (Participants) | 6
  Malaise, Week 37 | 0
  Malaise, Week 38: number analyzed (Participants) | 1275
  Malaise, Week 38 | 0
  Malaise, Week 39: number analyzed (Participants) | 3901
  Malaise, Week 39 | 0
  Malaise, Week 40: number analyzed (Participants) | 6047
  Malaise, Week 40 | 0
  Malaise, Week 41: number analyzed (Participants) | 8505
  Malaise, Week 41 | 0
  Malaise, Week 42: number analyzed (Participants) | 9867
  Malaise, Week 42 | 0
  Malaise, Week 43: number analyzed (Participants) | 10605
  Malaise, Week 43 | 0
  Malaise, Week 44: number analyzed (Participants) | 11374
  Malaise, Week 44 | 0
  Malaise, Week 45: number analyzed (Participants) | 12078
  Malaise, Week 45 | 0
  Malaise, Week 46: number analyzed (Participants) | 13023
  Malaise, Week 46 | 0
  Malaise, Week 47: number analyzed (Participants) | 13497
  Malaise, Week 47 | 0
  Malaise, Week 48 | 0

9. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Respiratory/Miscellaneous Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis.
Description: Respiratory/Miscellaneous AE include any respiratory/miscellaneous AE, conjunctivitis, coryza, cough, epistaxis, hoarseness, nasal congestion, oropharyngeal pain, rhinorrhoea and wheezing. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1269
  Any, Week 38 | 30
  Any, Week 39: number analyzed (Participants) | 2626
  Any, Week 39 | 100
  Any, Week 40: number analyzed (Participants) | 2146
  Any, Week 40 | 95
  Any, Week 41: number analyzed (Participants) | 2458
  Any, Week 41 | 64
  Any, Week 42: number analyzed (Participants) | 1362
  Any, Week 42 | 58
  Any, Week 43: number analyzed (Participants) | 738
  Any, Week 43 | 22
  Any, Week 44: number analyzed (Participants) | 769
  Any, Week 44 | 13
  Any, Week 45: number analyzed (Participants) | 704
  Any, Week 45 | 19
  Any, Week 46: number analyzed (Participants) | 945
  Any, Week 46 | 5
  Any, Week 47: number analyzed (Participants) | 474
  Any, Week 47 | 2
  Any, Week 48: number analyzed (Participants) | 364
  Any, Week 48 | 0
  Conjunctivitis, Week 37: number analyzed (Participants) | 6
  Conjunctivitis, Week 37 | 0
  Conjunctivitis, Week 38: number analyzed (Participants) | 1269
  Conjunctivitis, Week 38 | 3
  Conjunctivitis, Week 39: number analyzed (Participants) | 2626
  Conjunctivitis, Week 39 | 7
  Conjunctivitis, Week 40: number analyzed (Participants) | 2146
  Conjunctivitis, Week 40 | 2
  Conjunctivitis, Week 41: number analyzed (Participants) | 2458
  Conjunctivitis, Week 41 | 3
  Conjunctivitis, Week 42: number analyzed (Participants) | 1362
  Conjunctivitis, Week 42 | 1
  Conjunctivitis, Week 43: number analyzed (Participants) | 738
  Conjunctivitis, Week 43 | 1
  Conjunctivitis, Week 44: number analyzed (Participants) | 769
  Conjunctivitis, Week 44 | 3
  Conjunctivitis, Week 45: number analyzed (Participants) | 704
  Conjunctivitis, Week 45 | 1
  Conjunctivitis, Week 46: number analyzed (Participants) | 945
  Conjunctivitis, Week 46 | 0
  Conjunctivitis, Week 47: number analyzed (Participants) | 474
  Conjunctivitis, Week 47 | 0
  Conjunctivitis, Week 48: number analyzed (Participants) | 364
  Conjunctivitis, Week 48 | 0
  Coryza, Week 37: number analyzed (Participants) | 6
  Coryza, Week 37 | 0
  Coryza, Week 38: number analyzed (Participants) | 1269
  Coryza, Week 38 | 3
  Coryza, Week 39: number analyzed (Participants) | 2626
  Coryza, Week 39 | 19
  Coryza, Week 40: number analyzed (Participants) | 2146
  Coryza, Week 40 | 26
  Coryza, Week 41: number analyzed (Participants) | 2458
  Coryza, Week 41 | 11
  Coryza, Week 42: number analyzed (Participants) | 1362
  Coryza, Week 42 | 20
  Coryza, Week 43: number analyzed (Participants) | 738
  Coryza, Week 43 | 4
  Coryza, Week 44: number analyzed (Participants) | 769
  Coryza, Week 44 | 3
  Coryza, Week 45: number analyzed (Participants) | 704
  Coryza, Week 45 | 7
  Coryza, Week 46: number analyzed (Participants) | 945
  Coryza, Week 46 | 2
  Coryza, Week 47: number analyzed (Participants) | 474
  Coryza, Week 47 | 0
  Coryza, Week 48: number analyzed (Participants) | 364
  Coryza, Week 48 | 0
  Cough, Week 37: number analyzed (Participants) | 6
  Cough, Week 37 | 0
  Cough, Week 38: number analyzed (Participants) | 1269
  Cough, Week 38 | 9
  Cough, Week 39: number analyzed (Participants) | 2626
  Cough, Week 39 | 29
  Cough, Week 40: number analyzed (Participants) | 2146
  Cough, Week 40 | 33
  Cough, Week 41: number analyzed (Participants) | 2458
  Cough, Week 41 | 22
  Cough, Week 42: number analyzed (Participants) | 1362
  Cough, Week 42 | 25
  Cough, Week 43: number analyzed (Participants) | 738
  Cough, Week 43 | 4
  Cough, Week 44: number analyzed (Participants) | 769
  Cough, Week 44 | 5
  Cough, Week 45: number analyzed (Participants) | 704
  Cough, Week 45 | 6
  Cough, Week 46: number analyzed (Participants) | 945
  Cough, Week 46 | 3
  Cough, Week 47: number analyzed (Participants) | 474
  Cough, Week 47 | 0
  Cough, Week 48: number analyzed (Participants) | 364
  Cough, Week 48 | 0
  Epistaxis, Week 37: number analyzed (Participants) | 6
  Epistaxis, Week 37 | 0
  Epistaxis, Week 38: number analyzed (Participants) | 1269
  Epistaxis, Week 38 | 0
  Epistaxis, Week 39: number analyzed (Participants) | 2626
  Epistaxis, Week 39 | 1
  Epistaxis, Week 40: number analyzed (Participants) | 2146
  Epistaxis, Week 40 | 2
  Epistaxis, Week 41: number analyzed (Participants) | 2458
  Epistaxis, Week 41 | 3
  Epistaxis, Week 42: number analyzed (Participants) | 1362
  Epistaxis, Week 42 | 1
  Epistaxis, Week 43: number analyzed (Participants) | 738
  Epistaxis, Week 43 | 0
  Epistaxis, Week 44: number analyzed (Participants) | 769
  Epistaxis, Week 44 | 0
  Epistaxis, Week 45: number analyzed (Participants) | 704
  Epistaxis, Week 45 | 2
  Epistaxis, Week 46: number analyzed (Participants) | 945
  Epistaxis, Week 46 | 0
  Epistaxis, Week 47: number analyzed (Participants) | 474
  Epistaxis, Week 47 | 0
  Epistaxis, Week 48: number analyzed (Participants) | 364
  Epistaxis, Week 48 | 0
  Hoarseness, Week 37: number analyzed (Participants) | 6
  Hoarseness, Week 37 | 0
  Hoarseness, Week 38: number analyzed (Participants) | 1269
  Hoarseness, Week 38 | 6
  Hoarseness, Week 39: number analyzed (Participants) | 2626
  Hoarseness, Week 39 | 15
  Hoarseness, Week 40: number analyzed (Participants) | 2146
  Hoarseness, Week 40 | 16
  Hoarseness, Week 41: number analyzed (Participants) | 2458
  Hoarseness, Week 41 | 14
  Hoarseness, Week 42: number analyzed (Participants) | 1362
  Hoarseness, Week 42 | 8
  Hoarseness, Week 43: number analyzed (Participants) | 738
  Hoarseness, Week 43 | 2
  Hoarseness, Week 44: number analyzed (Participants) | 769
  Hoarseness, Week 44 | 2
  Hoarseness, Week 45: number analyzed (Participants) | 704
  Hoarseness, Week 45 | 3
  Hoarseness, Week 46: number analyzed (Participants) | 945
  Hoarseness, Week 46 | 3
  Hoarseness, Week 47: number analyzed (Participants) | 474
  Hoarseness, Week 47 | 0
  Hoarseness, Week 48: number analyzed (Participants) | 364
  Hoarseness, Week 48 | 0
  Nasal congestion, Week 37: number analyzed (Participants) | 6
  Nasal congestion, Week 37 | 0
  Nasal congestion, Week 38: number analyzed (Participants) | 1269
  Nasal congestion, Week 38 | 21
  Nasal congestion, Week 39: number analyzed (Participants) | 2626
  Nasal congestion, Week 39 | 69
  Nasal congestion, Week 40: number analyzed (Participants) | 2146
  Nasal congestion, Week 40 | 54
  Nasal congestion, Week 41: number analyzed (Participants) | 2458
  Nasal congestion, Week 41 | 45
  Nasal congestion, Week 42: number analyzed (Participants) | 1362
  Nasal congestion, Week 42 | 33
  Nasal congestion, Week 43: number analyzed (Participants) | 738
  Nasal congestion, Week 43 | 18
  Nasal congestion, Week 44: number analyzed (Participants) | 769
  Nasal congestion, Week 44 | 7
  Nasal congestion, Week 45: number analyzed (Participants) | 704
  Nasal congestion, Week 45 | 15
  Nasal congestion, Week 46: number analyzed (Participants) | 945
  Nasal congestion, Week 46 | 4
  Nasal congestion, Week 47: number analyzed (Participants) | 474
  Nasal congestion, Week 47 | 1
  Nasal congestion, Week 48: number analyzed (Participants) | 364
  Nasal congestion, Week 48 | 0
  Oropharyngeal pain, Week 37: number analyzed (Participants) | 6
  Oropharyngeal pain, Week 37 | 0
  Oropharyngeal pain, Week 38: number analyzed (Participants) | 1269
  Oropharyngeal pain, Week 38 | 9
  Oropharyngeal pain, Week 39: number analyzed (Participants) | 2626
  Oropharyngeal pain, Week 39 | 32
  Oropharyngeal pain, Week 40: number analyzed (Participants) | 2146
  Oropharyngeal pain, Week 40 | 38
  Oropharyngeal pain, Week 41: number analyzed (Participants) | 2458
  Oropharyngeal pain, Week 41 | 21
  Oropharyngeal pain, Week 42: number analyzed (Participants) | 1362
  Oropharyngeal pain, Week 42 | 25
  Oropharyngeal pain, Week 43: number analyzed (Participants) | 738
  Oropharyngeal pain, Week 43 | 9
  Oropharyngeal pain, Week 44: number analyzed (Participants) | 769
  Oropharyngeal pain, Week 44 | 5
  Oropharyngeal pain, Week 45: number analyzed (Participants) | 704
  Oropharyngeal pain, Week 45 | 7
  Oropharyngeal pain, Week 46: number analyzed (Participants) | 945
  Oropharyngeal pain, Week 46 | 2
  Oropharyngeal pain, Week 47: number analyzed (Participants) | 474
  Oropharyngeal pain, Week 47 | 2
  Oropharyngeal pain, Week 48: number analyzed (Participants) | 364
  Oropharyngeal pain, Week 48 | 0
  Rhinorrhoea, Week 37: number analyzed (Participants) | 6
  Rhinorrhoea, Week 37 | 0
  Rhinorrhoea, Week 38: number analyzed (Participants) | 1269
  Rhinorrhoea, Week 38 | 17
  Rhinorrhoea, Week 39: number analyzed (Participants) | 2626
  Rhinorrhoea, Week 39 | 58
  Rhinorrhoea, Week 40: number analyzed (Participants) | 2146
  Rhinorrhoea, Week 40 | 53
  Rhinorrhoea, Week 41: number analyzed (Participants) | 2458
  Rhinorrhoea, Week 41 | 44
  Rhinorrhoea, Week 42: number analyzed (Participants) | 1362
  Rhinorrhoea, Week 42 | 27
  Rhinorrhoea, Week 43: number analyzed (Participants) | 738
  Rhinorrhoea, Week 43 | 17
  Rhinorrhoea, Week 44: number analyzed (Participants) | 769
  Rhinorrhoea, Week 44 | 5
  Rhinorrhoea, Week 45: number analyzed (Participants) | 704
  Rhinorrhoea, Week 45 | 14
  Rhinorrhoea, Week 46: number analyzed (Participants) | 945
  Rhinorrhoea, Week 46 | 4
  Rhinorrhoea, Week 47: number analyzed (Participants) | 474
  Rhinorrhoea, Week 47 | 1
  Rhinorrhoea, Week 48: number analyzed (Participants) | 364
  Rhinorrhoea, Week 48 | 0
  Wheezing, Week 37: number analyzed (Participants) | 6
  Wheezing, Week 37 | 0
  Wheezing, Week 38: number analyzed (Participants) | 1269
  Wheezing, Week 38 | 2
  Wheezing, Week 39: number analyzed (Participants) | 2626
  Wheezing, Week 39 | 9
  Wheezing, Week 40: number analyzed (Participants) | 2146
  Wheezing, Week 40 | 11
  Wheezing, Week 41: number analyzed (Participants) | 2458
  Wheezing, Week 41 | 7
  Wheezing, Week 42: number analyzed (Participants) | 1362
  Wheezing, Week 42 | 12
  Wheezing, Week 43: number analyzed (Participants) | 738
  Wheezing, Week 43 | 2
  Wheezing, Week 44: number analyzed (Participants) | 769
  Wheezing, Week 44 | 5
  Wheezing, Week 45: number analyzed (Participants) | 704
  Wheezing, Week 45 | 3
  Wheezing, Week 46: number analyzed (Participants) | 945
  Wheezing, Week 46 | 2
  Wheezing, Week 47: number analyzed (Participants) | 474
  Wheezing, Week 47 | 0
  Wheezing, Week 48: number analyzed (Participants) | 364
  Wheezing, Week 48 | 0

10. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Respiratory/Miscellaneous Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis (Cumulative).
Description: as for outcome 9
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1275
  Any, Week 38 | 30
  Any, Week 39: number analyzed (Participants) | 3901
  Any, Week 39 | 130
  Any, Week 40: number analyzed (Participants) | 6047
  Any, Week 40 | 225
  Any, Week 41: number analyzed (Participants) | 8505
  Any, Week 41 | 289
  Any, Week 42: number analyzed (Participants) | 9867
  Any, Week 42 | 347
  Any, Week 43: number analyzed (Participants) | 10605
  Any, Week 43 | 369
  Any, Week 44: number analyzed (Participants) | 11374
  Any, Week 44 | 382
  Any, Week 45: number analyzed (Participants) | 12078
  Any, Week 45 | 401
  Any, Week 46: number analyzed (Participants) | 13023
  Any, Week 46 | 406
  Any, Week 47: number analyzed (Participants) | 13497
  Any, Week 47 | 408
  Any, Week 48 | 408
  Conjunctivitis, Week 37: number analyzed (Participants) | 6
  Conjunctivitis, Week 37 | 0
  Conjunctivitis, Week 38: number analyzed (Participants) | 1275
  Conjunctivitis, Week 38 | 3
  Conjunctivitis, Week 39: number analyzed (Participants) | 3901
  Conjunctivitis, Week 39 | 10
  Conjunctivitis, Week 40: number analyzed (Participants) | 6047
  Conjunctivitis, Week 40 | 12
  Conjunctivitis, Week 41: number analyzed (Participants) | 8505
  Conjunctivitis, Week 41 | 15
  Conjunctivitis, Week 42: number analyzed (Participants) | 9867
  Conjunctivitis, Week 42 | 16
  Conjunctivitis, Week 43: number analyzed (Participants) | 10605
  Conjunctivitis, Week 43 | 17
  Conjunctivitis, Week 44: number analyzed (Participants) | 11374
  Conjunctivitis, Week 44 | 20
  Conjunctivitis, Week 45: number analyzed (Participants) | 12078
  Conjunctivitis, Week 45 | 21
  Conjunctivitis, Week 46: number analyzed (Participants) | 13023
  Conjunctivitis, Week 46 | 21
  Conjunctivitis, Week 47: number analyzed (Participants) | 13497
  Conjunctivitis, Week 47 | 21
  Conjunctivitis, Week 48 | 21
  Coryza, Week 37: number analyzed (Participants) | 6
  Coryza, Week 37 | 0
  Coryza, Week 38: number analyzed (Participants) | 1275
  Coryza, Week 38 | 3
  Coryza, Week 39: number analyzed (Participants) | 3901
  Coryza, Week 39 | 22
  Coryza, Week 40: number analyzed (Participants) | 6047
  Coryza, Week 40 | 48
  Coryza, Week 41: number analyzed (Participants) | 8505
  Coryza, Week 41 | 59
  Coryza, Week 42: number analyzed (Participants) | 9867
  Coryza, Week 42 | 79
  Coryza, Week 43: number analyzed (Participants) | 10605
  Coryza, Week 43 | 83
  Coryza, Week 44: number analyzed (Participants) | 11374
  Coryza, Week 44 | 86
  Coryza, Week 45: number analyzed (Participants) | 12078
  Coryza, Week 45 | 93
  Coryza, Week 46: number analyzed (Participants) | 13023
  Coryza, Week 46 | 95
  Coryza, Week 47: number analyzed (Participants) | 13497
  Coryza, Week 47 | 95
  Coryza, Week 48 | 95
  Cough, Week 37: number analyzed (Participants) | 6
  Cough, Week 37 | 0
  Cough, Week 38: number analyzed (Participants) | 1275
  Cough, Week 38 | 9
  Cough, Week 39: number analyzed (Participants) | 3901
  Cough, Week 39 | 38
  Cough, Week 40: number analyzed (Participants) | 6047
  Cough, Week 40 | 71
  Cough, Week 41: number analyzed (Participants) | 8505
  Cough, Week 41 | 93
  Cough, Week 42: number analyzed (Participants) | 9867
  Cough, Week 42 | 118
  Cough, Week 43: number analyzed (Participants) | 10605
  Cough, Week 43 | 122
  Cough, Week 44: number analyzed (Participants) | 11374
  Cough, Week 44 | 127
  Cough, Week 45: number analyzed (Participants) | 12078
  Cough, Week 45 | 133
  Cough, Week 46: number analyzed (Participants) | 13023
  Cough, Week 46 | 136
  Cough, Week 47: number analyzed (Participants) | 13497
  Cough, Week 47 | 136
  Cough, Week 48 | 136
  Epistaxis, Week 37: number analyzed (Participants) | 6
  Epistaxis, Week 37 | 0
  Epistaxis, Week 38: number analyzed (Participants) | 1275
  Epistaxis, Week 38 | 0
  Epistaxis, Week 39: number analyzed (Participants) | 3901
  Epistaxis, Week 39 | 1
  Epistaxis, Week 40: number analyzed (Participants) | 6047
  Epistaxis, Week 40 | 3
  Epistaxis, Week 41: number analyzed (Participants) | 8505
  Epistaxis, Week 41 | 6
  Epistaxis, Week 42: number analyzed (Participants) | 9867
  Epistaxis, Week 42 | 7
  Epistaxis, Week 43: number analyzed (Participants) | 10605
  Epistaxis, Week 43 | 7
  Epistaxis, Week 44: number analyzed (Participants) | 11374
  Epistaxis, Week 44 | 7
  Epistaxis, Week 45: number analyzed (Participants) | 12078
  Epistaxis, Week 45 | 9
  Epistaxis, Week 46: number analyzed (Participants) | 13023
  Epistaxis, Week 46 | 9
  Epistaxis, Week 47: number analyzed (Participants) | 13497
  Epistaxis, Week 47 | 9
  Epistaxis, Week 48 | 9
  Hoarseness, Week 37: number analyzed (Participants) | 6
  Hoarseness, Week 37 | 0
  Hoarseness, Week 38: number analyzed (Participants) | 1275
  Hoarseness, Week 38 | 6
  Hoarseness, Week 39: number analyzed (Participants) | 3901
  Hoarseness, Week 39 | 21
  Hoarseness, Week 40: number analyzed (Participants) | 6047
  Hoarseness, Week 40 | 37
  Hoarseness, Week 41: number analyzed (Participants) | 8505
  Hoarseness, Week 41 | 51
  Hoarseness, Week 42: number analyzed (Participants) | 9867
  Hoarseness, Week 42 | 59
  Hoarseness, Week 43: number analyzed (Participants) | 10605
  Hoarseness, Week 43 | 61
  Hoarseness, Week 44: number analyzed (Participants) | 11374
  Hoarseness, Week 44 | 63
  Hoarseness, Week 45: number analyzed (Participants) | 12078
  Hoarseness, Week 45 | 66
  Hoarseness, Week 46: number analyzed (Participants) | 13023
  Hoarseness, Week 46 | 69
  Hoarseness, Week 47: number analyzed (Participants) | 13497
  Hoarseness, Week 47 | 69
  Hoarseness, Week 48 | 69
  Nasal congestion, Week 37: number analyzed (Participants) | 6
  Nasal congestion, Week 37 | 0
  Nasal congestion, Week 38: number analyzed (Participants) | 1275
  Nasal congestion, Week 38 | 21
  Nasal congestion, Week 39: number analyzed (Participants) | 3901
  Nasal congestion, Week 39 | 90
  Nasal congestion, Week 40: number analyzed (Participants) | 6047
  Nasal congestion, Week 40 | 144
  Nasal congestion, Week 41: number analyzed (Participants) | 8505
  Nasal congestion, Week 41 | 189
  Nasal congestion, Week 42: number analyzed (Participants) | 9867
  Nasal congestion, Week 42 | 222
  Nasal congestion, Week 43: number analyzed (Participants) | 10605
  Nasal congestion, Week 43 | 240
  Nasal congestion, Week 44: number analyzed (Participants) | 11374
  Nasal congestion, Week 44 | 247
  Nasal congestion, Week 45: number analyzed (Participants) | 12078
  Nasal congestion, Week 45 | 262
  Nasal congestion, Week 46: number analyzed (Participants) | 13023
  Nasal congestion, Week 46 | 266
  Nasal congestion, Week 47: number analyzed (Participants) | 13497
  Nasal congestion, Week 47 | 267
  Nasal congestion, Week 48 | 267
  Oropharyngeal pain, Week 37: number analyzed (Participants) | 6
  Oropharyngeal pain, Week 37 | 0
  Oropharyngeal pain, Week 38: number analyzed (Participants) | 1275
  Oropharyngeal pain, Week 38 | 9
  Oropharyngeal pain, Week 39: number analyzed (Participants) | 3901
  Oropharyngeal pain, Week 39 | 41
  Oropharyngeal pain, Week 40: number analyzed (Participants) | 6047
  Oropharyngeal pain, Week 40 | 79
  Oropharyngeal pain, Week 41: number analyzed (Participants) | 8505
  Oropharyngeal pain, Week 41 | 100
  Oropharyngeal pain, Week 42: number analyzed (Participants) | 9867
  Oropharyngeal pain, Week 42 | 125
  Oropharyngeal pain, Week 43: number analyzed (Participants) | 10605
  Oropharyngeal pain, Week 43 | 134
  Oropharyngeal pain, Week 44: number analyzed (Participants) | 11374
  Oropharyngeal pain, Week 44 | 139
  Oropharyngeal pain, Week 45: number analyzed (Participants) | 12078
  Oropharyngeal pain, Week 45 | 146
  Oropharyngeal pain, Week 46: number analyzed (Participants) | 13023
  Oropharyngeal pain, Week 46 | 148
  Oropharyngeal pain, Week 47: number analyzed (Participants) | 13497
  Oropharyngeal pain, Week 47 | 150
  Oropharyngeal pain, Week 48 | 150
  Rhinorrhoea, Week 37: number analyzed (Participants) | 6
  Rhinorrhoea, Week 37 | 0
  Rhinorrhoea, Week 38: number analyzed (Participants) | 1275
  Rhinorrhoea, Week 38 | 17
  Rhinorrhoea, Week 39: number analyzed (Participants) | 3901
  Rhinorrhoea, Week 39 | 75
  Rhinorrhoea, Week 40: number analyzed (Participants) | 6047
  Rhinorrhoea, Week 40 | 128
  Rhinorrhoea, Week 41: number analyzed (Participants) | 8505
  Rhinorrhoea, Week 41 | 172
  Rhinorrhoea, Week 42: number analyzed (Participants) | 9867
  Rhinorrhoea, Week 42 | 199
  Rhinorrhoea, Week 43: number analyzed (Participants) | 10605
  Rhinorrhoea, Week 43 | 216
  Rhinorrhoea, Week 44: number analyzed (Participants) | 11374
  Rhinorrhoea, Week 44 | 221
  Rhinorrhoea, Week 45: number analyzed (Participants) | 12078
  Rhinorrhoea, Week 45 | 235
  Rhinorrhoea, Week 46: number analyzed (Participants) | 13023
  Rhinorrhoea, Week 46 | 239
  Rhinorrhoea, Week 47: number analyzed (Participants) | 13497
  Rhinorrhoea, Week 47 | 240
  Rhinorrhoea, Week 48 | 240
  Wheezing, Week 37: number analyzed (Participants) | 6
  Wheezing, Week 37 | 0
  Wheezing, Week 38: number analyzed (Participants) | 1275
  Wheezing, Week 38 | 2
  Wheezing, Week 39: number analyzed (Participants) | 3901
  Wheezing, Week 39 | 11
  Wheezing, Week 40: number analyzed (Participants) | 6047
  Wheezing, Week 40 | 22
  Wheezing, Week 41: number analyzed (Participants) | 8505
  Wheezing, Week 41 | 29
  Wheezing, Week 42: number analyzed (Participants) | 9867
  Wheezing, Week 42 | 41
  Wheezing, Week 43: number analyzed (Participants) | 10605
  Wheezing, Week 43 | 43
  Wheezing, Week 44: number analyzed (Participants) | 11374
  Wheezing, Week 44 | 48
  Wheezing, Week 45: number analyzed (Participants) | 12078
  Wheezing, Week 45 | 51
  Wheezing, Week 46: number analyzed (Participants) | 13023
  Wheezing, Week 46 | 53
  Wheezing, Week 47: number analyzed (Participants) | 13497
  Wheezing, Week 47 | 53
  Wheezing, Week 48 | 53

11. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Gastrointestinal Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis.
Description: Gastrointestinal AEs include any gastrointestinal AEs, decreased appetite, diarrhoea, nausea and vomiting. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1269
  Any, Week 38 | 15
  Any, Week 39: number analyzed (Participants) | 2626
  Any, Week 39 | 29
  Any, Week 40: number analyzed (Participants) | 2146
  Any, Week 40 | 29
  Any, Week 41: number analyzed (Participants) | 2458
  Any, Week 41 | 21
  Any, Week 42: number analyzed (Participants) | 1362
  Any, Week 42 | 18
  Any, Week 43: number analyzed (Participants) | 738
  Any, Week 43 | 6
  Any, Week 44: number analyzed (Participants) | 769
  Any, Week 44 | 4
  Any, Week 45: number analyzed (Participants) | 704
  Any, Week 45 | 5
  Any, Week 46: number analyzed (Participants) | 945
  Any, Week 46 | 3
  Any, Week 47: number analyzed (Participants) | 474
  Any, Week 47 | 0
  Any, Week 48: number analyzed (Participants) | 364
  Any, Week 48 | 1
  Decreased appetite, Week 37: number analyzed (Participants) | 6
  Decreased appetite, Week 37 | 0
  Decreased appetite, Week 38: number analyzed (Participants) | 1269
  Decreased appetite, Week 38 | 7
  Decreased appetite, Week 39: number analyzed (Participants) | 2626
  Decreased appetite, Week 39 | 11
  Decreased appetite, Week 40: number analyzed (Participants) | 2146
  Decreased appetite, Week 40 | 11
  Decreased appetite, Week 41: number analyzed (Participants) | 2458
  Decreased appetite, Week 41 | 7
  Decreased appetite, Week 42: number analyzed (Participants) | 1362
  Decreased appetite, Week 42 | 6
  Decreased appetite, Week 43: number analyzed (Participants) | 738
  Decreased appetite, Week 43 | 2
  Decreased appetite, Week 44: number analyzed (Participants) | 769
  Decreased appetite, Week 44 | 1
  Decreased appetite, Week 45: number analyzed (Participants) | 704
  Decreased appetite, Week 45 | 2
  Decreased appetite, Week 46: number analyzed (Participants) | 945
  Decreased appetite, Week 46 | 2
  Decreased appetite, Week 47: number analyzed (Participants) | 474
  Decreased appetite, Week 47 | 0
  Decreased appetite, Week 48: number analyzed (Participants) | 364
  Decreased appetite, Week 48 | 0
  Diarrhoea, Week 37: number analyzed (Participants) | 6
  Diarrhoea, Week 37 | 0
  Diarrhoea, Week 38: number analyzed (Participants) | 1269
  Diarrhoea, Week 38 | 5
  Diarrhoea, Week 39: number analyzed (Participants) | 2626
  Diarrhoea, Week 39 | 10
  Diarrhoea, Week 40: number analyzed (Participants) | 2146
  Diarrhoea, Week 40 | 12
  Diarrhoea, Week 41: number analyzed (Participants) | 2458
  Diarrhoea, Week 41 | 8
  Diarrhoea, Week 42: number analyzed (Participants) | 1362
  Diarrhoea, Week 42 | 5
  Diarrhoea, Week 43: number analyzed (Participants) | 738
  Diarrhoea, Week 43 | 3
  Diarrhoea, Week 44: number analyzed (Participants) | 769
  Diarrhoea, Week 44 | 3
  Diarrhoea, Week 45: number analyzed (Participants) | 704
  Diarrhoea, Week 45 | 2
  Diarrhoea, Week 46: number analyzed (Participants) | 945
  Diarrhoea, Week 46 | 0
  Diarrhoea, Week 47: number analyzed (Participants) | 474
  Diarrhoea, Week 47 | 0
  Diarrhoea, Week 48: number analyzed (Participants) | 364
  Diarrhoea, Week 48 | 0
  Nausea, Week 37: number analyzed (Participants) | 6
  Nausea, Week 37 | 0
  Nausea, Week 38: number analyzed (Participants) | 1269
  Nausea, Week 38 | 11
  Nausea, Week 39: number analyzed (Participants) | 2626
  Nausea, Week 39 | 17
  Nausea, Week 40: number analyzed (Participants) | 2146
  Nausea, Week 40 | 14
  Nausea, Week 41: number analyzed (Participants) | 2458
  Nausea, Week 41 | 8
  Nausea, Week 42: number analyzed (Participants) | 1362
  Nausea, Week 42 | 9
  Nausea, Week 43: number analyzed (Participants) | 738
  Nausea, Week 43 | 2
  Nausea, Week 44: number analyzed (Participants) | 769
  Nausea, Week 44 | 0
  Nausea, Week 45: number analyzed (Participants) | 704
  Nausea, Week 45 | 4
  Nausea, Week 46: number analyzed (Participants) | 945
  Nausea, Week 46 | 1
  Nausea, Week 47: number analyzed (Participants) | 474
  Nausea, Week 47 | 0
  Nausea, Week 48: number analyzed (Participants) | 364
  Nausea, Week 48 | 1
  Vomiting, Week 37: number analyzed (Participants) | 6
  Vomiting, Week 37 | 0
  Vomiting, Week 38: number analyzed (Participants) | 1269
  Vomiting, Week 38 | 2
  Vomiting, Week 39: number analyzed (Participants) | 2626
  Vomiting, Week 39 | 2
  Vomiting, Week 40: number analyzed (Participants) | 2146
  Vomiting, Week 40 | 6
  Vomiting, Week 41: number analyzed (Participants) | 2458
  Vomiting, Week 41 | 1
  Vomiting, Week 42: number analyzed (Participants) | 1362
  Vomiting, Week 42 | 3
  Vomiting, Week 43: number analyzed (Participants) | 738
  Vomiting, Week 43 | 0
  Vomiting, Week 44: number analyzed (Participants) | 769
  Vomiting, Week 44 | 0
  Vomiting, Week 45: number analyzed (Participants) | 704
  Vomiting, Week 45 | 2
  Vomiting, Week 46: number analyzed (Participants) | 945
  Vomiting, Week 46 | 0
  Vomiting, Week 47: number analyzed (Participants) | 474
  Vomiting, Week 47 | 0
  Vomiting, Week 48: number analyzed (Participants) | 364
  Vomiting, Week 48 | 0

12. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Gastrointestinal Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis (Cumulative).
Description: as for outcome 11
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1275
  Any, Week 38 | 15
  Any, Week 39: number analyzed (Participants) | 3901
  Any, Week 39 | 44
  Any, Week 40: number analyzed (Participants) | 6047
  Any, Week 40 | 73
  Any, Week 41: number analyzed (Participants) | 8505
  Any, Week 41 | 94
  Any, Week 42: number analyzed (Participants) | 9867
  Any, Week 42 | 112
  Any, Week 43: number analyzed (Participants) | 10605
  Any, Week 43 | 118
  Any, Week 44: number analyzed (Participants) | 11374
  Any, Week 44 | 122
  Any, Week 45: number analyzed (Participants) | 12078
  Any, Week 45 | 127
  Any, Week 46: number analyzed (Participants) | 13023
  Any, Week 46 | 130
  Any, Week 47: number analyzed (Participants) | 13497
  Any, Week 47 | 130
  Any, Week 48 | 131
  Decreased appetite, Week 37: number analyzed (Participants) | 6
  Decreased appetite, Week 37 | 0
  Decreased appetite, Week 38: number analyzed (Participants) | 1275
  Decreased appetite, Week 38 | 7
  Decreased appetite, Week 39: number analyzed (Participants) | 3901
  Decreased appetite, Week 39 | 18
  Decreased appetite, Week 40: number analyzed (Participants) | 6047
  Decreased appetite, Week 40 | 29
  Decreased appetite, Week 41: number analyzed (Participants) | 8505
  Decreased appetite, Week 41 | 36
  Decreased appetite, Week 42: number analyzed (Participants) | 9867
  Decreased appetite, Week 42 | 42
  Decreased appetite, Week 43: number analyzed (Participants) | 10605
  Decreased appetite, Week 43 | 44
  Decreased appetite, Week 44: number analyzed (Participants) | 11374
  Decreased appetite, Week 44 | 45
  Decreased appetite, Week 45: number analyzed (Participants) | 12078
  Decreased appetite, Week 45 | 47
  Decreased appetite, Week 46: number analyzed (Participants) | 13023
  Decreased appetite, Week 46 | 49
  Decreased appetite, Week 47: number analyzed (Participants) | 13497
  Decreased appetite, Week 47 | 49
  Decreased appetite, Week 48 | 49
  Diarrhoea, Week 37: number analyzed (Participants) | 6
  Diarrhoea, Week 37 | 0
  Diarrhoea, Week 38: number analyzed (Participants) | 1275
  Diarrhoea, Week 38 | 5
  Diarrhoea, Week 39: number analyzed (Participants) | 3901
  Diarrhoea, Week 39 | 15
  Diarrhoea, Week 40: number analyzed (Participants) | 6047
  Diarrhoea, Week 40 | 27
  Diarrhoea, Week 41: number analyzed (Participants) | 8505
  Diarrhoea, Week 41 | 35
  Diarrhoea, Week 42: number analyzed (Participants) | 9867
  Diarrhoea, Week 42 | 40
  Diarrhoea, Week 43: number analyzed (Participants) | 10605
  Diarrhoea, Week 43 | 43
  Diarrhoea, Week 44: number analyzed (Participants) | 11374
  Diarrhoea, Week 44 | 46
  Diarrhoea, Week 45: number analyzed (Participants) | 12078
  Diarrhoea, Week 45 | 48
  Diarrhoea, Week 46: number analyzed (Participants) | 13023
  Diarrhoea, Week 46 | 48
  Diarrhoea, Week 47: number analyzed (Participants) | 13497
  Diarrhoea, Week 47 | 48
  Diarrhoea, Week 48 | 48
  Nausea, Week 37: number analyzed (Participants) | 6
  Nausea, Week 37 | 0
  Nausea, Week 38: number analyzed (Participants) | 1275
  Nausea, Week 38 | 11
  Nausea, Week 39: number analyzed (Participants) | 3901
  Nausea, Week 39 | 28
  Nausea, Week 40: number analyzed (Participants) | 6047
  Nausea, Week 40 | 42
  Nausea, Week 41: number analyzed (Participants) | 8505
  Nausea, Week 41 | 50
  Nausea, Week 42: number analyzed (Participants) | 9867
  Nausea, Week 42 | 59
  Nausea, Week 43: number analyzed (Participants) | 10605
  Nausea, Week 43 | 61
  Nausea, Week 44: number analyzed (Participants) | 11374
  Nausea, Week 44 | 61
  Nausea, Week 45: number analyzed (Participants) | 12078
  Nausea, Week 45 | 65
  Nausea, Week 46: number analyzed (Participants) | 13023
  Nausea, Week 46 | 66
  Nausea, Week 47: number analyzed (Participants) | 13497
  Nausea, Week 47 | 66
  Nausea, Week 48 | 67
  Vomiting, Week 37: number analyzed (Participants) | 6
  Vomiting, Week 37 | 0
  Vomiting, Week 38: number analyzed (Participants) | 1275
  Vomiting, Week 38 | 2
  Vomiting, Week 39: number analyzed (Participants) | 3901
  Vomiting, Week 39 | 4
  Vomiting, Week 40: number analyzed (Participants) | 6047
  Vomiting, Week 40 | 10
  Vomiting, Week 41: number analyzed (Participants) | 8505
  Vomiting, Week 41 | 11
  Vomiting, Week 42: number analyzed (Participants) | 9867
  Vomiting, Week 42 | 14
  Vomiting, Week 43: number analyzed (Participants) | 10605
  Vomiting, Week 43 | 14
  Vomiting, Week 44: number analyzed (Participants) | 11374
  Vomiting, Week 44 | 14
  Vomiting, Week 45: number analyzed (Participants) | 12078
  Vomiting, Week 45 | 16
  Vomiting, Week 46: number analyzed (Participants) | 13023
  Vomiting, Week 46 | 16
  Vomiting, Week 47: number analyzed (Participants) | 13497
  Vomiting, Week 47 | 16
  Vomiting, Week 48 | 16

13. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Sensitivity/Anaphylaxis) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis.
Description: Sensitivity/anaphylaxis AEs include any sensitivity/anaphylaxis AEs, anaphylactic reactions, facial oedema and hypersensitivity reactions. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1269
  Any, Week 38 | 0
  Any, Week 39: number analyzed (Participants) | 2626
  Any, Week 39 | 0
  Any, Week 40: number analyzed (Participants) | 2146
  Any, Week 40 | 3
  Any, Week 41: number analyzed (Participants) | 2458
  Any, Week 41 | 0
  Any, Week 42: number analyzed (Participants) | 1362
  Any, Week 42 | 2
  Any, Week 43: number analyzed (Participants) | 738
  Any, Week 43 | 0
  Any, Week 44: number analyzed (Participants) | 769
  Any, Week 44 | 1
  Any, Week 45: number analyzed (Participants) | 704
  Any, Week 45 | 1
  Any, Week 46: number analyzed (Participants) | 945
  Any, Week 46 | 0
  Any, Week 47: number analyzed (Participants) | 474
  Any, Week 47 | 0
  Any, Week 48: number analyzed (Participants) | 364
  Any, Week 48 | 0
  Anaphylactic reactions, Week 37: number analyzed (Participants) | 6
  Anaphylactic reactions, Week 37 | 0
  Anaphylactic reactions, Week 38: number analyzed (Participants) | 1269
  Anaphylactic reactions, Week 38 | 0
  Anaphylactic reactions, Week 39: number analyzed (Participants) | 2626
  Anaphylactic reactions, Week 39 | 0
  Anaphylactic reactions, Week 40: number analyzed (Participants) | 2146
  Anaphylactic reactions, Week 40 | 0
  Anaphylactic reactions, Week 41: number analyzed (Participants) | 2458
  Anaphylactic reactions, Week 41 | 0
  Anaphylactic reactions, Week 42: number analyzed (Participants) | 1362
  Anaphylactic reactions, Week 42 | 0
  Anaphylactic reactions, Week 43: number analyzed (Participants) | 738
  Anaphylactic reactions, Week 43 | 0
  Anaphylactic reactions, Week 44: number analyzed (Participants) | 769
  Anaphylactic reactions, Week 44 | 0
  Anaphylactic reactions, Week 45: number analyzed (Participants) | 704
  Anaphylactic reactions, Week 45 | 0
  Anaphylactic reactions, Week 46: number analyzed (Participants) | 945
  Anaphylactic reactions, Week 46 | 0
  Anaphylactic reactions, Week 47: number analyzed (Participants) | 474
  Anaphylactic reactions, Week 47 | 0
  Anaphylactic reactions, Week 48: number analyzed (Participants) | 364
  Anaphylactic reactions, Week 48 | 0
  Facial oedema, Week 37: number analyzed (Participants) | 6
  Facial oedema, Week 37 | 0
  Facial oedema, Week 38: number analyzed (Participants) | 1269
  Facial oedema, Week 38 | 0
  Facial oedema, Week 39: number analyzed (Participants) | 2626
  Facial oedema, Week 39 | 0
  Facial oedema, Week 40: number analyzed (Participants) | 2146
  Facial oedema, Week 40 | 1
  Facial oedema, Week 41: number analyzed (Participants) | 2458
  Facial oedema, Week 41 | 0
  Facial oedema, Week 42: number analyzed (Participants) | 1362
  Facial oedema, Week 42 | 0
  Facial oedema, Week 43: number analyzed (Participants) | 738
  Facial oedema, Week 43 | 0
  Facial oedema, Week 44: number analyzed (Participants) | 769
  Facial oedema, Week 44 | 0
  Facial oedema, Week 45: number analyzed (Participants) | 704
  Facial oedema, Week 45 | 0
  Facial oedema, Week 46: number analyzed (Participants) | 945
  Facial oedema, Week 46 | 0
  Facial oedema, Week 47: number analyzed (Participants) | 474
  Facial oedema, Week 47 | 0
  Facial oedema, Week 48: number analyzed (Participants) | 364
  Facial oedema, Week 48 | 0
  Hypersensitivity reactions, Week 37: number analyzed (Participants) | 6
  Hypersensitivity reactions, Week 37 | 0
  Hypersensitivity reactions, Week 38: number analyzed (Participants) | 1269
  Hypersensitivity reactions, Week 38 | 0
  Hypersensitivity reactions, Week 39: number analyzed (Participants) | 2626
  Hypersensitivity reactions, Week 39 | 0
  Hypersensitivity reactions, Week 40: number analyzed (Participants) | 2146
  Hypersensitivity reactions, Week 40 | 2
  Hypersensitivity reactions, Week 41: number analyzed (Participants) | 2458
  Hypersensitivity reactions, Week 41 | 0
  Hypersensitivity reactions, Week 42: number analyzed (Participants) | 1362
  Hypersensitivity reactions, Week 42 | 2
  Hypersensitivity reactions, Week 43: number analyzed (Participants) | 738
  Hypersensitivity reactions, Week 43 | 0
  Hypersensitivity reactions, Week 44: number analyzed (Participants) | 769
  Hypersensitivity reactions, Week 44 | 1
  Hypersensitivity reactions, Week 45: number analyzed (Participants) | 704
  Hypersensitivity reactions, Week 45 | 1
  Hypersensitivity reactions, Week 46: number analyzed (Participants) | 945
  Hypersensitivity reactions, Week 46 | 0
  Hypersensitivity reactions, Week 47: number analyzed (Participants) | 474
  Hypersensitivity reactions, Week 47 | 0
  Hypersensitivity reactions, Week 48: number analyzed (Participants) | 364
  Hypersensitivity reactions, Week 48 | 0

14. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Sensitivity/Anaphylaxis) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis (Cumulative).
Description: as for outcome 13
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1275
  Any, Week 38 | 0
  Any, Week 39: number analyzed (Participants) | 3901
  Any, Week 39 | 0
  Any, Week 40: number analyzed (Participants) | 6047
  Any, Week 40 | 3
  Any, Week 41: number analyzed (Participants) | 8505
  Any, Week 41 | 3
  Any, Week 42: number analyzed (Participants) | 9867
  Any, Week 42 | 5
  Any, Week 43: number analyzed (Participants) | 10605
  Any, Week 43 | 5
  Any, Week 44: number analyzed (Participants) | 11374
  Any, Week 44 | 6
  Any, Week 45: number analyzed (Participants) | 12078
  Any, Week 45 | 7
  Any, Week 46: number analyzed (Participants) | 13023
  Any, Week 46 | 7
  Any, Week 47: number analyzed (Participants) | 13497
  Any, Week 47 | 7
  Any, Week 48 | 7
  Anaphylactic reactions, Week 37: number analyzed (Participants) | 6
  Anaphylactic reactions, Week 37 | 0
  Anaphylactic reactions, Week 38: number analyzed (Participants) | 1275
  Anaphylactic reactions, Week 38 | 0
  Anaphylactic reactions, Week 39: number analyzed (Participants) | 3901
  Anaphylactic reactions, Week 39 | 0
  Anaphylactic reactions, Week 40: number analyzed (Participants) | 6047
  Anaphylactic reactions, Week 40 | 0
  Anaphylactic reactions, Week 41: number analyzed (Participants) | 8505
  Anaphylactic reactions, Week 41 | 0
  Anaphylactic reactions, Week 42: number analyzed (Participants) | 9867
  Anaphylactic reactions, Week 42 | 0
  Anaphylactic reactions, Week 43: number analyzed (Participants) | 10605
  Anaphylactic reactions, Week 43 | 0
  Anaphylactic reactions, Week 44: number analyzed (Participants) | 11374
  Anaphylactic reactions, Week 44 | 0
  Anaphylactic reactions, Week 45: number analyzed (Participants) | 12078
  Anaphylactic reactions, Week 45 | 0
  Anaphylactic reactions, Week 46: number analyzed (Participants) | 13023
  Anaphylactic reactions, Week 46 | 0
  Anaphylactic reactions, Week 47: number analyzed (Participants) | 13497
  Anaphylactic reactions, Week 47 | 0
  Anaphylactic reactions, Week 48 | 0
  Facial oedema, Week 37: number analyzed (Participants) | 6
  Facial oedema, Week 37 | 0
  Facial oedema, Week 38: number analyzed (Participants) | 1275
  Facial oedema, Week 38 | 0
  Facial oedema, Week 39: number analyzed (Participants) | 3901
  Facial oedema, Week 39 | 0
  Facial oedema, Week 40: number analyzed (Participants) | 6047
  Facial oedema, Week 40 | 1
  Facial oedema, Week 41: number analyzed (Participants) | 8505
  Facial oedema, Week 41 | 1
  Facial oedema, Week 42: number analyzed (Participants) | 9867
  Facial oedema, Week 42 | 1
  Facial oedema, Week 43: number analyzed (Participants) | 10605
  Facial oedema, Week 43 | 1
  Facial oedema, Week 44: number analyzed (Participants) | 11374
  Facial oedema, Week 44 | 1
  Facial oedema, Week 45: number analyzed (Participants) | 12078
  Facial oedema, Week 45 | 1
  Facial oedema, Week 46: number analyzed (Participants) | 13023
  Facial oedema, Week 46 | 1
  Facial oedema, Week 47: number analyzed (Participants) | 13497
  Facial oedema, Week 47 | 1
  Facial oedema, Week 48 | 1
  Hypersensitivity reactions, Week 37: number analyzed (Participants) | 6
  Hypersensitivity reactions, Week 37 | 0
  Hypersensitivity reactions, Week 38: number analyzed (Participants) | 1275
  Hypersensitivity reactions, Week 38 | 0
  Hypersensitivity reactions, Week 39: number analyzed (Participants) | 3901
  Hypersensitivity reactions, Week 39 | 0
  Hypersensitivity reactions, Week 40: number analyzed (Participants) | 6047
  Hypersensitivity reactions, Week 40 | 2
  Hypersensitivity reactions, Week 41: number analyzed (Participants) | 8505
  Hypersensitivity reactions, Week 41 | 2
  Hypersensitivity reactions, Week 42: number analyzed (Participants) | 9867
  Hypersensitivity reactions, Week 42 | 4
  Hypersensitivity reactions, Week 43: number analyzed (Participants) | 10605
  Hypersensitivity reactions, Week 43 | 4
  Hypersensitivity reactions, Week 44: number analyzed (Participants) | 11374
  Hypersensitivity reactions, Week 44 | 5
  Hypersensitivity reactions, Week 45: number analyzed (Participants) | 12078
  Hypersensitivity reactions, Week 45 | 6
  Hypersensitivity reactions, Week 46: number analyzed (Participants) | 13023
  Hypersensitivity reactions, Week 46 | 6
  Hypersensitivity reactions, Week 47: number analyzed (Participants) | 13497
  Hypersensitivity reactions, Week 47 | 6
  Hypersensitivity reactions, Week 48 | 6

15. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis.
Description: Rash AEs include any rash AEs, generalised rash and rash. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1269
  Any, Week 38 | 1
  Any, Week 39: number analyzed (Participants) | 2626
  Any, Week 39 | 0
  Any, Week 40: number analyzed (Participants) | 2146
  Any, Week 40 | 5
  Any, Week 41: number analyzed (Participants) | 2458
  Any, Week 41 | 1
  Any, Week 42: number analyzed (Participants) | 1362
  Any, Week 42 | 3
  Any, Week 43: number analyzed (Participants) | 738
  Any, Week 43 | 3
  Any, Week 44: number analyzed (Participants) | 769
  Any, Week 44 | 1
  Any, Week 45: number analyzed (Participants) | 704
  Any, Week 45 | 1
  Any, Week 46: number analyzed (Participants) | 945
  Any, Week 46 | 2
  Any, Week 47: number analyzed (Participants) | 474
  Any, Week 47 | 0
  Any, Week 48: number analyzed (Participants) | 364
  Any, Week 48 | 0
  Generalised rash, Week 37: number analyzed (Participants) | 6
  Generalised rash, Week 37 | 0
  Generalised rash, Week 38: number analyzed (Participants) | 1269
  Generalised rash, Week 38 | 0
  Generalised rash, Week 39: number analyzed (Participants) | 2626
  Generalised rash, Week 39 | 0
  Generalised rash, Week 40: number analyzed (Participants) | 2146
  Generalised rash, Week 40 | 1
  Generalised rash, Week 41: number analyzed (Participants) | 2458
  Generalised rash, Week 41 | 0
  Generalised rash, Week 42: number analyzed (Participants) | 1362
  Generalised rash, Week 42 | 0
  Generalised rash, Week 43: number analyzed (Participants) | 738
  Generalised rash, Week 43 | 0
  Generalised rash, Week 44: number analyzed (Participants) | 769
  Generalised rash, Week 44 | 0
  Generalised rash, Week 45: number analyzed (Participants) | 704
  Generalised rash, Week 45 | 0
  Generalised rash, Week 46: number analyzed (Participants) | 945
  Generalised rash, Week 46 | 0
  Generalised rash, Week 47: number analyzed (Participants) | 474
  Generalised rash, Week 47 | 0
  Generalised rash, Week 48: number analyzed (Participants) | 364
  Generalised rash, Week 48 | 0
  Rash, Week 37: number analyzed (Participants) | 6
  Rash, Week 37 | 0
  Rash, Week 38: number analyzed (Participants) | 1269
  Rash, Week 38 | 1
  Rash, Week 39: number analyzed (Participants) | 2626
  Rash, Week 39 | 0
  Rash, Week 40: number analyzed (Participants) | 2146
  Rash, Week 40 | 4
  Rash, Week 41: number analyzed (Participants) | 2458
  Rash, Week 41 | 1
  Rash, Week 42: number analyzed (Participants) | 1362
  Rash, Week 42 | 3
  Rash, Week 43: number analyzed (Participants) | 738
  Rash, Week 43 | 3
  Rash, Week 44: number analyzed (Participants) | 769
  Rash, Week 44 | 1
  Rash, Week 45: number analyzed (Participants) | 704
  Rash, Week 45 | 1
  Rash, Week 46: number analyzed (Participants) | 945
  Rash, Week 46 | 2
  Rash, Week 47: number analyzed (Participants) | 474
  Rash, Week 47 | 0
  Rash, Week 48: number analyzed (Participants) | 364
  Rash, Week 48 | 0

16. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis (Cumulative).
Description: as for outcome 15
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1275
  Any, Week 38 | 1
  Any, Week 39: number analyzed (Participants) | 3901
  Any, Week 39 | 1
  Any, Week 40: number analyzed (Participants) | 6047
  Any, Week 40 | 6
  Any, Week 41: number analyzed (Participants) | 8505
  Any, Week 41 | 7
  Any, Week 42: number analyzed (Participants) | 9867
  Any, Week 42 | 10
  Any, Week 43: number analyzed (Participants) | 10605
  Any, Week 43 | 13
  Any, Week 44: number analyzed (Participants) | 11374
  Any, Week 44 | 14
  Any, Week 45: number analyzed (Participants) | 12078
  Any, Week 45 | 15
  Any, Week 46: number analyzed (Participants) | 13023
  Any, Week 46 | 17
  Any, Week 47: number analyzed (Participants) | 13497
  Any, Week 47 | 17
  Any, Week 48 | 17
  Generalised rash, Week 37: number analyzed (Participants) | 6
  Generalised rash, Week 37 | 0
  Generalised rash, Week 38: number analyzed (Participants) | 1275
  Generalised rash, Week 38 | 0
  Generalised rash, Week 39: number analyzed (Participants) | 3901
  Generalised rash, Week 39 | 0
  Generalised rash, Week 40: number analyzed (Participants) | 6047
  Generalised rash, Week 40 | 1
  Generalised rash, Week 41: number analyzed (Participants) | 8505
  Generalised rash, Week 41 | 1
  Generalised rash, Week 42: number analyzed (Participants) | 9867
  Generalised rash, Week 42 | 1
  Generalised rash, Week 43: number analyzed (Participants) | 10605
  Generalised rash, Week 43 | 1
  Generalised rash, Week 44: number analyzed (Participants) | 11374
  Generalised rash, Week 44 | 1
  Generalised rash, Week 45: number analyzed (Participants) | 12078
  Generalised rash, Week 45 | 1
  Generalised rash, Week 46: number analyzed (Participants) | 13023
  Generalised rash, Week 46 | 1
  Generalised rash, Week 47: number analyzed (Participants) | 13497
  Generalised rash, Week 47 | 1
  Generalised rash, Week 48 | 1
  Rash, Week 37: number analyzed (Participants) | 6
  Rash, Week 37 | 0
  Rash, Week 38: number analyzed (Participants) | 1275
  Rash, Week 38 | 1
  Rash, Week 39: number analyzed (Participants) | 3901
  Rash, Week 39 | 1
  Rash, Week 40: number analyzed (Participants) | 6047
  Rash, Week 40 | 5
  Rash, Week 41: number analyzed (Participants) | 8505
  Rash, Week 41 | 6
  Rash, Week 42: number analyzed (Participants) | 9867
  Rash, Week 42 | 9
  Rash, Week 43: number analyzed (Participants) | 10605
  Rash, Week 43 | 12
  Rash, Week 44: number analyzed (Participants) | 11374
  Rash, Week 44 | 13
  Rash, Week 45: number analyzed (Participants) | 12078
  Rash, Week 45 | 14
  Rash, Week 46: number analyzed (Participants) | 13023
  Rash, Week 46 | 16
  Rash, Week 47: number analyzed (Participants) | 13497
  Rash, Week 47 | 16
  Rash, Week 48 | 16

17. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis.
Description: Musculoskeletal AEs include any musculoskeletal AEs, arthropathy and muscle aches/myalgia. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1269
  Any, Week 38 | 27
  Any, Week 39: number analyzed (Participants) | 2626
  Any, Week 39 | 60
  Any, Week 40: number analyzed (Participants) | 2146
  Any, Week 40 | 64
  Any, Week 41: number analyzed (Participants) | 2458
  Any, Week 41 | 32
  Any, Week 42: number analyzed (Participants) | 1362
  Any, Week 42 | 33
  Any, Week 43: number analyzed (Participants) | 738
  Any, Week 43 | 7
  Any, Week 44: number analyzed (Participants) | 769
  Any, Week 44 | 9
  Any, Week 45: number analyzed (Participants) | 704
  Any, Week 45 | 13
  Any, Week 46: number analyzed (Participants) | 945
  Any, Week 46 | 7
  Any, Week 47: number analyzed (Participants) | 474
  Any, Week 47 | 2
  Any, Week 48: number analyzed (Participants) | 364
  Any, Week 48 | 1
  Arthropathy, Week 37: number analyzed (Participants) | 6
  Arthropathy, Week 37 | 0
  Arthropathy, Week 38: number analyzed (Participants) | 1269
  Arthropathy, Week 38 | 8
  Arthropathy, Week 39: number analyzed (Participants) | 2626
  Arthropathy, Week 39 | 17
  Arthropathy, Week 40: number analyzed (Participants) | 2146
  Arthropathy, Week 40 | 24
  Arthropathy, Week 41: number analyzed (Participants) | 2458
  Arthropathy, Week 41 | 9
  Arthropathy, Week 42: number analyzed (Participants) | 1362
  Arthropathy, Week 42 | 11
  Arthropathy, Week 43: number analyzed (Participants) | 738
  Arthropathy, Week 43 | 2
  Arthropathy, Week 44: number analyzed (Participants) | 769
  Arthropathy, Week 44 | 2
  Arthropathy, Week 45: number analyzed (Participants) | 704
  Arthropathy, Week 45 | 5
  Arthropathy, Week 46: number analyzed (Participants) | 945
  Arthropathy, Week 46 | 1
  Arthropathy, Week 47: number analyzed (Participants) | 474
  Arthropathy, Week 47 | 0
  Arthropathy, Week 48: number analyzed (Participants) | 364
  Arthropathy, Week 48 | 0
  Muscle aches/myalgia, Week 37: number analyzed (Participants) | 6
  Muscle aches/myalgia, Week 37 | 0
  Muscle aches/myalgia, Week 38: number analyzed (Participants) | 1269
  Muscle aches/myalgia, Week 38 | 25
  Muscle aches/myalgia, Week 39: number analyzed (Participants) | 2626
  Muscle aches/myalgia, Week 39 | 58
  Muscle aches/myalgia, Week 40: number analyzed (Participants) | 2146
  Muscle aches/myalgia, Week 40 | 57
  Muscle aches/myalgia, Week 41: number analyzed (Participants) | 2458
  Muscle aches/myalgia, Week 41 | 30
  Muscle aches/myalgia, Week 42: number analyzed (Participants) | 1362
  Muscle aches/myalgia, Week 42 | 29
  Muscle aches/myalgia, Week 43: number analyzed (Participants) | 738
  Muscle aches/myalgia, Week 43 | 7
  Muscle aches/myalgia, Week 44: number analyzed (Participants) | 769
  Muscle aches/myalgia, Week 44 | 7
  Muscle aches/myalgia, Week 45: number analyzed (Participants) | 704
  Muscle aches/myalgia, Week 45 | 13
  Muscle aches/myalgia, Week 46: number analyzed (Participants) | 945
  Muscle aches/myalgia, Week 46 | 6
  Muscle aches/myalgia, Week 47: number analyzed (Participants) | 474
  Muscle aches/myalgia, Week 47 | 2
  Muscle aches/myalgia, Week 48: number analyzed (Participants) | 364
  Muscle aches/myalgia, Week 48 | 1

18. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis (Cumulative).
Description: as for outcome 17
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1275
  Any, Week 38 | 27
  Any, Week 39: number analyzed (Participants) | 3901
  Any, Week 39 | 87
  Any, Week 40: number analyzed (Participants) | 6047
  Any, Week 40 | 151
  Any, Week 41: number analyzed (Participants) | 8505
  Any, Week 41 | 183
  Any, Week 42: number analyzed (Participants) | 9867
  Any, Week 42 | 216
  Any, Week 43: number analyzed (Participants) | 10605
  Any, Week 43 | 223
  Any, Week 44: number analyzed (Participants) | 11374
  Any, Week 44 | 232
  Any, Week 45: number analyzed (Participants) | 12078
  Any, Week 45 | 245
  Any, Week 46: number analyzed (Participants) | 13023
  Any, Week 46 | 252
  Any, Week 47: number analyzed (Participants) | 13497
  Any, Week 47 | 254
  Any, Week 48 | 255
  Arthropathy, Week 37: number analyzed (Participants) | 6
  Arthropathy, Week 37 | 0
  Arthropathy, Week 38: number analyzed (Participants) | 1275
  Arthropathy, Week 38 | 8
  Arthropathy, Week 39: number analyzed (Participants) | 3901
  Arthropathy, Week 39 | 25
  Arthropathy, Week 40: number analyzed (Participants) | 6047
  Arthropathy, Week 40 | 49
  Arthropathy, Week 41: number analyzed (Participants) | 8505
  Arthropathy, Week 41 | 58
  Arthropathy, Week 42: number analyzed (Participants) | 9867
  Arthropathy, Week 42 | 69
  Arthropathy, Week 43: number analyzed (Participants) | 10605
  Arthropathy, Week 43 | 71
  Arthropathy, Week 44: number analyzed (Participants) | 11374
  Arthropathy, Week 44 | 73
  Arthropathy, Week 45: number analyzed (Participants) | 12078
  Arthropathy, Week 45 | 78
  Arthropathy, Week 46: number analyzed (Participants) | 13023
  Arthropathy, Week 46 | 79
  Arthropathy, Week 47: number analyzed (Participants) | 13497
  Arthropathy, Week 47 | 79
  Arthropathy, Week 48 | 79
  Muscle aches/myalgia, Week 37: number analyzed (Participants) | 6
  Muscle aches/myalgia, Week 37 | 0
  Muscle aches/myalgia, Week 38: number analyzed (Participants) | 1275
  Muscle aches/myalgia, Week 38 | 25
  Muscle aches/myalgia, Week 39: number analyzed (Participants) | 3901
  Muscle aches/myalgia, Week 39 | 83
  Muscle aches/myalgia, Week 40: number analyzed (Participants) | 6047
  Muscle aches/myalgia, Week 40 | 140
  Muscle aches/myalgia, Week 41: number analyzed (Participants) | 8505
  Muscle aches/myalgia, Week 41 | 170
  Muscle aches/myalgia, Week 42: number analyzed (Participants) | 9867
  Muscle aches/myalgia, Week 42 | 199
  Muscle aches/myalgia, Week 43: number analyzed (Participants) | 10605
  Muscle aches/myalgia, Week 43 | 206
  Muscle aches/myalgia, Week 44: number analyzed (Participants) | 11374
  Muscle aches/myalgia, Week 44 | 213
  Muscle aches/myalgia, Week 45: number analyzed (Participants) | 12078
  Muscle aches/myalgia, Week 45 | 226
  Muscle aches/myalgia, Week 46: number analyzed (Participants) | 13023
  Muscle aches/myalgia, Week 46 | 232
  Muscle aches/myalgia, Week 47: number analyzed (Participants) | 13497
  Muscle aches/myalgia, Week 47 | 234
  Muscle aches/myalgia, Week 48 | 235

19. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis.
Description: Neurological AEs include any neurological AEs, Bell's palsy, Guillain-Barre syndrome, headache, peripheral tremor and seizure/febrile convulsions. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1269
  Any, Week 38 | 19
  Any, Week 39: number analyzed (Participants) | 2626
  Any, Week 39 | 48
  Any, Week 40: number analyzed (Participants) | 2146
  Any, Week 40 | 42
  Any, Week 41: number analyzed (Participants) | 2458
  Any, Week 41 | 25
  Any, Week 42: number analyzed (Participants) | 1362
  Any, Week 42 | 15
  Any, Week 43: number analyzed (Participants) | 738
  Any, Week 43 | 10
  Any, Week 44: number analyzed (Participants) | 769
  Any, Week 44 | 5
  Any, Week 45: number analyzed (Participants) | 704
  Any, Week 45 | 10
  Any, Week 46: number analyzed (Participants) | 945
  Any, Week 46 | 3
  Any, Week 47: number analyzed (Participants) | 474
  Any, Week 47 | 0
  Any, Week 48: number analyzed (Participants) | 364
  Any, Week 48 | 1
  Bell's palsy, Week 37: number analyzed (Participants) | 6
  Bell's palsy, Week 37 | 0
  Bell's palsy, Week 38: number analyzed (Participants) | 1269
  Bell's palsy, Week 38 | 0
  Bell's palsy, Week 39: number analyzed (Participants) | 2626
  Bell's palsy, Week 39 | 0
  Bell's palsy, Week 40: number analyzed (Participants) | 2146
  Bell's palsy, Week 40 | 0
  Bell's palsy, Week 41: number analyzed (Participants) | 2458
  Bell's palsy, Week 41 | 0
  Bell's palsy, Week 42: number analyzed (Participants) | 1362
  Bell's palsy, Week 42 | 0
  Bell's palsy, Week 43: number analyzed (Participants) | 738
  Bell's palsy, Week 43 | 0
  Bell's palsy, Week 44: number analyzed (Participants) | 769
  Bell's palsy, Week 44 | 0
  Bell's palsy, Week 45: number analyzed (Participants) | 704
  Bell's palsy, Week 45 | 0
  Bell's palsy, Week 46: number analyzed (Participants) | 945
  Bell's palsy, Week 46 | 0
  Bell's palsy, Week 47: number analyzed (Participants) | 474
  Bell's palsy, Week 47 | 0
  Bell's palsy, Week 48: number analyzed (Participants) | 364
  Bell's palsy, Week 48 | 0
  Guillain-Barre Syndrome, Week 37: number analyzed (Participants) | 6
  Guillain-Barre Syndrome, Week 37 | 0
  Guillain-Barre Syndrome, Week 38: number analyzed (Participants) | 1269
  Guillain-Barre Syndrome, Week 38 | 0
  Guillain-Barre Syndrome, Week 39: number analyzed (Participants) | 2626
  Guillain-Barre Syndrome, Week 39 | 0
  Guillain-Barre Syndrome, Week 40: number analyzed (Participants) | 2146
  Guillain-Barre Syndrome, Week 40 | 0
  Guillain-Barre Syndrome, Week 41: number analyzed (Participants) | 2458
  Guillain-Barre Syndrome, Week 41 | 0
  Guillain-Barre Syndrome, Week 42: number analyzed (Participants) | 1362
  Guillain-Barre Syndrome, Week 42 | 0
  Guillain-Barre Syndrome, Week 43: number analyzed (Participants) | 738
  Guillain-Barre Syndrome, Week 43 | 0
  Guillain-Barre Syndrome, Week 44: number analyzed (Participants) | 769
  Guillain-Barre Syndrome, Week 44 | 0
  Guillain-Barre Syndrome, Week 45: number analyzed (Participants) | 704
  Guillain-Barre Syndrome, Week 45 | 0
  Guillain-Barre Syndrome, Week 46: number analyzed (Participants) | 945
  Guillain-Barre Syndrome, Week 46 | 0
  Guillain-Barre Syndrome, Week 47: number analyzed (Participants) | 474
  Guillain-Barre Syndrome, Week 47 | 0
  Guillain-Barre Syndrome, Week 48: number analyzed (Participants) | 364
  Guillain-Barre Syndrome, Week 48 | 0
  Headache, Week 37: number analyzed (Participants) | 6
  Headache, Week 37 | 0
  Headache, Week 38: number analyzed (Participants) | 1269
  Headache, Week 38 | 17
  Headache, Week 39: number analyzed (Participants) | 2626
  Headache, Week 39 | 48
  Headache, Week 40: number analyzed (Participants) | 2146
  Headache, Week 40 | 40
  Headache, Week 41: number analyzed (Participants) | 2458
  Headache, Week 41 | 23
  Headache, Week 42: number analyzed (Participants) | 1362
  Headache, Week 42 | 13
  Headache, Week 43: number analyzed (Participants) | 738
  Headache, Week 43 | 8
  Headache, Week 44: number analyzed (Participants) | 769
  Headache, Week 44 | 5
  Headache, Week 45: number analyzed (Participants) | 704
  Headache, Week 45 | 9
  Headache, Week 46: number analyzed (Participants) | 945
  Headache, Week 46 | 3
  Headache, Week 47: number analyzed (Participants) | 474
  Headache, Week 47 | 0
  Headache, Week 48: number analyzed (Participants) | 364
  Headache, Week 48 | 1
  Peripheral tremor, Week 37: number analyzed (Participants) | 6
  Peripheral tremor, Week 37 | 0
  Peripheral tremor, Week 38: number analyzed (Participants) | 1269
  Peripheral tremor, Week 38 | 3
  Peripheral tremor, Week 39: number analyzed (Participants) | 2626
  Peripheral tremor, Week 39 | 5
  Peripheral tremor, Week 40: number analyzed (Participants) | 2146
  Peripheral tremor, Week 40 | 1
  Peripheral tremor, Week 41: number analyzed (Participants) | 2458
  Peripheral tremor, Week 41 | 7
  Peripheral tremor, Week 42: number analyzed (Participants) | 1362
  Peripheral tremor, Week 42 | 3
  Peripheral tremor, Week 43: number analyzed (Participants) | 738
  Peripheral tremor, Week 43 | 2
  Peripheral tremor, Week 44: number analyzed (Participants) | 769
  Peripheral tremor, Week 44 | 0
  Peripheral tremor, Week 45: number analyzed (Participants) | 704
  Peripheral tremor, Week 45 | 1
  Peripheral tremor, Week 46: number analyzed (Participants) | 945
  Peripheral tremor, Week 46 | 0
  Peripheral tremor, Week 47: number analyzed (Participants) | 474
  Peripheral tremor, Week 47 | 0
  Peripheral tremor, Week 48: number analyzed (Participants) | 364
  Peripheral tremor, Week 48 | 0
  Seizure/Febrile convulsions, Week 37: number analyzed (Participants) | 6
  Seizure/Febrile convulsions, Week 37 | 0
  Seizure/Febrile convulsions, Week 38: number analyzed (Participants) | 1269
  Seizure/Febrile convulsions, Week 38 | 0
  Seizure/Febrile convulsions, Week 39: number analyzed (Participants) | 2626
  Seizure/Febrile convulsions, Week 39 | 0
  Seizure/Febrile convulsions, Week 40: number analyzed (Participants) | 2146
  Seizure/Febrile convulsions, Week 40 | 1
  Seizure/Febrile convulsions, Week 41: number analyzed (Participants) | 2458
  Seizure/Febrile convulsions, Week 41 | 0
  Seizure/Febrile convulsions, Week 42: number analyzed (Participants) | 1362
  Seizure/Febrile convulsions, Week 42 | 0
  Seizure/Febrile convulsions, Week 43: number analyzed (Participants) | 738
  Seizure/Febrile convulsions, Week 43 | 0
  Seizure/Febrile convulsions, Week 44: number analyzed (Participants) | 769
  Seizure/Febrile convulsions, Week 44 | 0
  Seizure/Febrile convulsions, Week 45: number analyzed (Participants) | 704
  Seizure/Febrile convulsions, Week 45 | 0
  Seizure/Febrile convulsions, Week 46: number analyzed (Participants) | 945
  Seizure/Febrile convulsions, Week 46 | 0
  Seizure/Febrile convulsions, Week 47: number analyzed (Participants) | 474
  Seizure/Febrile convulsions, Week 47 | 0
  Seizure/Febrile convulsions, Week 48: number analyzed (Participants) | 364
  Seizure/Febrile convulsions, Week 48 | 0

20. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group, on a Weekly Basis (Cumulative).
Description: as for outcome 19
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  Any, Week 37: number analyzed (Participants) | 6
  Any, Week 37 | 0
  Any, Week 38: number analyzed (Participants) | 1275
  Any, Week 38 | 19
  Any, Week 39: number analyzed (Participants) | 3901
  Any, Week 39 | 67
  Any, Week 40: number analyzed (Participants) | 6047
  Any, Week 40 | 109
  Any, Week 41: number analyzed (Participants) | 8505
  Any, Week 41 | 134
  Any, Week 42: number analyzed (Participants) | 9867
  Any, Week 42 | 149
  Any, Week 43: number analyzed (Participants) | 10605
  Any, Week 43 | 159
  Any, Week 44: number analyzed (Participants) | 11374
  Any, Week 44 | 164
  Any, Week 45: number analyzed (Participants) | 12078
  Any, Week 45 | 174
  Any, Week 46: number analyzed (Participants) | 13023
  Any, Week 46 | 177
  Any, Week 47: number analyzed (Participants) | 13023
  Any, Week 47 | 177
  Any, Week 48 | 178
  Bell's palsy, Week 37: number analyzed (Participants) | 6
  Bell's palsy, Week 37 | 0
  Bell's palsy, Week 38: number analyzed (Participants) | 1275
  Bell's palsy, Week 38 | 0
  Bell's palsy, Week 39: number analyzed (Participants) | 3901
  Bell's palsy, Week 39 | 0
  Bell's palsy, Week 40: number analyzed (Participants) | 6047
  Bell's palsy, Week 40 | 0
  Bell's palsy, Week 41: number analyzed (Participants) | 8505
  Bell's palsy, Week 41 | 0
  Bell's palsy, Week 42: number analyzed (Participants) | 9867
  Bell's palsy, Week 42 | 0
  Bell's palsy, Week 43: number analyzed (Participants) | 10605
  Bell's palsy, Week 43 | 0
  Bell's palsy, Week 44: number analyzed (Participants) | 11374
  Bell's palsy, Week 44 | 0
  Bell's palsy, Week 45: number analyzed (Participants) | 12078
  Bell's palsy, Week 45 | 0
  Bell's palsy, Week 46: number analyzed (Participants) | 13023
  Bell's palsy, Week 46 | 0
  Bell's palsy, Week 47: number analyzed (Participants) | 13497
  Bell's palsy, Week 47 | 0
  Bell's palsy, Week 48 | 0
  Guillain-Barre Syndrome, Week 37: number analyzed (Participants) | 6
  Guillain-Barre Syndrome, Week 37 | 0
  Guillain-Barre Syndrome, Week 38: number analyzed (Participants) | 1275
  Guillain-Barre Syndrome, Week 38 | 0
  Guillain-Barre Syndrome, Week 39: number analyzed (Participants) | 3901
  Guillain-Barre Syndrome, Week 39 | 0
  Guillain-Barre Syndrome, Week 40: number analyzed (Participants) | 6047
  Guillain-Barre Syndrome, Week 40 | 0
  Guillain-Barre Syndrome, Week 41: number analyzed (Participants) | 8505
  Guillain-Barre Syndrome, Week 41 | 0
  Guillain-Barre Syndrome, Week 42: number analyzed (Participants) | 9867
  Guillain-Barre Syndrome, Week 42 | 0
  Guillain-Barre Syndrome, Week 43: number analyzed (Participants) | 10605
  Guillain-Barre Syndrome, Week 43 | 0
  Guillain-Barre Syndrome, Week 44: number analyzed (Participants) | 11374
  Guillain-Barre Syndrome, Week 44 | 0
  Guillain-Barre Syndrome, Week 45: number analyzed (Participants) | 12078
  Guillain-Barre Syndrome, Week 45 | 0
  Guillain-Barre Syndrome, Week 46: number analyzed (Participants) | 13023
  Guillain-Barre Syndrome, Week 46 | 0
  Guillain-Barre Syndrome, Week 47: number analyzed (Participants) | 13497
  Guillain-Barre Syndrome, Week 47 | 0
  Guillain-Barre Syndrome, Week 48 | 0
  Headache, Week 37: number analyzed (Participants) | 6
  Headache, Week 37 | 0
  Headache, Week 38: number analyzed (Participants) | 1275
  Headache, Week 38 | 17
  Headache, Week 39: number analyzed (Participants) | 3901
  Headache, Week 39 | 65
  Headache, Week 40: number analyzed (Participants) | 6047
  Headache, Week 40 | 105
  Headache, Week 41: number analyzed (Participants) | 8505
  Headache, Week 41 | 128
  Headache, Week 42: number analyzed (Participants) | 9867
  Headache, Week 42 | 141
  Headache, Week 43: number analyzed (Participants) | 10605
  Headache, Week 43 | 149
  Headache, Week 44: number analyzed (Participants) | 11374
  Headache, Week 44 | 154
  Headache, Week 45: number analyzed (Participants) | 12078
  Headache, Week 45 | 163
  Headache, Week 46: number analyzed (Participants) | 13023
  Headache, Week 46 | 166
  Headache, Week 47: number analyzed (Participants) | 13497
  Headache, Week 47 | 166
  Headache, Week 48 | 167
  Peripheral tremor, Week 37: number analyzed (Participants) | 6
  Peripheral tremor, Week 37 | 0
  Peripheral tremor, Week 38: number analyzed (Participants) | 1275
  Peripheral tremor, Week 38 | 3
  Peripheral tremor, Week 39: number analyzed (Participants) | 3901
  Peripheral tremor, Week 39 | 8
  Peripheral tremor, Week 40: number analyzed (Participants) | 6047
  Peripheral tremor, Week 40 | 9
  Peripheral tremor, Week 41: number analyzed (Participants) | 8505
  Peripheral tremor, Week 41 | 16
  Peripheral tremor, Week 42: number analyzed (Participants) | 9867
  Peripheral tremor, Week 42 | 19
  Peripheral tremor, Week 43: number analyzed (Participants) | 10605
  Peripheral tremor, Week 43 | 21
  Peripheral tremor, Week 44: number analyzed (Participants) | 11374
  Peripheral tremor, Week 44 | 21
  Peripheral tremor, Week 45: number analyzed (Participants) | 12078
  Peripheral tremor, Week 45 | 22
  Peripheral tremor, Week 46: number analyzed (Participants) | 13023
  Peripheral tremor, Week 46 | 22
  Peripheral tremor, Week 47: number analyzed (Participants) | 13497
  Peripheral tremor, Week 47 | 22
  Peripheral tremor, Week 48 | 22
  Seizure/Febrile convulsions, Week 37: number analyzed (Participants) | 6
  Seizure/Febrile convulsions, Week 37 | 0
  Seizure/Febrile convulsions, Week 38: number analyzed (Participants) | 1275
  Seizure/Febrile convulsions, Week 38 | 0
  Seizure/Febrile convulsions, Week 39: number analyzed (Participants) | 3901
  Seizure/Febrile convulsions, Week 39 | 0
  Seizure/Febrile convulsions, Week 40: number analyzed (Participants) | 6047
  Seizure/Febrile convulsions, Week 40 | 1
  Seizure/Febrile convulsions, Week 41: number analyzed (Participants) | 8505
  Seizure/Febrile convulsions, Week 41 | 1
  Seizure/Febrile convulsions, Week 42: number analyzed (Participants) | 9867
  Seizure/Febrile convulsions, Week 42 | 1
  Seizure/Febrile convulsions, Week 43: number analyzed (Participants) | 10605
  Seizure/Febrile convulsions, Week 43 | 1
  Seizure/Febrile convulsions, Week 44: number analyzed (Participants) | 11374
  Seizure/Febrile convulsions, Week 44 | 1
  Seizure/Febrile convulsions, Week 45: number analyzed (Participants) | 12078
  Seizure/Febrile convulsions, Week 45 | 1
  Seizure/Febrile convulsions, Week 46: number analyzed (Participants) | 13023
  Seizure/Febrile convulsions, Week 46 | 1
  Seizure/Febrile convulsions, Week 47: number analyzed (Participants) | 13497
  Seizure/Febrile convulsions, Week 47 | 1
  Seizure/Febrile convulsions, Week 48 | 1

21. Primary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Any) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis.
Description: The age strata analysed were 6 months to 5 years; 6 to 12 years; 13 to 18 years; greater than or equal to (≥) 18-65 years and >65 years. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0
  6 months - 5 years, Week 37 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0
  6 months - 5 years, Week 38 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1
  6 months - 5 years, Week 39 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2
  6 months - 5 years, Week 40 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3
  6 months - 5 years, Week 41 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2
  6 months - 5 years, Week 42 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5
  6 months - 5 years, Week 43 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0
  6 months - 5 years, Week 44 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 0
  6 months - 5 years, Week 45 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 1
  6 months - 5 years, Week 46 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2
  6 months - 5 years, Week 47 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0
  6 months - 5 years, Week 48 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0
  6-12 years, Week 37 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1
  6-12 years, Week 38 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2
  6-12 years, Week 39 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4
  6-12 years, Week 40 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2
  6-12 years, Week 41 | 0
  6-12 years, Week 42: number analyzed (Participants) | 4
  6-12 years, Week 42 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3
  6-12 years, Week 43 | 0
  6-12 years, Week 44: number analyzed (Participants) | 2
  6-12 years, Week 44 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0
  6-12 years, Week 45 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5
  6-12 years, Week 46 | 0
  6-12 years, Week 47: number analyzed (Participants) | 0
  6-12 years, Week 47 | 0
  6-12 years, Week 48: number analyzed (Participants) | 1
  6-12 years, Week 48 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0
  13-17 years, Week 37 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7
  13-17 years, Week 38 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5
  13-17 years, Week 39 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6
  13-17 years, Week 40 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9
  13-17 years, Week 41 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6
  13-17 years, Week 42 | 1
  13-17 years, Week 43: number analyzed (Participants) | 0
  13-17 years, Week 43 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5
  13-17 years, Week 44 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4
  13-17 years, Week 45 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6
  13-17 years, Week 46 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1
  13-17 years, Week 47 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5
  13-17 years, Week 48 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2
  18-65 years, Week 37 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363
  18-65 years, Week 38 | 21
  18-65 years, Week 39: number analyzed (Participants) | 781
  18-65 years, Week 39 | 45
  18-65 years, Week 40: number analyzed (Participants) | 675
  18-65 years, Week 40 | 57
  18-65 years, Week 41: number analyzed (Participants) | 815
  18-65 years, Week 41 | 36
  18-65 years, Week 42: number analyzed (Participants) | 486
  18-65 years, Week 42 | 38
  18-65 years, Week 43: number analyzed (Participants) | 273
  18-65 years, Week 43 | 10
  18-65 years, Week 44: number analyzed (Participants) | 278
  18-65 years, Week 44 | 12
  18-65 years, Week 45: number analyzed (Participants) | 304
  18-65 years, Week 45 | 12
  18-65 years, Week 46: number analyzed (Participants) | 425
  18-65 years, Week 46 | 5
  18-65 years, Week 47: number analyzed (Participants) | 217
  18-65 years, Week 47 | 1
  18-65 years, Week 48: number analyzed (Participants) | 175
  18-65 years, Week 48 | 1
  >65 years, Week 37: number analyzed (Participants) | 4
  >65 years, Week 37 | 0
  >65 years, Week 38: number analyzed (Participants) | 898
  >65 years, Week 38 | 46
  >65 years, Week 39: number analyzed (Participants) | 1837
  >65 years, Week 39 | 124
  >65 years, Week 40: number analyzed (Participants) | 1459
  >65 years, Week 40 | 107
  >65 years, Week 41: number analyzed (Participants) | 1629
  >65 years, Week 41 | 76
  >65 years, Week 42: number analyzed (Participants) | 864
  >65 years, Week 42 | 46
  >65 years, Week 43: number analyzed (Participants) | 457
  >65 years, Week 43 | 19
  >65 years, Week 44: number analyzed (Participants) | 484
  >65 years, Week 44 | 19
  >65 years, Week 45: number analyzed (Participants) | 396
  >65 years, Week 45 | 16
  >65 years, Week 46: number analyzed (Participants) | 508
  >65 years, Week 46 | 8
  >65 years, Week 47: number analyzed (Participants) | 254
  >65 years, Week 47 | 2
  >65 years, Week 48: number analyzed (Participants) | 183
  >65 years, Week 48 | 1

22. Primary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Any) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis (Cumulative).
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: Cumulative weekly safety vaccinated cohorts (for each calendar Week 38 to 48) included subjects who were vaccinated at any point from study start up to the week before the week of interest (i.e . cumulatively since the beginning of the study) and were registered during the safety follow-up period (from vaccination up to 7 days post vaccination).
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0
  6 months - 5 years, Week 37 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0
  6 months - 5 years, Week 38 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1
  6 months - 5 years, Week 39 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3
  6 months - 5 years, Week 40 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6
  6 months - 5 years, Week 41 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8
  6 months - 5 years, Week 42 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13
  6 months - 5 years, Week 43 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13
  6 months - 5 years, Week 44 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 13
  6 months - 5 years, Week 45 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 14
  6 months - 5 years, Week 46 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 16
  6 months - 5 years, Week 47 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 16
  6 months - 5 years, Week 48 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0
  6-12 years, Week 37 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1
  6-12 years, Week 38 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3
  6-12 years, Week 39 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7
  6-12 years, Week 40 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9
  6-12 years, Week 41 | 0
  6-12 years, Week 42: number analyzed (Participants) | 13
  6-12 years, Week 42 | 0
  6-12 years, Week 43: number analyzed (Participants) | 16
  6-12 years, Week 43 | 0
  6-12 years, Week 44: number analyzed (Participants) | 18
  6-12 years, Week 44 | 0
  6-12 years, Week 45: number analyzed (Participants) | 18
  6-12 years, Week 45 | 0
  6-12 years, Week 46: number analyzed (Participants) | 23
  6-12 years, Week 46 | 0
  6-12 years, Week 47: number analyzed (Participants) | 23
  6-12 years, Week 47 | 0
  6-12 years, Week 48: number analyzed (Participants) | 24
  6-12 years, Week 48 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0
  13-17 years, Week 37 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7
  13-17 years, Week 38 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12
  13-17 years, Week 39 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18
  13-17 years, Week 40 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27
  13-17 years, Week 41 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33
  13-17 years, Week 42 | 1
  13-17 years, Week 43: number analyzed (Participants) | 33
  13-17 years, Week 43 | 1
  13-17 years, Week 44: number analyzed (Participants) | 38
  13-17 years, Week 44 | 1
  13-17 years, Week 45: number analyzed (Participants) | 42
  13-17 years, Week 45 | 1
  13-17 years, Week 46: number analyzed (Participants) | 48
  13-17 years, Week 46 | 1
  13-17 years, Week 47: number analyzed (Participants) | 49
  13-17 years, Week 47 | 1
  13-17 years, Week 48: number analyzed (Participants) | 54
  13-17 years, Week 48 | 1
  18-65 years, Week 37: number analyzed (Participants) | 2
  18-65 years, Week 37 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365
  18-65 years, Week 38 | 21
  18-65 years, Week 39: number analyzed (Participants) | 1146
  18-65 years, Week 39 | 66
  18-65 years, Week 40: number analyzed (Participants) | 1821
  18-65 years, Week 40 | 123
  18-65 years, Week 41: number analyzed (Participants) | 2636
  18-65 years, Week 41 | 159
  18-65 years, Week 42: number analyzed (Participants) | 3122
  18-65 years, Week 42 | 197
  18-65 years, Week 43: number analyzed (Participants) | 3395
  18-65 years, Week 43 | 207
  18-65 years, Week 44: number analyzed (Participants) | 3673
  18-65 years, Week 44 | 219
  18-65 years, Week 45: number analyzed (Participants) | 3977
  18-65 years, Week 45 | 231
  18-65 years, Week 46: number analyzed (Participants) | 4402
  18-65 years, Week 46 | 236
  18-65 years, Week 47: number analyzed (Participants) | 4619
  18-65 years, Week 47 | 237
  18-65 years, Week 48: number analyzed (Participants) | 4794
  18-65 years, Week 48 | 238
  >65 years, Week 37: number analyzed (Participants) | 4
  >65 years, Week 37 | 0
  >65 years, Week 38: number analyzed (Participants) | 902
  >65 years, Week 38 | 46
  >65 years, Week 39: number analyzed (Participants) | 2739
  >65 years, Week 39 | 170
  >65 years, Week 40: number analyzed (Participants) | 4198
  >65 years, Week 40 | 277
  >65 years, Week 41: number analyzed (Participants) | 5827
  >65 years, Week 41 | 353
  >65 years, Week 42: number analyzed (Participants) | 6691
  >65 years, Week 42 | 399
  >65 years, Week 43: number analyzed (Participants) | 7148
  >65 years, Week 43 | 418
  >65 years, Week 44: number analyzed (Participants) | 7632
  >65 years, Week 44 | 437
  >65 years, Week 45: number analyzed (Participants) | 8028
  >65 years, Week 45 | 453
  >65 years, Week 46: number analyzed (Participants) | 8536
  >65 years, Week 46 | 461
  >65 years, Week 47: number analyzed (Participants) | 8790
  >65 years, Week 47 | 463
  >65 years, Week 48: number analyzed (Participants) | 8973
  >65 years, Week 48 | 464

23. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis.
Description: The age strata analysed were 6 months to 5 years; 6 to 12 years; 13 to 18 years; greater than or equal to (≥) 18-65 years and >65 years. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR .
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0
  6 months - 5 years, Week 37 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0
  6 months - 5 years, Week 38 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1
  6 months - 5 years, Week 39 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2
  6 months - 5 years, Week 40 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3
  6 months - 5 years, Week 41 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2
  6 months - 5 years, Week 42 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5
  6 months - 5 years, Week 43 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0
  6 months - 5 years, Week 44 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 0
  6 months - 5 years, Week 45 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 1
  6 months - 5 years, Week 46 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2
  6 months - 5 years, Week 47 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0
  6 months - 5 years, Week 48 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0
  6-12 years, Week 37 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1
  6-12 years, Week 38 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2
  6-12 years, Week 39 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4
  6-12 years, Week 40 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2
  6-12 years, Week 41 | 0
  6-12 years, Week 42: number analyzed (Participants) | 4
  6-12 years, Week 42 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3
  6-12 years, Week 43 | 0
  6-12 years, Week 44: number analyzed (Participants) | 2
  6-12 years, Week 44 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0
  6-12 years, Week 45 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5
  6-12 years, Week 46 | 0
  6-12 years, Week 47: number analyzed (Participants) | 0
  6-12 years, Week 47 | 0
  6-12 years, Week 48: number analyzed (Participants) | 1
  6-12 years, Week 48 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0
  13-17 years, Week 37 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7
  13-17 years, Week 38 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5
  13-17 years, Week 39 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6
  13-17 years, Week 40 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9
  13-17 years, Week 41 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6
  13-17 years, Week 42 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0
  13-17 years, Week 43 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5
  13-17 years, Week 44 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4
  13-17 years, Week 45 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6
  13-17 years, Week 46 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1
  13-17 years, Week 47 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5
  13-17 years, Week 48 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2
  18-65 years, Week 37 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363
  18-65 years, Week 38 | 1
  18-65 years, Week 39: number analyzed (Participants) | 781
  18-65 years, Week 39 | 6
  18-65 years, Week 40: number analyzed (Participants) | 675
  18-65 years, Week 40 | 3
  18-65 years, Week 41: number analyzed (Participants) | 815
  18-65 years, Week 41 | 4
  18-65 years, Week 42: number analyzed (Participants) | 486
  18-65 years, Week 42 | 5
  18-65 years, Week 43: number analyzed (Participants) | 273
  18-65 years, Week 43 | 1
  18-65 years, Week 44: number analyzed (Participants) | 278
  18-65 years, Week 44 | 1
  18-65 years, Week 45: number analyzed (Participants) | 304
  18-65 years, Week 45 | 1
  18-65 years, Week 46: number analyzed (Participants) | 425
  18-65 years, Week 46 | 1
  18-65 years, Week 47: number analyzed (Participants) | 217
  18-65 years, Week 47 | 0
  18-65 years, Week 48: number analyzed (Participants) | 175
  18-65 years, Week 48 | 0
  >65 years, Week 37: number analyzed (Participants) | 4
  >65 years, Week 37 | 0
  >65 years, Week 38: number analyzed (Participants) | 898
  >65 years, Week 38 | 3
  >65 years, Week 39: number analyzed (Participants) | 1837
  >65 years, Week 39 | 9
  >65 years, Week40: number analyzed (Participants) | 1459
  >65 years, Week40 | 5
  >65 years, Week 41: number analyzed (Participants) | 1629
  >65 years, Week 41 | 6
  >65 years, Week 42: number analyzed (Participants) | 864
  >65 years, Week 42 | 4
  >65 years, Week 43: number analyzed (Participants) | 457
  >65 years, Week 43 | 2
  >65 years, Week 44: number analyzed (Participants) | 484
  >65 years, Week 44 | 1
  >65 years, Week 45: number analyzed (Participants) | 396
  >65 years, Week 45 | 2
  >65 years, Week 46: number analyzed (Participants) | 508
  >65 years, Week 46 | 3
  >65 years, Week 47: number analyzed (Participants) | 254
  >65 years, Week 47 | 0
  >65 years, Week 48: number analyzed (Participants) | 183
  >65 years, Week 48 | 0

24. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis (Cumulative).
Description: The age strata analysed were 6 months to 5 years; 6 to 12 years; 13 to 18 years; greater than or equal to (≥) 18-65 years and >65 years. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who receive d the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR .
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016).
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0
  6 months - 5 years, Week 37 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0
  6 months - 5 years, Week 38 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1
  6 months - 5 years, Week 39 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3
  6 months - 5 years, Week 40 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6
  6 months - 5 years, Week 41 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8
  6 months - 5 years, Week 42 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13
  6 months - 5 years, Week 43 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13
  6 months - 5 years, Week 44 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 13
  6 months - 5 years, Week 45 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 14
  6 months - 5 years, Week 46 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 16
  6 months - 5 years, Week 47 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 16
  6 months - 5 years, Week 48 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0
  6-12 years, Week 37 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1
  6-12 years, Week 38 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3
  6-12 years, Week 39 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7
  6-12 years, Week 40 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9
  6-12 years, Week 41 | 0
  6-12 years, Week 42: number analyzed (Participants) | 13
  6-12 years, Week 42 | 0
  6-12 years, Week 43: number analyzed (Participants) | 16
  6-12 years, Week 43 | 0
  6-12 years, Week 44: number analyzed (Participants) | 18
  6-12 years, Week 44 | 0
  6-12 years, Week 45: number analyzed (Participants) | 18
  6-12 years, Week 45 | 0
  6-12 years, Week 46: number analyzed (Participants) | 23
  6-12 years, Week 46 | 0
  6-12 years, Week 47: number analyzed (Participants) | 23
  6-12 years, Week 47 | 0
  6-12 years, Week 48: number analyzed (Participants) | 24
  6-12 years, Week 48 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0
  13-17 years, Week 37 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7
  13-17 years, Week 38 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12
  13-17 years, Week 39 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18
  13-17 years, Week 40 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27
  13-17 years, Week 41 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33
  13-17 years, Week 42 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33
  13-17 years, Week 43 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38
  13-17 years, Week 44 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42
  13-17 years, Week 45 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48
  13-17 years, Week 46 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49
  13-17 years, Week 47 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54
  13-17 years, Week 48 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2
  18-65 years, Week 37 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365
  18-65 years, Week 38 | 1
  18-65 years, Week 39: number analyzed (Participants) | 1146
  18-65 years, Week 39 | 7
  18-65 years, Week 40: number analyzed (Participants) | 1821
  18-65 years, Week 40 | 10
  18-65 years, Week 41: number analyzed (Participants) | 2636
  18-65 years, Week 41 | 14
  18-65 years, Week 42: number analyzed (Participants) | 3122
  18-65 years, Week 42 | 19
  18-65 years, Week 43: number analyzed (Participants) | 3395
  18-65 years, Week 43 | 20
  18-65 years, Week 44: number analyzed (Participants) | 3673
  18-65 years, Week 44 | 21
  18-65 years, Week 45: number analyzed (Participants) | 3977
  18-65 years, Week 45 | 22
  18-65 years, Week 46: number analyzed (Participants) | 4402
  18-65 years, Week 46 | 23
  18-65 years, Week 47: number analyzed (Participants) | 4619
  18-65 years, Week 47 | 23
  18-65 years, Week 48: number analyzed (Participants) | 4794
  18-65 years, Week 48 | 23
  >65 years, Week 37: number analyzed (Participants) | 4
  >65 years, Week 37 | 0
  >65 years, Week 38: number analyzed (Participants) | 902
  >65 years, Week 38 | 3
  >65 years, Week 39: number analyzed (Participants) | 2739
  >65 years, Week 39 | 12
  >65 years, Week 40: number analyzed (Participants) | 4198
  >65 years, Week 40 | 17
  >65 years, Week 41: number analyzed (Participants) | 5827
  >65 years, Week 41 | 23
  >65 years, Week 42: number analyzed (Participants) | 6691
  >65 years, Week 42 | 27
  >65 years, Week 43: number analyzed (Participants) | 7148
  >65 years, Week 43 | 29
  >65 years, Week 44: number analyzed (Participants) | 7632
  >65 years, Week 44 | 30
  >65 years, Week 45: number analyzed (Participants) | 8028
  >65 years, Week 45 | 32
  >65 years, Week 46: number analyzed (Participants) | 8536
  >65 years, Week 46 | 35
  >65 years, Week 47: number analyzed (Participants) | 8790
  >65 years, Week 47 | 35
  >65 years, Week 48: number analyzed (Participants) | 8973
  >65 years, Week 48 | 35

25. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis.
Description: Local symptoms included local erythema. The age strata analysed were 6 months to 5 years; 6 to 12 years; 13 to 18 years; greater than or equal to (≥) 18-65 years and >65 years. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Vaccinated_Fluarix Tetra Group: Volunteered subjects who received GlaxoSmithKline 's (GSK's) influenza vaccination (Fluarix Tetra ) in 10 volunteer practices.
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 2
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 3
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 2
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 5
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 0
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 0
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 1
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 2
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 0
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 2
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 4
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 2
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 4
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 3
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 2
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 0
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 5
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 0
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 1
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 5
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 6
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 9
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 6
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 0
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 5
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 4
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 6
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 1
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 5
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 363
  18-65 years: Week 38 | 9
  18-65 years: Week 39: number analyzed (Participants) | 781
  18-65 years: Week 39 | 8
  18-65 years: Week 40: number analyzed (Participants) | 675
  18-65 years: Week 40 | 10
  18-65 years: Week 41: number analyzed (Participants) | 815
  18-65 years: Week 41 | 12
  18-65 years: Week 42: number analyzed (Participants) | 486
  18-65 years: Week 42 | 9
  18-65 years: Week 43: number analyzed (Participants) | 273
  18-65 years: Week 43 | 1
  18-65 years: Week 44: number analyzed (Participants) | 278
  18-65 years: Week 44 | 4
  18-65 years: Week 45: number analyzed (Participants) | 304
  18-65 years: Week 45 | 3
  18-65 years: Week 46: number analyzed (Participants) | 425
  18-65 years: Week 46 | 3
  18-65 years: Week 47: number analyzed (Participants) | 217
  18-65 years: Week 47 | 0
  18-65 years: Week 48: number analyzed (Participants) | 175
  18-65 years: Week 48 | 0
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 898
  >65 years: Week 38 | 7
  >65 years: Week 39: number analyzed (Participants) | 1837
  >65 years: Week 39 | 12
  >65 years: Week 40: number analyzed (Participants) | 1459
  >65 years: Week 40 | 14
  >65 years: Week 41: number analyzed (Participants) | 1629
  >65 years: Week 41 | 16
  >65 years: Week 42: number analyzed (Participants) | 864
  >65 years: Week 42 | 6
  >65 years: Week 43: number analyzed (Participants) | 457
  >65 years: Week 43 | 5
  >65 years: Week 44: number analyzed (Participants) | 484
  >65 years: Week 44 | 3
  >65 years: Week 45: number analyzed (Participants) | 396
  >65 years: Week 45 | 5
  >65 years: Week 46: number analyzed (Participants) | 508
  >65 years: Week 46 | 0
  >65 years: Week 47: number analyzed (Participants) | 254
  >65 years: Week 47 | 0
  >65 years: Week 48: number analyzed (Participants) | 183
  >65 years: Week 48 | 0

26. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis (Cumulative).
Description: Local symptoms included local erythema. The age strata analysed were 6 months to 5 years; 6 to 12 years; 13 to 18 years; greater than or equal to (≥) 18-65 years and >65 years. The primary analysis included all subjects vaccinated with GSK vaccine instead of the subjects who received the ADR card as the information whether or not subjects received the ADR card was not encoded in EHR .
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 3
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 6
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 8
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 13
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 13
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 13
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 14
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 16
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 16
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 3
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 7
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 9
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 13
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 16
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 18
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 18
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 23
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 23
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 24
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 12
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 18
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 27
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 33
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 33
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 38
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 42
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 48
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 49
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 54
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 365
  18-65 years: Week 38 | 9
  18-65 years: Week 39: number analyzed (Participants) | 1146
  18-65 years: Week 39 | 17
  18-65 years: Week 40: number analyzed (Participants) | 1821
  18-65 years: Week 40 | 27
  18-65 years: Week 41: number analyzed (Participants) | 2636
  18-65 years: Week 41 | 39
  18-65 years: Week 42: number analyzed (Participants) | 3122
  18-65 years: Week 42 | 48
  18-65 years: Week 43: number analyzed (Participants) | 3395
  18-65 years: Week 43 | 49
  18-65 years: Week 44: number analyzed (Participants) | 3673
  18-65 years: Week 44 | 53
  18-65 years: Week 45: number analyzed (Participants) | 3977
  18-65 years: Week 45 | 56
  18-65 years: Week 46: number analyzed (Participants) | 4402
  18-65 years: Week 46 | 59
  18-65 years: Week 47: number analyzed (Participants) | 4619
  18-65 years: Week 47 | 59
  18-65 years: Week 48: number analyzed (Participants) | 4794
  18-65 years: Week 48 | 59
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 902
  >65 years: Week 38 | 7
  >65 years: Week 39: number analyzed (Participants) | 2739
  >65 years: Week 39 | 19
  >65 years: Week 40: number analyzed (Participants) | 4198
  >65 years: Week 40 | 33
  >65 years: Week 41: number analyzed (Participants) | 5827
  >65 years: Week 41 | 49
  >65 years: Week 42: number analyzed (Participants) | 6691
  >65 years: Week 42 | 55
  >65 years: Week 43: number analyzed (Participants) | 7148
  >65 years: Week 43 | 60
  >65 years: Week 44: number analyzed (Participants) | 7632
  >65 years: Week 44 | 63
  >65 years: Week 45: number analyzed (Participants) | 8028
  >65 years: Week 45 | 68
  >65 years: Week 46: number analyzed (Participants) | 8536
  >65 years: Week 46 | 68
  >65 years: Week 47: number analyzed (Participants) | 8790
  >65 years: Week 47 | 68
  >65 years: Week 48: number analyzed (Participants) | 8973
  >65 years: Week 48 | 68

27. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (General Non-specific Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis.
Description: as for outcome 23
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 2
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 3
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 2
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 5
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 0
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 0
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 1
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 2
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 0
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 2
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 4
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 2
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 4
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 3
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 2
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 0
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 5
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 0
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 1
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 5
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 6
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 9
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 6
  13-17 years: Week 42 | 1
  13-17 years: Week 43: number analyzed (Participants) | 0
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 5
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 4
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 6
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 1
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 5
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 363
  18-65 years: Week 38 | 6
  18-65 years: Week 39: number analyzed (Participants) | 781
  18-65 years: Week 39 | 15
  18-65 years: Week 40: number analyzed (Participants) | 675
  18-65 years: Week 40 | 17
  18-65 years: Week 41: number analyzed (Participants) | 815
  18-65 years: Week 41 | 3
  18-65 years: Week 42: number analyzed (Participants) | 486
  18-65 years: Week 42 | 9
  18-65 years: Week 43: number analyzed (Participants) | 273
  18-65 years: Week 43 | 0
  18-65 years: Week 44: number analyzed (Participants) | 278
  18-65 years: Week 44 | 2
  18-65 years: Week 45: number analyzed (Participants) | 304
  18-65 years: Week 45 | 5
  18-65 years: Week 46: number analyzed (Participants) | 425
  18-65 years: Week 46 | 2
  18-65 years: Week 47: number analyzed (Participants) | 217
  18-65 years: Week 47 | 0
  18-65 years: Week 48: number analyzed (Participants) | 175
  18-65 years: Week 48 | 1
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 898
  >65 years: Week 38 | 14
  >65 years: Week 39: number analyzed (Participants) | 1837
  >65 years: Week 39 | 32
  >65 years: Week 40: number analyzed (Participants) | 1459
  >65 years: Week 40 | 26
  >65 years: Week 41: number analyzed (Participants) | 1629
  >65 years: Week 41 | 22
  >65 years: Week 42: number analyzed (Participants) | 864
  >65 years: Week 42 | 10
  >65 years: Week 43: number analyzed (Participants) | 457
  >65 years: Week 43 | 3
  >65 years: Week 44: number analyzed (Participants) | 484
  >65 years: Week 44 | 4
  >65 years: Week 45: number analyzed (Participants) | 396
  >65 years: Week 45 | 4
  >65 years: Week 46: number analyzed (Participants) | 508
  >65 years: Week 46 | 4
  >65 years: Week 47: number analyzed (Participants) | 254
  >65 years: Week 47 | 2
  >65 years: Week 48: number analyzed (Participants) | 183
  >65 years: Week 48 | 0

28. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (General Non-specific Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis (Cumulative).
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 3
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 6
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 8
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 13
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 13
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 13
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 14
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 16
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 16
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 3
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 7
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 9
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 13
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 16
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 18
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 18
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 23
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 23
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 24
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 12
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 18
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 27
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 33
  13-17 years: Week 42 | 1
  13-17 years: Week 43: number analyzed (Participants) | 33
  13-17 years: Week 43 | 1
  13-17 years: Week 44: number analyzed (Participants) | 38
  13-17 years: Week 44 | 1
  13-17 years: Week 45: number analyzed (Participants) | 42
  13-17 years: Week 45 | 1
  13-17 years: Week 46: number analyzed (Participants) | 48
  13-17 years: Week 46 | 1
  13-17 years: Week 47: number analyzed (Participants) | 49
  13-17 years: Week 47 | 1
  13-17 years: Week 48: number analyzed (Participants) | 54
  13-17 years: Week 48 | 1
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 365
  18-65 years: Week 38 | 6
  18-65 years: Week 39: number analyzed (Participants) | 1146
  18-65 years: Week 39 | 21
  18-65 years: Week 40: number analyzed (Participants) | 1821
  18-65 years: Week 40 | 38
  18-65 years: Week 41: number analyzed (Participants) | 2636
  18-65 years: Week 41 | 41
  18-65 years: Week 42: number analyzed (Participants) | 3122
  18-65 years: Week 42 | 50
  18-65 years: Week 43: number analyzed (Participants) | 3395
  18-65 years: Week 43 | 50
  18-65 years: Week 44: number analyzed (Participants) | 3673
  18-65 years: Week 44 | 52
  18-65 years: Week 45: number analyzed (Participants) | 3977
  18-65 years: Week 45 | 57
  18-65 years: Week 46: number analyzed (Participants) | 4402
  18-65 years: Week 46 | 59
  18-65 years: Week 47: number analyzed (Participants) | 4619
  18-65 years: Week 47 | 59
  18-65 years: Week 48: number analyzed (Participants) | 4794
  18-65 years: Week 48 | 60
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 902
  >65 years: Week 38 | 14
  >65 years: Week 39: number analyzed (Participants) | 2739
  >65 years: Week 39 | 46
  >65 years: Week 40: number analyzed (Participants) | 4198
  >65 years: Week 40 | 72
  >65 years: Week 41: number analyzed (Participants) | 5827
  >65 years: Week 41 | 94
  >65 years: Week 42: number analyzed (Participants) | 6691
  >65 years: Week 42 | 104
  >65 years: Week 43: number analyzed (Participants) | 7148
  >65 years: Week 43 | 107
  >65 years: Week 44: number analyzed (Participants) | 7632
  >65 years: Week 44 | 111
  >65 years: Week 45: number analyzed (Participants) | 8028
  >65 years: Week 45 | 115
  >65 years: Week 46: number analyzed (Participants) | 8536
  >65 years: Week 46 | 119
  >65 years: Week 47: number analyzed (Participants) | 8790
  >65 years: Week 47 | 121
  >65 years: Week 48: number analyzed (Participants) | 8973
  >65 years: Week 48 | 121

29. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Respiratory/Miscellaneous Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis.
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 2
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 3
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 2
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 5
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 0
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 0
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 1
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 2
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 0
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 2
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 4
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 2
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 4
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 3
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 2
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 0
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 5
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 0
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 1
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 5
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 6
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 9
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 6
  13-17 years: Week 42 | 1
  13-17 years: Week 43: number analyzed (Participants) | 0
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 5
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 4
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 6
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 1
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 5
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 363
  18-65 years: Week 38 | 8
  18-65 years: Week 39: number analyzed (Participants) | 781
  18-65 years: Week 39 | 25
  18-65 years: Week 40: number analyzed (Participants) | 675
  18-65 years: Week 40 | 32
  18-65 years: Week 41: number analyzed (Participants) | 815
  18-65 years: Week 41 | 17
  18-65 years: Week 42: number analyzed (Participants) | 486
  18-65 years: Week 42 | 27
  18-65 years: Week 43: number analyzed (Participants) | 273
  18-65 years: Week 43 | 9
  18-65 years: Week 44: number analyzed (Participants) | 278
  18-65 years: Week 44 | 4
  18-65 years: Week 45: number analyzed (Participants) | 304
  18-65 years: Week 45 | 10
  18-65 years: Week 46: number analyzed (Participants) | 425
  18-65 years: Week 46 | 2
  18-65 years: Week 47: number analyzed (Participants) | 217
  18-65 years: Week 47 | 1
  18-65 years: Week 48: number analyzed (Participants) | 175
  18-65 years: Week 48 | 0
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 898
  >65 years: Week 38 | 22
  >65 years: Week 39: number analyzed (Participants) | 1837
  >65 years: Week 39 | 75
  >65 years: Week 40: number analyzed (Participants) | 1459
  >65 years: Week 40 | 63
  >65 years: Week 41: number analyzed (Participants) | 1629
  >65 years: Week 41 | 47
  >65 years: Week 42: number analyzed (Participants) | 864
  >65 years: Week 42 | 30
  >65 years: Week 43: number analyzed (Participants) | 457
  >65 years: Week 43 | 13
  >65 years: Week 44: number analyzed (Participants) | 484
  >65 years: Week 44 | 9
  >65 years: Week 45: number analyzed (Participants) | 396
  >65 years: Week 45 | 9
  >65 years: Week 46: number analyzed (Participants) | 508
  >65 years: Week 46 | 3
  >65 years: Week 47: number analyzed (Participants) | 254
  >65 years: Week 47 | 1
  >65 years: Week 48: number analyzed (Participants) | 183
  >65 years: Week 48 | 0

30. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Respiratory/Miscellaneous Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis (Cumulative).
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 3
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 6
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 8
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 13
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 13
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 13
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 14
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 16
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 16
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 3
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 7
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 9
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 13
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 16
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 18
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 18
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 23
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 23
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 24
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 12
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 18
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 27
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 33
  13-17 years: Week 42 | 1
  13-17 years: Week 43: number analyzed (Participants) | 33
  13-17 years: Week 43 | 1
  13-17 years: Week 44: number analyzed (Participants) | 38
  13-17 years: Week 44 | 1
  13-17 years: Week 45: number analyzed (Participants) | 42
  13-17 years: Week 45 | 1
  13-17 years: Week 46: number analyzed (Participants) | 48
  13-17 years: Week 46 | 1
  13-17 years: Week 47: number analyzed (Participants) | 49
  13-17 years: Week 47 | 1
  13-17 years: Week 48: number analyzed (Participants) | 54
  13-17 years: Week 48 | 1
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 365
  18-65 years: Week 38 | 8
  18-65 years: Week 39: number analyzed (Participants) | 1146
  18-65 years: Week 39 | 33
  18-65 years: Week 40: number analyzed (Participants) | 1821
  18-65 years: Week 40 | 65
  18-65 years: Week 41: number analyzed (Participants) | 2636
  18-65 years: Week 41 | 82
  18-65 years: Week 42: number analyzed (Participants) | 3122
  18-65 years: Week 42 | 109
  18-65 years: Week 43: number analyzed (Participants) | 3395
  18-65 years: Week 43 | 118
  18-65 years: Week 44: number analyzed (Participants) | 3673
  18-65 years: Week 44 | 122
  18-65 years: Week 45: number analyzed (Participants) | 3977
  18-65 years: Week 45 | 132
  18-65 years: Week 46: number analyzed (Participants) | 4402
  18-65 years: Week 46 | 134
  18-65 years: Week 47: number analyzed (Participants) | 4619
  18-65 years: Week 47 | 135
  18-65 years: Week 48: number analyzed (Participants) | 4794
  18-65 years: Week 48 | 135
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 902
  >65 years: Week 38 | 22
  >65 years: Week 39: number analyzed (Participants) | 2739
  >65 years: Week 39 | 97
  >65 years: Week 40: number analyzed (Participants) | 4198
  >65 years: Week 40 | 160
  >65 years: Week 41: number analyzed (Participants) | 5827
  >65 years: Week 41 | 207
  >65 years: Week 42: number analyzed (Participants) | 6691
  >65 years: Week 42 | 237
  >65 years: Week 43: number analyzed (Participants) | 7148
  >65 years: Week 43 | 250
  >65 years: Week 44: number analyzed (Participants) | 7632
  >65 years: Week 44 | 259
  >65 years: Week 45: number analyzed (Participants) | 8028
  >65 years: Week 45 | 268
  >65 years: Week 46: number analyzed (Participants) | 8536
  >65 years: Week 46 | 271
  >65 years: Week 47: number analyzed (Participants) | 8790
  >65 years: Week 47 | 272
  >65 years: Week 48: number analyzed (Participants) | 8973
  >65 years: Week 48 | 272

31. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Gastrointestinal Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis.
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 2
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 3
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 2
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 5
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 0
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 0
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 1
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 2
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 0
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 2
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 4
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 2
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 4
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 3
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 2
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 0
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 5
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 0
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 1
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 5
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 6
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 9
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 6
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 0
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 5
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 4
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 6
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 1
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 5
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 363
  18-65 years: Week 38 | 7
  18-65 years: Week 39: number analyzed (Participants) | 781
  18-65 years: Week 39 | 9
  18-65 years: Week 40: number analyzed (Participants) | 675
  18-65 years: Week 40 | 10
  18-65 years: Week 41: number analyzed (Participants) | 815
  18-65 years: Week 41 | 7
  18-65 years: Week 42: number analyzed (Participants) | 486
  18-65 years: Week 42 | 7
  18-65 years: Week 43: number analyzed (Participants) | 273
  18-65 years: Week 43 | 3
  18-65 years: Week 44: number analyzed (Participants) | 278
  18-65 years: Week 44 | 2
  18-65 years: Week 45: number analyzed (Participants) | 304
  18-65 years: Week 45 | 3
  18-65 years: Week 46: number analyzed (Participants) | 425
  18-65 years: Week 46 | 2
  18-65 years: Week 47: number analyzed (Participants) | 217
  18-65 years: Week 47 | 0
  18-65 years: Week 48: number analyzed (Participants) | 175
  18-65 years: Week 48 | 1
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 898
  >65 years: Week 38 | 8
  >65 years: Week 39: number analyzed (Participants) | 1837
  >65 years: Week 39 | 20
  >65 years: Week 40: number analyzed (Participants) | 1459
  >65 years: Week 40 | 19
  >65 years: Week 41: number analyzed (Participants) | 1629
  >65 years: Week 41 | 14
  >65 years: Week 42: number analyzed (Participants) | 864
  >65 years: Week 42 | 11
  >65 years: Week 43: number analyzed (Participants) | 457
  >65 years: Week 43 | 3
  >65 years: Week 44: number analyzed (Participants) | 484
  >65 years: Week 44 | 2
  >65 years: Week 45: number analyzed (Participants) | 396
  >65 years: Week 45 | 2
  >65 years: Week 46: number analyzed (Participants) | 508
  >65 years: Week 46 | 1
  >65 years: Week 47: number analyzed (Participants) | 254
  >65 years: Week 47 | 0
  >65 years: Week 48: number analyzed (Participants) | 183
  >65 years: Week 48 | 0

32. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Gastrointestinal Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis (Cumulative).
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 3
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 6
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 8
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 13
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 13
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 13
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 14
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 16
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 16
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 3
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 7
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 9
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 13
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 16
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 18
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 18
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 23
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 23
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 24
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 12
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 18
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 27
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 33
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 33
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 38
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 42
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 48
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 49
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 54
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 365
  18-65 years: Week 38 | 7
  18-65 years: Week 39: number analyzed (Participants) | 1146
  18-65 years: Week 39 | 16
  18-65 years: Week 40: number analyzed (Participants) | 1821
  18-65 years: Week 40 | 26
  18-65 years: Week 41: number analyzed (Participants) | 2636
  18-65 years: Week 41 | 33
  18-65 years: Week 42: number analyzed (Participants) | 3122
  18-65 years: Week 42 | 40
  18-65 years: Week 43: number analyzed (Participants) | 3395
  18-65 years: Week 43 | 43
  18-65 years: Week 44: number analyzed (Participants) | 3673
  18-65 years: Week 44 | 45
  18-65 years: Week 45: number analyzed (Participants) | 3977
  18-65 years: Week 45 | 48
  18-65 years: Week 46: number analyzed (Participants) | 4402
  18-65 years: Week 46 | 50
  18-65 years: Week 47: number analyzed (Participants) | 4619
  18-65 years: Week 47 | 50
  18-65 years: Week 48: number analyzed (Participants) | 4794
  18-65 years: Week 48 | 51
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 902
  >65 years: Week 38 | 8
  >65 years: Week 39: number analyzed (Participants) | 2739
  >65 years: Week 39 | 28
  >65 years: Week 40: number analyzed (Participants) | 4198
  >65 years: Week 40 | 47
  >65 years: Week 41: number analyzed (Participants) | 5827
  >65 years: Week 41 | 61
  >65 years: Week 42: number analyzed (Participants) | 6691
  >65 years: Week 42 | 72
  >65 years: Week 43: number analyzed (Participants) | 7148
  >65 years: Week 43 | 75
  >65 years: Week 44: number analyzed (Participants) | 7632
  >65 years: Week 44 | 77
  >65 years: Week 45: number analyzed (Participants) | 8028
  >65 years: Week 45 | 79
  >65 years: Week 46: number analyzed (Participants) | 8536
  >65 years: Week 46 | 80
  >65 years: Week 47: number analyzed (Participants) | 8790
  >65 years: Week 47 | 80
  >65 years: Week 48: number analyzed (Participants) | 8973
  >65 years: Week 48 | 80

33. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Sesnsitivity/Anapylaxis) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis.
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 2
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 3
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 2
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 5
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 0
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 0
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 1
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 2
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 0
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 2
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 4
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 2
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 4
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 3
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 2
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 0
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 5
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 0
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 1
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 5
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 6
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 9
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 6
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 0
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 5
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 4
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 6
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 1
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 5
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 363
  18-65 years: Week 38 | 0
  18-65 years: Week 39: number analyzed (Participants) | 781
  18-65 years: Week 39 | 0
  18-65 years: Week 40: number analyzed (Participants) | 675
  18-65 years: Week 40 | 2
  18-65 years: Week 41: number analyzed (Participants) | 815
  18-65 years: Week 41 | 0
  18-65 years: Week 42: number analyzed (Participants) | 486
  18-65 years: Week 42 | 1
  18-65 years: Week 43: number analyzed (Participants) | 273
  18-65 years: Week 43 | 0
  18-65 years: Week 44: number analyzed (Participants) | 278
  18-65 years: Week 44 | 1
  18-65 years: Week 45: number analyzed (Participants) | 304
  18-65 years: Week 45 | 0
  18-65 years: Week 46: number analyzed (Participants) | 425
  18-65 years: Week 46 | 0
  18-65 years: Week 47: number analyzed (Participants) | 217
  18-65 years: Week 47 | 0
  18-65 years: Week 48: number analyzed (Participants) | 175
  18-65 years: Week 48 | 0
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 898
  >65 years: Week 38 | 0
  >65 years: Week 39: number analyzed (Participants) | 1837
  >65 years: Week 39 | 0
  >65 years: Week 40: number analyzed (Participants) | 1459
  >65 years: Week 40 | 1
  >65 years: Week 41: number analyzed (Participants) | 1629
  >65 years: Week 41 | 0
  >65 years: Week 42: number analyzed (Participants) | 864
  >65 years: Week 42 | 1
  >65 years: Week 43: number analyzed (Participants) | 457
  >65 years: Week 43 | 0
  >65 years: Week 44: number analyzed (Participants) | 484
  >65 years: Week 44 | 0
  >65 years: Week 45: number analyzed (Participants) | 396
  >65 years: Week 45 | 1
  >65 years: Week 46: number analyzed (Participants) | 508
  >65 years: Week 46 | 0
  >65 years: Week 47: number analyzed (Participants) | 254
  >65 years: Week 47 | 0
  >65 years: Week 48: number analyzed (Participants) | 183
  >65 years: Week 48 | 0

34. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Sesnsitivity/Anapylaxis) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis (Cumulative).
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 3
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 6
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 8
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 13
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 13
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 13
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 14
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 16
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 16
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 3
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 7
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 9
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 13
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 16
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 18
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 18
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 23
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 23
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 24
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 12
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 18
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 27
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 33
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 33
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 38
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 42
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 48
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 49
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 54
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 365
  18-65 years: Week 38 | 0
  18-65 years: Week 39: number analyzed (Participants) | 1146
  18-65 years: Week 39 | 0
  18-65 years: Week 40: number analyzed (Participants) | 1821
  18-65 years: Week 40 | 2
  18-65 years: Week 41: number analyzed (Participants) | 2636
  18-65 years: Week 41 | 2
  18-65 years: Week 42: number analyzed (Participants) | 3122
  18-65 years: Week 42 | 3
  18-65 years: Week 43: number analyzed (Participants) | 3395
  18-65 years: Week 43 | 3
  18-65 years: Week 44: number analyzed (Participants) | 3673
  18-65 years: Week 44 | 4
  18-65 years: Week 45: number analyzed (Participants) | 3977
  18-65 years: Week 45 | 4
  18-65 years: Week 46: number analyzed (Participants) | 4402
  18-65 years: Week 46 | 4
  18-65 years: Week 47: number analyzed (Participants) | 4619
  18-65 years: Week 47 | 4
  18-65 years: Week 48: number analyzed (Participants) | 4794
  18-65 years: Week 48 | 4
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 902
  >65 years: Week 38 | 0
  >65 years: Week 39: number analyzed (Participants) | 2739
  >65 years: Week 39 | 0
  >65 years: Week 40: number analyzed (Participants) | 4198
  >65 years: Week 40 | 1
  >65 years: Week 41: number analyzed (Participants) | 5827
  >65 years: Week 41 | 1
  >65 years: Week 42: number analyzed (Participants) | 6691
  >65 years: Week 42 | 2
  >65 years: Week 43: number analyzed (Participants) | 7148
  >65 years: Week 43 | 2
  >65 years: Week 44: number analyzed (Participants) | 7632
  >65 years: Week 44 | 2
  >65 years: Week 45: number analyzed (Participants) | 8028
  >65 years: Week 45 | 3
  >65 years: Week 46: number analyzed (Participants) | 8536
  >65 years: Week 46 | 3
  >65 years: Week 47: number analyzed (Participants) | 8790
  >65 years: Week 47 | 3
  >65 years: Week 48: number analyzed (Participants) | 8973
  >65 years: Week 48 | 3

35. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis.
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 2
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 3
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 2
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 5
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 0
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 0
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 1
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 2
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 0
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 2
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 4
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 2
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 4
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 3
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 2
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 0
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 5
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 0
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 1
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 5
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 6
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 9
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 6
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 0
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 5
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 4
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 6
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 1
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 5
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 363
  18-65 years: Week 38 | 0
  18-65 years: Week 39: number analyzed (Participants) | 781
  18-65 years: Week 39 | 0
  18-65 years: Week 40: number analyzed (Participants) | 675
  18-65 years: Week 40 | 2
  18-65 years: Week 41: number analyzed (Participants) | 815
  18-65 years: Week 41 | 0
  18-65 years: Week 42: number analyzed (Participants) | 486
  18-65 years: Week 42 | 2
  18-65 years: Week 43: number analyzed (Participants) | 273
  18-65 years: Week 43 | 1
  18-65 years: Week 44: number analyzed (Participants) | 278
  18-65 years: Week 44 | 0
  18-65 years: Week 45: number analyzed (Participants) | 304
  18-65 years: Week 45 | 0
  18-65 years: Week 46: number analyzed (Participants) | 425
  18-65 years: Week 46 | 1
  18-65 years: Week 47: number analyzed (Participants) | 217
  18-65 years: Week 47 | 0
  18-65 years: Week 48: number analyzed (Participants) | 175
  18-65 years: Week 48 | 0
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 898
  >65 years: Week 38 | 1
  >65 years: Week 39: number analyzed (Participants) | 1837
  >65 years: Week 39 | 0
  >65 years: Week 40: number analyzed (Participants) | 1459
  >65 years: Week 40 | 3
  >65 years: Week 41: number analyzed (Participants) | 1629
  >65 years: Week 41 | 1
  >65 years: Week 42: number analyzed (Participants) | 864
  >65 years: Week 42 | 1
  >65 years: Week 43: number analyzed (Participants) | 457
  >65 years: Week 43 | 2
  >65 years: Week 44: number analyzed (Participants) | 484
  >65 years: Week 44 | 1
  >65 years: Week 45: number analyzed (Participants) | 396
  >65 years: Week 45 | 1
  >65 years: Week 46: number analyzed (Participants) | 508
  >65 years: Week 46 | 1
  >65 years: Week 47: number analyzed (Participants) | 254
  >65 years: Week 47 | 0
  >65 years: Week 48: number analyzed (Participants) | 183
  >65 years: Week 48 | 0

36. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis (Cumulative).
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 3
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 6
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 8
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 13
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 13
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 13
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 14
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 16
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 16
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 3
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 7
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 9
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 13
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 16
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 18
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 18
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 23
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 23
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 24
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 12
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 18
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 27
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 33
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 33
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 38
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 42
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 48
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 49
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 54
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 365
  18-65 years: Week 38 | 0
  18-65 years: Week 39: number analyzed (Participants) | 1146
  18-65 years: Week 39 | 0
  18-65 years: Week 40: number analyzed (Participants) | 1821
  18-65 years: Week 40 | 2
  18-65 years: Week 41: number analyzed (Participants) | 2636
  18-65 years: Week 41 | 2
  18-65 years: Week 42: number analyzed (Participants) | 3122
  18-65 years: Week 42 | 4
  18-65 years: Week 43: number analyzed (Participants) | 3395
  18-65 years: Week 43 | 5
  18-65 years: Week 44: number analyzed (Participants) | 3673
  18-65 years: Week 44 | 5
  18-65 years: Week 45: number analyzed (Participants) | 3977
  18-65 years: Week 45 | 5
  18-65 years: Week 46: number analyzed (Participants) | 4402
  18-65 years: Week 46 | 6
  18-65 years: Week 47: number analyzed (Participants) | 4619
  18-65 years: Week 47 | 6
  18-65 years: Week 48: number analyzed (Participants) | 4794
  18-65 years: Week 48 | 6
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 902
  >65 years: Week 38 | 1
  >65 years: Week 39: number analyzed (Participants) | 2739
  >65 years: Week 39 | 1
  >65 years: Week 40: number analyzed (Participants) | 4198
  >65 years: Week 40 | 4
  >65 years: Week 41: number analyzed (Participants) | 5827
  >65 years: Week 41 | 5
  >65 years: Week 42: number analyzed (Participants) | 6691
  >65 years: Week 42 | 6
  >65 years: Week 43: number analyzed (Participants) | 7148
  >65 years: Week 43 | 8
  >65 years: Week 44: number analyzed (Participants) | 7632
  >65 years: Week 44 | 9
  >65 years: Week 45: number analyzed (Participants) | 8028
  >65 years: Week 45 | 10
  >65 years: Week 46: number analyzed (Participants) | 8536
  >65 years: Week 46 | 11
  >65 years: Week 47: number analyzed (Participants) | 8790
  >65 years: Week 47 | 11
  >65 years: Week 48: number analyzed (Participants) | 8973
  >65 years: Week 48 | 11

37. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis.
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 2
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 3
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 2
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 5
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 0
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 0
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 1
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 2
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 0
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 2
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 4
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 2
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 4
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 3
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 2
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 0
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 5
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 0
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 1
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 5
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 6
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 9
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 6
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 0
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 5
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 4
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 6
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 1
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 5
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 363
  18-65 years: Week 38 | 11
  18-65 years: Week 39: number analyzed (Participants) | 781
  18-65 years: Week 39 | 18
  18-65 years: Week 40: number analyzed (Participants) | 675
  18-65 years: Week 40 | 22
  18-65 years: Week 41: number analyzed (Participants) | 815
  18-65 years: Week 41 | 12
  18-65 years: Week 42: number analyzed (Participants) | 486
  18-65 years: Week 42 | 18
  18-65 years: Week 43: number analyzed (Participants) | 273
  18-65 years: Week 43 | 5
  18-65 years: Week 44: number analyzed (Participants) | 278
  18-65 years: Week 44 | 3
  18-65 years: Week 45: number analyzed (Participants) | 304
  18-65 years: Week 45 | 7
  18-65 years: Week 46: number analyzed (Participants) | 425
  18-65 years: Week 46 | 3
  18-65 years: Week 47: number analyzed (Participants) | 217
  18-65 years: Week 47 | 1
  18-65 years: Week 48: number analyzed (Participants) | 175
  18-65 years: Week 48 | 0
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 898
  >65 years: Week 38 | 16
  >65 years: Week 39: number analyzed (Participants) | 1837
  >65 years: Week 39 | 42
  >65 years: Week 40: number analyzed (Participants) | 1459
  >65 years: Week 40 | 42
  >65 years: Week 41: number analyzed (Participants) | 1629
  >65 years: Week 41 | 20
  >65 years: Week 42: number analyzed (Participants) | 864
  >65 years: Week 42 | 15
  >65 years: Week 43: number analyzed (Participants) | 457
  >65 years: Week 43 | 2
  >65 years: Week 44: number analyzed (Participants) | 484
  >65 years: Week 44 | 6
  >65 years: Week 45: number analyzed (Participants) | 396
  >65 years: Week 45 | 6
  >65 years: Week 46: number analyzed (Participants) | 508
  >65 years: Week 46 | 4
  >65 years: Week 47: number analyzed (Participants) | 254
  >65 years: Week 47 | 1
  >65 years: Week 48: number analyzed (Participants) | 183
  >65 years: Week 48 | 1

38. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis (Cumulative).
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 3
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 6
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 8
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 13
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 13
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 13
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 14
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 16
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 16
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 3
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 7
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 9
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 13
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 16
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 18
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 18
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 23
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 23
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 24
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 12
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 18
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 27
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 33
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 33
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 38
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 42
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 48
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 49
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 54
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 365
  18-65 years: Week 38 | 11
  18-65 years: Week 39: number analyzed (Participants) | 1146
  18-65 years: Week 39 | 29
  18-65 years: Week 40: number analyzed (Participants) | 1821
  18-65 years: Week 40 | 51
  18-65 years: Week 41: number analyzed (Participants) | 2636
  18-65 years: Week 41 | 63
  18-65 years: Week 42: number analyzed (Participants) | 3122
  18-65 years: Week 42 | 81
  18-65 years: Week 43: number analyzed (Participants) | 3395
  18-65 years: Week 43 | 86
  18-65 years: Week 44: number analyzed (Participants) | 3673
  18-65 years: Week 44 | 89
  18-65 years: Week 45: number analyzed (Participants) | 3977
  18-65 years: Week 45 | 96
  18-65 years: Week 46: number analyzed (Participants) | 4402
  18-65 years: Week 46 | 99
  18-65 years: Week 47: number analyzed (Participants) | 4619
  18-65 years: Week 47 | 100
  18-65 years: Week 48: number analyzed (Participants) | 4794
  18-65 years: Week 48 | 100
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 902
  >65 years: Week 38 | 16
  >65 years: Week 39: number analyzed (Participants) | 2739
  >65 years: Week 39 | 58
  >65 years: Week 40: number analyzed (Participants) | 4198
  >65 years: Week 40 | 100
  >65 years: Week 41: number analyzed (Participants) | 5827
  >65 years: Week 41 | 120
  >65 years: Week 42: number analyzed (Participants) | 6691
  >65 years: Week 42 | 135
  >65 years: Week 43: number analyzed (Participants) | 7148
  >65 years: Week 43 | 137
  >65 years: Week 44: number analyzed (Participants) | 7632
  >65 years: Week 44 | 143
  >65 years: Week 45: number analyzed (Participants) | 8028
  >65 years: Week 45 | 149
  >65 years: Week 46: number analyzed (Participants) | 8536
  >65 years: Week 46 | 153
  >65 years: Week 47: number analyzed (Participants) | 8790
  >65 years: Week 47 | 154
  >65 years: Week 48: number analyzed (Participants) | 8973
  >65 years: Week 48 | 155

39. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis.
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 2
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 3
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 2
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 5
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 0
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 0
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 1
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 2
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 0
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 2
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 4
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 2
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 4
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 3
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 2
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 0
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 5
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 0
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 1
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 5
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 6
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 9
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 6
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 0
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 5
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 4
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 6
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 1
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 5
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 363
  18-65 years: Week 38 | 9
  18-65 years: Week 39: number analyzed (Participants) | 781
  18-65 years: Week 39 | 20
  18-65 years: Week 40: number analyzed (Participants) | 675
  18-65 years: Week 40 | 17
  18-65 years: Week 41: number analyzed (Participants) | 815
  18-65 years: Week 41 | 8
  18-65 years: Week 42: number analyzed (Participants) | 486
  18-65 years: Week 42 | 8
  18-65 years: Week 43: number analyzed (Participants) | 273
  18-65 years: Week 43 | 6
  18-65 years: Week 44: number analyzed (Participants) | 278
  18-65 years: Week 44 | 1
  18-65 years: Week 45: number analyzed (Participants) | 304
  18-65 years: Week 45 | 7
  18-65 years: Week 46: number analyzed (Participants) | 425
  18-65 years: Week 46 | 1
  18-65 years: Week 47: number analyzed (Participants) | 217
  18-65 years: Week 47 | 0
  18-65 years: Week 48: number analyzed (Participants) | 175
  18-65 years: Week 48 | 1
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 898
  >65 years: Week 38 | 10
  >65 years: Week 39: number analyzed (Participants) | 1837
  >65 years: Week 39 | 28
  >65 years: Week 40: number analyzed (Participants) | 1459
  >65 years: Week 40 | 25
  >65 years: Week 41: number analyzed (Participants) | 1629
  >65 years: Week 41 | 17
  >65 years: Week 42: number analyzed (Participants) | 864
  >65 years: Week 42 | 7
  >65 years: Week 43: number analyzed (Participants) | 457
  >65 years: Week 43 | 4
  >65 years: Week 44: number analyzed (Participants) | 484
  >65 years: Week 44 | 4
  >65 years: Week 45: number analyzed (Participants) | 396
  >65 years: Week 45 | 3
  >65 years: Week 46: number analyzed (Participants) | 508
  >65 years: Week 46 | 2
  >65 years: Week 47: number analyzed (Participants) | 254
  >65 years: Week 47 | 0
  >65 years: Week 48: number analyzed (Participants) | 183
  >65 years: Week 48 | 0

40. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Age-strata, on a Weekly Basis (Cumulative).
Description: as for outcome 21
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  6 months - 5 years: Week 37: number analyzed (Participants) | 0
  6 months - 5 years: Week 37 | 0
  6 months - 5 years: Week 38: number analyzed (Participants) | 0
  6 months - 5 years: Week 38 | 0
  6 months - 5 years: Week 39: number analyzed (Participants) | 1
  6 months - 5 years: Week 39 | 0
  6 months - 5 years: Week 40: number analyzed (Participants) | 3
  6 months - 5 years: Week 40 | 0
  6 months - 5 years: Week 41: number analyzed (Participants) | 6
  6 months - 5 years: Week 41 | 0
  6 months - 5 years: Week 42: number analyzed (Participants) | 8
  6 months - 5 years: Week 42 | 0
  6 months - 5 years: Week 43: number analyzed (Participants) | 13
  6 months - 5 years: Week 43 | 0
  6 months - 5 years: Week 44: number analyzed (Participants) | 13
  6 months - 5 years: Week 44 | 0
  6 months - 5 years: Week 45: number analyzed (Participants) | 13
  6 months - 5 years: Week 45 | 0
  6 months - 5 years: Week 46: number analyzed (Participants) | 14
  6 months - 5 years: Week 46 | 0
  6 months - 5 years: Week 47: number analyzed (Participants) | 16
  6 months - 5 years: Week 47 | 0
  6 months - 5 years: Week 48: number analyzed (Participants) | 16
  6 months - 5 years: Week 48 | 0
  6-12 years: Week 37: number analyzed (Participants) | 0
  6-12 years: Week 37 | 0
  6-12 years: Week 38: number analyzed (Participants) | 1
  6-12 years: Week 38 | 0
  6-12 years: Week 39: number analyzed (Participants) | 3
  6-12 years: Week 39 | 0
  6-12 years: Week 40: number analyzed (Participants) | 7
  6-12 years: Week 40 | 0
  6-12 years: Week 41: number analyzed (Participants) | 9
  6-12 years: Week 41 | 0
  6-12 years: Week 42: number analyzed (Participants) | 13
  6-12 years: Week 42 | 0
  6-12 years: Week 43: number analyzed (Participants) | 16
  6-12 years: Week 43 | 0
  6-12 years: Week 44: number analyzed (Participants) | 18
  6-12 years: Week 44 | 0
  6-12 years: Week 45: number analyzed (Participants) | 18
  6-12 years: Week 45 | 0
  6-12 years: Week 46: number analyzed (Participants) | 23
  6-12 years: Week 46 | 0
  6-12 years: Week 47: number analyzed (Participants) | 23
  6-12 years: Week 47 | 0
  6-12 years: Week 48: number analyzed (Participants) | 24
  6-12 years: Week 48 | 0
  13-17 years: Week 37: number analyzed (Participants) | 0
  13-17 years: Week 37 | 0
  13-17 years: Week 38: number analyzed (Participants) | 7
  13-17 years: Week 38 | 0
  13-17 years: Week 39: number analyzed (Participants) | 12
  13-17 years: Week 39 | 0
  13-17 years: Week 40: number analyzed (Participants) | 18
  13-17 years: Week 40 | 0
  13-17 years: Week 41: number analyzed (Participants) | 27
  13-17 years: Week 41 | 0
  13-17 years: Week 42: number analyzed (Participants) | 33
  13-17 years: Week 42 | 0
  13-17 years: Week 43: number analyzed (Participants) | 33
  13-17 years: Week 43 | 0
  13-17 years: Week 44: number analyzed (Participants) | 38
  13-17 years: Week 44 | 0
  13-17 years: Week 45: number analyzed (Participants) | 42
  13-17 years: Week 45 | 0
  13-17 years: Week 46: number analyzed (Participants) | 48
  13-17 years: Week 46 | 0
  13-17 years: Week 47: number analyzed (Participants) | 49
  13-17 years: Week 47 | 0
  13-17 years: Week 48: number analyzed (Participants) | 54
  13-17 years: Week 48 | 0
  18-65 years: Week 37: number analyzed (Participants) | 2
  18-65 years: Week 37 | 0
  18-65 years: Week 38: number analyzed (Participants) | 365
  18-65 years: Week 38 | 9
  18-65 years: Week 39: number analyzed (Participants) | 1146
  18-65 years: Week 39 | 29
  18-65 years: Week 40: number analyzed (Participants) | 1821
  18-65 years: Week 40 | 46
  18-65 years: Week 41: number analyzed (Participants) | 2636
  18-65 years: Week 41 | 54
  18-65 years: Week 42: number analyzed (Participants) | 3122
  18-65 years: Week 42 | 62
  18-65 years: Week 43: number analyzed (Participants) | 3395
  18-65 years: Week 43 | 68
  18-65 years: Week 44: number analyzed (Participants) | 3673
  18-65 years: Week 44 | 69
  18-65 years: Week 45: number analyzed (Participants) | 3977
  18-65 years: Week 45 | 76
  18-65 years: Week 46: number analyzed (Participants) | 4402
  18-65 years: Week 46 | 77
  18-65 years: Week 47: number analyzed (Participants) | 4619
  18-65 years: Week 47 | 77
  18-65 years: Week 48: number analyzed (Participants) | 4794
  18-65 years: Week 48 | 78
  >65 years: Week 37: number analyzed (Participants) | 4
  >65 years: Week 37 | 0
  >65 years: Week 38: number analyzed (Participants) | 902
  >65 years: Week 38 | 10
  >65 years: Week 39: number analyzed (Participants) | 2739
  >65 years: Week 39 | 38
  >65 years: Week 40: number analyzed (Participants) | 4198
  >65 years: Week 40 | 63
  >65 years: Week 41: number analyzed (Participants) | 5827
  >65 years: Week 41 | 80
  >65 years: Week 42: number analyzed (Participants) | 6691
  >65 years: Week 42 | 87
  >65 years: Week 43: number analyzed (Participants) | 7148
  >65 years: Week 43 | 91
  >65 years: Week 44: number analyzed (Participants) | 7632
  >65 years: Week 44 | 95
  >65 years: Week 45: number analyzed (Participants) | 8028
  >65 years: Week 45 | 98
  >65 years: Week 46: number analyzed (Participants) | 8536
  >65 years: Week 46 | 100
  >65 years: Week 47: number analyzed (Participants) | 8790
  >65 years: Week 47 | 100
  >65 years: Week 48: number analyzed (Participants) | 8973
  >65 years: Week 48 | 100

41. Primary Outcome: Number of Subjects Reporting EMA Defined Any AEIs and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis.
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At Risk: Week 37: number analyzed (Participants) | 6
  At Risk: Week 37 | 0
  At Risk: Week 38: number analyzed (Participants) | 1188
  At Risk: Week 38 | 62
  At Risk: Week 39: number analyzed (Participants) | 2432
  At Risk: Week 39 | 159
  At Risk: Week 40: number analyzed (Participants) | 1980
  At Risk: Week 40 | 151
  At Risk: Week 41: number analyzed (Participants) | 2246
  At Risk: Week 41 | 102
  At Risk: Week 42: number analyzed (Participants) | 1230
  At Risk: Week 42 | 74
  At Risk: Week 43: number analyzed (Participants) | 669
  At Risk: Week 43 | 29
  At Risk: Week 44: number analyzed (Participants) | 692
  At Risk: Week 44 | 28
  At Risk: Week 45: number analyzed (Participants) | 613
  At Risk: Week 45 | 25
  At Risk: Week 46: number analyzed (Participants) | 820
  At Risk: Week 46 | 11
  At Risk: Week 47: number analyzed (Participants) | 401
  At Risk: Week 47 | 2
  At Risk: Week 48: number analyzed (Participants) | 314
  At Risk: Week 48 | 1
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 5
  Not at risk: Week 39: number analyzed (Participants) | 194
  Not at risk: Week 39 | 10
  Not at risk: Week 40: number analyzed (Participants) | 166
  Not at risk: Week 40 | 13
  Not at risk: Week 41: number analyzed (Participants) | 212
  Not at risk: Week 41 | 10
  Not at risk: Week 42: number analyzed (Participants) | 132
  Not at risk: Week 42 | 11
  Not at risk: Week 43: number analyzed (Participants) | 69
  Not at risk: Week 43 | 0
  Not at risk: Week 44: number analyzed (Participants) | 77
  Not at risk: Week 44 | 3
  Not at risk: Week 45: number analyzed (Participants) | 91
  Not at risk: Week 45 | 3
  Not at risk: Week 46: number analyzed (Participants) | 125
  Not at risk: Week 46 | 2
  Not at risk: Week 47: number analyzed (Participants) | 73
  Not at risk: Week 47 | 1
  Not at risk: Week 48: number analyzed (Participants) | 50
  Not at risk: Week 48 | 1

42. Primary Outcome: Number of Subjects Reporting EMA Defined Any AEIs and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1194
  At risk: Week 38 | 62
  At risk: Week 39: number analyzed (Participants) | 3626
  At risk: Week 39 | 221
  At risk: Week 40: number analyzed (Participants) | 5606
  At risk: Week 40 | 372
  At risk: Week 41: number analyzed (Participants) | 7852
  At risk: Week 41 | 474
  At risk: Week 42: number analyzed (Participants) | 9082
  At risk: Week 42 | 548
  At risk: Week 43: number analyzed (Participants) | 9751
  At risk: Week 43 | 577
  At risk: Week 44: number analyzed (Participants) | 10443
  At risk: Week 44 | 605
  At risk: Week 45: number analyzed (Participants) | 11056
  At risk: Week 45 | 630
  At risk: Week 46: number analyzed (Participants) | 11876
  At risk: Week 46 | 641
  At risk: Week 47: number analyzed (Participants) | 12277
  At risk: Week 47 | 643
  At risk: Week 48: number analyzed (Participants) | 12591
  At risk: Week 48 | 644
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 5
  Not at risk: Week 39: number analyzed (Participants) | 275
  Not at risk: Week 39 | 15
  Not at risk: Week 40: number analyzed (Participants) | 441
  Not at risk: Week 40 | 28
  Not at risk: Week 41: number analyzed (Participants) | 653
  Not at risk: Week 41 | 38
  Not at risk: Week 42: number analyzed (Participants) | 785
  Not at risk: Week 42 | 49
  Not at risk: Week 43: number analyzed (Participants) | 854
  Not at risk: Week 43 | 49
  Not at risk: Week 44: number analyzed (Participants) | 931
  Not at risk: Week 44 | 52
  Not at risk: Week 45: number analyzed (Participants) | 1022
  Not at risk: Week 45 | 55
  Not at risk: Week 46: number analyzed (Participants) | 1147
  Not at risk: Week 46 | 57
  Not at risk: Week 47: number analyzed (Participants) | 1220
  Not at risk: Week 47 | 58
  Not at risk: Week 48: number analyzed (Participants) | 1270
  Not at risk: Week 48 | 59

43. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis.
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1188
  At risk: Week 38 | 4
  At risk: Week 39: number analyzed (Participants) | 2432
  At risk: Week 39 | 15
  At risk: Week 40: number analyzed (Participants) | 1980
  At risk: Week 40 | 8
  At risk: Week 41: number analyzed (Participants) | 2246
  At risk: Week 41 | 8
  At risk: Week 42: number analyzed (Participants) | 1230
  At risk: Week 42 | 8
  At risk: Week 43: number analyzed (Participants) | 669
  At risk: Week 43 | 3
  At risk: Week 44: number analyzed (Participants) | 692
  At risk: Week 44 | 2
  At risk: Week 45: number analyzed (Participants) | 613
  At risk: Week 45 | 3
  At risk: Week 46: number analyzed (Participants) | 820
  At risk: Week 46 | 4
  At risk: Week 47: number analyzed (Participants) | 401
  At risk: Week 47 | 0
  At risk: Week 48: number analyzed (Participants) | 314
  At risk: Week 48 | 0
  Not at risk: Week 37: number analyzed (Participants) | 37
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 0
  Not at risk: Week 39: number analyzed (Participants) | 194
  Not at risk: Week 39 | 0
  Not at risk: Week 40: number analyzed (Participants) | 166
  Not at risk: Week 40 | 0
  Not at risk: Week 41: number analyzed (Participants) | 212
  Not at risk: Week 41 | 2
  Not at risk: Week 42: number analyzed (Participants) | 132
  Not at risk: Week 42 | 1
  Not at risk: Week 43: number analyzed (Participants) | 69
  Not at risk: Week 43 | 0
  Not at risk: Week 44: number analyzed (Participants) | 77
  Not at risk: Week 44 | 0
  Not at risk: Week 45: number analyzed (Participants) | 91
  Not at risk: Week 45 | 0
  Not at risk: Week 46: number analyzed (Participants) | 125
  Not at risk: Week 46 | 0
  Not at risk: Week 47: number analyzed (Participants) | 73
  Not at risk: Week 47 | 0
  Not at risk: Week 48: number analyzed (Participants) | 50
  Not at risk: Week 48 | 0

44. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1194
  At risk: Week 38 | 4
  At risk: Week 39: number analyzed (Participants) | 3626
  At risk: Week 39 | 19
  At risk: Week 40: number analyzed (Participants) | 5606
  At risk: Week 40 | 27
  At risk: Week 41: number analyzed (Participants) | 7852
  At risk: Week 41 | 35
  At risk: Week 42: number analyzed (Participants) | 9082
  At risk: Week 42 | 43
  At risk: Week 43: number analyzed (Participants) | 9751
  At risk: Week 43 | 46
  At risk: Week 44: number analyzed (Participants) | 10443
  At risk: Week 44 | 48
  At risk: Week 45: number analyzed (Participants) | 11056
  At risk: Week 45 | 51
  At risk: Week 46: number analyzed (Participants) | 11876
  At risk: Week 46 | 55
  At risk: Week 47: number analyzed (Participants) | 12277
  At risk: Week 47 | 55
  At risk: Week 48: number analyzed (Participants) | 12591
  At risk: Week 48 | 55
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 0
  Not at risk: Week 39: number analyzed (Participants) | 275
  Not at risk: Week 39 | 0
  Not at risk: Week 40: number analyzed (Participants) | 441
  Not at risk: Week 40 | 0
  Not at risk: Week 41: number analyzed (Participants) | 653
  Not at risk: Week 41 | 2
  Not at risk: Week 42: number analyzed (Participants) | 785
  Not at risk: Week 42 | 3
  Not at risk: Week 43: number analyzed (Participants) | 854
  Not at risk: Week 43 | 3
  Not at risk: Week 44: number analyzed (Participants) | 931
  Not at risk: Week 44 | 3
  Not at risk: Week 45: number analyzed (Participants) | 1022
  Not at risk: Week 45 | 3
  Not at risk: Week 46: number analyzed (Participants) | 1147
  Not at risk: Week 46 | 3
  Not at risk: Week 47: number analyzed (Participants) | 1220
  Not at risk: Week 47 | 3
  Not at risk: Week 48: number analyzed (Participants) | 1270
  Not at risk: Week 48 | 3

45. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis.
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1188
  At risk: Week 38 | 14
  At risk: Week 39: number analyzed (Participants) | 2432
  At risk: Week 39 | 19
  At risk: Week 40: number analyzed (Participants) | 1980
  At risk: Week 40 | 21
  At risk: Week 41: number analyzed (Participants) | 2246
  At risk: Week 41 | 26
  At risk: Week 42: number analyzed (Participants) | 1230
  At risk: Week 42 | 13
  At risk: Week 43: number analyzed (Participants) | 669
  At risk: Week 43 | 6
  At risk: Week 44: number analyzed (Participants) | 692
  At risk: Week 44 | 5
  At risk: Week 45: number analyzed (Participants) | 613
  At risk: Week 45 | 8
  At risk: Week 46: number analyzed (Participants) | 820
  At risk: Week 46 | 2
  At risk: Week 47: number analyzed (Participants) | 401
  At risk: Week 47 | 0
  At risk: Week 48: number analyzed (Participants) | 314
  At risk: Week 48 | 0
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 2
  Not at risk: Week 39: number analyzed (Participants) | 194
  Not at risk: Week 39 | 1
  Not at risk: Week 40: number analyzed (Participants) | 166
  Not at risk: Week 40 | 3
  Not at risk: Week 41: number analyzed (Participants) | 212
  Not at risk: Week 41 | 2
  Not at risk: Week 42: number analyzed (Participants) | 132
  Not at risk: Week 42 | 2
  Not at risk: Week 43: number analyzed (Participants) | 69
  Not at risk: Week 43 | 0
  Not at risk: Week 44: number analyzed (Participants) | 77
  Not at risk: Week 44 | 2
  Not at risk: Week 45: number analyzed (Participants) | 91
  Not at risk: Week 45 | 0
  Not at risk: Week 46: number analyzed (Participants) | 125
  Not at risk: Week 46 | 1
  Not at risk: Week 47: number analyzed (Participants) | 73
  Not at risk: Week 47 | 0
  Not at risk: Week 48: number analyzed (Participants) | 50
  Not at risk: Week 48 | 0

46. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1194
  At risk: Week 38 | 14
  At risk: Week 39: number analyzed (Participants) | 3626
  At risk: Week 39 | 33
  At risk: Week 40: number analyzed (Participants) | 5606
  At risk: Week 40 | 54
  At risk: Week 41: number analyzed (Participants) | 7852
  At risk: Week 41 | 80
  At risk: Week 42: number analyzed (Participants) | 9082
  At risk: Week 42 | 93
  At risk: Week 43: number analyzed (Participants) | 9751
  At risk: Week 43 | 99
  At risk: Week 44: number analyzed (Participants) | 10443
  At risk: Week 44 | 104
  At risk: Week 45: number analyzed (Participants) | 11056
  At risk: Week 45 | 112
  At risk: Week 46: number analyzed (Participants) | 11876
  At risk: Week 46 | 114
  At risk: Week 47: number analyzed (Participants) | 12277
  At risk: Week 47 | 114
  At risk: Week 48: number analyzed (Participants) | 12591
  At risk: Week 48 | 114
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 2
  Not at risk: Week 39: number analyzed (Participants) | 275
  Not at risk: Week 39 | 3
  Not at risk: Week 40: number analyzed (Participants) | 441
  Not at risk: Week 40 | 6
  Not at risk: Week 41: number analyzed (Participants) | 653
  Not at risk: Week 41 | 8
  Not at risk: Week 42: number analyzed (Participants) | 785
  Not at risk: Week 42 | 10
  Not at risk: Week 43: number analyzed (Participants) | 854
  Not at risk: Week 43 | 10
  Not at risk: Week 44: number analyzed (Participants) | 931
  Not at risk: Week 44 | 12
  Not at risk: Week 45: number analyzed (Participants) | 1022
  Not at risk: Week 45 | 12
  Not at risk: Week 46: number analyzed (Participants) | 1147
  Not at risk: Week 46 | 13
  Not at risk: Week 47: number analyzed (Participants) | 1220
  Not at risk: Week 47 | 13
  Not at risk: Week 48: number analyzed (Participants) | 1270
  Not at risk: Week 48 | 13

47. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (General Non-specific Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis.
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1188
  At risk: Week 38 | 18
  At risk: Week 39: number analyzed (Participants) | 2432
  At risk: Week 39 | 42
  At risk: Week 40: number analyzed (Participants) | 1980
  At risk: Week 40 | 41
  At risk: Week 41: number analyzed (Participants) | 2246
  At risk: Week 41 | 25
  At risk: Week 42: number analyzed (Participants) | 1230
  At risk: Week 42 | 18
  At risk: Week 43: number analyzed (Participants) | 669
  At risk: Week 43 | 3
  At risk: Week 44: number analyzed (Participants) | 692
  At risk: Week 44 | 6
  At risk: Week 45: number analyzed (Participants) | 613
  At risk: Week 45 | 7
  At risk: Week 46: number analyzed (Participants) | 820
  At risk: Week 46 | 5
  At risk: Week 47: number analyzed (Participants) | 401
  At risk: Week 47 | 2
  At risk: Week 48: number analyzed (Participants) | 314
  At risk: Week 48 | 0
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 2
  Not at risk: Week 39: number analyzed (Participants) | 194
  Not at risk: Week 39 | 5
  Not at risk: Week 40: number analyzed (Participants) | 166
  Not at risk: Week 40 | 2
  Not at risk: Week 41: number analyzed (Participants) | 212
  Not at risk: Week 41 | 0
  Not at risk: Week 42: number analyzed (Participants) | 132
  Not at risk: Week 42 | 2
  Not at risk: Week 43: number analyzed (Participants) | 69
  Not at risk: Week 43 | 0
  Not at risk: Week 44: number analyzed (Participants) | 77
  Not at risk: Week 44 | 0
  Not at risk: Week 45: number analyzed (Participants) | 91
  Not at risk: Week 45 | 2
  Not at risk: Week 46: number analyzed (Participants) | 125
  Not at risk: Week 46 | 1
  Not at risk: Week 47: number analyzed (Participants) | 73
  Not at risk: Week 47 | 0
  Not at risk: Week 48: number analyzed (Participants) | 50
  Not at risk: Week 48 | 1

48. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (General Non-specific Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis (Cumulative)
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1194
  At risk: Week 38 | 18
  At risk: Week 39: number analyzed (Participants) | 3626
  At risk: Week 39 | 60
  At risk: Week 40: number analyzed (Participants) | 5606
  At risk: Week 40 | 101
  At risk: Week 41: number analyzed (Participants) | 7852
  At risk: Week 41 | 126
  At risk: Week 42: number analyzed (Participants) | 9082
  At risk: Week 42 | 144
  At risk: Week 43: number analyzed (Participants) | 9751
  At risk: Week 43 | 147
  At risk: Week 44: number analyzed (Participants) | 10443
  At risk: Week 44 | 153
  At risk: Week 45: number analyzed (Participants) | 11056
  At risk: Week 45 | 160
  At risk: Week 46: number analyzed (Participants) | 11876
  At risk: Week 46 | 165
  At risk: Week 47: number analyzed (Participants) | 12277
  At risk: Week 47 | 167
  At risk: Week 48: number analyzed (Participants) | 12591
  At risk: Week 48 | 167
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 2
  Not at risk: Week 39: number analyzed (Participants) | 275
  Not at risk: Week 39 | 7
  Not at risk: Week 40: number analyzed (Participants) | 441
  Not at risk: Week 40 | 9
  Not at risk: Week 41: number analyzed (Participants) | 653
  Not at risk: Week 41 | 9
  Not at risk: Week 42: number analyzed (Participants) | 785
  Not at risk: Week 42 | 11
  Not at risk: Week 43: number analyzed (Participants) | 854
  Not at risk: Week 43 | 11
  Not at risk: Week 44: number analyzed (Participants) | 931
  Not at risk: Week 44 | 11
  Not at risk: Week 45: number analyzed (Participants) | 1022
  Not at risk: Week 45 | 13
  Not at risk: Week 46: number analyzed (Participants) | 1147
  Not at risk: Week 46 | 14
  Not at risk: Week 47: number analyzed (Participants) | 1220
  Not at risk: Week 47 | 14
  Not at risk: Week 48: number analyzed (Participants) | 1270
  Not at risk: Week 48 | 15

49. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Respiratory/Miscellaneous AEs) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis.
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1188
  At risk: Week 38 | 28
  At risk: Week 39: number analyzed (Participants) | 2432
  At risk: Week 39 | 94
  At risk: Week 40: number analyzed (Participants) | 1980
  At risk: Week 40 | 88
  At risk: Week 41: number analyzed (Participants) | 2246
  At risk: Week 41 | 62
  At risk: Week 42: number analyzed (Participants) | 1230
  At risk: Week 42 | 49
  At risk: Week 43: number analyzed (Participants) | 669
  At risk: Week 43 | 22
  At risk: Week 44: number analyzed (Participants) | 692
  At risk: Week 44 | 12
  At risk: Week 45: number analyzed (Participants) | 613
  At risk: Week 45 | 16
  At risk: Week 46: number analyzed (Participants) | 820
  At risk: Week 46 | 5
  At risk: Week 47: number analyzed (Participants) | 401
  At risk: Week 47 | 1
  At risk: Week 48: number analyzed (Participants) | 314
  At risk: Week 48 | 0
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 2
  Not at risk: Week 39: number analyzed (Participants) | 194
  Not at risk: Week 39 | 6
  Not at risk: Week 40: number analyzed (Participants) | 166
  Not at risk: Week 40 | 7
  Not at risk: Week 41: number analyzed (Participants) | 212
  Not at risk: Week 41 | 2
  Not at risk: Week 42: number analyzed (Participants) | 132
  Not at risk: Week 42 | 9
  Not at risk: Week 43: number analyzed (Participants) | 69
  Not at risk: Week 43 | 0
  Not at risk: Week 44: number analyzed (Participants) | 77
  Not at risk: Week 44 | 1
  Not at risk: Week 45: number analyzed (Participants) | 91
  Not at risk: Week 45 | 3
  Not at risk: Week 46: number analyzed (Participants) | 125
  Not at risk: Week 46 | 0
  Not at risk: Week 47: number analyzed (Participants) | 73
  Not at risk: Week 47 | 1
  Not at risk: Week 48: number analyzed (Participants) | 50
  Not at risk: Week 48 | 0

50. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Respiratory/Miscellaneous AEs) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1194
  At risk: Week 38 | 28
  At risk: Week 39: number analyzed (Participants) | 3626
  At risk: Week 39 | 122
  At risk: Week 40: number analyzed (Participants) | 5606
  At risk: Week 40 | 210
  At risk: Week 41: number analyzed (Participants) | 7852
  At risk: Week 41 | 272
  At risk: Week 42: number analyzed (Participants) | 9082
  At risk: Week 42 | 321
  At risk: Week 43: number analyzed (Participants) | 9751
  At risk: Week 43 | 343
  At risk: Week 44: number analyzed (Participants) | 10443
  At risk: Week 44 | 355
  At risk: Week 45: number analyzed (Participants) | 11056
  At risk: Week 45 | 371
  At risk: Week 46: number analyzed (Participants) | 11876
  At risk: Week 46 | 376
  At risk: Week 47: number analyzed (Participants) | 12277
  At risk: Week 47 | 377
  At risk: Week 48: number analyzed (Participants) | 12591
  At risk: Week 48 | 377
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 2
  Not at risk: Week 39: number analyzed (Participants) | 275
  Not at risk: Week 39 | 8
  Not at risk: Week 40: number analyzed (Participants) | 441
  Not at risk: Week 40 | 15
  Not at risk: Week 41: number analyzed (Participants) | 653
  Not at risk: Week 41 | 17
  Not at risk: Week 42: number analyzed (Participants) | 785
  Not at risk: Week 42 | 26
  Not at risk: Week 43: number analyzed (Participants) | 854
  Not at risk: Week 43 | 26
  Not at risk: Week 44: number analyzed (Participants) | 931
  Not at risk: Week 44 | 27
  Not at risk: Week 45: number analyzed (Participants) | 1022
  Not at risk: Week 45 | 30
  Not at risk: Week 46: number analyzed (Participants) | 1147
  Not at risk: Week 46 | 30
  Not at risk: Week 47: number analyzed (Participants) | 1220
  Not at risk: Week 47 | 31
  Not at risk: Week 48: number analyzed (Participants) | 1270
  Not at risk: Week 48 | 31

51. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Gastrointestinal AEs) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis.
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1188
  At risk: Week 38 | 13
  At risk: Week 39: number analyzed (Participants) | 2432
  At risk: Week 39 | 27
  At risk: Week 40: number analyzed (Participants) | 1980
  At risk: Week 40 | 28
  At risk: Week 41: number analyzed (Participants) | 2246
  At risk: Week 41 | 18
  At risk: Week 42: number analyzed (Participants) | 1230
  At risk: Week 42 | 17
  At risk: Week 43: number analyzed (Participants) | 669
  At risk: Week 43 | 6
  At risk: Week 44: number analyzed (Participants) | 692
  At risk: Week 44 | 4
  At risk: Week 45: number analyzed (Participants) | 613
  At risk: Week 45 | 5
  At risk: Week 46: number analyzed (Participants) | 820
  At risk: Week 46 | 3
  At risk: Week 47: number analyzed (Participants) | 401
  At risk: Week 47 | 0
  At risk: Week 48: number analyzed (Participants) | 314
  At risk: Week 48 | 0
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 2
  Not at risk: Week 39: number analyzed (Participants) | 194
  Not at risk: Week 39 | 2
  Not at risk: Week 40: number analyzed (Participants) | 166
  Not at risk: Week 40 | 1
  Not at risk: Week 41: number analyzed (Participants) | 212
  Not at risk: Week 41 | 3
  Not at risk: Week 42: number analyzed (Participants) | 132
  Not at risk: Week 42 | 1
  Not at risk: Week 43: number analyzed (Participants) | 69
  Not at risk: Week 43 | 0
  Not at risk: Week 44: number analyzed (Participants) | 77
  Not at risk: Week 44 | 0
  Not at risk: Week 45: number analyzed (Participants) | 91
  Not at risk: Week 45 | 0
  Not at risk: Week 46: number analyzed (Participants) | 125
  Not at risk: Week 46 | 0
  Not at risk: Week 47: number analyzed (Participants) | 73
  Not at risk: Week 47 | 0
  Not at risk: Week 48: number analyzed (Participants) | 50
  Not at risk: Week 48 | 1

52. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Gastrointestinal AEs) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1194
  At risk: Week 38 | 13
  At risk: Week 39: number analyzed (Participants) | 3626
  At risk: Week 39 | 40
  At risk: Week 40: number analyzed (Participants) | 5606
  At risk: Week 40 | 68
  At risk: Week 41: number analyzed (Participants) | 7852
  At risk: Week 41 | 86
  At risk: Week 42: number analyzed (Participants) | 9082
  At risk: Week 42 | 103
  At risk: Week 43: number analyzed (Participants) | 9751
  At risk: Week 43 | 109
  At risk: Week 44: number analyzed (Participants) | 10443
  At risk: Week 44 | 113
  At risk: Week 45: number analyzed (Participants) | 11056
  At risk: Week 45 | 118
  At risk: Week 46: number analyzed (Participants) | 11876
  At risk: Week 46 | 121
  At risk: Week 47: number analyzed (Participants) | 12277
  At risk: Week 47 | 121
  At risk: Week 48: number analyzed (Participants) | 12591
  At risk: Week 48 | 121
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 2
  Not at risk: Week 39: number analyzed (Participants) | 275
  Not at risk: Week 39 | 4
  Not at risk: Week 40: number analyzed (Participants) | 441
  Not at risk: Week 40 | 5
  Not at risk: Week 41: number analyzed (Participants) | 653
  Not at risk: Week 41 | 8
  Not at risk: Week 42: number analyzed (Participants) | 785
  Not at risk: Week 42 | 9
  Not at risk: Week 43: number analyzed (Participants) | 854
  Not at risk: Week 43 | 9
  Not at risk: Week 44: number analyzed (Participants) | 931
  Not at risk: Week 44 | 9
  Not at risk: Week 45: number analyzed (Participants) | 1022
  Not at risk: Week 45 | 9
  Not at risk: Week 46: number analyzed (Participants) | 1147
  Not at risk: Week 46 | 9
  Not at risk: Week 47: number analyzed (Participants) | 1220
  Not at risk: Week 47 | 9
  Not at risk: Week 48: number analyzed (Participants) | 1270
  Not at risk: Week 48 | 10

53. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Sensitivity/Anaphylaxis AEs) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis.
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1188
  At risk: Week 38 | 0
  At risk: Week 39: number analyzed (Participants) | 2432
  At risk: Week 39 | 0
  At risk: Week 40: number analyzed (Participants) | 1980
  At risk: Week 40 | 3
  At risk: Week 41: number analyzed (Participants) | 2246
  At risk: Week 41 | 0
  At risk: Week 42: number analyzed (Participants) | 1230
  At risk: Week 42 | 1
  At risk: Week 43: number analyzed (Participants) | 669
  At risk: Week 43 | 0
  At risk: Week 44: number analyzed (Participants) | 692
  At risk: Week 44 | 1
  At risk: Week 45: number analyzed (Participants) | 613
  At risk: Week 45 | 1
  At risk: Week 46: number analyzed (Participants) | 820
  At risk: Week 46 | 0
  At risk: Week 47: number analyzed (Participants) | 401
  At risk: Week 47 | 0
  At risk: Week 48: number analyzed (Participants) | 314
  At risk: Week 48 | 0
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 0
  Not at risk: Week 39: number analyzed (Participants) | 194
  Not at risk: Week 39 | 0
  Not at risk: Week 40: number analyzed (Participants) | 166
  Not at risk: Week 40 | 0
  Not at risk: Week 41: number analyzed (Participants) | 212
  Not at risk: Week 41 | 0
  Not at risk: Week 42: number analyzed (Participants) | 132
  Not at risk: Week 42 | 1
  Not at risk: Week 43: number analyzed (Participants) | 69
  Not at risk: Week 43 | 0
  Not at risk: Week 44: number analyzed (Participants) | 77
  Not at risk: Week 44 | 0
  Not at risk: Week 45: number analyzed (Participants) | 91
  Not at risk: Week 45 | 0
  Not at risk: Week 46: number analyzed (Participants) | 125
  Not at risk: Week 46 | 0
  Not at risk: Week 47: number analyzed (Participants) | 73
  Not at risk: Week 47 | 0
  Not at risk: Week 48: number analyzed (Participants) | 50
  Not at risk: Week 48 | 0

54. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Sensitivity/Anaphylaxis AEs) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1194
  At risk: Week 38 | 0
  At risk: Week 39: number analyzed (Participants) | 3626
  At risk: Week 39 | 0
  At risk: Week 40: number analyzed (Participants) | 5606
  At risk: Week 40 | 3
  At risk: Week 41: number analyzed (Participants) | 7852
  At risk: Week 41 | 3
  At risk: Week 42: number analyzed (Participants) | 9082
  At risk: Week 42 | 4
  At risk: Week 43: number analyzed (Participants) | 9751
  At risk: Week 43 | 4
  At risk: Week 44: number analyzed (Participants) | 10443
  At risk: Week 44 | 5
  At risk: Week 45: number analyzed (Participants) | 11056
  At risk: Week 45 | 6
  At risk: Week 46: number analyzed (Participants) | 11876
  At risk: Week 46 | 6
  At risk: Week 47: number analyzed (Participants) | 12277
  At risk: Week 47 | 6
  At risk: Week 48: number analyzed (Participants) | 12591
  At risk: Week 48 | 6
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 0
  Not at risk: Week 39: number analyzed (Participants) | 275
  Not at risk: Week 39 | 0
  Not at risk: Week 40: number analyzed (Participants) | 441
  Not at risk: Week 40 | 0
  Not at risk: Week 41: number analyzed (Participants) | 653
  Not at risk: Week 41 | 0
  Not at risk: Week 42: number analyzed (Participants) | 785
  Not at risk: Week 42 | 1
  Not at risk: Week 43: number analyzed (Participants) | 854
  Not at risk: Week 43 | 1
  Not at risk: Week 44: number analyzed (Participants) | 931
  Not at risk: Week 44 | 1
  Not at risk: Week 45: number analyzed (Participants) | 1022
  Not at risk: Week 45 | 1
  Not at risk: Week 46: number analyzed (Participants) | 1147
  Not at risk: Week 46 | 1
  Not at risk: Week 47: number analyzed (Participants) | 1220
  Not at risk: Week 47 | 1
  Not at risk: Week 48: number analyzed (Participants) | 1270
  Not at risk: Week 48 | 1

55. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis.
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1188
  At risk: Week 38 | 1
  At risk: Week 39: number analyzed (Participants) | 2432
  At risk: Week 39 | 0
  At risk: Week 40: number analyzed (Participants) | 1980
  At risk: Week 40 | 5
  At risk: Week 41: number analyzed (Participants) | 2246
  At risk: Week 41 | 1
  At risk: Week 42: number analyzed (Participants) | 1230
  At risk: Week 42 | 2
  At risk: Week 43: number analyzed (Participants) | 669
  At risk: Week 43 | 3
  At risk: Week 44: number analyzed (Participants) | 692
  At risk: Week 44 | 1
  At risk: Week 45: number analyzed (Participants) | 613
  At risk: Week 45 | 1
  At risk: Week 46: number analyzed (Participants) | 820
  At risk: Week 46 | 2
  At risk: Week 47: number analyzed (Participants) | 401
  At risk: Week 47 | 0
  At risk: Week 48: number analyzed (Participants) | 314
  At risk: Week 48 | 0
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 0
  Not at risk: Week 39: number analyzed (Participants) | 194
  Not at risk: Week 39 | 0
  Not at risk: Week 40: number analyzed (Participants) | 166
  Not at risk: Week 40 | 0
  Not at risk: Week 41: number analyzed (Participants) | 212
  Not at risk: Week 41 | 0
  Not at risk: Week 42: number analyzed (Participants) | 132
  Not at risk: Week 42 | 1
  Not at risk: Week 43: number analyzed (Participants) | 69
  Not at risk: Week 43 | 0
  Not at risk: Week 44: number analyzed (Participants) | 77
  Not at risk: Week 44 | 0
  Not at risk: Week 45: number analyzed (Participants) | 91
  Not at risk: Week 45 | 0
  Not at risk: Week 46: number analyzed (Participants) | 125
  Not at risk: Week 46 | 0
  Not at risk: Week 47: number analyzed (Participants) | 73
  Not at risk: Week 47 | 0
  Not at risk: Week 48: number analyzed (Participants) | 50
  Not at risk: Week 48 | 0

56. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1194
  At risk: Week 38 | 1
  At risk: Week 39: number analyzed (Participants) | 3626
  At risk: Week 39 | 1
  At risk: Week 40: number analyzed (Participants) | 5606
  At risk: Week 40 | 6
  At risk: Week 41: number analyzed (Participants) | 7852
  At risk: Week 41 | 7
  At risk: Week 42: number analyzed (Participants) | 9082
  At risk: Week 42 | 9
  At risk: Week 43: number analyzed (Participants) | 9751
  At risk: Week 43 | 12
  At risk: Week 44: number analyzed (Participants) | 10443
  At risk: Week 44 | 13
  At risk: Week 45: number analyzed (Participants) | 11056
  At risk: Week 45 | 14
  At risk: Week 46: number analyzed (Participants) | 11876
  At risk: Week 46 | 16
  At risk: Week 47: number analyzed (Participants) | 12277
  At risk: Week 47 | 16
  At risk: Week 48: number analyzed (Participants) | 12591
  At risk: Week 48 | 16
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 0
  Not at risk: Week 39: number analyzed (Participants) | 275
  Not at risk: Week 39 | 0
  Not at risk: Week 40: number analyzed (Participants) | 441
  Not at risk: Week 40 | 0
  Not at risk: Week 41: number analyzed (Participants) | 653
  Not at risk: Week 41 | 0
  Not at risk: Week 42: number analyzed (Participants) | 785
  Not at risk: Week 42 | 1
  Not at risk: Week 43: number analyzed (Participants) | 854
  Not at risk: Week 43 | 1
  Not at risk: Week 44: number analyzed (Participants) | 931
  Not at risk: Week 44 | 1
  Not at risk: Week 45: number analyzed (Participants) | 1022
  Not at risk: Week 45 | 1
  Not at risk: Week 46: number analyzed (Participants) | 1147
  Not at risk: Week 46 | 1
  Not at risk: Week 47: number analyzed (Participants) | 1220
  Not at risk: Week 47 | 1
  Not at risk: Week 48: number analyzed (Participants) | 1270
  Not at risk: Week 48 | 1

57. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis.
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1188
  At risk: Week 38 | 24
  At risk: Week 39: number analyzed (Participants) | 2432
  At risk: Week 39 | 54
  At risk: Week 40: number analyzed (Participants) | 1980
  At risk: Week 40 | 61
  At risk: Week 41: number analyzed (Participants) | 2246
  At risk: Week 41 | 29
  At risk: Week 42: number analyzed (Participants) | 1230
  At risk: Week 42 | 31
  At risk: Week 43: number analyzed (Participants) | 669
  At risk: Week 43 | 7
  At risk: Week 44: number analyzed (Participants) | 692
  At risk: Week 44 | 9
  At risk: Week 45: number analyzed (Participants) | 613
  At risk: Week 45 | 11
  At risk: Week 46: number analyzed (Participants) | 820
  At risk: Week 46 | 5
  At risk: Week 47: number analyzed (Participants) | 401
  At risk: Week 47 | 1
  At risk: Week 48: number analyzed (Participants) | 314
  At risk: Week 48 | 1
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 3
  Not at risk: Week 39: number analyzed (Participants) | 194
  Not at risk: Week 39 | 6
  Not at risk: Week 40: number analyzed (Participants) | 166
  Not at risk: Week 40 | 3
  Not at risk: Week 41: number analyzed (Participants) | 212
  Not at risk: Week 41 | 3
  Not at risk: Week 42: number analyzed (Participants) | 132
  Not at risk: Week 42 | 2
  Not at risk: Week 43: number analyzed (Participants) | 69
  Not at risk: Week 43 | 0
  Not at risk: Week 44: number analyzed (Participants) | 77
  Not at risk: Week 44 | 0
  Not at risk: Week 45: number analyzed (Participants) | 91
  Not at risk: Week 45 | 2
  Not at risk: Week 46: number analyzed (Participants) | 125
  Not at risk: Week 46 | 2
  Not at risk: Week 47: number analyzed (Participants) | 73
  Not at risk: Week 47 | 1
  Not at risk: Week 48: number analyzed (Participants) | 50
  Not at risk: Week 48 | 0

58. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1194
  At risk: Week 38 | 24
  At risk: Week 39: number analyzed (Participants) | 3626
  At risk: Week 39 | 78
  At risk: Week 40: number analyzed (Participants) | 5606
  At risk: Week 40 | 139
  At risk: Week 41: number analyzed (Participants) | 7852
  At risk: Week 41 | 168
  At risk: Week 42: number analyzed (Participants) | 9082
  At risk: Week 42 | 199
  At risk: Week 43: number analyzed (Participants) | 9751
  At risk: Week 43 | 206
  At risk: Week 44: number analyzed (Participants) | 10443
  At risk: Week 44 | 215
  At risk: Week 45: number analyzed (Participants) | 11056
  At risk: Week 45 | 226
  At risk: Week 46: number analyzed (Participants) | 11876
  At risk: Week 46 | 231
  At risk: Week 47: number analyzed (Participants) | 12277
  At risk: Week 47 | 232
  At risk: Week 48: number analyzed (Participants) | 12591
  At risk: Week 48 | 233
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 3
  Not at risk: Week 39: number analyzed (Participants) | 275
  Not at risk: Week 39 | 9
  Not at risk: Week 40: number analyzed (Participants) | 441
  Not at risk: Week 40 | 12
  Not at risk: Week 41: number analyzed (Participants) | 653
  Not at risk: Week 41 | 15
  Not at risk: Week 42: number analyzed (Participants) | 785
  Not at risk: Week 42 | 17
  Not at risk: Week 43: number analyzed (Participants) | 854
  Not at risk: Week 43 | 17
  Not at risk: Week 44: number analyzed (Participants) | 931
  Not at risk: Week 44 | 17
  Not at risk: Week 45: number analyzed (Participants) | 1022
  Not at risk: Week 45 | 19
  Not at risk: Week 46: number analyzed (Participants) | 1147
  Not at risk: Week 46 | 21
  Not at risk: Week 47: number analyzed (Participants) | 1220
  Not at risk: Week 47 | 22
  Not at risk: Week 48: number analyzed (Participants) | 1270
  Not at risk: Week 48 | 22

59. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis.
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1188
  At risk: Week 38 | 17
  At risk: Week 39: number analyzed (Participants) | 2432
  At risk: Week 39 | 44
  At risk: Week 40: number analyzed (Participants) | 1980
  At risk: Week 40 | 37
  At risk: Week 41: number analyzed (Participants) | 2246
  At risk: Week 41 | 24
  At risk: Week 42: number analyzed (Participants) | 1230
  At risk: Week 42 | 13
  At risk: Week 43: number analyzed (Participants) | 669
  At risk: Week 43 | 10
  At risk: Week 44: number analyzed (Participants) | 692
  At risk: Week 44 | 5
  At risk: Week 45: number analyzed (Participants) | 613
  At risk: Week 45 | 8
  At risk: Week 46: number analyzed (Participants) | 820
  At risk: Week 46 | 3
  At risk: Week 47: number analyzed (Participants) | 401
  At risk: Week 47 | 0
  At risk: Week 48: number analyzed (Participants) | 314
  At risk: Week 48 | 0
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 2
  Not at risk: Week 39: number analyzed (Participants) | 194
  Not at risk: Week 39 | 4
  Not at risk: Week 40: number analyzed (Participants) | 166
  Not at risk: Week 40 | 5
  Not at risk: Week 41: number analyzed (Participants) | 212
  Not at risk: Week 41 | 1
  Not at risk: Week 42: number analyzed (Participants) | 132
  Not at risk: Week 42 | 2
  Not at risk: Week 43: number analyzed (Participants) | 69
  Not at risk: Week 43 | 0
  Not at risk: Week 44: number analyzed (Participants) | 77
  Not at risk: Week 44 | 0
  Not at risk: Week 45: number analyzed (Participants) | 91
  Not at risk: Week 45 | 2
  Not at risk: Week 46: number analyzed (Participants) | 125
  Not at risk: Week 46 | 0
  Not at risk: Week 47: number analyzed (Participants) | 73
  Not at risk: Week 47 | 0
  Not at risk: Week 48: number analyzed (Participants) | 50
  Not at risk: Week 48 | 1

60. Primary Outcome: Number of Subjects Reporting EMA Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System in the Vaccinated_Fluarix Tetra Group by CMO-specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 3
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group
Number analyzed (Participants) | 13861
Participants
  At risk: Week 37: number analyzed (Participants) | 6
  At risk: Week 37 | 0
  At risk: Week 38: number analyzed (Participants) | 1194
  At risk: Week 38 | 17
  At risk: Week 39: number analyzed (Participants) | 3626
  At risk: Week 39 | 61
  At risk: Week 40: number analyzed (Participants) | 5606
  At risk: Week 40 | 98
  At risk: Week 41: number analyzed (Participants) | 7852
  At risk: Week 41 | 122
  At risk: Week 42: number analyzed (Participants) | 9082
  At risk: Week 42 | 135
  At risk: Week 43: number analyzed (Participants) | 9751
  At risk: Week 43 | 145
  At risk: Week 44: number analyzed (Participants) | 10443
  At risk: Week 44 | 150
  At risk: Week 45: number analyzed (Participants) | 11056
  At risk: Week 45 | 158
  At risk: Week 46: number analyzed (Participants) | 11876
  At risk: Week 46 | 161
  At risk: Week 47: number analyzed (Participants) | 12277
  At risk: Week 47 | 161
  At risk: Week 48: number analyzed (Participants) | 12591
  At risk: Week 48 | 161
  Not at risk: Week 37: number analyzed (Participants) | 0
  Not at risk: Week 37 | 0
  Not at risk: Week 38: number analyzed (Participants) | 81
  Not at risk: Week 38 | 2
  Not at risk: Week 39: number analyzed (Participants) | 275
  Not at risk: Week 39 | 6
  Not at risk: Week 40: number analyzed (Participants) | 441
  Not at risk: Week 40 | 11
  Not at risk: Week 41: number analyzed (Participants) | 653
  Not at risk: Week 41 | 12
  Not at risk: Week 42: number analyzed (Participants) | 785
  Not at risk: Week 42 | 14
  Not at risk: Week 43: number analyzed (Participants) | 854
  Not at risk: Week 43 | 14
  Not at risk: Week 44: number analyzed (Participants) | 931
  Not at risk: Week 44 | 14
  Not at risk: Week 45: number analyzed (Participants) | 1022
  Not at risk: Week 45 | 16
  Not at risk: Week 46: number analyzed (Participants) | 1147
  Not at risk: Week 46 | 16
  Not at risk: Week 47: number analyzed (Participants) | 1220
  Not at risk: Week 47 | 16
  Not at risk: Week 48: number analyzed (Participants) | 1270
  Not at risk: Week 48 | 17

61. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Any) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis.
Description: AEIs were presented by categories depending of the nature of the event. - Fever or other febrile illness; - Local reaction; - General reaction (fatigue, myalgia, etc.); - All other presentations that were reported following vaccination (e.g., Bell's palsy, Guillain-Barre syndrome).
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Week 37: number analyzed (Participants) | 6 | 0 | 88
  Week 37 | 0 | 0 | 0
  Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Week 38 | 87 | 4 | 7
  Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Week 39 | 227 | 10 | 3
  Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Week 40 | 218 | 11 | 4
  Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Week 41 | 172 | 5 | 7
  Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Week 42 | 118 | 10 | 8
  Week 43: number analyzed (Participants) | 738 | 140 | 356
  Week 43 | 57 | 4 | 10
  Week 44: number analyzed (Participants) | 769 | 179 | 204
  Week 44 | 52 | 6 | 4
  Week 45: number analyzed (Participants) | 704 | 113 | 242
  Week 45 | 54 | 2 | 4
  Week 46: number analyzed (Participants) | 945 | 272 | 141
  Week 46 | 37 | 6 | 2
  Week 47: number analyzed (Participants) | 474 | 132 | 149
  Week 47 | 14 | 2 | 3
  Week 48: number analyzed (Participants) | 364 | 80 | 103
  Week 48 | 13 | 2 | 2

62. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Any) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis (Cumulative).
Description: as for outcome 61
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Week 37: number analyzed (Participants) | 6 | 0 | 88
  Week 37 | 0 | 0 | 0
  Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Week 38 | 87 | 4 | 7
  Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Week 39 | 314 | 14 | 10
  Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Week 40 | 532 | 25 | 14
  Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Week 41 | 704 | 30 | 21
  Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Week 42 | 822 | 40 | 29
  Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Week 43 | 879 | 44 | 39
  Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Week 44 | 931 | 50 | 43
  Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Week 45 | 985 | 52 | 47
  Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Week 46 | 1022 | 58 | 49
  Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Week 47 | 1036 | 60 | 52
  Week 48 | 1049 | 62 | 54

63. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis.
Description: as for outcome 61
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Week 37: number analyzed (Participants) | 6 | 0 | 88
  Week 37 | 0 | 0 | 0
  Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Week 38 | 8 | 2 | 2
  Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Week 39 | 23 | 5 | 0
  Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Week 40 | 22 | 5 | 0
  Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Week 41 | 20 | 3 | 1
  Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Week 42 | 15 | 4 | 2
  Week 43: number analyzed (Participants) | 738 | 140 | 356
  Week 43 | 13 | 0 | 3
  Week 44: number analyzed (Participants) | 769 | 179 | 204
  Week 44 | 6 | 2 | 3
  Week 45: number analyzed (Participants) | 704 | 113 | 242
  Week 45 | 8 | 2 | 2
  Week 46: number analyzed (Participants) | 945 | 272 | 141
  Week 46 | 11 | 1 | 0
  Week 47: number analyzed (Participants) | 474 | 132 | 149
  Week 47 | 2 | 0 | 1
  Week 48: number analyzed (Participants) | 364 | 80 | 103
  Week 48 | 5 | 1 | 2

64. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis in a (Cumulative).
Description: as for outcome 61
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Week 37: number analyzed (Participants) | 6 | 0 | 88
  Week 37 | 0 | 0 | 0
  Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Week 38 | 8 | 2 | 2
  Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Week 39 | 31 | 7 | 2
  Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Week 40 | 53 | 12 | 2
  Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Week 41 | 73 | 15 | 3
  Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Week 42 | 88 | 19 | 5
  Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Week 43 | 101 | 19 | 8
  Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Week 44 | 107 | 21 | 11
  Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Week 45 | 115 | 23 | 13
  Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Week 46 | 126 | 24 | 13
  Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Week 47 | 128 | 24 | 14
  Week 48 | 133 | 25 | 16

65. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis.
Description: as for outcome 61
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Week 37: number analyzed (Participants) | 6 | 0 | 88
  Week 37 | 0 | 0 | 0
  Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Week 38 | 16 | 0 | 0
  Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Week 39 | 20 | 0 | 0
  Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Week 40 | 24 | 0 | 0
  Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Week 41 | 28 | 0 | 0
  Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Week 42 | 15 | 0 | 0
  Week 43: number analyzed (Participants) | 738 | 140 | 356
  Week 43 | 6 | 0 | 0
  Week 44: number analyzed (Participants) | 769 | 179 | 204
  Week 44 | 7 | 0 | 0
  Week 45: number analyzed (Participants) | 704 | 113 | 242
  Week 45 | 8 | 0 | 0
  Week 46: number analyzed (Participants) | 945 | 272 | 141
  Week 46 | 3 | 0 | 0
  Week 47: number analyzed (Participants) | 474 | 132 | 149
  Week 47 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 364 | 80 | 103
  Week 48 | 0 | 0 | 0

66. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis in a (Cumulative).
Description: as for outcome 61
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Week 37: number analyzed (Participants) | 6 | 0 | 88
  Week 37 | 0 | 0 | 0
  Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Week 38 | 16 | 0 | 0
  Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Week 39 | 36 | 0 | 0
  Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Week 40 | 60 | 0 | 0
  Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Week 41 | 88 | 0 | 0
  Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Week 42 | 103 | 0 | 0
  Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Week 43 | 109 | 0 | 0
  Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Week 44 | 116 | 0 | 0
  Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Week 45 | 124 | 0 | 0
  Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Week 46 | 127 | 0 | 0
  Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Week 47 | 127 | 0 | 0
  Week 48 | 127 | 0 | 0

67. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (General Non-specific Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis.
Description: as for outcome 61
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Any, Week 38 | 21 | 0 | 0
  Any, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Any, Week 39 | 51 | 1 | 0
  Any, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Any, Week 40 | 48 | 0 | 0
  Any, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Any, Week 41 | 28 | 0 | 0
  Any, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Any, Week 42 | 22 | 0 | 1
  Any, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Any, Week 43 | 5 | 0 | 0
  Any, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Any, Week 44 | 7 | 0 | 0
  Any, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Any, Week 45 | 10 | 0 | 0
  Any, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Any, Week 46 | 7 | 0 | 0
  Any, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Any, Week 47 | 2 | 0 | 0
  Any, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Any, Week 48 | 1 | 0 | 0
  Drowsiness, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Drowsiness, Week 37 | 0 | 0 | 0
  Drowsiness, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Drowsiness, Week 38 | 8 | 0 | 0
  Drowsiness, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Drowsiness, Week 39 | 20 | 0 | 0
  Drowsiness, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Drowsiness, Week 40 | 18 | 0 | 0
  Drowsiness, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Drowsiness, Week 41 | 10 | 0 | 0
  Drowsiness, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Drowsiness, Week 42 | 9 | 0 | 0
  Drowsiness, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Drowsiness, Week 43 | 1 | 0 | 0
  Drowsiness, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Drowsiness, Week 44 | 1 | 0 | 0
  Drowsiness, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Drowsiness, Week 45 | 2 | 0 | 0
  Drowsiness, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Drowsiness, Week 46 | 2 | 0 | 0
  Drowsiness, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Drowsiness, Week 47 | 1 | 0 | 0
  Drowsiness, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Drowsiness, Week 48 | 0 | 0 | 0
  Fatigue, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Fatigue, Week 37 | 0 | 0 | 0
  Fatigue, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Fatigue, Week 38 | 20 | 0 | 0
  Fatigue, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Fatigue, Week 39 | 44 | 0 | 0
  Fatigue, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Fatigue, Week 40 | 39 | 0 | 0
  Fatigue, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Fatigue, Week 41 | 22 | 0 | 0
  Fatigue, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Fatigue, Week 42 | 15 | 0 | 1
  Fatigue, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Fatigue, Week 43 | 5 | 0 | 0
  Fatigue, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Fatigue, Week 44 | 6 | 0 | 0
  Fatigue, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Fatigue, Week 45 | 9 | 0 | 0
  Fatigue, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Fatigue, Week 46 | 7 | 0 | 0
  Fatigue, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Fatigue, Week 47 | 1 | 0 | 0
  Fatigue, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Fatigue, Week 48 | 1 | 0 | 0
  Irritability, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Irritability, Week 37 | 0 | 0 | 0
  Irritability, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Irritability, Week 38 | 3 | 0 | 0
  Irritability, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Irritability, Week 39 | 2 | 0 | 0
  Irritability, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Irritability, Week 40 | 7 | 0 | 0
  Irritability, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Irritability, Week 41 | 1 | 0 | 0
  Irritability, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Irritability, Week 42 | 1 | 0 | 0
  Irritability, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Irritability, Week 43 | 1 | 0 | 0
  Irritability, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Irritability, Week 44 | 1 | 0 | 0
  Irritability, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Irritability, Week 45 | 1 | 0 | 0
  Irritability, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Irritability, Week 46 | 0 | 0 | 0
  Irritability, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Irritability, Week 47 | 0 | 0 | 0
  Irritability, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Irritability, Week 48 | 0 | 0 | 0
  Malaise, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Malaise, Week 37 | 0 | 0 | 0
  Malaise, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Malaise, Week 38 | 1 | 0 | 0
  Malaise, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Malaise, Week 39 | 0 | 1 | 0
  Malaise, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Malaise, Week 40 | 0 | 0 | 0
  Malaise, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Malaise, Week 41 | 1 | 0 | 0
  Malaise, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Malaise, Week 42 | 0 | 0 | 0
  Malaise, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Malaise, Week 43 | 0 | 0 | 0
  Malaise, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Malaise, Week 44 | 1 | 0 | 0
  Malaise, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Malaise, Week 45 | 1 | 0 | 0
  Malaise, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Malaise, Week 46 | 0 | 0 | 0
  Malaise, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Malaise, Week 47 | 0 | 0 | 0
  Malaise, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Malaise, Week 48 | 0 | 0 | 0

68. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (General Non-specific Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis (Cumulative).
Description: as for outcome 61
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Any, Week 38 | 21 | 0 | 0
  Any, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Any, Week 39 | 72 | 1 | 0
  Any, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Any, Week 40 | 120 | 1 | 0
  Any, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Any, Week 41 | 148 | 1 | 0
  Any, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Any, Week 42 | 170 | 1 | 1
  Any, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Any, Week 43 | 175 | 1 | 1
  Any, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Any, Week 44 | 182 | 1 | 1
  Any, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Any, Week 45 | 192 | 1 | 1
  Any, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Any, Week 46 | 199 | 1 | 1
  Any, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Any, Week 47 | 201 | 1 | 1
  Any, Week 48 | 202 | 1 | 1
  Drowsiness, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Drowsiness, Week 37 | 0 | 0 | 0
  Drowsiness, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Drowsiness, Week 38 | 8 | 0 | 0
  Drowsiness, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Drowsiness, Week 39 | 28 | 0 | 0
  Drowsiness, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Drowsiness, Week 40 | 46 | 0 | 0
  Drowsiness, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Drowsiness, Week 41 | 56 | 0 | 0
  Drowsiness, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Drowsiness, Week 42 | 65 | 0 | 0
  Drowsiness, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Drowsiness, Week 43 | 66 | 0 | 0
  Drowsiness, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Drowsiness, Week 44 | 67 | 0 | 0
  Drowsiness, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Drowsiness, Week 45 | 69 | 0 | 0
  Drowsiness, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Drowsiness, Week 46 | 71 | 0 | 0
  Drowsiness, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Drowsiness, Week 47 | 72 | 0 | 0
  Drowsiness, Week 48 | 72 | 0 | 0
  Fatigue, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Fatigue, Week 37 | 0 | 0 | 0
  Fatigue, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Fatigue, Week 38 | 20 | 0 | 0
  Fatigue, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Fatigue, Week 39 | 64 | 0 | 0
  Fatigue, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Fatigue, Week 40 | 103 | 0 | 0
  Fatigue, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Fatigue, Week 41 | 125 | 0 | 0
  Fatigue, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Fatigue, Week 42 | 140 | 0 | 1
  Fatigue, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Fatigue, Week 43 | 145 | 0 | 1
  Fatigue, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Fatigue, Week 44 | 151 | 0 | 1
  Fatigue, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Fatigue, Week 45 | 160 | 0 | 1
  Fatigue, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Fatigue, Week 46 | 167 | 0 | 1
  Fatigue, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Fatigue, Week 47 | 168 | 0 | 1
  Fatigue, Week 48 | 169 | 0 | 1
  Irritability, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Irritability, Week 37 | 0 | 0 | 0
  Irritability, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Irritability, Week 38 | 3 | 0 | 0
  Irritability, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Irritability, Week 39 | 5 | 0 | 0
  Irritability, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Irritability, Week 40 | 12 | 0 | 0
  Irritability, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Irritability, Week 41 | 13 | 0 | 0
  Irritability, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Irritability, Week 42 | 14 | 0 | 0
  Irritability, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Irritability, Week 43 | 15 | 0 | 0
  Irritability, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Irritability, Week 44 | 16 | 0 | 0
  Irritability, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Irritability, Week 45 | 17 | 0 | 0
  Irritability, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Irritability, Week 46 | 17 | 0 | 0
  Irritability, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Irritability, Week 47 | 17 | 0 | 0
  Irritability, Week 48 | 17 | 0 | 0
  Malaise, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Malaise, Week 37 | 0 | 0 | 0
  Malaise, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Malaise, Week 38 | 1 | 0 | 0
  Malaise, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Malaise, Week 39 | 1 | 1 | 0
  Malaise, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Malaise, Week 40 | 1 | 1 | 0
  Malaise, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Malaise, Week 41 | 2 | 1 | 0
  Malaise, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Malaise, Week 42 | 2 | 1 | 0
  Malaise, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Malaise, Week 43 | 2 | 1 | 0
  Malaise, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Malaise, Week 44 | 3 | 1 | 0
  Malaise, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Malaise, Week 45 | 4 | 1 | 0
  Malaise, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Malaise, Week 46 | 4 | 1 | 0
  Malaise, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Malaise, Week 47 | 4 | 1 | 0
  Malaise, Week 48 | 4 | 1 | 0

69. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Respiratory/Miscellaneous Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis.
Description: Respiratory/Miscellaneous AE include any respiratory/miscellaneous AE, conjunctivitis, epistaxis, hoarseness, nasal congestion, oropharyngeal pain, rhinorrhoea and wheezing.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Any, Week 38 | 34 | 1 | 1
  Any, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Any, Week 39 | 120 | 3 | 0
  Any, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Any, Week 40 | 111 | 2 | 1
  Any, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Any, Week 41 | 82 | 2 | 2
  Any, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Any, Week 42 | 65 | 4 | 3
  Any, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Any, Week 43 | 29 | 1 | 5
  Any, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Any, Week 44 | 20 | 4 | 1
  Any, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Any, Week 45 | 29 | 0 | 0
  Any, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Any, Week 46 | 14 | 3 | 0
  Any, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Any, Week 47 | 7 | 2 | 0
  Any, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Any, Week 48 | 2 | 1 | 0
  Conjunctivitis, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Conjunctivitis, Week 37 | 0 | 0 | 0
  Conjunctivitis, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Conjunctivitis, Week 38 | 4 | 0 | 0
  Conjunctivitis, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Conjunctivitis, Week 39 | 10 | 0 | 0
  Conjunctivitis, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Conjunctivitis, Week 40 | 2 | 1 | 0
  Conjunctivitis, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Conjunctivitis, Week 41 | 5 | 0 | 0
  Conjunctivitis, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Conjunctivitis, Week 42 | 2 | 0 | 0
  Conjunctivitis, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Conjunctivitis, Week 43 | 1 | 0 | 0
  Conjunctivitis, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Conjunctivitis, Week 44 | 3 | 0 | 0
  Conjunctivitis, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Conjunctivitis, Week 45 | 1 | 0 | 0
  Conjunctivitis, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Conjunctivitis, Week 46 | 0 | 0 | 0
  Conjunctivitis, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Conjunctivitis, Week 47 | 0 | 0 | 0
  Conjunctivitis, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Conjunctivitis, Week 48 | 0 | 1 | 0
  Coryza, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Coryza, Week 37 | 0 | 0 | 0
  Coryza, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Coryza, Week 38 | 3 | 0 | 0
  Coryza, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Coryza, Week 39 | 19 | 0 | 0
  Coryza, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Coryza, Week 40 | 26 | 0 | 0
  Coryza, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Coryza, Week 41 | 11 | 0 | 0
  Coryza, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Coryza, Week 42 | 20 | 0 | 0
  Coryza, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Coryza, Week 43 | 4 | 0 | 0
  Coryza, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Coryza, Week 44 | 3 | 0 | 0
  Coryza, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Coryza, Week 45 | 7 | 0 | 0
  Coryza, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Coryza, Week 46 | 2 | 0 | 0
  Coryza, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Coryza, Week 47 | 0 | 0 | 0
  Coryza, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Coryza, Week 48 | 1 | 0 | 0
  Cough, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Cough, Week 37 | 0 | 0 | 0
  Cough, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Cough, Week 38 | 11 | 1 | 1
  Cough, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Cough, Week 39 | 43 | 2 | 0
  Cough, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Cough, Week 40 | 45 | 0 | 1
  Cough, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Cough, Week 41 | 33 | 2 | 2
  Cough, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Cough, Week 42 | 30 | 2 | 3
  Cough, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Cough, Week 43 | 8 | 1 | 5
  Cough, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Cough, Week 44 | 12 | 4 | 1
  Cough, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Cough, Week 45 | 14 | 0 | 0
  Cough, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Cough, Week 46 | 10 | 3 | 0
  Cough, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Cough, Week 47 | 3 | 2 | 0
  Cough, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Cough, Week 48 | 1 | 0 | 0
  Epistaxis, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Epistaxis, Week 37 | 0 | 0 | 0
  Epistaxis, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Epistaxis, Week 38 | 0 | 0 | 0
  Epistaxis, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Epistaxis, Week 39 | 2 | 1 | 0
  Epistaxis, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Epistaxis, Week 40 | 2 | 0 | 0
  Epistaxis, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Epistaxis, Week 41 | 4 | 0 | 0
  Epistaxis, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Epistaxis, Week 42 | 2 | 0 | 0
  Epistaxis, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Epistaxis, Week 43 | 0 | 0 | 0
  Epistaxis, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Epistaxis, Week 44 | 0 | 0 | 0
  Epistaxis, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Epistaxis, Week 45 | 2 | 0 | 0
  Epistaxis, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Epistaxis, Week 46 | 0 | 0 | 0
  Epistaxis, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Epistaxis, Week 47 | 0 | 0 | 0
  Epistaxis, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Epistaxis, Week 48 | 0 | 0 | 0
  Hoarseness, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Hoarseness, Week 37 | 0 | 0 | 0
  Hoarseness, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Hoarseness, Week 38 | 6 | 0 | 0
  Hoarseness, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Hoarseness, Week 39 | 15 | 0 | 0
  Hoarseness, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Hoarseness, Week 40 | 16 | 0 | 0
  Hoarseness, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Hoarseness, Week 41 | 15 | 0 | 0
  Hoarseness, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Hoarseness, Week 42 | 8 | 0 | 0
  Hoarseness, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Hoarseness, Week 43 | 3 | 0 | 0
  Hoarseness, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Hoarseness, Week 44 | 2 | 0 | 0
  Hoarseness, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Hoarseness, Week 45 | 3 | 0 | 0
  Hoarseness, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Hoarseness, Week 46 | 3 | 0 | 0
  Hoarseness, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Hoarseness, Week 47 | 0 | 0 | 0
  Hoarseness, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Hoarseness, Week 48 | 0 | 0 | 0
  Nasal congestion, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Nasal congestion, Week 37 | 0 | 0 | 0
  Nasal congestion, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Nasal congestion, Week 38 | 22 | 0 | 0
  Nasal congestion, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Nasal congestion, Week 39 | 70 | 0 | 0
  Nasal congestion, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Nasal congestion, Week 40 | 57 | 1 | 0
  Nasal congestion, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Nasal congestion, Week 41 | 46 | 0 | 0
  Nasal congestion, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Nasal congestion, Week 42 | 33 | 2 | 0
  Nasal congestion, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Nasal congestion, Week 43 | 19 | 0 | 0
  Nasal congestion, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Nasal congestion, Week 44 | 7 | 0 | 0
  Nasal congestion, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Nasal congestion, Week 45 | 15 | 0 | 0
  Nasal congestion, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Nasal congestion, Week 46 | 5 | 0 | 0
  Nasal congestion, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Nasal congestion, Week 47 | 2 | 0 | 0
  Nasal congestion, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Nasal congestion, Week 48 | 0 | 0 | 0
  Oropharyngeal pain, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Oropharyngeal pain, Week 37 | 0 | 0 | 0
  Oropharyngeal pain, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Oropharyngeal pain, Week 38 | 9 | 0 | 0
  Oropharyngeal pain, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Oropharyngeal pain, Week 39 | 33 | 0 | 0
  Oropharyngeal pain, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Oropharyngeal pain, Week 40 | 39 | 0 | 0
  Oropharyngeal pain, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Oropharyngeal pain, Week 41 | 21 | 0 | 0
  Oropharyngeal pain, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Oropharyngeal pain, Week 42 | 25 | 2 | 0
  Oropharyngeal pain, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Oropharyngeal pain, Week 43 | 10 | 0 | 0
  Oropharyngeal pain, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Oropharyngeal pain, Week 44 | 5 | 0 | 0
  Oropharyngeal pain, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Oropharyngeal pain, Week 45 | 8 | 0 | 0
  Oropharyngeal pain, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Oropharyngeal pain, Week 46 | 2 | 0 | 0
  Oropharyngeal pain, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Oropharyngeal pain, Week 47 | 3 | 0 | 0
  Oropharyngeal pain, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Oropharyngeal pain, Week 48 | 0 | 0 | 0
  Rhinorrhoea, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Rhinorrhoea, Week 37 | 0 | 0 | 0
  Rhinorrhoea, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Rhinorrhoea, Week 38 | 17 | 0 | 0
  Rhinorrhoea, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Rhinorrhoea, Week 39 | 58 | 0 | 0
  Rhinorrhoea, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Rhinorrhoea, Week 40 | 54 | 0 | 0
  Rhinorrhoea, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Rhinorrhoea, Week 41 | 45 | 0 | 0
  Rhinorrhoea, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Rhinorrhoea, Week 42 | 27 | 2 | 0
  Rhinorrhoea, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Rhinorrhoea, Week 43 | 17 | 0 | 0
  Rhinorrhoea, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Rhinorrhoea, Week 44 | 5 | 0 | 0
  Rhinorrhoea, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Rhinorrhoea, Week 45 | 15 | 0 | 0
  Rhinorrhoea, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Rhinorrhoea, Week 46 | 4 | 0 | 0
  Rhinorrhoea, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Rhinorrhoea, Week 47 | 1 | 0 | 0
  Rhinorrhoea, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Rhinorrhoea, Week 48 | 0 | 0 | 0
  Wheezing, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Wheezing, Week 37 | 0 | 0 | 0
  Wheezing, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Wheezing, Week 38 | 2 | 0 | 0
  Wheezing, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Wheezing, Week 39 | 11 | 0 | 0
  Wheezing, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Wheezing, Week 40 | 13 | 0 | 1
  Wheezing, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Wheezing, Week 41 | 10 | 0 | 0
  Wheezing, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Wheezing, Week 42 | 12 | 0 | 0
  Wheezing, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Wheezing, Week 43 | 2 | 0 | 0
  Wheezing, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Wheezing, Week 44 | 6 | 0 | 0
  Wheezing, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Wheezing, Week 45 | 3 | 0 | 0
  Wheezing, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Wheezing, Week 46 | 4 | 0 | 0
  Wheezing, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Wheezing, Week 47 | 0 | 0 | 0
  Wheezing, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Wheezing, Week 48 | 0 | 0 | 0

70. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Respiratory/Miscellaneous Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis (Cumulative).
Description: as for outcome 69
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Any, Week 38 | 34 | 1 | 1
  Any, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Any, Week 39 | 154 | 4 | 1
  Any, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Any, Week 40 | 265 | 6 | 2
  Any, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Any, Week 41 | 347 | 8 | 4
  Any, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Any, Week 42 | 412 | 12 | 7
  Any, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Any, Week 43 | 441 | 13 | 12
  Any, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Any, Week 44 | 461 | 17 | 13
  Any, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Any, Week 45 | 490 | 17 | 13
  Any, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Any, Week 46 | 504 | 20 | 13
  Any, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Any, Week 47 | 511 | 22 | 13
  Any, Week 48 | 513 | 23 | 13
  Conjunctivitis, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Conjunctivitis, Week 37 | 0 | 0 | 0
  Conjunctivitis, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Conjunctivitis, Week 38 | 4 | 0 | 0
  Conjunctivitis, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Conjunctivitis, Week 39 | 14 | 0 | 0
  Conjunctivitis, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Conjunctivitis, Week 40 | 16 | 1 | 0
  Conjunctivitis, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Conjunctivitis, Week 41 | 21 | 1 | 0
  Conjunctivitis, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Conjunctivitis, Week 42 | 23 | 1 | 0
  Conjunctivitis, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Conjunctivitis, Week 43 | 24 | 1 | 0
  Conjunctivitis, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Conjunctivitis, Week 44 | 27 | 1 | 0
  Conjunctivitis, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Conjunctivitis, Week 45 | 28 | 1 | 0
  Conjunctivitis, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Conjunctivitis, Week 46 | 28 | 1 | 0
  Conjunctivitis, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Conjunctivitis, Week 47 | 28 | 1 | 0
  Conjunctivitis, Week 48 | 28 | 2 | 0
  Coryza, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Coryza, Week 37 | 0 | 0 | 0
  Coryza, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Coryza, Week 38 | 3 | 0 | 0
  Coryza, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Coryza, Week 39 | 22 | 0 | 0
  Coryza, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Coryza, Week 40 | 48 | 0 | 0
  Coryza, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Coryza, Week 41 | 59 | 0 | 0
  Coryza, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Coryza, Week 42 | 79 | 0 | 0
  Coryza, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Coryza, Week 43 | 83 | 0 | 0
  Coryza, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Coryza, Week 44 | 86 | 0 | 0
  Coryza, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Coryza, Week 45 | 93 | 0 | 0
  Coryza, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Coryza, Week 46 | 95 | 0 | 0
  Coryza, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Coryza, Week 47 | 95 | 0 | 0
  Coryza, Week 48 | 96 | 0 | 0
  Cough, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Cough, Week 37 | 0 | 0 | 0
  Cough, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Cough, Week 38 | 11 | 1 | 1
  Cough, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Cough, Week 39 | 54 | 3 | 1
  Cough, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Cough, Week 40 | 99 | 3 | 2
  Cough, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Cough, Week 41 | 132 | 5 | 4
  Cough, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Cough, Week 42 | 162 | 7 | 7
  Cough, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Cough, Week 43 | 170 | 8 | 12
  Cough, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Cough, Week 44 | 182 | 12 | 13
  Cough, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Cough, Week 45 | 196 | 12 | 13
  Cough, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Cough, Week 46 | 206 | 15 | 13
  Cough, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Cough, Week 47 | 209 | 17 | 13
  Cough, Week 48 | 210 | 17 | 13
  Epistaxis, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Epistaxis, Week 37 | 0 | 0 | 0
  Epistaxis, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Epistaxis, Week 38 | 0 | 0 | 0
  Epistaxis, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Epistaxis, Week 39 | 2 | 1 | 0
  Epistaxis, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Epistaxis, Week 40 | 4 | 1 | 0
  Epistaxis, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Epistaxis, Week 41 | 8 | 1 | 0
  Epistaxis, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Epistaxis, Week 42 | 10 | 1 | 0
  Epistaxis, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Epistaxis, Week 43 | 10 | 1 | 0
  Epistaxis, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Epistaxis, Week 44 | 10 | 1 | 0
  Epistaxis, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Epistaxis, Week 45 | 12 | 1 | 0
  Epistaxis, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Epistaxis, Week 46 | 12 | 1 | 0
  Epistaxis, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Epistaxis, Week 47 | 12 | 1 | 0
  Epistaxis, Week 48 | 12 | 1 | 0
  Hoarseness, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Hoarseness, Week 37 | 0 | 0 | 0
  Hoarseness, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Hoarseness, Week 38 | 6 | 0 | 0
  Hoarseness, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Hoarseness, Week 39 | 21 | 0 | 0
  Hoarseness, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Hoarseness, Week 40 | 37 | 0 | 0
  Hoarseness, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Hoarseness, Week 41 | 52 | 0 | 0
  Hoarseness, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Hoarseness, Week 42 | 60 | 0 | 0
  Hoarseness, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Hoarseness, Week 43 | 63 | 0 | 0
  Hoarseness, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Hoarseness, Week 44 | 65 | 0 | 0
  Hoarseness, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Hoarseness, Week 45 | 68 | 0 | 0
  Hoarseness, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Hoarseness, Week 46 | 71 | 0 | 0
  Hoarseness, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Hoarseness, Week 47 | 71 | 0 | 0
  Hoarseness, Week 48 | 71 | 0 | 0
  Nasal congestion, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Nasal congestion, Week 37 | 0 | 0 | 0
  Nasal congestion, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Nasal congestion, Week 38 | 22 | 0 | 0
  Nasal congestion, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Nasal congestion, Week 39 | 92 | 0 | 0
  Nasal congestion, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Nasal congestion, Week 40 | 149 | 1 | 0
  Nasal congestion, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Nasal congestion, Week 41 | 195 | 1 | 0
  Nasal congestion, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Nasal congestion, Week 42 | 228 | 3 | 0
  Nasal congestion, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Nasal congestion, Week 43 | 247 | 3 | 0
  Nasal congestion, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Nasal congestion, Week 44 | 254 | 3 | 0
  Nasal congestion, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Nasal congestion, Week 45 | 269 | 3 | 0
  Nasal congestion, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Nasal congestion, Week 46 | 274 | 3 | 0
  Nasal congestion, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Nasal congestion, Week 47 | 276 | 3 | 0
  Nasal congestion, Week 48 | 276 | 3 | 0
  Oropharyngeal pain, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Oropharyngeal pain, Week 37 | 0 | 0 | 0
  Oropharyngeal pain, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Oropharyngeal pain, Week 38 | 9 | 0 | 0
  Oropharyngeal pain, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Oropharyngeal pain, Week 39 | 42 | 0 | 0
  Oropharyngeal pain, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Oropharyngeal pain, Week 40 | 81 | 0 | 0
  Oropharyngeal pain, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Oropharyngeal pain, Week 41 | 102 | 0 | 0
  Oropharyngeal pain, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Oropharyngeal pain, Week 42 | 127 | 2 | 0
  Oropharyngeal pain, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Oropharyngeal pain, Week 43 | 137 | 2 | 0
  Oropharyngeal pain, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Oropharyngeal pain, Week 44 | 142 | 2 | 0
  Oropharyngeal pain, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Oropharyngeal pain, Week 45 | 150 | 2 | 0
  Oropharyngeal pain, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Oropharyngeal pain, Week 46 | 152 | 2 | 0
  Oropharyngeal pain, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Oropharyngeal pain, Week 47 | 155 | 2 | 0
  Oropharyngeal pain, Week 48 | 155 | 2 | 0
  Rhinorrhoea, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Rhinorrhoea, Week 37 | 0 | 0 | 0
  Rhinorrhoea, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Rhinorrhoea, Week 38 | 17 | 0 | 0
  Rhinorrhoea, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Rhinorrhoea, Week 39 | 75 | 0 | 0
  Rhinorrhoea, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Rhinorrhoea, Week 40 | 129 | 0 | 0
  Rhinorrhoea, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Rhinorrhoea, Week 41 | 174 | 0 | 0
  Rhinorrhoea, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Rhinorrhoea, Week 42 | 201 | 2 | 0
  Rhinorrhoea, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Rhinorrhoea, Week 43 | 218 | 2 | 0
  Rhinorrhoea, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Rhinorrhoea, Week 44 | 223 | 2 | 0
  Rhinorrhoea, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Rhinorrhoea, Week 45 | 238 | 2 | 0
  Rhinorrhoea, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Rhinorrhoea, Week 46 | 242 | 2 | 0
  Rhinorrhoea, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Rhinorrhoea, Week 47 | 243 | 2 | 0
  Rhinorrhoea, Week 48 | 243 | 2 | 0
  Wheezing, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Wheezing, Week 37 | 0 | 0 | 0
  Wheezing, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Wheezing, Week 38 | 2 | 0 | 0
  Wheezing, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Wheezing, Week 39 | 13 | 0 | 0
  Wheezing, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Wheezing, Week 40 | 26 | 0 | 1
  Wheezing, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Wheezing, Week 41 | 36 | 0 | 1
  Wheezing, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Wheezing, Week 42 | 48 | 0 | 1
  Wheezing, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Wheezing, Week 43 | 50 | 0 | 1
  Wheezing, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Wheezing, Week 44 | 56 | 0 | 1
  Wheezing, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Wheezing, Week 45 | 59 | 0 | 1
  Wheezing, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Wheezing, Week 46 | 63 | 0 | 1
  Wheezing, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Wheezing, Week 47 | 63 | 0 | 1
  Wheezing, Week 48 | 63 | 0 | 1

71. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Gastrointestinal Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis.
Description: Gastrointestinal AEs include any gastrointestinal AEs, decreased appetite, diarrhoea, nausea and vomiting.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Any, Week 38 | 18 | 0 | 0
  Any, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Any, Week 39 | 32 | 0 | 0
  Any, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Any, Week 40 | 34 | 0 | 1
  Any, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Any, Week 41 | 25 | 0 | 1
  Any, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Any, Week 42 | 19 | 2 | 0
  Any, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Any, Week 43 | 9 | 0 | 0
  Any, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Any, Week 44 | 5 | 0 | 0
  Any, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Any, Week 45 | 6 | 0 | 0
  Any, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Any, Week 46 | 4 | 0 | 1
  Any, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Any, Week 47 | 1 | 0 | 0
  Any, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Any, Week 48 | 1 | 0 | 0
  Decreased appetite, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Decreased appetite, Week 37 | 0 | 0 | 0
  Decreased appetite, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Decreased appetite, Week 38 | 7 | 0 | 0
  Decreased appetite, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Decreased appetite, Week 39 | 11 | 0 | 0
  Decreased appetite, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Decreased appetite, Week 40 | 12 | 0 | 1
  Decreased appetite, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Decreased appetite, Week 41 | 7 | 0 | 0
  Decreased appetite, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Decreased appetite, Week 42 | 6 | 1 | 0
  Decreased appetite, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Decreased appetite, Week 43 | 2 | 0 | 0
  Decreased appetite, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Decreased appetite, Week 44 | 1 | 0 | 0
  Decreased appetite, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Decreased appetite, Week 45 | 2 | 0 | 0
  Decreased appetite, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Decreased appetite, Week 46 | 2 | 0 | 0
  Decreased appetite, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Decreased appetite, Week 47 | 0 | 0 | 0
  Decreased appetite, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Decreased appetite, Week 48 | 0 | 0 | 0
  Diarrhoea, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Diarrhoea, Week 37 | 0 | 0 | 0
  Diarrhoea, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Diarrhoea, Week 38 | 6 | 0 | 0
  Diarrhoea, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Diarrhoea, Week 39 | 12 | 0 | 0
  Diarrhoea, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Diarrhoea, Week 40 | 14 | 0 | 0
  Diarrhoea, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Diarrhoea, Week 41 | 12 | 0 | 1
  Diarrhoea, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Diarrhoea, Week 42 | 6 | 0 | 0
  Diarrhoea, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Diarrhoea, Week 43 | 5 | 0 | 0
  Diarrhoea, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Diarrhoea, Week 44 | 4 | 0 | 0
  Diarrhoea, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Diarrhoea, Week 45 | 3 | 0 | 0
  Diarrhoea, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Diarrhoea, Week 46 | 1 | 0 | 1
  Diarrhoea, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Diarrhoea, Week 47 | 1 | 0 | 0
  Diarrhoea, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Diarrhoea, Week 48 | 0 | 0 | 0
  Nausea, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Nausea, Week 37 | 0 | 0 | 0
  Nausea, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Nausea, Week 38 | 12 | 0 | 0
  Nausea, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Nausea, Week 39 | 18 | 0 | 0
  Nausea, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Nausea, Week 40 | 15 | 0 | 0
  Nausea, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Nausea, Week 41 | 8 | 0 | 0
  Nausea, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Nausea, Week 42 | 9 | 0 | 0
  Nausea, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Nausea, Week 43 | 3 | 0 | 0
  Nausea, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Nausea, Week 44 | 0 | 0 | 0
  Nausea, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Nausea, Week 45 | 4 | 0 | 0
  Nausea, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Nausea, Week 46 | 1 | 0 | 0
  Nausea, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Nausea, Week 47 | 0 | 0 | 0
  Nausea, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Nausea, Week 48 | 1 | 0 | 0
  Vomiting, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Vomiting, Week 37 | 0 | 0 | 0
  Vomiting, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Vomiting, Week 38 | 3 | 0 | 0
  Vomiting, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Vomiting, Week 39 | 2 | 0 | 0
  Vomiting, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Vomiting, Week 40 | 7 | 0 | 0
  Vomiting, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Vomiting, Week 41 | 1 | 0 | 0
  Vomiting, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Vomiting, Week 42 | 3 | 1 | 0
  Vomiting, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Vomiting, Week 43 | 1 | 0 | 0
  Vomiting, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Vomiting, Week 44 | 0 | 0 | 0
  Vomiting, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Vomiting, Week 45 | 2 | 0 | 0
  Vomiting, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Vomiting, Week 46 | 0 | 0 | 0
  Vomiting, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Vomiting, Week 47 | 0 | 0 | 0
  Vomiting, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Vomiting, Week 48 | 0 | 0 | 0

72. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Gastrointestinal Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis (Cumulative).
Description: Gastrointestinal AEs include any gastrointestinal AEs, decreased appetite, diarrhoea, nausea and vomiting.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Any, Week 38 | 18 | 0 | 0
  Any, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Any, Week 39 | 50 | 0 | 0
  Any, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Any, Week 40 | 84 | 0 | 1
  Any, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Any, Week 41 | 109 | 0 | 2
  Any, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Any, Week 42 | 128 | 2 | 2
  Any, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Any, Week 43 | 137 | 2 | 2
  Any, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Any, Week 44 | 142 | 2 | 2
  Any, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Any, Week 45 | 148 | 2 | 2
  Any, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Any, Week 46 | 152 | 2 | 3
  Any, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Any, Week 47 | 153 | 2 | 3
  Any, Week 48 | 154 | 2 | 3
  Decreased appetite, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Decreased appetite, Week 37 | 0 | 0 | 0
  Decreased appetite, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Decreased appetite, Week 38 | 7 | 0 | 0
  Decreased appetite, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Decreased appetite, Week 39 | 18 | 0 | 0
  Decreased appetite, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Decreased appetite, Week 40 | 30 | 0 | 1
  Decreased appetite, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Decreased appetite, Week 41 | 37 | 0 | 1
  Decreased appetite, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Decreased appetite, Week 42 | 43 | 1 | 1
  Decreased appetite, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Decreased appetite, Week 43 | 45 | 1 | 1
  Decreased appetite, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Decreased appetite, Week 44 | 46 | 1 | 1
  Decreased appetite, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Decreased appetite, Week 45 | 48 | 1 | 1
  Decreased appetite, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Decreased appetite, Week 46 | 50 | 1 | 1
  Decreased appetite, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Decreased appetite, Week 47 | 50 | 1 | 1
  Decreased appetite, Week 48 | 50 | 1 | 1
  Diarrhoea, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Diarrhoea, Week 37 | 0 | 0 | 0
  Diarrhoea, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Diarrhoea, Week 38 | 6 | 0 | 0
  Diarrhoea, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Diarrhoea, Week 39 | 18 | 0 | 0
  Diarrhoea, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Diarrhoea, Week 40 | 32 | 0 | 0
  Diarrhoea, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Diarrhoea, Week 41 | 44 | 0 | 1
  Diarrhoea, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Diarrhoea, Week 42 | 50 | 0 | 1
  Diarrhoea, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Diarrhoea, Week 43 | 55 | 0 | 1
  Diarrhoea, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Diarrhoea, Week 44 | 59 | 0 | 1
  Diarrhoea, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Diarrhoea, Week 45 | 62 | 0 | 1
  Diarrhoea, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Diarrhoea, Week 46 | 63 | 0 | 2
  Diarrhoea, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Diarrhoea, Week 47 | 64 | 0 | 2
  Diarrhoea, Week 48 | 64 | 0 | 2
  Nausea, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Nausea, Week 37 | 0 | 0 | 0
  Nausea, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Nausea, Week 38 | 12 | 0 | 0
  Nausea, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Nausea, Week 39 | 30 | 0 | 0
  Nausea, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Nausea, Week 40 | 45 | 0 | 0
  Nausea, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Nausea, Week 41 | 53 | 0 | 0
  Nausea, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Nausea, Week 42 | 62 | 0 | 0
  Nausea, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Nausea, Week 43 | 65 | 0 | 0
  Nausea, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Nausea, Week 44 | 65 | 0 | 0
  Nausea, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Nausea, Week 45 | 69 | 0 | 0
  Nausea, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Nausea, Week 46 | 70 | 0 | 0
  Nausea, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Nausea, Week 47 | 70 | 0 | 0
  Nausea, Week 48 | 71 | 0 | 0
  Vomiting, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Vomiting, Week 37 | 0 | 0 | 0
  Vomiting, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Vomiting, Week 38 | 3 | 0 | 0
  Vomiting, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Vomiting, Week 39 | 5 | 0 | 0
  Vomiting, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Vomiting, Week 40 | 12 | 0 | 0
  Vomiting, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Vomiting, Week 41 | 13 | 0 | 0
  Vomiting, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Vomiting, Week 42 | 16 | 1 | 0
  Vomiting, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Vomiting, Week 43 | 17 | 1 | 0
  Vomiting, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Vomiting, Week 44 | 17 | 1 | 0
  Vomiting, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Vomiting, Week 45 | 19 | 1 | 0
  Vomiting, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Vomiting, Week 46 | 19 | 1 | 0
  Vomiting, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Vomiting, Week 47 | 19 | 1 | 0
  Vomiting, Week 48 | 19 | 1 | 0

73. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Sensitivity/Anaphylaxis) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis.
Description: Sensitivity/anaphylaxis AEs include any sensitivity/anaphylaxis AEs, anaphylactic reactions, facial oedema and hypersensitivity reactions.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Any, Week 38 | 1 | 1 | 0
  Any, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Any, Week 39 | 2 | 0 | 0
  Any, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Any, Week 40 | 3 | 0 | 0
  Any, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Any, Week 41 | 0 | 0 | 0
  Any, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Any, Week 42 | 3 | 0 | 0
  Any, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Any, Week 43 | 2 | 0 | 0
  Any, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Any, Week 44 | 1 | 0 | 0
  Any, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Any, Week 45 | 1 | 0 | 0
  Any, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Any, Week 46 | 1 | 0 | 0
  Any, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Any, Week 47 | 0 | 0 | 0
  Any, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Any, Week 48 | 1 | 0 | 0
  Anaphylactic reactions, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Anaphylactic reactions, Week 37 | 0 | 0 | 0
  Anaphylactic reactions, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Anaphylactic reactions, Week 38 | 0 | 0 | 0
  Anaphylactic reactions, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Anaphylactic reactions, Week 39 | 0 | 0 | 0
  Anaphylactic reactions, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Anaphylactic reactions, Week 40 | 0 | 0 | 0
  Anaphylactic reactions, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Anaphylactic reactions, Week 41 | 0 | 0 | 0
  Anaphylactic reactions, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Anaphylactic reactions, Week 42 | 0 | 0 | 0
  Anaphylactic reactions, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Anaphylactic reactions, Week 43 | 0 | 0 | 0
  Anaphylactic reactions, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Anaphylactic reactions, Week 44 | 0 | 0 | 0
  Anaphylactic reactions, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Anaphylactic reactions, Week 45 | 0 | 0 | 0
  Anaphylactic reactions, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Anaphylactic reactions, Week 46 | 0 | 0 | 0
  Anaphylactic reactions, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Anaphylactic reactions, Week 47 | 0 | 0 | 0
  Anaphylactic reactions, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Anaphylactic reactions, Week 48 | 0 | 0 | 0
  Facial oedema, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Facial oedema, Week 37 | 0 | 0 | 0
  Facial oedema, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Facial oedema, Week 38 | 0 | 0 | 0
  Facial oedema, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Facial oedema, Week 39 | 0 | 0 | 0
  Facial oedema, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Facial oedema, Week 40 | 1 | 0 | 0
  Facial oedema, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Facial oedema, Week 41 | 0 | 0 | 0
  Facial oedema, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Facial oedema, Week 42 | 0 | 0 | 0
  Facial oedema, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Facial oedema, Week 43 | 0 | 0 | 0
  Facial oedema, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Facial oedema, Week 44 | 0 | 0 | 0
  Facial oedema, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Facial oedema, Week 45 | 0 | 0 | 0
  Facial oedema, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Facial oedema, Week 46 | 0 | 0 | 0
  Facial oedema, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Facial oedema, Week 47 | 0 | 0 | 0
  Facial oedema, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Facial oedema, Week 48 | 0 | 0 | 0
  Hypersensitivity reactions, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Hypersensitivity reactions, Week 37 | 0 | 0 | 0
  Hypersensitivity reactions, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Hypersensitivity reactions, Week 38 | 1 | 1 | 0
  Hypersensitivity reactions, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Hypersensitivity reactions, Week 39 | 2 | 0 | 0
  Hypersensitivity reactions, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Hypersensitivity reactions, Week 40 | 2 | 0 | 0
  Hypersensitivity reactions, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Hypersensitivity reactions, Week 41 | 0 | 0 | 0
  Hypersensitivity reactions, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Hypersensitivity reactions, Week 42 | 3 | 0 | 0
  Hypersensitivity reactions, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Hypersensitivity reactions, Week 43 | 2 | 0 | 0
  Hypersensitivity reactions, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Hypersensitivity reactions, Week 44 | 1 | 0 | 0
  Hypersensitivity reactions, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Hypersensitivity reactions, Week 45 | 1 | 0 | 0
  Hypersensitivity reactions, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Hypersensitivity reactions, Week 46 | 1 | 0 | 0
  Hypersensitivity reactions, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Hypersensitivity reactions, Week 47 | 0 | 0 | 0
  Hypersensitivity reactions, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Hypersensitivity reactions, Week 48 | 1 | 0 | 0

74. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Sensitivity/Anaphylaxis) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis (Cumulative).
Description: as for outcome 73
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Any, Week 38 | 1 | 1 | 0
  Any, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Any, Week 39 | 3 | 1 | 0
  Any, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Any, Week 40 | 6 | 1 | 0
  Any, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Any, Week 41 | 6 | 1 | 0
  Any, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Any, Week 42 | 9 | 1 | 0
  Any, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Any, Week 43 | 11 | 1 | 0
  Any, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Any, Week 44 | 12 | 1 | 0
  Any, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Any, Week 45 | 13 | 1 | 0
  Any, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Any, Week 46 | 14 | 1 | 0
  Any, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Any, Week 47 | 14 | 1 | 0
  Any, Week 48 | 15 | 1 | 0
  Anaphylactic reactions, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Anaphylactic reactions, Week 37 | 0 | 0 | 0
  Anaphylactic reactions, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Anaphylactic reactions, Week 38 | 0 | 0 | 0
  Anaphylactic reactions, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Anaphylactic reactions, Week 39 | 0 | 0 | 0
  Anaphylactic reactions, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Anaphylactic reactions, Week 40 | 0 | 0 | 0
  Anaphylactic reactions, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Anaphylactic reactions, Week 41 | 0 | 0 | 0
  Anaphylactic reactions, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Anaphylactic reactions, Week 42 | 0 | 0 | 0
  Anaphylactic reactions, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Anaphylactic reactions, Week 43 | 0 | 0 | 0
  Anaphylactic reactions, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Anaphylactic reactions, Week 44 | 0 | 0 | 0
  Anaphylactic reactions, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Anaphylactic reactions, Week 45 | 0 | 0 | 0
  Anaphylactic reactions, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Anaphylactic reactions, Week 46 | 0 | 0 | 0
  Anaphylactic reactions, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Anaphylactic reactions, Week 47 | 0 | 0 | 0
  Anaphylactic reactions, Week 48 | 0 | 0 | 0
  Facial oedema, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Facial oedema, Week 37 | 0 | 0 | 0
  Facial oedema, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Facial oedema, Week 38 | 0 | 0 | 0
  Facial oedema, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Facial oedema, Week 39 | 0 | 0 | 0
  Facial oedema, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Facial oedema, Week 40 | 1 | 0 | 0
  Facial oedema, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Facial oedema, Week 41 | 1 | 0 | 0
  Facial oedema, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Facial oedema, Week 42 | 1 | 0 | 0
  Facial oedema, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Facial oedema, Week 43 | 1 | 0 | 0
  Facial oedema, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Facial oedema, Week 44 | 1 | 0 | 0
  Facial oedema, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Facial oedema, Week 45 | 1 | 0 | 0
  Facial oedema, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Facial oedema, Week 46 | 1 | 0 | 0
  Facial oedema, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Facial oedema, Week 47 | 1 | 0 | 0
  Facial oedema, Week 48 | 1 | 0 | 0
  Hypersensitivity reactions, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Hypersensitivity reactions, Week 37 | 0 | 0 | 0
  Hypersensitivity reactions, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Hypersensitivity reactions, Week 38 | 1 | 1 | 0
  Hypersensitivity reactions, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Hypersensitivity reactions, Week 39 | 3 | 1 | 0
  Hypersensitivity reactions, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Hypersensitivity reactions, Week 40 | 5 | 1 | 0
  Hypersensitivity reactions, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Hypersensitivity reactions, Week 41 | 5 | 1 | 0
  Hypersensitivity reactions, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Hypersensitivity reactions, Week 42 | 8 | 1 | 0
  Hypersensitivity reactions, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Hypersensitivity reactions, Week 43 | 10 | 1 | 0
  Hypersensitivity reactions, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Hypersensitivity reactions, Week 44 | 11 | 1 | 0
  Hypersensitivity reactions, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Hypersensitivity reactions, Week 45 | 12 | 1 | 0
  Hypersensitivity reactions, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Hypersensitivity reactions, Week 46 | 13 | 1 | 0
  Hypersensitivity reactions, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Hypersensitivity reactions, Week 47 | 13 | 1 | 0
  Hypersensitivity reactions, Week 48 | 14 | 1 | 0

75. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis.
Description: Rash AEs include any rash AEs, generalised rash and rash.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Any, Week 38 | 2 | 0 | 0
  Any, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Any, Week 39 | 10 | 0 | 0
  Any, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Any, Week 40 | 7 | 3 | 0
  Any, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Any, Week 41 | 7 | 0 | 0
  Any, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Any, Week 42 | 5 | 2 | 0
  Any, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Any, Week 43 | 4 | 1 | 0
  Any, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Any, Week 44 | 3 | 0 | 0
  Any, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Any, Week 45 | 2 | 0 | 0
  Any, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Any, Week 46 | 4 | 0 | 1
  Any, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Any, Week 47 | 3 | 0 | 1
  Any, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Any, Week 48 | 0 | 0 | 0
  Generalised rash, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Generalised rash, Week 37 | 0 | 0 | 0
  Generalised rash, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Generalised rash, Week 38 | 1 | 0 | 0
  Generalised rash, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Generalised rash, Week 39 | 10 | 0 | 0
  Generalised rash, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Generalised rash, Week 40 | 3 | 3 | 0
  Generalised rash, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Generalised rash, Week 41 | 6 | 0 | 0
  Generalised rash, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Generalised rash, Week 42 | 2 | 2 | 0
  Generalised rash, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Generalised rash, Week 43 | 1 | 1 | 0
  Generalised rash, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Generalised rash, Week 44 | 2 | 0 | 0
  Generalised rash, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Generalised rash, Week 45 | 1 | 0 | 0
  Generalised rash, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Generalised rash, Week 46 | 2 | 0 | 1
  Generalised rash, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Generalised rash, Week 47 | 3 | 0 | 1
  Generalised rash, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Generalised rash, Week 48 | 0 | 0 | 0
  Rash, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Rash, Week 37 | 0 | 0 | 0
  Rash, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Rash, Week 38 | 1 | 0 | 0
  Rash, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Rash, Week 39 | 0 | 0 | 0
  Rash, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Rash, Week 40 | 4 | 0 | 0
  Rash, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Rash, Week 41 | 1 | 0 | 0
  Rash, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Rash, Week 42 | 3 | 0 | 0
  Rash, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Rash, Week 43 | 3 | 0 | 0
  Rash, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Rash, Week 44 | 1 | 0 | 0
  Rash, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Rash, Week 45 | 1 | 0 | 0
  Rash, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Rash, Week 46 | 2 | 0 | 0
  Rash, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Rash, Week 47 | 0 | 0 | 0
  Rash, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Rash, Week 48 | 0 | 0 | 0

76. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis (Cumulative)
Description: Rash AEs include any rash AEs, generalised rash and rash.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Any, Week 38 | 2 | 0 | 0
  Any, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Any, Week 39 | 12 | 0 | 0
  Any, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Any, Week 40 | 19 | 3 | 0
  Any, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Any, Week 41 | 26 | 3 | 0
  Any, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Any, Week 42 | 31 | 5 | 0
  Any, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Any, Week 43 | 35 | 6 | 0
  Any, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Any, Week 44 | 38 | 6 | 0
  Any, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Any, Week 45 | 40 | 6 | 0
  Any, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Any, Week 46 | 44 | 6 | 1
  Any, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Any, Week 47 | 47 | 6 | 2
  Any, Week 48 | 47 | 6 | 2
  Generalised rash, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Generalised rash, Week 37 | 0 | 0 | 0
  Generalised rash, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Generalised rash, Week 38 | 1 | 0 | 0
  Generalised rash, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Generalised rash, Week 39 | 11 | 0 | 0
  Generalised rash, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Generalised rash, Week 40 | 14 | 3 | 0
  Generalised rash, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Generalised rash, Week 41 | 20 | 3 | 0
  Generalised rash, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Generalised rash, Week 42 | 22 | 5 | 0
  Generalised rash, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Generalised rash, Week 43 | 23 | 6 | 0
  Generalised rash, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Generalised rash, Week 44 | 25 | 6 | 0
  Generalised rash, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Generalised rash, Week 45 | 26 | 6 | 0
  Generalised rash, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Generalised rash, Week 46 | 28 | 6 | 1
  Generalised rash, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Generalised rash, Week 47 | 31 | 6 | 2
  Generalised rash, Week 48 | 31 | 6 | 2
  Rash, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Rash, Week 37 | 0 | 0 | 0
  Rash, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Rash, Week 38 | 1 | 0 | 0
  Rash, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Rash, Week 39 | 1 | 0 | 0
  Rash, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Rash, Week 40 | 5 | 0 | 0
  Rash, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Rash, Week 41 | 6 | 0 | 0
  Rash, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Rash, Week 42 | 9 | 0 | 0
  Rash, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Rash, Week 43 | 12 | 0 | 0
  Rash, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Rash, Week 44 | 13 | 0 | 0
  Rash, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Rash, Week 45 | 14 | 0 | 0
  Rash, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Rash, Week 46 | 16 | 0 | 0
  Rash, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Rash, Week 47 | 16 | 0 | 0
  Rash, Week 48 | 16 | 0 | 0

77. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis.
Description: Musculoskeletal AEs include any musculoskeletal AEs, arthropathy and muscle aches/myalgia.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Any, Week 38 | 32 | 1 | 4
  Any, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Any, Week 39 | 71 | 2 | 3
  Any, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Any, Week 40 | 75 | 1 | 3
  Any, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Any, Week 41 | 48 | 1 | 0
  Any, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Any, Week 42 | 46 | 0 | 2
  Any, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Any, Week 43 | 8 | 1 | 0
  Any, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Any, Week 44 | 15 | 0 | 0
  Any, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Any, Week 45 | 18 | 0 | 2
  Any, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Any, Week 46 | 12 | 1 | 0
  Any, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Any, Week 47 | 2 | 0 | 1
  Any, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Any, Week 48 | 4 | 0 | 0
  Arthropathy, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Arthropathy, Week 37 | 0 | 0 | 0
  Arthropathy, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Arthropathy, Week 38 | 8 | 0 | 0
  Arthropathy, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Arthropathy, Week 39 | 17 | 0 | 0
  Arthropathy, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Arthropathy, Week 40 | 24 | 0 | 0
  Arthropathy, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Arthropathy, Week 41 | 9 | 0 | 0
  Arthropathy, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Arthropathy, Week 42 | 11 | 0 | 0
  Arthropathy, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Arthropathy, Week 43 | 2 | 0 | 0
  Arthropathy, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Arthropathy, Week 44 | 2 | 0 | 0
  Arthropathy, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Arthropathy, Week 45 | 5 | 0 | 0
  Arthropathy, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Arthropathy, Week 46 | 1 | 0 | 0
  Arthropathy, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Arthropathy, Week 47 | 0 | 0 | 0
  Arthropathy, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Arthropathy, Week 48 | 0 | 0 | 0
  Muscle aches/myalgia, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Muscle aches/myalgia, Week 37 | 0 | 0 | 0
  Muscle aches/myalgia, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Muscle aches/myalgia, Week 38 | 30 | 1 | 4
  Muscle aches/myalgia, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Muscle aches/myalgia, Week 39 | 69 | 2 | 3
  Muscle aches/myalgia, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Muscle aches/myalgia, Week 40 | 68 | 1 | 3
  Muscle aches/myalgia, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Muscle aches/myalgia, Week 41 | 46 | 1 | 0
  Muscle aches/myalgia, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Muscle aches/myalgia, Week 42 | 42 | 0 | 2
  Muscle aches/myalgia, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Muscle aches/myalgia, Week 43 | 8 | 1 | 0
  Muscle aches/myalgia, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Muscle aches/myalgia, Week 44 | 13 | 0 | 0
  Muscle aches/myalgia, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Muscle aches/myalgia, Week 45 | 18 | 0 | 2
  Muscle aches/myalgia, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Muscle aches/myalgia, Week 46 | 11 | 1 | 0
  Muscle aches/myalgia, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Muscle aches/myalgia, Week 47 | 2 | 0 | 1
  Muscle aches/myalgia, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Muscle aches/myalgia, Week 48 | 4 | 0 | 0

78. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis (Cumulative).
Description: Musculoskeletal AEs include any musculoskeletal AEs, arthropathy and muscle aches/myalgia.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Any, Week 38 | 32 | 1 | 4
  Any, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Any, Week 39 | 103 | 3 | 7
  Any, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Any, Week 40 | 178 | 4 | 10
  Any, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Any, Week 41 | 226 | 5 | 10
  Any, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Any, Week 42 | 272 | 5 | 12
  Any, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Any, Week 43 | 280 | 6 | 12
  Any, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Any, Week 44 | 295 | 6 | 12
  Any, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Any, Week 45 | 313 | 6 | 14
  Any, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Any, Week 46 | 325 | 7 | 14
  Any, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Any, Week 47 | 327 | 7 | 15
  Any, Week 48 | 331 | 7 | 15
  Arthropathy, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Arthropathy, Week 37 | 0 | 0 | 0
  Arthropathy, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Arthropathy, Week 38 | 8 | 0 | 0
  Arthropathy, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Arthropathy, Week 39 | 25 | 0 | 0
  Arthropathy, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Arthropathy, Week 40 | 49 | 0 | 0
  Arthropathy, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Arthropathy, Week 41 | 58 | 0 | 0
  Arthropathy, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Arthropathy, Week 42 | 69 | 0 | 0
  Arthropathy, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Arthropathy, Week 43 | 71 | 0 | 0
  Arthropathy, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Arthropathy, Week 44 | 73 | 0 | 0
  Arthropathy, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Arthropathy, Week 45 | 78 | 0 | 0
  Arthropathy, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Arthropathy, Week 46 | 79 | 0 | 0
  Arthropathy, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Arthropathy, Week 47 | 79 | 0 | 0
  Arthropathy, Week 48 | 79 | 0 | 0
  Muscle aches/myalgia, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Muscle aches/myalgia, Week 37 | 0 | 0 | 0
  Muscle aches/myalgia, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Muscle aches/myalgia, Week 38 | 30 | 1 | 4
  Muscle aches/myalgia, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Muscle aches/myalgia, Week 39 | 99 | 3 | 7
  Muscle aches/myalgia, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Muscle aches/myalgia, Week 40 | 167 | 4 | 10
  Muscle aches/myalgia, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Muscle aches/myalgia, Week 41 | 213 | 5 | 10
  Muscle aches/myalgia, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Muscle aches/myalgia, Week 42 | 255 | 5 | 12
  Muscle aches/myalgia, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Muscle aches/myalgia, Week 43 | 263 | 6 | 12
  Muscle aches/myalgia, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Muscle aches/myalgia, Week 44 | 276 | 6 | 12
  Muscle aches/myalgia, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Muscle aches/myalgia, Week 45 | 294 | 6 | 14
  Muscle aches/myalgia, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Muscle aches/myalgia, Week 46 | 305 | 7 | 14
  Muscle aches/myalgia, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Muscle aches/myalgia, Week 47 | 307 | 7 | 15
  Muscle aches/myalgia, Week 48 | 311 | 7 | 15

79. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis.
Description: Neurological AEs include any neurological AEs, Bell's palsy, Guillain-Barre syndrome, headache, peripheral tremor and seizure/febrile convulsions.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Any, Week 38 | 22 | 0 | 0
  Any, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Any, Week 39 | 52 | 1 | 0
  Any, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Any, Week 40 | 46 | 1 | 0
  Any, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Any, Week 41 | 31 | 0 | 3
  Any, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Any, Week 42 | 17 | 1 | 0
  Any, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Any, Week 43 | 13 | 1 | 2
  Any, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Any, Week 44 | 7 | 1 | 0
  Any, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Any, Week 45 | 13 | 0 | 0
  Any, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Any, Week 46 | 3 | 1 | 0
  Any, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Any, Week 47 | 1 | 0 | 0
  Any, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Any, Week 48 | 1 | 0 | 0
  Bell's palsy, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Bell's palsy, Week 37 | 0 | 0 | 0
  Bell's palsy, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Bell's palsy, Week 38 | 0 | 0 | 0
  Bell's palsy, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Bell's palsy, Week 39 | 0 | 0 | 0
  Bell's palsy, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Bell's palsy, Week 40 | 0 | 0 | 0
  Bell's palsy, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Bell's palsy, Week 41 | 0 | 0 | 0
  Bell's palsy, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Bell's palsy, Week 42 | 0 | 0 | 0
  Bell's palsy, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Bell's palsy, Week 43 | 0 | 0 | 0
  Bell's palsy, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Bell's palsy, Week 44 | 0 | 0 | 0
  Bell's palsy, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Bell's palsy, Week 45 | 0 | 0 | 0
  Bell's palsy, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Bell's palsy, Week 46 | 0 | 0 | 0
  Bell's palsy, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Bell's palsy, Week 47 | 0 | 0 | 0
  Bell's palsy, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Bell's palsy, Week 48 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Guillain-Barre Syndrome, Week 37 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Guillain-Barre Syndrome, Week 38 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Guillain-Barre Syndrome, Week 39 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Guillain-Barre Syndrome, Week 40 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Guillain-Barre Syndrome, Week 41 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Guillain-Barre Syndrome, Week 42 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Guillain-Barre Syndrome, Week 43 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Guillain-Barre Syndrome, Week 44 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Guillain-Barre Syndrome, Week 45 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Guillain-Barre Syndrome, Week 46 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Guillain-Barre Syndrome, Week 47 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Guillain-Barre Syndrome, Week 48 | 0 | 0 | 0
  Headache, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Headache, Week 37 | 0 | 0 | 0
  Headache, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Headache, Week 38 | 20 | 0 | 0
  Headache, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Headache, Week 39 | 52 | 1 | 0
  Headache, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Headache, Week 40 | 44 | 1 | 0
  Headache, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Headache, Week 41 | 28 | 0 | 3
  Headache, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Headache, Week 42 | 15 | 1 | 0
  Headache, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Headache, Week 43 | 11 | 1 | 2
  Headache, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Headache, Week 44 | 6 | 1 | 0
  Headache, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Headache, Week 45 | 11 | 0 | 0
  Headache, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Headache, Week 46 | 3 | 1 | 0
  Headache, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Headache, Week 47 | 1 | 0 | 0
  Headache, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Headache, Week 48 | 1 | 0 | 0
  Peripheral tremor, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Peripheral tremor, Week 37 | 0 | 0 | 0
  Peripheral tremor, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Peripheral tremor, Week 38 | 3 | 0 | 0
  Peripheral tremor, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Peripheral tremor, Week 39 | 5 | 0 | 0
  Peripheral tremor, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Peripheral tremor, Week 40 | 1 | 0 | 0
  Peripheral tremor, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Peripheral tremor, Week 41 | 8 | 0 | 0
  Peripheral tremor, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Peripheral tremor, Week 42 | 3 | 0 | 0
  Peripheral tremor, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Peripheral tremor, Week 43 | 2 | 0 | 0
  Peripheral tremor, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Peripheral tremor, Week 44 | 1 | 0 | 0
  Peripheral tremor, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Peripheral tremor, Week 45 | 1 | 0 | 0
  Peripheral tremor, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Peripheral tremor, Week 46 | 0 | 0 | 0
  Peripheral tremor, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Peripheral tremor, Week 47 | 0 | 0 | 0
  Peripheral tremor, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Peripheral tremor, Week 48 | 0 | 0 | 0
  Seizure/Febrile convulsions, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Seizure/Febrile convulsions, Week 37 | 0 | 0 | 0
  Seizure/Febrile convulsions, Week 38: number analyzed (Participants) | 1269 | 312 | 252
  Seizure/Febrile convulsions, Week 38 | 0 | 0 | 0
  Seizure/Febrile convulsions, Week 39: number analyzed (Participants) | 2626 | 169 | 430
  Seizure/Febrile convulsions, Week 39 | 0 | 0 | 0
  Seizure/Febrile convulsions, Week 40: number analyzed (Participants) | 2146 | 325 | 357
  Seizure/Febrile convulsions, Week 40 | 1 | 0 | 0
  Seizure/Febrile convulsions, Week 41: number analyzed (Participants) | 2458 | 334 | 424
  Seizure/Febrile convulsions, Week 41 | 0 | 0 | 0
  Seizure/Febrile convulsions, Week 42: number analyzed (Participants) | 1362 | 239 | 432
  Seizure/Febrile convulsions, Week 42 | 0 | 0 | 0
  Seizure/Febrile convulsions, Week 43: number analyzed (Participants) | 738 | 140 | 356
  Seizure/Febrile convulsions, Week 43 | 0 | 0 | 0
  Seizure/Febrile convulsions, Week 44: number analyzed (Participants) | 769 | 179 | 204
  Seizure/Febrile convulsions, Week 44 | 0 | 0 | 0
  Seizure/Febrile convulsions, Week 45: number analyzed (Participants) | 704 | 113 | 242
  Seizure/Febrile convulsions, Week 45 | 1 | 0 | 0
  Seizure/Febrile convulsions, Week 46: number analyzed (Participants) | 945 | 272 | 141
  Seizure/Febrile convulsions, Week 46 | 0 | 0 | 0
  Seizure/Febrile convulsions, Week 47: number analyzed (Participants) | 474 | 132 | 149
  Seizure/Febrile convulsions, Week 47 | 0 | 0 | 0
  Seizure/Febrile convulsions, Week 48: number analyzed (Participants) | 364 | 80 | 103
  Seizure/Febrile convulsions, Week 48 | 0 | 0 | 0

80. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Vaccine Group, on a Weekly Basis (Cumulative),
Description: as for outcome 79
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  Any, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Any, Week 37 | 0 | 0 | 0
  Any, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Any, Week 38 | 22 | 0 | 0
  Any, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Any, Week 39 | 74 | 1 | 0
  Any, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Any, Week 40 | 120 | 2 | 0
  Any, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Any, Week 41 | 151 | 2 | 3
  Any, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Any, Week 42 | 168 | 3 | 3
  Any, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Any, Week 43 | 181 | 4 | 5
  Any, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Any, Week 44 | 188 | 5 | 5
  Any, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Any, Week 45 | 201 | 5 | 5
  Any, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Any, Week 46 | 204 | 6 | 5
  Any, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Any, Week 47 | 205 | 6 | 5
  Any, Week 48 | 206 | 6 | 5
  Bell's palsy, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Bell's palsy, Week 37 | 0 | 0 | 0
  Bell's palsy, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Bell's palsy, Week 38 | 0 | 0 | 0
  Bell's palsy, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Bell's palsy, Week 39 | 0 | 0 | 0
  Bell's palsy, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Bell's palsy, Week 40 | 0 | 0 | 0
  Bell's palsy, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Bell's palsy, Week 41 | 0 | 0 | 0
  Bell's palsy, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Bell's palsy, Week 42 | 0 | 0 | 0
  Bell's palsy, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Bell's palsy, Week 43 | 0 | 0 | 0
  Bell's palsy, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Bell's palsy, Week 44 | 0 | 0 | 0
  Bell's palsy, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Bell's palsy, Week 45 | 0 | 0 | 0
  Bell's palsy, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Bell's palsy, Week 46 | 0 | 0 | 0
  Bell's palsy, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Bell's palsy, Week 47 | 0 | 0 | 0
  Bell's palsy, Week 48 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Guillain-Barre Syndrome, Week 37 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Guillain-Barre Syndrome, Week 38 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Guillain-Barre Syndrome, Week 39 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Guillain-Barre Syndrome, Week 40 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Guillain-Barre Syndrome, Week 41 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Guillain-Barre Syndrome, Week 42 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Guillain-Barre Syndrome, Week 43 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Guillain-Barre Syndrome, Week 44 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Guillain-Barre Syndrome, Week 45 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Guillain-Barre Syndrome, Week 46 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Guillain-Barre Syndrome, Week 47 | 0 | 0 | 0
  Guillain-Barre Syndrome, Week 48 | 0 | 0 | 0
  Headache, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Headache, Week 37 | 0 | 0 | 0
  Headache, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Headache, Week 38 | 20 | 0 | 0
  Headache, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Headache, Week 39 | 72 | 1 | 0
  Headache, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Headache, Week 40 | 116 | 2 | 0
  Headache, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Headache, Week 41 | 144 | 2 | 3
  Headache, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Headache, Week 42 | 159 | 3 | 3
  Headache, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Headache, Week 43 | 170 | 4 | 5
  Headache, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Headache, Week 44 | 176 | 5 | 5
  Headache, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Headache, Week 45 | 187 | 5 | 5
  Headache, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Headache, Week 46 | 190 | 6 | 5
  Headache, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Headache, Week 47 | 191 | 6 | 5
  Headache, Week 48 | 192 | 6 | 5
  Peripheral tremor, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Peripheral tremor, Week 37 | 0 | 0 | 0
  Peripheral tremor, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Peripheral tremor, Week 38 | 3 | 0 | 0
  Peripheral tremor, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Peripheral tremor, Week 39 | 8 | 0 | 0
  Peripheral tremor, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Peripheral tremor, Week 40 | 9 | 0 | 0
  Peripheral tremor, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Peripheral tremor, Week 41 | 17 | 0 | 0
  Peripheral tremor, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Peripheral tremor, Week 42 | 20 | 0 | 0
  Peripheral tremor, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Peripheral tremor, Week 43 | 22 | 0 | 0
  Peripheral tremor, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Peripheral tremor, Week 44 | 23 | 0 | 0
  Peripheral tremor, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Peripheral tremor, Week 45 | 24 | 0 | 0
  Peripheral tremor, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Peripheral tremor, Week 46 | 24 | 0 | 0
  Peripheral tremor, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Peripheral tremor, Week 47 | 24 | 0 | 0
  Peripheral tremor, Week 48 | 24 | 0 | 0
  Seizure / Febrile convulsions, Week 37: number analyzed (Participants) | 6 | 0 | 88
  Seizure / Febrile convulsions, Week 37 | 0 | 0 | 0
  Seizure / Febrile convulsions, Week 38: number analyzed (Participants) | 1275 | 312 | 340
  Seizure / Febrile convulsions, Week 38 | 0 | 0 | 0
  Seizure / Febrile convulsions, Week 39: number analyzed (Participants) | 3901 | 481 | 770
  Seizure / Febrile convulsions, Week 39 | 0 | 0 | 0
  Seizure / Febrile convulsions, Week 40: number analyzed (Participants) | 6047 | 806 | 1127
  Seizure / Febrile convulsions, Week 40 | 1 | 0 | 0
  Seizure / Febrile convulsions, Week 41: number analyzed (Participants) | 8505 | 1140 | 1551
  Seizure / Febrile convulsions, Week 41 | 1 | 0 | 0
  Seizure / Febrile convulsions, Week 42: number analyzed (Participants) | 9867 | 1379 | 1983
  Seizure / Febrile convulsions, Week 42 | 1 | 0 | 0
  Seizure / Febrile convulsions, Week 43: number analyzed (Participants) | 10605 | 1519 | 2339
  Seizure / Febrile convulsions, Week 43 | 1 | 0 | 0
  Seizure / Febrile convulsions, Week 44: number analyzed (Participants) | 11374 | 1698 | 2543
  Seizure / Febrile convulsions, Week 44 | 1 | 0 | 0
  Seizure / Febrile convulsions, Week 45: number analyzed (Participants) | 12078 | 1811 | 2785
  Seizure / Febrile convulsions, Week 45 | 2 | 0 | 0
  Seizure / Febrile convulsions, Week 46: number analyzed (Participants) | 13023 | 2083 | 2926
  Seizure / Febrile convulsions, Week 46 | 2 | 0 | 0
  Seizure / Febrile convulsions, Week 47: number analyzed (Participants) | 13497 | 2215 | 3075
  Seizure / Febrile convulsions, Week 47 | 2 | 0 | 0
  Seizure / Febrile convulsions, Week 48 | 2 | 0 | 0

81. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Any) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis.
Description: The age strata analysed were 6 months to 5 years; 6 to 12 years; 13 to 18 years; greater than or equal to (≥) 18-65 years and >65 years.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2 | 149 | 2
  6 months - 5 years, Week 40 | 0 | 2 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3 | 214 | 23
  6 months - 5 years, Week 41 | 0 | 3 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2 | 143 | 17
  6 months - 5 years, Week 42 | 1 | 6 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5 | 80 | 31
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0 | 116 | 5
  6 months - 5 years, Week 44 | 0 | 4 | 1
  6 months - 5 years, Week 45: number analyzed (Participants) | 0 | 87 | 38
  6 months - 5 years, Week 45 | 0 | 2 | 2
  6 months - 5 years, Week 46: number analyzed (Participants) | 1 | 221 | 13
  6 months - 5 years, Week 46 | 0 | 4 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2 | 89 | 13
  6 months - 5 years, Week 47 | 1 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0 | 60 | 9
  6 months - 5 years, Week 48 | 0 | 2 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4 | 28 | 3
  6-12 years, Week 40 | 1 | 2 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2 | 51 | 84
  6-12 years, Week 41 | 0 | 0 | 1
  6-12 years, Week 42: number analyzed (Participants) | 4 | 34 | 35
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3 | 30 | 45
  6-12 years, Week 43 | 1 | 1 | 1
  6-12 years, Week 44: number analyzed (Participants) | 2 | 30 | 2
  6-12 years, Week 44 | 0 | 1 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0 | 13 | 27
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5 | 34 | 15
  6-12 years, Week 46 | 1 | 0 | 1
  6-12 years, Week 47: number analyzed (Participants) | 0 | 37 | 35
  6-12 years, Week 47 | 0 | 2 | 1
  6-12 years, Week 48: number analyzed (Participants) | 1 | 13 | 23
  6-12 years, Week 48 | 0 | 0 | 2
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5 | 3 | 0
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6 | 5 | 3
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9 | 11 | 1
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6 | 16 | 3
  13-17 years, Week 42 | 1 | 2 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0 | 6 | 1
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5 | 13 | 0
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4 | 5 | 4
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6 | 11 | 3
  13-17 years, Week 46 | 0 | 1 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1 | 6 | 1
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5 | 6 | 1
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363 | 183 | 104
  18-65 years, Week 38 | 28 | 3 | 2
  18-65 years, Week 39: number analyzed (Participants) | 781 | 63 | 140
  18-65 years, Week 39 | 67 | 6 | 1
  18-65 years, Week 40: number analyzed (Participants) | 675 | 54 | 117
  18-65 years, Week 40 | 77 | 5 | 1
  18-65 years, Week 41: number analyzed (Participants) | 815 | 15 | 98
  18-65 years, Week 41 | 60 | 1 | 3
  18-65 years, Week 42: number analyzed (Participants) | 486 | 25 | 163
  18-65 years, Week 42 | 49 | 1 | 3
  18-65 years, Week 43: number analyzed (Participants) | 273 | 12 | 105
  18-65 years, Week 43 | 23 | 1 | 4
  18-65 years, Week 44: number analyzed (Participants) | 278 | 9 | 86
  18-65 years, Week 44 | 21 | 0 | 2
  18-65 years, Week 45: number analyzed (Participants) | 304 | 5 | 83
  18-65 years, Week 45 | 27 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 425 | 4 | 57
  18-65 years, Week 46 | 21 | 1 | 1
  18-65 years, Week 47: number analyzed (Participants) | 217 | 0 | 54
  18-65 years, Week 47 | 5 | 0 | 1
  18-65 years, Week 48: number analyzed (Participants) | 175 | 0 | 33
  18-65 years, Week 48 | 6 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 898 | 128 | 147
  >65 years, Week 38 | 59 | 1 | 5
  >65 years, Week 39: number analyzed (Participants) | 1837 | 89 | 289
  >65 years, Week 39 | 160 | 4 | 2
  >65 years, Week 40: number analyzed (Participants) | 1459 | 89 | 232
  >65 years, Week 40 | 140 | 2 | 3
  >65 years, Week 41: number analyzed (Participants) | 1629 | 43 | 218
  >65 years, Week 41 | 112 | 1 | 3
  >65 years, Week 42: number analyzed (Participants) | 864 | 21 | 214
  >65 years, Week 42 | 67 | 1 | 5
  >65 years, Week 43: number analyzed (Participants) | 457 | 12 | 174
  >65 years, Week 43 | 33 | 2 | 5
  >65 years, Week 44: number analyzed (Participants) | 484 | 11 | 111
  >65 years, Week 44 | 31 | 1 | 1
  >65 years, Week 45: number analyzed (Participants) | 396 | 3 | 90
  >65 years, Week 45 | 27 | 0 | 2
  >65 years, Week 46: number analyzed (Participants) | 508 | 2 | 53
  >65 years, Week 46 | 15 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 254 | 0 | 40
  >65 years, Week 47 | 8 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 183 | 1 | 37
  >65 years, Week 48 | 7 | 0 | 0

82. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Any) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis (Cumulative).
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3 | 158 | 2
  6 months - 5 years, Week 40 | 0 | 2 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6 | 372 | 25
  6 months - 5 years, Week 41 | 0 | 5 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8 | 515 | 42
  6 months - 5 years, Week 42 | 1 | 11 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13 | 595 | 73
  6 months - 5 years, Week 43 | 1 | 11 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13 | 711 | 78
  6 months - 5 years, Week 44 | 1 | 15 | 1
  6 months - 5 years, Week 45: number analyzed (Participants) | 13 | 798 | 116
  6 months - 5 years, Week 45 | 1 | 17 | 3
  6 months - 5 years, Week 46: number analyzed (Participants) | 14 | 1019 | 129
  6 months - 5 years, Week 46 | 1 | 21 | 3
  6 months - 5 years, Week 47: number analyzed (Participants) | 16 | 1108 | 148
  6 months - 5 years, Week 47 | 2 | 21 | 4
  6 months - 5 years, Week 48: number analyzed (Participants) | 16 | 1168 | 157
  6 months - 5 years, Week 48 | 2 | 23 | 4
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7 | 33 | 4
  6-12 years, Week 40 | 1 | 2 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9 | 84 | 88
  6-12 years, Week 41 | 1 | 2 | 1
  6-12 years, Week 42: number analyzed (Participants) | 13 | 118 | 123
  6-12 years, Week 42 | 1 | 2 | 1
  6-12 years, Week 43: number analyzed (Participants) | 16 | 148 | 168
  6-12 years, Week 43 | 2 | 3 | 2
  6-12 years, Week 44: number analyzed (Participants) | 18 | 178 | 170
  6-12 years, Week 44 | 2 | 4 | 2
  6-12 years, Week 45: number analyzed (Participants) | 18 | 191 | 197
  6-12 years, Week 45 | 2 | 4 | 2
  6-12 years, Week 46: number analyzed (Participants) | 23 | 225 | 212
  6-12 years, Week 46 | 3 | 4 | 3
  6-12 years, Week 47: number analyzed (Participants) | 23 | 262 | 274
  6-12 years, Week 47 | 3 | 6 | 2
  6-12 years, Week 48: number analyzed (Participants) | 24 | 275 | 270
  6-12 years, Week 48 | 3 | 6 | 6
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12 | 4 | 1
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18 | 9 | 4
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27 | 20 | 5
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33 | 36 | 8
  13-17 years, Week 42 | 1 | 2 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33 | 42 | 9
  13-17 years, Week 43 | 1 | 2 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38 | 55 | 9
  13-17 years, Week 44 | 1 | 2 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42 | 60 | 13
  13-17 years, Week 45 | 1 | 2 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48 | 71 | 16
  13-17 years, Week 46 | 1 | 3 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49 | 77 | 17
  13-17 years, Week 47 | 1 | 3 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54 | 83 | 18
  13-17 years, Week 48 | 1 | 3 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365 | 183 | 134
  18-65 years, Week 38 | 28 | 3 | 2
  18-65 years, Week 39: number analyzed (Participants) | 1146 | 246 | 274
  18-65 years, Week 39 | 95 | 9 | 3
  18-65 years, Week 40: number analyzed (Participants) | 1821 | 300 | 391
  18-65 years, Week 40 | 172 | 14 | 4
  18-65 years, Week 41: number analyzed (Participants) | 2636 | 315 | 489
  18-65 years, Week 41 | 232 | 15 | 7
  18-65 years, Week 42: number analyzed (Participants) | 3122 | 340 | 652
  18-65 years, Week 42 | 281 | 16 | 10
  18-65 years, Week 43: number analyzed (Participants) | 3395 | 352 | 757
  18-65 years, Week 43 | 304 | 17 | 14
  18-65 years, Week 44: number analyzed (Participants) | 3673 | 361 | 843
  18-65 years, Week 44 | 325 | 17 | 16
  18-65 years, Week 45: number analyzed (Participants) | 3977 | 366 | 926
  18-65 years, Week 45 | 352 | 17 | 16
  18-65 years, Week 46: number analyzed (Participants) | 4402 | 370 | 983
  18-65 years, Week 46 | 373 | 18 | 17
  18-65 years, Week 47: number analyzed (Participants) | 4619 | 370 | 1037
  18-65 years, Week 47 | 378 | 18 | 18
  18-65 years, Week 48: number analyzed (Participants) | 4794 | 370 | 1070
  18-65 years, Week 48 | 384 | 18 | 18
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 902 | 128 | 205
  >65 years, Week 38 | 59 | 1 | 5
  >65 years, Week 39: number analyzed (Participants) | 2739 | 217 | 494
  >65 years, Week 39 | 219 | 5 | 7
  >65 years, Week 40: number analyzed (Participants) | 4198 | 306 | 726
  >65 years, Week 40 | 359 | 7 | 10
  >65 years, Week 41: number analyzed (Participants) | 5827 | 349 | 944
  >65 years, Week 41 | 471 | 8 | 13
  >65 years, Week 42: number analyzed (Participants) | 6691 | 370 | 1158
  >65 years, Week 42 | 538 | 9 | 18
  >65 years, Week 43: number analyzed (Participants) | 7148 | 382 | 1332
  >65 years, Week 43 | 571 | 11 | 23
  >65 years, Week 44: number analyzed (Participants) | 7632 | 393 | 1443
  >65 years, Week 44 | 602 | 12 | 24
  >65 years, Week 45: number analyzed (Participants) | 8028 | 396 | 1533
  >65 years, Week 45 | 629 | 12 | 26
  >65 years, Week 46: number analyzed (Participants) | 8536 | 398 | 1586
  >65 years, Week 46 | 644 | 12 | 26
  >65 years, Week 47: number analyzed (Participants) | 8790 | 398 | 1626
  >65 years, Week 47 | 652 | 12 | 26
  >65 years, Week 48: number analyzed (Participants) | 8973 | 398 | 1663
  >65 years, Week 48 | 659 | 12 | 26

83. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis.
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2 | 149 | 2
  6 months - 5 years, Week 40 | 0 | 1 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3 | 214 | 23
  6 months - 5 years, Week 41 | 0 | 3 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2 | 143 | 17
  6 months - 5 years, Week 42 | 1 | 3 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5 | 80 | 31
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0 | 116 | 5
  6 months - 5 years, Week 44 | 0 | 1 | 1
  6 months - 5 years, Week 45: number analyzed (Participants) | 0 | 87 | 38
  6 months - 5 years, Week 45 | 0 | 2 | 2
  6 months - 5 years, Week 46: number analyzed (Participants) | 1 | 221 | 13
  6 months - 5 years, Week 46 | 0 | 1 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2 | 89 | 19
  6 months - 5 years, Week 47 | 0 | 0 | 1
  6 months - 5 years, Week 48: number analyzed (Participants) | 0 | 60 | 9
  6 months - 5 years, Week 48 | 0 | 1 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4 | 28 | 3
  6-12 years, Week 40 | 1 | 1 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2 | 51 | 84
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 4 | 34 | 35
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3 | 30 | 45
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 2 | 30 | 2
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0 | 13 | 27
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5 | 34 | 15
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 0 | 37 | 35
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 1 | 13 | 23
  6-12 years, Week 48 | 0 | 0 | 2
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5 | 3 | 0
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6 | 5 | 3
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 0 | 11 | 1
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6 | 16 | 3
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0 | 6 | 1
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5 | 13 | 0
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4 | 5 | 4
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6 | 11 | 3
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1 | 6 | 1
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5 | 6 | 1
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363 | 183 | 104
  18-65 years, Week 38 | 3 | 2 | 0
  18-65 years, Week 39: number analyzed (Participants) | 781 | 63 | 140
  18-65 years, Week 39 | 13 | 4 | 0
  18-65 years, Week 40: number analyzed (Participants) | 675 | 54 | 117
  18-65 years, Week 40 | 7 | 2 | 0
  18-65 years, Week 41: number analyzed (Participants) | 815 | 15 | 98
  18-65 years, Week 41 | 8 | 0 | 1
  18-65 years, Week 42: number analyzed (Participants) | 486 | 25 | 163
  18-65 years, Week 42 | 7 | 0 | 1
  18-65 years, Week 43: number analyzed (Participants) | 273 | 12 | 105
  18-65 years, Week 43 | 5 | 0 | 1
  18-65 years, Week 44: number analyzed (Participants) | 278 | 9 | 86
  18-65 years, Week 44 | 4 | 0 | 2
  18-65 years, Week 45: number analyzed (Participants) | 304 | 5 | 83
  18-65 years, Week 45 | 3 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 425 | 4 | 57
  18-65 years, Week 46 | 6 | 0 | 0
  18-65 years, Week 47: number analyzed (Participants) | 217 | 0 | 54
  18-65 years, Week 47 | 1 | 0 | 0
  18-65 years, Week 48: number analyzed (Participants) | 175 | 0 | 33
  18-65 years, Week 48 | 3 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 898 | 128 | 147
  >65 years, Week 38 | 5 | 0 | 2
  >65 years, Week 39: number analyzed (Participants) | 1837 | 89 | 289
  >65 years, Week 39 | 10 | 1 | 0
  >65 years, Week 40: number analyzed (Participants) | 1459 | 89 | 232
  >65 years, Week 40 | 14 | 1 | 0
  >65 years, Week 41: number analyzed (Participants) | 1629 | 43 | 218
  >65 years, Week 41 | 12 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 864 | 21 | 214
  >65 years, Week 42 | 7 | 0 | 1
  >65 years, Week 43: number analyzed (Participants) | 457 | 12 | 174
  >65 years, Week 43 | 8 | 0 | 2
  >65 years, Week 44: number analyzed (Participants) | 484 | 11 | 111
  >65 years, Week 44 | 2 | 1 | 0
  >65 years, Week 45: number analyzed (Participants) | 396 | 3 | 90
  >65 years, Week 45 | 5 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 508 | 2 | 53
  >65 years, Week 46 | 5 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 254 | 0 | 40
  >65 years, Week 47 | 1 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 183 | 1 | 37
  >65 years, Week 48 | 2 | 0 | 0

84. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Fever/Pyrexia ) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis (Cumulative).
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3 | 158 | 2
  6 months - 5 years, Week 40 | 0 | 1 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6 | 372 | 25
  6 months - 5 years, Week 41 | 0 | 4 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8 | 515 | 42
  6 months - 5 years, Week 42 | 1 | 8 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13 | 595 | 73
  6 months - 5 years, Week 43 | 1 | 8 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13 | 711 | 78
  6 months - 5 years, Week 44 | 1 | 9 | 1
  6 months - 5 years, Week 45: number analyzed (Participants) | 13 | 798 | 116
  6 months - 5 years, Week 45 | 1 | 11 | 3
  6 months - 5 years, Week 46: number analyzed (Participants) | 14 | 1019 | 129
  6 months - 5 years, Week 46 | 1 | 12 | 3
  6 months - 5 years, Week 47: number analyzed (Participants) | 16 | 1108 | 148
  6 months - 5 years, Week 47 | 1 | 12 | 4
  6 months - 5 years, Week 48: number analyzed (Participants) | 16 | 1168 | 157
  6 months - 5 years, Week 48 | 1 | 13 | 4
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7 | 33 | 4
  6-12 years, Week 40 | 1 | 1 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9 | 84 | 88
  6-12 years, Week 41 | 1 | 1 | 0
  6-12 years, Week 42: number analyzed (Participants) | 13 | 118 | 123
  6-12 years, Week 42 | 1 | 1 | 0
  6-12 years, Week 43: number analyzed (Participants) | 16 | 148 | 168
  6-12 years, Week 43 | 1 | 1 | 0
  6-12 years, Week 44: number analyzed (Participants) | 18 | 178 | 170
  6-12 years, Week 44 | 1 | 1 | 0
  6-12 years, Week 45: number analyzed (Participants) | 18 | 191 | 197
  6-12 years, Week 45 | 1 | 1 | 0
  6-12 years, Week 46: number analyzed (Participants) | 23 | 225 | 212
  6-12 years, Week 46 | 1 | 1 | 0
  6-12 years, Week 47: number analyzed (Participants) | 23 | 262 | 247
  6-12 years, Week 47 | 1 | 1 | 0
  6-12 years, Week 48: number analyzed (Participants) | 24 | 275 | 270
  6-12 years, Week 48 | 1 | 1 | 2
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12 | 4 | 1
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18 | 9 | 4
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27 | 20 | 5
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33 | 36 | 8
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33 | 42 | 9
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38 | 55 | 9
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42 | 60 | 13
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48 | 71 | 16
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49 | 77 | 17
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54 | 83 | 18
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365 | 183 | 134
  18-65 years, Week 38 | 3 | 2 | 0
  18-65 years, Week 39: number analyzed (Participants) | 1146 | 246 | 274
  18-65 years, Week 39 | 16 | 6 | 0
  18-65 years, Week 40: number analyzed (Participants) | 1821 | 300 | 391
  18-65 years, Week 40 | 23 | 8 | 0
  18-65 years, Week 41: number analyzed (Participants) | 2636 | 315 | 489
  18-65 years, Week 41 | 31 | 8 | 1
  18-65 years, Week 42: number analyzed (Participants) | 3122 | 340 | 652
  18-65 years, Week 42 | 38 | 8 | 2
  18-65 years, Week 43: number analyzed (Participants) | 3395 | 352 | 757
  18-65 years, Week 43 | 43 | 8 | 3
  18-65 years, Week 44: number analyzed (Participants) | 3673 | 361 | 843
  18-65 years, Week 44 | 47 | 8 | 5
  18-65 years, Week 45: number analyzed (Participants) | 3977 | 366 | 926
  18-65 years, Week 45 | 50 | 8 | 5
  18-65 years, Week 46: number analyzed (Participants) | 4402 | 370 | 983
  18-65 years, Week 46 | 56 | 8 | 5
  18-65 years, Week 47: number analyzed (Participants) | 4619 | 370 | 1037
  18-65 years, Week 47 | 57 | 8 | 5
  18-65 years, Week 48: number analyzed (Participants) | 4794 | 370 | 1070
  18-65 years, Week 48 | 60 | 8 | 5
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 902 | 128 | 205
  >65 years, Week 38 | 5 | 0 | 2
  >65 years, Week 39: number analyzed (Participants) | 2739 | 217 | 494
  >65 years, Week 39 | 15 | 1 | 2
  >65 years, Week 40: number analyzed (Participants) | 4198 | 306 | 726
  >65 years, Week 40 | 29 | 2 | 2
  >65 years, Week 41: number analyzed (Participants) | 5827 | 349 | 944
  >65 years, Week 41 | 41 | 2 | 2
  >65 years, Week 42: number analyzed (Participants) | 6691 | 370 | 1158
  >65 years, Week 42 | 48 | 2 | 3
  >65 years, Week 43: number analyzed (Participants) | 7148 | 382 | 1332
  >65 years, Week 43 | 56 | 2 | 5
  >65 years, Week 44: number analyzed (Participants) | 7632 | 393 | 1443
  >65 years, Week 44 | 58 | 3 | 5
  >65 years, Week 45: number analyzed (Participants) | 8028 | 396 | 1533
  >65 years, Week 45 | 63 | 3 | 5
  >65 years, Week 46: number analyzed (Participants) | 8536 | 398 | 1586
  >65 years, Week 46 | 68 | 3 | 5
  >65 years, Week 47: number analyzed (Participants) | 8790 | 398 | 1626
  >65 years, Week 47 | 69 | 3 | 5
  >65 years, Week 48: number analyzed (Participants) | 8973 | 399 | 1663
  >65 years, Week 48 | 71 | 3 | 5

85. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis.
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2 | 149 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3 | 214 | 23
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2 | 143 | 17
  6 months - 5 years, Week 42 | 0 | 0 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5 | 80 | 31
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0 | 116 | 5
  6 months - 5 years, Week 44 | 0 | 0 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 0 | 87 | 38
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 1 | 221 | 13
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2 | 89 | 19
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0 | 60 | 9
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4 | 28 | 3
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2 | 51 | 84
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 4 | 34 | 35
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3 | 30 | 45
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 2 | 30 | 2
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0 | 13 | 27
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5 | 34 | 15
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 0 | 37 | 35
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 1 | 13 | 23
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5 | 3 | 0
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6 | 5 | 3
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9 | 11 | 1
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6 | 16 | 3
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0 | 6 | 1
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5 | 13 | 0
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4 | 5 | 4
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6 | 11 | 3
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1 | 6 | 1
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5 | 6 | 1
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363 | 183 | 104
  18-65 years, Week 38 | 9 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 781 | 63 | 140
  18-65 years, Week 39 | 8 | 0 | 0
  18-65 years, Week 40: number analyzed (Participants) | 675 | 54 | 117
  18-65 years, Week 40 | 10 | 0 | 0
  18-65 years, Week 41: number analyzed (Participants) | 815 | 15 | 98
  18-65 years, Week 41 | 12 | 0 | 0
  18-65 years, Week 42: number analyzed (Participants) | 486 | 25 | 163
  18-65 years, Week 42 | 9 | 0 | 0
  18-65 years, Week 43: number analyzed (Participants) | 273 | 12 | 105
  18-65 years, Week 43 | 1 | 0 | 0
  18-65 years, Week 44: number analyzed (Participants) | 278 | 9 | 86
  18-65 years, Week 44 | 4 | 0 | 0
  18-65 years, Week 45: number analyzed (Participants) | 304 | 5 | 83
  18-65 years, Week 45 | 3 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 425 | 4 | 57
  18-65 years, Week 46 | 3 | 0 | 0
  18-65 years, Week 47: number analyzed (Participants) | 217 | 0 | 54
  18-65 years, Week 47 | 0 | 0 | 0
  18-65 years, Week 48: number analyzed (Participants) | 175 | 0 | 33
  18-65 years, Week 48 | 0 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 898 | 128 | 147
  >65 years, Week 38 | 7 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 1837 | 89 | 289
  >65 years, Week 39 | 12 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 1459 | 89 | 232
  >65 years, Week 40 | 14 | 0 | 0
  >65 years, Week 41: number analyzed (Participants) | 1629 | 43 | 218
  >65 years, Week 41 | 16 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 864 | 21 | 214
  >65 years, Week 42 | 6 | 0 | 0
  >65 years, Week 43: number analyzed (Participants) | 457 | 12 | 174
  >65 years, Week 43 | 5 | 0 | 0
  >65 years, Week 44: number analyzed (Participants) | 484 | 11 | 111
  >65 years, Week 44 | 3 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 396 | 3 | 90
  >65 years, Week 45 | 5 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 508 | 2 | 53
  >65 years, Week 46 | 0 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 254 | 0 | 40
  >65 years, Week 47 | 0 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 183 | 1 | 37
  >65 years, Week 48 | 0 | 0 | 0

86. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis (Cumulative).
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3 | 158 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6 | 372 | 25
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8 | 515 | 42
  6 months - 5 years, Week 42 | 0 | 0 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13 | 595 | 73
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13 | 711 | 78
  6 months - 5 years, Week 44 | 0 | 0 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 13 | 798 | 116
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 14 | 1019 | 129
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 16 | 1108 | 148
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 16 | 1168 | 157
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7 | 33 | 4
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9 | 84 | 88
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 13 | 118 | 123
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 16 | 148 | 168
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 18 | 178 | 170
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 18 | 191 | 197
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 23 | 225 | 212
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 23 | 262 | 147
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 24 | 275 | 270
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12 | 4 | 1
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18 | 9 | 4
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27 | 20 | 5
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33 | 36 | 8
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33 | 42 | 9
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38 | 55 | 9
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42 | 60 | 13
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48 | 71 | 16
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49 | 77 | 17
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54 | 83 | 18
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365 | 183 | 134
  18-65 years, Week 38 | 9 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 1146 | 246 | 274
  18-65 years, Week 39 | 17 | 0 | 0
  18-65 years, Week 40: number analyzed (Participants) | 1821 | 300 | 391
  18-65 years, Week 40 | 27 | 0 | 0
  18-65 years, Week 41: number analyzed (Participants) | 2636 | 315 | 489
  18-65 years, Week 41 | 39 | 0 | 0
  18-65 years, Week 42: number analyzed (Participants) | 3122 | 340 | 652
  18-65 years, Week 42 | 48 | 0 | 0
  18-65 years, Week 43: number analyzed (Participants) | 3395 | 352 | 757
  18-65 years, Week 43 | 49 | 0 | 0
  18-65 years, Week 44: number analyzed (Participants) | 3673 | 361 | 843
  18-65 years, Week 44 | 53 | 0 | 0
  18-65 years, Week 45: number analyzed (Participants) | 3977 | 366 | 926
  18-65 years, Week 45 | 56 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 4402 | 370 | 983
  18-65 years, Week 46 | 59 | 0 | 0
  18-65 years, Week 47: number analyzed (Participants) | 4619 | 370 | 1037
  18-65 years, Week 47 | 59 | 0 | 0
  18-65 years, Week 48: number analyzed (Participants) | 4794 | 370 | 1070
  18-65 years, Week 48 | 59 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 902 | 128 | 205
  >65 years, Week 38 | 7 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 2739 | 217 | 494
  >65 years, Week 39 | 19 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 4198 | 306 | 726
  >65 years, Week 40 | 33 | 0 | 0
  >65 years, Week 41: number analyzed (Participants) | 5827 | 349 | 944
  >65 years, Week 41 | 49 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 6691 | 370 | 1158
  >65 years, Week 42 | 55 | 0 | 0
  >65 years, Week 43: number analyzed (Participants) | 7148 | 382 | 1332
  >65 years, Week 43 | 60 | 0 | 0
  >65 years, Week 44: number analyzed (Participants) | 7632 | 393 | 1443
  >65 years, Week 44 | 63 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 8028 | 396 | 1533
  >65 years, Week 45 | 68 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 8536 | 398 | 1586
  >65 years, Week 46 | 68 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 8790 | 398 | 1626
  >65 years, Week 47 | 68 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 8973 | 399 | 1663
  >65 years, Week 48 | 68 | 0 | 0

87. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (General Non-specific) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis.
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2 | 149 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3 | 214 | 23
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2 | 143 | 17
  6 months - 5 years, Week 42 | 0 | 0 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5 | 80 | 31
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0 | 116 | 5
  6 months - 5 years, Week 44 | 0 | 0 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 0 | 87 | 38
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 1 | 221 | 13
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2 | 89 | 19
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0 | 60 | 9
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4 | 28 | 3
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2 | 51 | 84
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 4 | 34 | 35
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3 | 30 | 45
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 2 | 30 | 2
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0 | 13 | 27
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5 | 34 | 15
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 0 | 37 | 35
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 1 | 13 | 23
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5 | 3 | 0
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6 | 5 | 3
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9 | 11 | 1
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6 | 16 | 3
  13-17 years, Week 42 | 1 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0 | 6 | 1
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5 | 13 | 0
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4 | 5 | 4
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6 | 11 | 3
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1 | 6 | 1
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5 | 6 | 1
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363 | 183 | 104
  18-65 years, Week 38 | 6 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 781 | 63 | 140
  18-65 years, Week 39 | 18 | 1 | 0
  18-65 years, Week 40: number analyzed (Participants) | 675 | 54 | 117
  18-65 years, Week 40 | 20 | 0 | 0
  18-65 years, Week 41: number analyzed (Participants) | 815 | 15 | 98
  18-65 years, Week 41 | 6 | 0 | 0
  18-65 years, Week 42: number analyzed (Participants) | 486 | 25 | 163
  18-65 years, Week 42 | 10 | 0 | 1
  18-65 years, Week 43: number analyzed (Participants) | 273 | 12 | 105
  18-65 years, Week 43 | 1 | 0 | 0
  18-65 years, Week 44: number analyzed (Participants) | 278 | 9 | 86
  18-65 years, Week 44 | 2 | 0 | 0
  18-65 years, Week 45: number analyzed (Participants) | 304 | 5 | 83
  18-65 years, Week 45 | 5 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 425 | 4 | 57
  18-65 years, Week 46 | 3 | 0 | 0
  18-65 years, Week 47: number analyzed (Participants) | 217 | 0 | 54
  18-65 years, Week 47 | 0 | 0 | 0
  18-65 years, Week 48: number analyzed (Participants) | 175 | 0 | 33
  18-65 years, Week 48 | 1 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 2295 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 898 | 128 | 147
  >65 years, Week 38 | 15 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 1837 | 89 | 289
  >65 years, Week 39 | 33 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 1459 | 89 | 232
  >65 years, Week 40 | 28 | 0 | 0
  >65 years, Week 41: number analyzed (Participants) | 1629 | 43 | 218
  >65 years, Week 41 | 22 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 864 | 21 | 214
  >65 years, Week 42 | 11 | 0 | 0
  >65 years, Week 43: number analyzed (Participants) | 457 | 12 | 174
  >65 years, Week 43 | 4 | 0 | 0
  >65 years, Week 44: number analyzed (Participants) | 484 | 11 | 111
  >65 years, Week 44 | 5 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 396 | 3 | 90
  >65 years, Week 45 | 5 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 508 | 2 | 53
  >65 years, Week 46 | 4 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 254 | 0 | 40
  >65 years, Week 47 | 2 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 183 | 1 | 37
  >65 years, Week 48 | 0 | 0 | 0

88. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (General Non-specific) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis (Cumulative).
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3 | 158 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6 | 372 | 25
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8 | 515 | 42
  6 months - 5 years, Week 42 | 0 | 0 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13 | 595 | 73
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13 | 711 | 78
  6 months - 5 years, Week 44 | 0 | 0 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 13 | 798 | 116
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 14 | 1019 | 129
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 16 | 1108 | 148
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 16 | 1168 | 157
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7 | 33 | 4
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9 | 84 | 88
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 13 | 118 | 123
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 16 | 148 | 168
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 18 | 178 | 170
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 18 | 191 | 197
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 23 | 225 | 212
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 23 | 262 | 247
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 24 | 275 | 270
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12 | 4 | 1
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18 | 9 | 4
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27 | 20 | 5
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33 | 36 | 8
  13-17 years, Week 42 | 1 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33 | 42 | 9
  13-17 years, Week 43 | 1 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38 | 55 | 9
  13-17 years, Week 44 | 1 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42 | 60 | 13
  13-17 years, Week 45 | 1 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48 | 71 | 16
  13-17 years, Week 46 | 1 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49 | 77 | 17
  13-17 years, Week 47 | 1 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54 | 83 | 18
  13-17 years, Week 48 | 1 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365 | 183 | 134
  18-65 years, Week 38 | 6 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 1146 | 246 | 274
  18-65 years, Week 39 | 24 | 1 | 0
  18-65 years, Week 40: number analyzed (Participants) | 1821 | 300 | 391
  18-65 years, Week 40 | 44 | 1 | 0
  18-65 years, Week 41: number analyzed (Participants) | 2636 | 315 | 489
  18-65 years, Week 41 | 50 | 1 | 0
  18-65 years, Week 42: number analyzed (Participants) | 3122 | 340 | 652
  18-65 years, Week 42 | 60 | 1 | 1
  18-65 years, Week 43: number analyzed (Participants) | 3395 | 352 | 757
  18-65 years, Week 43 | 61 | 1 | 1
  18-65 years, Week 44: number analyzed (Participants) | 3673 | 361 | 843
  18-65 years, Week 44 | 63 | 1 | 1
  18-65 years, Week 45: number analyzed (Participants) | 3977 | 366 | 926
  18-65 years, Week 45 | 68 | 1 | 1
  18-65 years, Week 46: number analyzed (Participants) | 4402 | 370 | 983
  18-65 years, Week 46 | 71 | 1 | 1
  18-65 years, Week 47: number analyzed (Participants) | 4619 | 370 | 1037
  18-65 years, Week 47 | 71 | 1 | 1
  18-65 years, Week 48: number analyzed (Participants) | 4794 | 370 | 1070
  18-65 years, Week 48 | 72 | 1 | 1
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 902 | 128 | 205
  >65 years, Week 38 | 15 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 2739 | 217 | 494
  >65 years, Week 39 | 48 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 4198 | 306 | 726
  >65 years, Week 40 | 76 | 0 | 0
  >65 years, Week 41: number analyzed (Participants) | 5827 | 349 | 944
  >65 years, Week 41 | 98 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 6691 | 370 | 1158
  >65 years, Week 42 | 109 | 0 | 0
  >65 years, Week 43: number analyzed (Participants) | 7148 | 382 | 1332
  >65 years, Week 43 | 113 | 0 | 0
  >65 years, Week 44: number analyzed (Participants) | 7632 | 393 | 1443
  >65 years, Week 44 | 118 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 8028 | 396 | 1533
  >65 years, Week 45 | 123 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 8536 | 398 | 1586
  >65 years, Week 46 | 127 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 8790 | 398 | 1626
  >65 years, Week 47 | 129 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 8973 | 399 | 1663
  >65 years, Week 48 | 129 | 0 | 0

89. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Respiratory/Miscellaneous) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis.
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2 | 149 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3 | 214 | 23
  6 months - 5 years, Week 41 | 0 | 1 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2 | 143 | 17
  6 months - 5 years, Week 42 | 0 | 1 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5 | 80 | 31
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0 | 116 | 5
  6 months - 5 years, Week 44 | 0 | 2 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 0 | 87 | 38
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 1 | 221 | 13
  6 months - 5 years, Week 46 | 0 | 3 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2 | 89 | 19
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0 | 60 | 9
  6 months - 5 years, Week 48 | 0 | 1 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4 | 28 | 3
  6-12 years, Week 40 | 0 | 1 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2 | 51 | 84
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 4 | 34 | 35
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3 | 30 | 45
  6-12 years, Week 43 | 0 | 0 | 1
  6-12 years, Week 44: number analyzed (Participants) | 2 | 30 | 2
  6-12 years, Week 44 | 0 | 1 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0 | 13 | 27
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5 | 34 | 15
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 0 | 37 | 35
  6-12 years, Week 47 | 0 | 2 | 0
  6-12 years, Week 48: number analyzed (Participants) | 1 | 13 | 23
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5 | 3 | 0
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6 | 5 | 3
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9 | 11 | 1
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6 | 16 | 3
  13-17 years, Week 42 | 1 | 2 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0 | 6 | 1
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5 | 13 | 0
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4 | 5 | 4
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6 | 11 | 3
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1 | 6 | 1
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5 | 6 | 1
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363 | 183 | 104
  18-65 years, Week 38 | 8 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 781 | 63 | 140
  18-65 years, Week 39 | 32 | 1 | 0
  18-65 years, Week 40: number analyzed (Participants) | 675 | 54 | 117
  18-65 years, Week 40 | 36 | 0 | 1
  18-65 years, Week 41: number analyzed (Participants) | 815 | 15 | 98
  18-65 years, Week 41 | 24 | 0 | 0
  18-65 years, Week 42: number analyzed (Participants) | 486 | 25 | 163
  18-65 years, Week 42 | 28 | 1 | 0
  18-65 years, Week 43: number analyzed (Participants) | 273 | 12 | 105
  18-65 years, Week 43 | 12 | 0 | 1
  18-65 years, Week 44: number analyzed (Participants) | 278 | 9 | 86
  18-65 years, Week 44 | 7 | 0 | 0
  18-65 years, Week 45: number analyzed (Participants) | 304 | 5 | 83
  18-65 years, Week 45 | 18 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 425 | 4 | 57
  18-65 years, Week 46 | 9 | 0 | 0
  18-65 years, Week 47: number analyzed (Participants) | 217 | 0 | 54
  18-65 years, Week 47 | 4 | 0 | 0
  18-65 years, Week 48: number analyzed (Participants) | 175 | 0 | 33
  18-65 years, Week 48 | 0 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 898 | 128 | 147
  >65 years, Week 38 | 26 | 1 | 1
  >65 years, Week 39: number analyzed (Participants) | 1837 | 89 | 289
  >65 years, Week 39 | 88 | 2 | 0
  >65 years, Week 40: number analyzed (Participants) | 1459 | 89 | 232
  >65 years, Week 40 | 75 | 1 | 0
  >65 years, Week 41: number analyzed (Participants) | 1629 | 43 | 218
  >65 years, Week 41 | 58 | 1 | 2
  >65 years, Week 42: number analyzed (Participants) | 864 | 21 | 214
  >65 years, Week 42 | 36 | 0 | 3
  >65 years, Week 43: number analyzed (Participants) | 457 | 12 | 174
  >65 years, Week 43 | 17 | 1 | 3
  >65 years, Week 44: number analyzed (Participants) | 484 | 11 | 111
  >65 years, Week 44 | 13 | 1 | 1
  >65 years, Week 45: number analyzed (Participants) | 396 | 3 | 90
  >65 years, Week 45 | 11 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 508 | 2 | 53
  >65 years, Week 46 | 4 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 254 | 0 | 40
  >65 years, Week 47 | 3 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 183 | 1 | 37
  >65 years, Week 48 | 2 | 0 | 0

90. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Respiratory/Miscellaneous) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis (Cumulative).
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3 | 158 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6 | 372 | 25
  6 months - 5 years, Week 41 | 0 | 1 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8 | 515 | 42
  6 months - 5 years, Week 42 | 0 | 2 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13 | 595 | 73
  6 months - 5 years, Week 43 | 0 | 2 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13 | 711 | 78
  6 months - 5 years, Week 44 | 0 | 4 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 13 | 798 | 116
  6 months - 5 years, Week 45 | 0 | 4 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 14 | 1019 | 129
  6 months - 5 years, Week 46 | 0 | 7 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 16 | 1108 | 148
  6 months - 5 years, Week 47 | 0 | 7 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 16 | 1168 | 157
  6 months - 5 years, Week 48 | 0 | 8 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 1
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7 | 33 | 4
  6-12 years, Week 40 | 0 | 1 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9 | 84 | 88
  6-12 years, Week 41 | 0 | 1 | 0
  6-12 years, Week 42: number analyzed (Participants) | 13 | 118 | 123
  6-12 years, Week 42 | 0 | 1 | 0
  6-12 years, Week 43: number analyzed (Participants) | 16 | 148 | 168
  6-12 years, Week 43 | 0 | 1 | 1
  6-12 years, Week 44: number analyzed (Participants) | 18 | 178 | 170
  6-12 years, Week 44 | 0 | 2 | 1
  6-12 years, Week 45: number analyzed (Participants) | 18 | 191 | 197
  6-12 years, Week 45 | 0 | 2 | 1
  6-12 years, Week 46: number analyzed (Participants) | 23 | 225 | 212
  6-12 years, Week 46 | 1 | 2 | 1
  6-12 years, Week 47: number analyzed (Participants) | 23 | 262 | 247
  6-12 years, Week 47 | 1 | 4 | 1
  6-12 years, Week 48: number analyzed (Participants) | 24 | 275 | 270
  6-12 years, Week 48 | 1 | 4 | 1
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12 | 4 | 1
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18 | 9 | 4
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27 | 20 | 5
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33 | 36 | 8
  13-17 years, Week 42 | 1 | 2 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33 | 42 | 9
  13-17 years, Week 43 | 1 | 2 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38 | 55 | 9
  13-17 years, Week 44 | 1 | 2 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42 | 60 | 13
  13-17 years, Week 45 | 1 | 2 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48 | 71 | 16
  13-17 years, Week 46 | 1 | 2 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49 | 77 | 17
  13-17 years, Week 47 | 1 | 2 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54 | 83 | 18
  13-17 years, Week 48 | 1 | 2 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365 | 183 | 134
  18-65 years, Week 38 | 8 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 1146 | 246 | 274
  18-65 years, Week 39 | 40 | 1 | 0
  18-65 years, Week 40: number analyzed (Participants) | 1821 | 300 | 391
  18-65 years, Week 40 | 76 | 1 | 1
  18-65 years, Week 41: number analyzed (Participants) | 2636 | 315 | 489
  18-65 years, Week 41 | 100 | 1 | 1
  18-65 years, Week 42: number analyzed (Participants) | 3122 | 340 | 652
  18-65 years, Week 42 | 128 | 2 | 1
  18-65 years, Week 43: number analyzed (Participants) | 3395 | 352 | 757
  18-65 years, Week 43 | 140 | 2 | 2
  18-65 years, Week 44: number analyzed (Participants) | 3673 | 361 | 843
  18-65 years, Week 44 | 147 | 2 | 2
  18-65 years, Week 45: number analyzed (Participants) | 3977 | 366 | 926
  18-65 years, Week 45 | 165 | 2 | 2
  18-65 years, Week 46: number analyzed (Participants) | 4402 | 370 | 983
  18-65 years, Week 46 | 174 | 2 | 2
  18-65 years, Week 47: number analyzed (Participants) | 4619 | 370 | 1037
  18-65 years, Week 47 | 178 | 2 | 2
  18-65 years, Week 48: number analyzed (Participants) | 4794 | 370 | 1070
  18-65 years, Week 48 | 178 | 2 | 2
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 902 | 128 | 205
  >65 years, Week 38 | 26 | 1 | 1
  >65 years, Week 39: number analyzed (Participants) | 2739 | 217 | 494
  >65 years, Week 39 | 114 | 3 | 1
  >65 years, Week 40: number analyzed (Participants) | 4198 | 306 | 726
  >65 years, Week 40 | 189 | 4 | 1
  >65 years, Week 41: number analyzed (Participants) | 5827 | 349 | 944
  >65 years, Week 41 | 247 | 5 | 3
  >65 years, Week 42: number analyzed (Participants) | 6691 | 370 | 1158
  >65 years, Week 42 | 283 | 5 | 6
  >65 years, Week 43: number analyzed (Participants) | 7148 | 382 | 1332
  >65 years, Week 43 | 300 | 6 | 9
  >65 years, Week 44: number analyzed (Participants) | 7632 | 393 | 1443
  >65 years, Week 44 | 313 | 7 | 10
  >65 years, Week 45: number analyzed (Participants) | 8028 | 396 | 1533
  >65 years, Week 45 | 324 | 7 | 10
  >65 years, Week 46: number analyzed (Participants) | 8536 | 398 | 1586
  >65 years, Week 46 | 328 | 7 | 10
  >65 years, Week 47: number analyzed (Participants) | 8790 | 398 | 1626
  >65 years, Week 47 | 331 | 7 | 10
  >65 years, Week 48: number analyzed (Participants) | 8973 | 399 | 1663
  >65 years, Week 48 | 333 | 7 | 10

91. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Gastrointestinal) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis.
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2 | 149 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3 | 214 | 23
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2 | 143 | 17
  6 months - 5 years, Week 42 | 0 | 2 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5 | 80 | 31
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0 | 116 | 5
  6 months - 5 years, Week 44 | 0 | 0 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 0 | 87 | 38
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 1 | 221 | 13
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2 | 89 | 19
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0 | 60 | 9
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4 | 28 | 3
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2 | 51 | 84
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 4 | 34 | 35
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3 | 30 | 45
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 2 | 30 | 2
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0 | 13 | 27
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5 | 34 | 15
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 0 | 37 | 35
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 1 | 13 | 23
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5 | 3 | 0
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6 | 5 | 3
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9 | 11 | 1
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6 | 16 | 3
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0 | 6 | 1
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5 | 13 | 0
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4 | 5 | 4
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6 | 11 | 3
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1 | 6 | 1
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5 | 6 | 1
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363 | 183 | 104
  18-65 years, Week 38 | 7 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 781 | 63 | 140
  18-65 years, Week 39 | 9 | 0 | 0
  18-65 years, Week 40: number analyzed (Participants) | 675 | 54 | 117
  18-65 years, Week 40 | 12 | 0 | 0
  18-65 years, Week 41: number analyzed (Participants) | 815 | 15 | 98
  18-65 years, Week 41 | 8 | 0 | 0
  18-65 years, Week 42: number analyzed (Participants) | 486 | 25 | 163
  18-65 years, Week 42 | 7 | 0 | 0
  18-65 years, Week 43: number analyzed (Participants) | 273 | 12 | 105
  18-65 years, Week 43 | 5 | 0 | 0
  18-65 years, Week 44: number analyzed (Participants) | 278 | 9 | 86
  18-65 years, Week 44 | 2 | 0 | 0
  18-65 years, Week 45: number analyzed (Participants) | 304 | 5 | 83
  18-65 years, Week 45 | 3 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 425 | 4 | 57
  18-65 years, Week 46 | 2 | 0 | 1
  18-65 years, Week 47: number analyzed (Participants) | 217 | 0 | 54
  18-65 years, Week 47 | 0 | 0 | 0
  18-65 years, Week 48: number analyzed (Participants) | 175 | 0 | 33
  18-65 years, Week 48 | 1 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 898 | 128 | 147
  >65 years, Week 38 | 11 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 1837 | 89 | 289
  >65 years, Week 39 | 23 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 1459 | 89 | 232
  >65 years, Week 40 | 22 | 0 | 1
  >65 years, Week 41: number analyzed (Participants) | 1629 | 43 | 218
  >65 years, Week 41 | 17 | 0 | 1
  >65 years, Week 42: number analyzed (Participants) | 864 | 21 | 214
  >65 years, Week 42 | 12 | 0 | 0
  >65 years, Week 43: number analyzed (Participants) | 457 | 12 | 174
  >65 years, Week 43 | 4 | 0 | 0
  >65 years, Week 44: number analyzed (Participants) | 484 | 11 | 111
  >65 years, Week 44 | 3 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 396 | 3 | 90
  >65 years, Week 45 | 3 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 508 | 2 | 53
  >65 years, Week 46 | 2 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 254 | 0 | 40
  >65 years, Week 47 | 1 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 183 | 1 | 37
  >65 years, Week 48 | 0 | 0 | 0

92. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Gastrointestinal) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis (Cumulative).
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3 | 158 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6 | 372 | 25
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8 | 515 | 42
  6 months - 5 years, Week 42 | 0 | 2 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13 | 595 | 73
  6 months - 5 years, Week 43 | 0 | 2 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13 | 711 | 78
  6 months - 5 years, Week 44 | 0 | 2 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 13 | 798 | 116
  6 months - 5 years, Week 45 | 0 | 2 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 14 | 1019 | 129
  6 months - 5 years, Week 46 | 0 | 2 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 16 | 1108 | 148
  6 months - 5 years, Week 47 | 0 | 2 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 16 | 1168 | 157
  6 months - 5 years, Week 48 | 0 | 2 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7 | 33 | 4
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9 | 84 | 88
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 13 | 118 | 123
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 16 | 148 | 168
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 18 | 178 | 170
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 18 | 191 | 197
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 23 | 225 | 212
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 23 | 262 | 247
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 24 | 275 | 270
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12 | 4 | 1
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18 | 9 | 4
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27 | 20 | 5
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33 | 36 | 8
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33 | 42 | 9
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38 | 55 | 9
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42 | 60 | 13
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48 | 71 | 16
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49 | 77 | 17
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54 | 83 | 18
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365 | 183 | 134
  18-65 years, Week 38 | 7 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 1146 | 246 | 274
  18-65 years, Week 39 | 16 | 0 | 0
  18-65 years, Week 40: number analyzed (Participants) | 1821 | 300 | 391
  18-65 years, Week 40 | 28 | 0 | 0
  18-65 years, Week 41: number analyzed (Participants) | 2636 | 315 | 489
  18-65 years, Week 41 | 36 | 0 | 0
  18-65 years, Week 42: number analyzed (Participants) | 3122 | 340 | 652
  18-65 years, Week 42 | 43 | 0 | 0
  18-65 years, Week 43: number analyzed (Participants) | 3395 | 352 | 757
  18-65 years, Week 43 | 48 | 0 | 0
  18-65 years, Week 44: number analyzed (Participants) | 3673 | 361 | 843
  18-65 years, Week 44 | 50 | 0 | 0
  18-65 years, Week 45: number analyzed (Participants) | 3977 | 366 | 926
  18-65 years, Week 45 | 53 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 4402 | 370 | 983
  18-65 years, Week 46 | 55 | 0 | 1
  18-65 years, Week 47: number analyzed (Participants) | 4619 | 370 | 1037
  18-65 years, Week 47 | 55 | 0 | 1
  18-65 years, Week 48: number analyzed (Participants) | 4794 | 370 | 1070
  18-65 years, Week 48 | 56 | 0 | 1
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 902 | 128 | 205
  >65 years, Week 38 | 11 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 2739 | 217 | 494
  >65 years, Week 39 | 34 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 4198 | 306 | 726
  >65 years, Week 40 | 56 | 0 | 1
  >65 years, Week 41: number analyzed (Participants) | 5827 | 349 | 944
  >65 years, Week 41 | 73 | 0 | 2
  >65 years, Week 42: number analyzed (Participants) | 6691 | 370 | 1158
  >65 years, Week 42 | 85 | 0 | 2
  >65 years, Week 43: number analyzed (Participants) | 7148 | 382 | 1332
  >65 years, Week 43 | 89 | 0 | 2
  >65 years, Week 44: number analyzed (Participants) | 7632 | 393 | 1443
  >65 years, Week 44 | 92 | 0 | 2
  >65 years, Week 45: number analyzed (Participants) | 8028 | 396 | 1533
  >65 years, Week 45 | 95 | 0 | 2
  >65 years, Week 46: number analyzed (Participants) | 8536 | 398 | 1586
  >65 years, Week 46 | 97 | 0 | 2
  >65 years, Week 47: number analyzed (Participants) | 8790 | 398 | 1626
  >65 years, Week 47 | 98 | 0 | 2
  >65 years, Week 48: number analyzed (Participants) | 8973 | 399 | 1663
  >65 years, Week 48 | 98 | 0 | 2

93. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Sensitivity/Anaphylaxis) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis.
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2 | 149 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3 | 214 | 23
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2 | 143 | 17
  6 months - 5 years, Week 42 | 0 | 0 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5 | 80 | 31
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0 | 116 | 5
  6 months - 5 years, Week 44 | 0 | 0 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 0 | 87 | 38
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 1 | 221 | 13
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2 | 89 | 19
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0 | 60 | 9
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4 | 28 | 3
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2 | 51 | 84
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 4 | 34 | 35
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3 | 30 | 45
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 2 | 30 | 2
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0 | 13 | 27
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5 | 34 | 15
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 0 | 37 | 35
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 1 | 13 | 23
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5 | 3 | 0
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6 | 5 | 3
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9 | 11 | 1
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6 | 16 | 3
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0 | 6 | 1
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5 | 13 | 0
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4 | 5 | 4
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6 | 11 | 3
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1 | 6 | 1
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5 | 6 | 1
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363 | 183 | 104
  18-65 years, Week 38 | 1 | 1 | 0
  18-65 years, Week 39: number analyzed (Participants) | 781 | 63 | 140
  18-65 years, Week 39 | 1 | 0 | 0
  18-65 years, Week 40: number analyzed (Participants) | 675 | 54 | 117
  18-65 years, Week 40 | 2 | 0 | 0
  18-65 years, Week 41: number analyzed (Participants) | 815 | 15 | 98
  18-65 years, Week 41 | 0 | 0 | 0
  18-65 years, Week 42: number analyzed (Participants) | 486 | 25 | 163
  18-65 years, Week 42 | 2 | 0 | 0
  18-65 years, Week 43: number analyzed (Participants) | 273 | 12 | 105
  18-65 years, Week 43 | 1 | 0 | 0
  18-65 years, Week 44: number analyzed (Participants) | 278 | 9 | 86
  18-65 years, Week 44 | 1 | 0 | 0
  18-65 years, Week 45: number analyzed (Participants) | 304 | 5 | 83
  18-65 years, Week 45 | 0 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 425 | 4 | 57
  18-65 years, Week 46 | 1 | 0 | 0
  18-65 years, Week 47: number analyzed (Participants) | 217 | 0 | 54
  18-65 years, Week 47 | 0 | 0 | 0
  18-65 years, Week 48: number analyzed (Participants) | 175 | 0 | 33
  18-65 years, Week 48 | 0 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 898 | 128 | 147
  >65 years, Week 38 | 0 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 1837 | 89 | 289
  >65 years, Week 39 | 1 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 1459 | 89 | 232
  >65 years, Week 40 | 1 | 0 | 0
  >65 years, Week 41: number analyzed (Participants) | 1629 | 43 | 218
  >65 years, Week 41 | 0 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 864 | 21 | 214
  >65 years, Week 42 | 1 | 0 | 0
  >65 years, Week 43: number analyzed (Participants) | 457 | 12 | 174
  >65 years, Week 43 | 1 | 0 | 0
  >65 years, Week 44: number analyzed (Participants) | 484 | 11 | 111
  >65 years, Week 44 | 0 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 396 | 3 | 90
  >65 years, Week 45 | 1 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 508 | 2 | 53
  >65 years, Week 46 | 0 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 254 | 0 | 40
  >65 years, Week 47 | 0 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 183 | 1 | 37
  >65 years, Week 48 | 1 | 0 | 0

94. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Sensitivity/Anaphylaxis) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis (Cumulative).
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3 | 158 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6 | 372 | 25
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8 | 515 | 42
  6 months - 5 years, Week 42 | 0 | 0 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13 | 595 | 73
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13 | 711 | 78
  6 months - 5 years, Week 44 | 0 | 0 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 13 | 798 | 116
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 14 | 1019 | 129
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 16 | 1108 | 148
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 16 | 1168 | 157
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7 | 33 | 4
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9 | 84 | 88
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 13 | 118 | 123
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 16 | 148 | 168
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 18 | 178 | 170
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 18 | 191 | 197
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 23 | 225 | 212
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 23 | 262 | 247
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 24 | 275 | 270
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12 | 4 | 1
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18 | 9 | 4
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27 | 20 | 5
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33 | 36 | 8
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33 | 42 | 9
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38 | 55 | 9
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42 | 60 | 13
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48 | 71 | 16
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49 | 77 | 17
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54 | 83 | 18
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365 | 183 | 134
  18-65 years, Week 38 | 1 | 1 | 0
  18-65 years, Week 39: number analyzed (Participants) | 1146 | 246 | 274
  18-65 years, Week 39 | 2 | 1 | 0
  18-65 years, Week 40: number analyzed (Participants) | 1821 | 300 | 391
  18-65 years, Week 40 | 4 | 1 | 0
  18-65 years, Week 41: number analyzed (Participants) | 2636 | 315 | 489
  18-65 years, Week 41 | 4 | 1 | 0
  18-65 years, Week 42: number analyzed (Participants) | 3122 | 340 | 652
  18-65 years, Week 42 | 6 | 1 | 0
  18-65 years, Week 43: number analyzed (Participants) | 3395 | 352 | 757
  18-65 years, Week 43 | 7 | 1 | 0
  18-65 years, Week 44: number analyzed (Participants) | 3673 | 361 | 843
  18-65 years, Week 44 | 8 | 1 | 0
  18-65 years, Week 45: number analyzed (Participants) | 3977 | 366 | 926
  18-65 years, Week 45 | 8 | 1 | 0
  18-65 years, Week 46: number analyzed (Participants) | 4402 | 370 | 983
  18-65 years, Week 46 | 9 | 1 | 0
  18-65 years, Week 47: number analyzed (Participants) | 4619 | 370 | 1037
  18-65 years, Week 47 | 9 | 1 | 0
  18-65 years, Week 48: number analyzed (Participants) | 4794 | 370 | 1070
  18-65 years, Week 48 | 9 | 1 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 902 | 128 | 205
  >65 years, Week 38 | 0 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 2739 | 217 | 494
  >65 years, Week 39 | 1 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 4198 | 306 | 726
  >65 years, Week 40 | 2 | 0 | 0
  >65 years, Week 41: number analyzed (Participants) | 5827 | 349 | 944
  >65 years, Week 41 | 2 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 6691 | 370 | 1158
  >65 years, Week 42 | 3 | 0 | 0
  >65 years, Week 43: number analyzed (Participants) | 7148 | 382 | 1332
  >65 years, Week 43 | 4 | 0 | 0
  >65 years, Week 44: number analyzed (Participants) | 7632 | 393 | 1443
  >65 years, Week 44 | 4 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 8028 | 396 | 1533
  >65 years, Week 45 | 5 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 8536 | 398 | 1586
  >65 years, Week 46 | 5 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 8790 | 398 | 1626
  >65 years, Week 47 | 5 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 8973 | 399 | 1663
  >65 years, Week 48 | 6 | 0 | 0

95. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis.
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2 | 149 | 2
  6 months - 5 years, Week 40 | 0 | 2 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3 | 214 | 23
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2 | 143 | 17
  6 months - 5 years, Week 42 | 0 | 1 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5 | 80 | 31
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0 | 116 | 5
  6 months - 5 years, Week 44 | 0 | 0 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 0 | 87 | 38
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 1 | 221 | 13
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2 | 89 | 19
  6 months - 5 years, Week 47 | 1 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0 | 60 | 9
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4 | 28 | 3
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2 | 51 | 84
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 4 | 34 | 35
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3 | 30 | 45
  6-12 years, Week 43 | 0 | 1 | 0
  6-12 years, Week 44: number analyzed (Participants) | 2 | 30 | 2
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0 | 13 | 27
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5 | 34 | 15
  6-12 years, Week 46 | 0 | 0 | 1
  6-12 years, Week 47: number analyzed (Participants) | 0 | 37 | 35
  6-12 years, Week 47 | 0 | 0 | 1
  6-12 years, Week 48: number analyzed (Participants) | 1 | 13 | 23
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5 | 3 | 0
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6 | 5 | 3
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9 | 11 | 1
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6 | 16 | 3
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0 | 6 | 1
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5 | 13 | 0
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4 | 5 | 4
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6 | 11 | 3
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1 | 6 | 1
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5 | 6 | 1
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363 | 183 | 104
  18-65 years, Week 38 | 0 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 781 | 63 | 140
  18-65 years, Week 39 | 2 | 0 | 0
  18-65 years, Week 40: number analyzed (Participants) | 675 | 54 | 117
  18-65 years, Week 40 | 4 | 1 | 0
  18-65 years, Week 41: number analyzed (Participants) | 815 | 15 | 98
  18-65 years, Week 41 | 2 | 0 | 0
  18-65 years, Week 42: number analyzed (Participants) | 486 | 25 | 163
  18-65 years, Week 42 | 2 | 0 | 0
  18-65 years, Week 43: number analyzed (Participants) | 273 | 12 | 105
  18-65 years, Week 43 | 2 | 0 | 0
  18-65 years, Week 44: number analyzed (Participants) | 278 | 9 | 86
  18-65 years, Week 44 | 1 | 0 | 0
  18-65 years, Week 45: number analyzed (Participants) | 304 | 5 | 83
  18-65 years, Week 45 | 1 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 425 | 4 | 57
  18-65 years, Week 46 | 2 | 0 | 0
  18-65 years, Week 47: number analyzed (Participants) | 217 | 0 | 54
  18-65 years, Week 47 | 0 | 0 | 0
  18-65 years, Week 48: number analyzed (Participants) | 175 | 0 | 33
  18-65 years, Week 48 | 0 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 898 | 128 | 147
  >65 years, Week 38 | 2 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 1837 | 89 | 289
  >65 years, Week 39 | 8 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 1459 | 89 | 232
  >65 years, Week 40 | 3 | 0 | 0
  >65 years, Week 41: number analyzed (Participants) | 1629 | 43 | 218
  >65 years, Week 41 | 5 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 864 | 43 | 218
  >65 years, Week 42 | 5 | 0 | 0
  >65 years, Week 43: number analyzed (Participants) | 457 | 12 | 174
  >65 years, Week 43 | 2 | 0 | 0
  >65 years, Week 44: number analyzed (Participants) | 484 | 11 | 111
  >65 years, Week 44 | 2 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 396 | 3 | 90
  >65 years, Week 45 | 1 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 508 | 2 | 53
  >65 years, Week 46 | 2 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 254 | 0 | 40
  >65 years, Week 47 | 2 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 183 | 1 | 37
  >65 years, Week 48 | 0 | 0 | 0

96. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis (Cumulative).
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3 | 158 | 2
  6 months - 5 years, Week 40 | 0 | 2 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6 | 372 | 25
  6 months - 5 years, Week 41 | 0 | 2 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8 | 515 | 42
  6 months - 5 years, Week 42 | 0 | 3 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13 | 595 | 73
  6 months - 5 years, Week 43 | 0 | 3 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13 | 711 | 78
  6 months - 5 years, Week 44 | 0 | 3 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 13 | 798 | 116
  6 months - 5 years, Week 45 | 0 | 3 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 14 | 1019 | 129
  6 months - 5 years, Week 46 | 0 | 3 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 16 | 1108 | 148
  6 months - 5 years, Week 47 | 1 | 3 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 16 | 1168 | 157
  6 months - 5 years, Week 48 | 1 | 3 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7 | 33 | 4
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9 | 84 | 88
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 13 | 118 | 123
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 16 | 148 | 168
  6-12 years, Week 43 | 0 | 1 | 0
  6-12 years, Week 44: number analyzed (Participants) | 18 | 178 | 170
  6-12 years, Week 44 | 0 | 1 | 0
  6-12 years, Week 45: number analyzed (Participants) | 18 | 191 | 197
  6-12 years, Week 45 | 0 | 1 | 0
  6-12 years, Week 46: number analyzed (Participants) | 23 | 225 | 212
  6-12 years, Week 46 | 0 | 1 | 1
  6-12 years, Week 47: number analyzed (Participants) | 23 | 262 | 247
  6-12 years, Week 47 | 0 | 1 | 2
  6-12 years, Week 48: number analyzed (Participants) | 24 | 275 | 270
  6-12 years, Week 48 | 0 | 1 | 2
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12 | 4 | 1
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18 | 9 | 4
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27 | 20 | 5
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33 | 36 | 8
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33 | 42 | 9
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38 | 55 | 9
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42 | 60 | 13
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48 | 71 | 16
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49 | 77 | 17
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54 | 83 | 18
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365 | 183 | 134
  18-65 years, Week 38 | 0 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 1146 | 246 | 274
  18-65 years, Week 39 | 2 | 0 | 0
  18-65 years, Week 40: number analyzed (Participants) | 1821 | 300 | 391
  18-65 years, Week 40 | 6 | 1 | 0
  18-65 years, Week 41: number analyzed (Participants) | 2636 | 315 | 489
  18-65 years, Week 41 | 8 | 1 | 0
  18-65 years, Week 42: number analyzed (Participants) | 3122 | 340 | 652
  18-65 years, Week 42 | 10 | 1 | 0
  18-65 years, Week 43: number analyzed (Participants) | 3395 | 352 | 757
  18-65 years, Week 43 | 12 | 1 | 0
  18-65 years, Week 44: number analyzed (Participants) | 3673 | 361 | 843
  18-65 years, Week 44 | 13 | 1 | 0
  18-65 years, Week 45: number analyzed (Participants) | 3977 | 366 | 926
  18-65 years, Week 45 | 14 | 1 | 0
  18-65 years, Week 46: number analyzed (Participants) | 4402 | 370 | 983
  18-65 years, Week 46 | 16 | 1 | 0
  18-65 years, Week 47: number analyzed (Participants) | 4619 | 370 | 1037
  18-65 years, Week 47 | 16 | 1 | 0
  18-65 years, Week 48: number analyzed (Participants) | 4794 | 370 | 1070
  18-65 years, Week 48 | 16 | 1 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 902 | 128 | 205
  >65 years, Week 38 | 2 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 2739 | 217 | 494
  >65 years, Week 39 | 10 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 4198 | 306 | 726
  >65 years, Week 40 | 13 | 6 | 0
  >65 years, Week 41: number analyzed (Participants) | 5827 | 349 | 944
  >65 years, Week 41 | 18 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 6691 | 370 | 1158
  >65 years, Week 42 | 21 | 1 | 0
  >65 years, Week 43: number analyzed (Participants) | 7148 | 382 | 1332
  >65 years, Week 43 | 23 | 1 | 0
  >65 years, Week 44: number analyzed (Participants) | 7632 | 393 | 1443
  >65 years, Week 44 | 25 | 1 | 0
  >65 years, Week 45: number analyzed (Participants) | 8028 | 396 | 1533
  >65 years, Week 45 | 26 | 1 | 0
  >65 years, Week 46: number analyzed (Participants) | 8536 | 398 | 1586
  >65 years, Week 46 | 28 | 1 | 0
  >65 years, Week 47: number analyzed (Participants) | 8790 | 398 | 1626
  >65 years, Week 47 | 30 | 1 | 0
  >65 years, Week 48: number analyzed (Participants) | 8973 | 399 | 1663
  >65 years, Week 48 | 30 | 1 | 0

97. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis.
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2 | 149 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3 | 214 | 23
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2 | 143 | 17
  6 months - 5 years, Week 42 | 0 | 0 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5 | 80 | 31
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0 | 116 | 5
  6 months - 5 years, Week 44 | 0 | 0 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 0 | 87 | 38
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 1 | 221 | 13
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2 | 89 | 19
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0 | 60 | 9
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4 | 28 | 3
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2 | 51 | 84
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 4 | 34 | 35
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3 | 30 | 45
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 2 | 30 | 2
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0 | 13 | 27
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5 | 34 | 15
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 0 | 37 | 35
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 1 | 13 | 23
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5 | 3 | 0
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6 | 5 | 3
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9 | 11 | 1
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6 | 16 | 3
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0 | 6 | 1
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5 | 13 | 0
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4 | 5 | 4
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6 | 11 | 3
  13-17 years, Week 46 | 0 | 1 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1 | 6 | 1
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5 | 6 | 1
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363 | 183 | 104
  18-65 years, Week 38 | 13 | 1 | 2
  18-65 years, Week 39: number analyzed (Participants) | 781 | 63 | 140
  18-65 years, Week 39 | 19 | 1 | 1
  18-65 years, Week 40: number analyzed (Participants) | 675 | 54 | 117
  18-65 years, Week 40 | 25 | 1 | 0
  18-65 years, Week 41: number analyzed (Participants) | 815 | 15 | 98
  18-65 years, Week 41 | 15 | 1 | 0
  18-65 years, Week 42: number analyzed (Participants) | 486 | 25 | 163
  18-65 years, Week 42 | 23 | 0 | 1
  18-65 years, Week 43: number analyzed (Participants) | 273 | 12 | 105
  18-65 years, Week 43 | 5 | 0 | 0
  18-65 years, Week 44: number analyzed (Participants) | 278 | 9 | 86
  18-65 years, Week 44 | 5 | 0 | 0
  18-65 years, Week 45: number analyzed (Participants) | 304 | 5 | 83
  18-65 years, Week 45 | 9 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 425 | 4 | 57
  18-65 years, Week 46 | 6 | 0 | 0
  18-65 years, Week 47: number analyzed (Participants) | 217 | 0 | 54
  18-65 years, Week 47 | 1 | 0 | 1
  18-65 years, Week 48: number analyzed (Participants) | 175 | 0 | 33
  18-65 years, Week 48 | 2 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 898 | 128 | 147
  >65 years, Week 38 | 19 | 0 | 2
  >65 years, Week 39: number analyzed (Participants) | 1837 | 89 | 289
  >65 years, Week 39 | 52 | 1 | 2
  >65 years, Week 40: number analyzed (Participants) | 1459 | 89 | 232
  >65 years, Week 40 | 50 | 0 | 3
  >65 years, Week 41: number analyzed (Participants) | 1629 | 43 | 218
  >65 years, Week 41 | 33 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 864 | 21 | 214
  >65 years, Week 42 | 23 | 0 | 1
  >65 years, Week 43: number analyzed (Participants) | 457 | 12 | 174
  >65 years, Week 43 | 3 | 1 | 0
  >65 years, Week 44: number analyzed (Participants) | 484 | 11 | 111
  >65 years, Week 44 | 10 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 396 | 3 | 90
  >65 years, Week 45 | 9 | 0 | 2
  >65 years, Week 46: number analyzed (Participants) | 508 | 2 | 53
  >65 years, Week 46 | 6 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 254 | 0 | 40
  >65 years, Week 47 | 1 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 183 | 1 | 37
  >65 years, Week 48 | 2 | 0 | 0

98. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis (Cumulative).
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3 | 158 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6 | 372 | 25
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8 | 515 | 42
  6 months - 5 years, Week 42 | 0 | 0 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13 | 595 | 73
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13 | 711 | 78
  6 months - 5 years, Week 44 | 0 | 0 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 13 | 798 | 116
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 14 | 1019 | 129
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 16 | 1108 | 148
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 16 | 1168 | 157
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7 | 33 | 4
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9 | 84 | 88
  6-12 years, Week 41 | 0 | 0 | 0
  6-12 years, Week 42: number analyzed (Participants) | 13 | 118 | 123
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 16 | 148 | 168
  6-12 years, Week 43 | 0 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 18 | 178 | 170
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 18 | 191 | 197
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 23 | 225 | 212
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 23 | 262 | 247
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 24 | 275 | 270
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12 | 4 | 1
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18 | 9 | 4
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27 | 20 | 5
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33 | 36 | 8
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33 | 42 | 9
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38 | 55 | 9
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42 | 60 | 13
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48 | 71 | 16
  13-17 years, Week 46 | 0 | 1 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49 | 77 | 17
  13-17 years, Week 47 | 0 | 1 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54 | 83 | 18
  13-17 years, Week 48 | 0 | 1 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365 | 183 | 134
  18-65 years, Week 38 | 13 | 1 | 2
  18-65 years, Week 39: number analyzed (Participants) | 1146 | 246 | 274
  18-65 years, Week 39 | 32 | 2 | 3
  18-65 years, Week 40: number analyzed (Participants) | 1821 | 300 | 391
  18-65 years, Week 40 | 57 | 3 | 3
  18-65 years, Week 41: number analyzed (Participants) | 2636 | 315 | 489
  18-65 years, Week 41 | 72 | 4 | 3
  18-65 years, Week 42: number analyzed (Participants) | 3122 | 340 | 652
  18-65 years, Week 42 | 95 | 4 | 4
  18-65 years, Week 43: number analyzed (Participants) | 3395 | 352 | 757
  18-65 years, Week 43 | 100 | 4 | 4
  18-65 years, Week 44: number analyzed (Participants) | 3673 | 361 | 843
  18-65 years, Week 44 | 105 | 4 | 4
  18-65 years, Week 45: number analyzed (Participants) | 3977 | 366 | 926
  18-65 years, Week 45 | 114 | 4 | 4
  18-65 years, Week 46: number analyzed (Participants) | 4402 | 370 | 983
  18-65 years, Week 46 | 120 | 4 | 4
  18-65 years, Week 47: number analyzed (Participants) | 4619 | 370 | 1037
  18-65 years, Week 47 | 121 | 4 | 5
  18-65 years, Week 48: number analyzed (Participants) | 4794 | 370 | 1070
  18-65 years, Week 48 | 123 | 4 | 5
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 902 | 128 | 205
  >65 years, Week 38 | 19 | 0 | 2
  >65 years, Week 39: number analyzed (Participants) | 2739 | 217 | 494
  >65 years, Week 39 | 71 | 1 | 4
  >65 years, Week 40: number analyzed (Participants) | 4198 | 306 | 726
  >65 years, Week 40 | 121 | 1 | 7
  >65 years, Week 41: number analyzed (Participants) | 5827 | 349 | 944
  >65 years, Week 41 | 154 | 1 | 7
  >65 years, Week 42: number analyzed (Participants) | 6691 | 370 | 1158
  >65 years, Week 42 | 177 | 1 | 8
  >65 years, Week 43: number analyzed (Participants) | 7148 | 382 | 1332
  >65 years, Week 43 | 180 | 2 | 8
  >65 years, Week 44: number analyzed (Participants) | 7632 | 393 | 1443
  >65 years, Week 44 | 190 | 2 | 8
  >65 years, Week 45: number analyzed (Participants) | 8028 | 396 | 1533
  >65 years, Week 45 | 199 | 2 | 10
  >65 years, Week 46: number analyzed (Participants) | 8536 | 398 | 1586
  >65 years, Week 46 | 205 | 2 | 10
  >65 years, Week 47: number analyzed (Participants) | 8790 | 398 | 1626
  >65 years, Week 47 | 206 | 2 | 10
  >65 years, Week 48: number analyzed (Participants) | 8973 | 399 | 1663
  >65 years, Week 48 | 208 | 2 | 10

99. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis.
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 2 | 149 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 3 | 214 | 23
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 2 | 143 | 17
  6 months - 5 years, Week 42 | 0 | 1 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 5 | 80 | 31
  6 months - 5 years, Week 43 | 0 | 0 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 0 | 116 | 5
  6 months - 5 years, Week 44 | 0 | 1 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 0 | 87 | 38
  6 months - 5 years, Week 45 | 0 | 0 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 1 | 221 | 13
  6 months - 5 years, Week 46 | 0 | 0 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 2 | 89 | 19
  6 months - 5 years, Week 47 | 0 | 0 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 0 | 60 | 9
  6 months - 5 years, Week 48 | 0 | 0 | 0
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 2 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 4 | 28 | 3
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 2 | 51 | 84
  6-12 years, Week 41 | 0 | 0 | 1
  6-12 years, Week 42: number analyzed (Participants) | 4 | 34 | 35
  6-12 years, Week 42 | 0 | 0 | 0
  6-12 years, Week 43: number analyzed (Participants) | 3 | 30 | 45
  6-12 years, Week 43 | 1 | 0 | 0
  6-12 years, Week 44: number analyzed (Participants) | 2 | 30 | 2
  6-12 years, Week 44 | 0 | 0 | 0
  6-12 years, Week 45: number analyzed (Participants) | 0 | 13 | 27
  6-12 years, Week 45 | 0 | 0 | 0
  6-12 years, Week 46: number analyzed (Participants) | 5 | 34 | 15
  6-12 years, Week 46 | 0 | 0 | 0
  6-12 years, Week 47: number analyzed (Participants) | 13861 | 37 | 35
  6-12 years, Week 47 | 0 | 0 | 0
  6-12 years, Week 48: number analyzed (Participants) | 1 | 13 | 23
  6-12 years, Week 48 | 0 | 0 | 0
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 5 | 3 | 0
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 6 | 5 | 3
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 9 | 11 | 1
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 6 | 16 | 3
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 0 | 6 | 1
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 5 | 13 | 0
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 4 | 5 | 4
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 6 | 11 | 3
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 1 | 6 | 1
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 5 | 6 | 1
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 363 | 183 | 104
  18-65 years, Week 38 | 12 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 781 | 63 | 140
  18-65 years, Week 39 | 22 | 1 | 0
  18-65 years, Week 40: number analyzed (Participants) | 675 | 54 | 117
  18-65 years, Week 40 | 20 | 1 | 0
  18-65 years, Week 41: number analyzed (Participants) | 815 | 15 | 98
  18-65 years, Week 41 | 13 | 0 | 2
  18-65 years, Week 42: number analyzed (Participants) | 486 | 25 | 163
  18-65 years, Week 42 | 9 | 0 | 0
  18-65 years, Week 43: number analyzed (Participants) | 273 | 12 | 105
  18-65 years, Week 43 | 8 | 1 | 2
  18-65 years, Week 44: number analyzed (Participants) | 278 | 9 | 86
  18-65 years, Week 44 | 2 | 0 | 0
  18-65 years, Week 45: number analyzed (Participants) | 304 | 5 | 83
  18-65 years, Week 45 | 9 | 0 | 0
  18-65 years, Week 46: number analyzed (Participants) | 425 | 4 | 57
  18-65 years, Week 46 | 1 | 1 | 0
  18-65 years, Week 47: number analyzed (Participants) | 217 | 0 | 54
  18-65 years, Week 47 | 1 | 0 | 0
  18-65 years, Week 48: number analyzed (Participants) | 175 | 0 | 33
  18-65 years, Week 48 | 1 | 0 | 0
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 898 | 128 | 147
  >65 years, Week 38 | 10 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 1837 | 89 | 289
  >65 years, Week 39 | 30 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 1459 | 89 | 232
  >65 years, Week 40 | 26 | 0 | 0
  >65 years, Week 41: number analyzed (Participants) | 1629 | 43 | 218
  >65 years, Week 41 | 18 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 864 | 21 | 214
  >65 years, Week 42 | 8 | 0 | 0
  >65 years, Week 43: number analyzed (Participants) | 457 | 12 | 174
  >65 years, Week 43 | 4 | 0 | 0
  >65 years, Week 44: number analyzed (Participants) | 484 | 11 | 111
  >65 years, Week 44 | 5 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 396 | 3 | 90
  >65 years, Week 45 | 4 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 508 | 2 | 53
  >65 years, Week 46 | 2 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 254 | 0 | 40
  >65 years, Week 47 | 0 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 183 | 1 | 37
  >65 years, Week 48 | 0 | 0 | 0

100. Secondary Outcome: Number of Subjects Reporting European Medical Agency (EMA) Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Age Strata, on a Weekly Basis (Cumulative).
Description: as for outcome 81
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  6 months - 5 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 37 | 0 | 0 | 0
  6 months - 5 years, Week 38: number analyzed (Participants) | 0 | 0 | 0
  6 months - 5 years, Week 38 | 0 | 0 | 0
  6 months - 5 years, Week 39: number analyzed (Participants) | 1 | 9 | 0
  6 months - 5 years, Week 39 | 0 | 0 | 0
  6 months - 5 years, Week 40: number analyzed (Participants) | 3 | 158 | 2
  6 months - 5 years, Week 40 | 0 | 0 | 0
  6 months - 5 years, Week 41: number analyzed (Participants) | 6 | 372 | 25
  6 months - 5 years, Week 41 | 0 | 0 | 0
  6 months - 5 years, Week 42: number analyzed (Participants) | 8 | 515 | 42
  6 months - 5 years, Week 42 | 0 | 1 | 0
  6 months - 5 years, Week 43: number analyzed (Participants) | 13 | 595 | 73
  6 months - 5 years, Week 43 | 0 | 1 | 0
  6 months - 5 years, Week 44: number analyzed (Participants) | 13 | 711 | 78
  6 months - 5 years, Week 44 | 0 | 2 | 0
  6 months - 5 years, Week 45: number analyzed (Participants) | 13 | 798 | 116
  6 months - 5 years, Week 45 | 0 | 2 | 0
  6 months - 5 years, Week 46: number analyzed (Participants) | 14 | 1019 | 129
  6 months - 5 years, Week 46 | 0 | 2 | 0
  6 months - 5 years, Week 47: number analyzed (Participants) | 16 | 1108 | 148
  6 months - 5 years, Week 47 | 0 | 2 | 0
  6 months - 5 years, Week 48: number analyzed (Participants) | 16 | 1168 | 157
  6 months - 5 years, Week 48 | 0 | 2 | 2
  6-12 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  6-12 years, Week 37 | 0 | 0 | 0
  6-12 years, Week 38: number analyzed (Participants) | 1 | 0 | 0
  6-12 years, Week 38 | 0 | 0 | 0
  6-12 years, Week 39: number analyzed (Participants) | 3 | 5 | 1
  6-12 years, Week 39 | 0 | 0 | 0
  6-12 years, Week 40: number analyzed (Participants) | 7 | 33 | 4
  6-12 years, Week 40 | 0 | 0 | 0
  6-12 years, Week 41: number analyzed (Participants) | 9 | 84 | 88
  6-12 years, Week 41 | 0 | 0 | 1
  6-12 years, Week 42: number analyzed (Participants) | 13 | 118 | 123
  6-12 years, Week 42 | 0 | 0 | 1
  6-12 years, Week 43: number analyzed (Participants) | 16 | 148 | 168
  6-12 years, Week 43 | 1 | 0 | 1
  6-12 years, Week 44: number analyzed (Participants) | 18 | 178 | 170
  6-12 years, Week 44 | 1 | 1 | 1
  6-12 years, Week 45: number analyzed (Participants) | 18 | 191 | 197
  6-12 years, Week 45 | 1 | 0 | 1
  6-12 years, Week 46: number analyzed (Participants) | 23 | 225 | 212
  6-12 years, Week 46 | 1 | 0 | 1
  6-12 years, Week 47: number analyzed (Participants) | 23 | 262 | 247
  6-12 years, Week 47 | 1 | 0 | 1
  6-12 years, Week 48: number analyzed (Participants) | 24 | 275 | 270
  6-12 years, Week 48 | 1 | 0 | 1
  13-17 years, Week 37: number analyzed (Participants) | 0 | 0 | 0
  13-17 years, Week 37 | 0 | 0 | 0
  13-17 years, Week 38: number analyzed (Participants) | 7 | 1 | 1
  13-17 years, Week 38 | 0 | 0 | 0
  13-17 years, Week 39: number analyzed (Participants) | 12 | 4 | 1
  13-17 years, Week 39 | 0 | 0 | 0
  13-17 years, Week 40: number analyzed (Participants) | 18 | 9 | 4
  13-17 years, Week 40 | 0 | 0 | 0
  13-17 years, Week 41: number analyzed (Participants) | 27 | 20 | 5
  13-17 years, Week 41 | 0 | 0 | 0
  13-17 years, Week 42: number analyzed (Participants) | 33 | 36 | 8
  13-17 years, Week 42 | 0 | 0 | 0
  13-17 years, Week 43: number analyzed (Participants) | 33 | 42 | 9
  13-17 years, Week 43 | 0 | 0 | 0
  13-17 years, Week 44: number analyzed (Participants) | 38 | 55 | 9
  13-17 years, Week 44 | 0 | 0 | 0
  13-17 years, Week 45: number analyzed (Participants) | 42 | 60 | 13
  13-17 years, Week 45 | 0 | 0 | 0
  13-17 years, Week 46: number analyzed (Participants) | 48 | 71 | 16
  13-17 years, Week 46 | 0 | 0 | 0
  13-17 years, Week 47: number analyzed (Participants) | 49 | 77 | 17
  13-17 years, Week 47 | 0 | 0 | 0
  13-17 years, Week 48: number analyzed (Participants) | 54 | 83 | 18
  13-17 years, Week 48 | 0 | 0 | 0
  18-65 years, Week 37: number analyzed (Participants) | 2 | 0 | 30
  18-65 years, Week 37 | 0 | 0 | 0
  18-65 years, Week 38: number analyzed (Participants) | 365 | 183 | 134
  18-65 years, Week 38 | 12 | 0 | 0
  18-65 years, Week 39: number analyzed (Participants) | 1146 | 246 | 274
  18-65 years, Week 39 | 34 | 1 | 0
  18-65 years, Week 40: number analyzed (Participants) | 1821 | 300 | 391
  18-65 years, Week 40 | 54 | 2 | 0
  18-65 years, Week 41: number analyzed (Participants) | 2636 | 315 | 489
  18-65 years, Week 41 | 67 | 2 | 2
  18-65 years, Week 42: number analyzed (Participants) | 3122 | 340 | 652
  18-65 years, Week 42 | 76 | 2 | 2
  18-65 years, Week 43: number analyzed (Participants) | 3395 | 352 | 757
  18-65 years, Week 43 | 84 | 3 | 4
  18-65 years, Week 44: number analyzed (Participants) | 3673 | 361 | 843
  18-65 years, Week 44 | 86 | 3 | 4
  18-65 years, Week 45: number analyzed (Participants) | 3977 | 366 | 926
  18-65 years, Week 45 | 95 | 3 | 4
  18-65 years, Week 46: number analyzed (Participants) | 4402 | 370 | 983
  18-65 years, Week 46 | 96 | 4 | 4
  18-65 years, Week 47: number analyzed (Participants) | 4619 | 370 | 1037
  18-65 years, Week 47 | 97 | 4 | 4
  18-65 years, Week 48: number analyzed (Participants) | 4794 | 370 | 1070
  18-65 years, Week 48 | 98 | 4 | 4
  >65 years, Week 37: number analyzed (Participants) | 4 | 0 | 58
  >65 years, Week 37 | 0 | 0 | 0
  >65 years, Week 38: number analyzed (Participants) | 902 | 128 | 205
  >65 years, Week 38 | 10 | 0 | 0
  >65 years, Week 39: number analyzed (Participants) | 2739 | 217 | 494
  >65 years, Week 39 | 40 | 0 | 0
  >65 years, Week 40: number analyzed (Participants) | 4198 | 306 | 726
  >65 years, Week 40 | 66 | 0 | 0
  >65 years, Week 41: number analyzed (Participants) | 5827 | 349 | 944
  >65 years, Week 41 | 84 | 0 | 0
  >65 years, Week 42: number analyzed (Participants) | 6691 | 370 | 1158
  >65 years, Week 42 | 92 | 0 | 0
  >65 years, Week 43: number analyzed (Participants) | 7148 | 382 | 1332
  >65 years, Week 43 | 96 | 0 | 0
  >65 years, Week 44: number analyzed (Participants) | 7632 | 393 | 1443
  >65 years, Week 44 | 101 | 0 | 0
  >65 years, Week 45: number analyzed (Participants) | 8028 | 396 | 1533
  >65 years, Week 45 | 105 | 0 | 0
  >65 years, Week 46: number analyzed (Participants) | 8536 | 398 | 1586
  >65 years, Week 46 | 107 | 0 | 0
  >65 years, Week 47: number analyzed (Participants) | 8790 | 398 | 1626
  >65 years, Week 47 | 107 | 0 | 0
  >65 years, Week 48: number analyzed (Participants) | 8973 | 399 | 1663
  >65 years, Week 48 | 107 | 0 | 0

101. Secondary Outcome: Number of Subjects Reporting EMA Defined Any AEIs and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis.
Description: AEIs were presented by categories depending of the nature of the event. -Fever or other febrile illness; - Local reaction; - General reaction (fatigue, myalgia,etc); - All other presentations that were reported following vaccination (e .g., Bell's palsy, Guillain-Barre syndrome).
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1188 | 222 | 214
  At risk, Week 38 | 81 | 4 | 7
  At risk, Week 39: number analyzed (Participants) | 2432 | 138 | 384
  At risk, Week 39 | 216 | 8 | 2
  At risk, Week 40: number analyzed (Participants) | 1980 | 262 | 320
  At risk, Week 40 | 203 | 10 | 4
  At risk, Week 41: number analyzed (Participants) | 2246 | 207 | 304
  At risk, Week 41 | 155 | 4 | 6
  At risk, Week 42: number analyzed (Participants) | 1230 | 172 | 349
  At risk, Week 42 | 105 | 7 | 7
  At risk, Week 43: number analyzed (Participants) | 669 | 106 | 259
  At risk, Week 43 | 49 | 4 | 9
  At risk, Week 44: number analyzed (Participants) | 692 | 134 | 168
  At risk, Week 44 | 47 | 4 | 3
  At risk, Week 45: number analyzed (Participants) | 613 | 88 | 167
  At risk, Week 45 | 49 | 1 | 3
  At risk, Week 46: number analyzed (Participants) | 820 | 183 | 108
  At risk, Week 46 | 29 | 5 | 2
  At risk, Week 47: number analyzed (Participants) | 401 | 71 | 101
  At risk, Week 47 | 11 | 2 | 3
  At risk, Week 48: number analyzed (Participants) | 314 | 56 | 61
  At risk, Week 48 | 11 | 1 | 1
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 38
  Not at risk, Week 38 | 6 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 194 | 31 | 46
  Not at risk, Week 39 | 11 | 2 | 1
  Not at risk, Week 40: number analyzed (Participants) | 166 | 63 | 37
  Not at risk, Week 40 | 15 | 1 | 0
  Not at risk, Week 41: number analyzed (Participants) | 212 | 127 | 120
  Not at risk, Week 41 | 17 | 1 | 1
  Not at risk, Week 42: number analyzed (Participants) | 132 | 67 | 83
  Not at risk, Week 42 | 13 | 3 | 1
  Not at risk, Week 43: number analyzed (Participants) | 69 | 34 | 97
  Not at risk, Week 43 | 8 | 0 | 1
  Not at risk, Week 44: number analyzed (Participants) | 77 | 45 | 36
  Not at risk, Week 44 | 5 | 2 | 1
  Not at risk, Week 45: number analyzed (Participants) | 91 | 25 | 75
  Not at risk, Week 45 | 5 | 1 | 1
  Not at risk, Week 46: number analyzed (Participants) | 125 | 89 | 33
  Not at risk, Week 46 | 8 | 1 | 0
  Not at risk, Week 47: number analyzed (Participants) | 73 | 61 | 48
  Not at risk, Week 47 | 3 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 50 | 24 | 42
  Not at risk, Week 48 | 2 | 1 | 1

102. Secondary Outcome: Number of Subjects Reporting EMA Defined Any AEIs and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 101
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1194 | 222 | 291
  At risk, Week 38 | 81 | 4 | 7
  At risk, Week 39: number analyzed (Participants) | 3626 | 360 | 675
  At risk, Week 39 | 297 | 12 | 9
  At risk, Week 40: number analyzed (Participants) | 5606 | 622 | 995
  At risk, Week 40 | 500 | 22 | 13
  At risk, Week 41: number analyzed (Participants) | 7852 | 829 | 1299
  At risk, Week 41 | 655 | 26 | 19
  At risk, Week 42: number analyzed (Participants) | 9082 | 1001 | 1648
  At risk, Week 42 | 760 | 33 | 26
  At risk, Week 43: number analyzed (Participants) | 9751 | 1107 | 1907
  At risk, Week 43 | 809 | 37 | 35
  At risk, Week 44: number analyzed (Participants) | 10443 | 1241 | 2075
  At risk, Week 44 | 856 | 41 | 38
  At risk, Week 45: number analyzed (Participants) | 11056 | 1329 | 2242
  At risk, Week 45 | 905 | 42 | 41
  At risk, Week 46: number analyzed (Participants) | 11876 | 1512 | 2350
  At risk, Week 46 | 934 | 47 | 43
  At risk, Week 47: number analyzed (Participants) | 12277 | 1583 | 2451
  At risk, Week 47 | 945 | 49 | 46
  At risk, Week 48: number analyzed (Participants) | 12591 | 1639 | 2512
  At risk, Week 48 | 956 | 50 | 47
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 49
  Not at risk, Week 38 | 6 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 275 | 121 | 95
  Not at risk, Week 39 | 17 | 2 | 1
  Not at risk, Week 40: number analyzed (Participants) | 441 | 184 | 132
  Not at risk, Week 40 | 32 | 3 | 1
  Not at risk, Week 41: number analyzed (Participants) | 653 | 311 | 252
  Not at risk, Week 41 | 49 | 4 | 2
  Not at risk, Week 42: number analyzed (Participants) | 785 | 378 | 335
  Not at risk, Week 42 | 62 | 7 | 3
  Not at risk, Week 43: number analyzed (Participants) | 854 | 412 | 432
  Not at risk, Week 43 | 70 | 7 | 4
  Not at risk, Week 44: number analyzed (Participants) | 931 | 457 | 468
  Not at risk, Week 44 | 75 | 9 | 5
  Not at risk, Week 45: number analyzed (Participants) | 1022 | 482 | 543
  Not at risk, Week 45 | 80 | 10 | 6
  Not at risk, Week 46: number analyzed (Participants) | 1147 | 571 | 576
  Not at risk, Week 46 | 88 | 11 | 6
  Not at risk, Week 47: number analyzed (Participants) | 1220 | 632 | 624
  Not at risk, Week 47 | 91 | 11 | 6
  Not at risk, Week 48: number analyzed (Participants) | 1270 | 656 | 666
  Not at risk, Week 48 | 93 | 12 | 7

103. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis.
Description: as for outcome 101
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1188 | 222 | 214
  At risk, Week 38 | 8 | 2 | 2
  At risk, Week 39: number analyzed (Participants) | 2432 | 138 | 384
  At risk, Week 39 | 23 | 3 | 0
  At risk, Week 40: number analyzed (Participants) | 1980 | 262 | 320
  At risk, Week 40 | 21 | 5 | 0
  At risk, Week 41: number analyzed (Participants) | 2246 | 207 | 304
  At risk, Week 41 | 18 | 2 | 1
  At risk, Week 42: number analyzed (Participants) | 1230 | 172 | 349
  At risk, Week 42 | 13 | 2 | 1
  At risk, Week 43: number analyzed (Participants) | 669 | 106 | 259
  At risk, Week 43 | 11 | 0 | 3
  At risk, Week 44: number analyzed (Participants) | 692 | 134 | 168
  At risk, Week 44 | 6 | 2 | 2
  At risk, Week 45: number analyzed (Participants) | 613 | 88 | 167
  At risk, Week 45 | 7 | 1 | 1
  At risk, Week 46: number analyzed (Participants) | 820 | 183 | 108
  At risk, Week 46 | 9 | 1 | 0
  At risk, Week 47: number analyzed (Participants) | 401 | 71 | 101
  At risk, Week 47 | 1 | 0 | 1
  At risk, Week 48: number analyzed (Participants) | 314 | 56 | 61
  At risk, Week 48 | 4 | 0 | 1
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 38
  Not at risk, Week 38 | 0 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 194 | 31 | 46
  Not at risk, Week 39 | 0 | 2 | 0
  Not at risk, Week 40: number analyzed (Participants) | 166 | 63 | 37
  Not at risk, Week 40 | 1 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 212 | 127 | 120
  Not at risk, Week 41 | 2 | 1 | 0
  Not at risk, Week 42: number analyzed (Participants) | 132 | 67 | 83
  Not at risk, Week 42 | 2 | 2 | 1
  Not at risk, Week 43: number analyzed (Participants) | 69 | 34 | 97
  Not at risk, Week 43 | 2 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 77 | 45 | 36
  Not at risk, Week 44 | 0 | 0 | 1
  Not at risk, Week 45: number analyzed (Participants) | 91 | 25 | 75
  Not at risk, Week 45 | 1 | 1 | 1
  Not at risk, Week 46: number analyzed (Participants) | 125 | 89 | 33
  Not at risk, Week 46 | 2 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 73 | 61 | 48
  Not at risk, Week 47 | 1 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 50 | 24 | 42
  Not at risk, Week 48 | 1 | 1 | 1

104. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Fever/Pyrexia) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 101
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1194 | 222 | 291
  At risk, Week 38 | 8 | 2 | 2
  At risk, Week 39: number analyzed (Participants) | 3626 | 360 | 675
  At risk, Week 39 | 31 | 5 | 2
  At risk, Week 40: number analyzed (Participants) | 5606 | 622 | 995
  At risk, Week 40 | 52 | 10 | 2
  At risk, Week 41: number analyzed (Participants) | 7852 | 829 | 1299
  At risk, Week 41 | 70 | 12 | 3
  At risk, Week 42: number analyzed (Participants) | 9082 | 1001 | 1648
  At risk, Week 42 | 83 | 14 | 4
  At risk, Week 43: number analyzed (Participants) | 9751 | 1107 | 1907
  At risk, Week 43 | 94 | 14 | 7
  At risk, Week 44: number analyzed (Participants) | 10443 | 1241 | 2075
  At risk, Week 44 | 100 | 16 | 9
  At risk, Week 45: number analyzed (Participants) | 11056 | 1329 | 2242
  At risk, Week 45 | 107 | 17 | 10
  At risk, Week 46: number analyzed (Participants) | 11876 | 1512 | 2350
  At risk, Week 46 | 116 | 18 | 10
  At risk, Week 47: number analyzed (Participants) | 12277 | 1583 | 2451
  At risk, Week 47 | 117 | 18 | 11
  At risk, Week 48: number analyzed (Participants) | 12591 | 1639 | 2512
  At risk, Week 48 | 121 | 18 | 12
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 49
  Not at risk, Week 38 | 0 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 275 | 121 | 95
  Not at risk, Week 39 | 0 | 2 | 0
  Not at risk, Week 40: number analyzed (Participants) | 441 | 184 | 132
  Not at risk, Week 40 | 1 | 2 | 0
  Not at risk, Week 41: number analyzed (Participants) | 653 | 311 | 252
  Not at risk, Week 41 | 3 | 3 | 0
  Not at risk, Week 42: number analyzed (Participants) | 785 | 378 | 335
  Not at risk, Week 42 | 5 | 5 | 1
  Not at risk, Week 43: number analyzed (Participants) | 854 | 412 | 432
  Not at risk, Week 43 | 7 | 5 | 1
  Not at risk, Week 44: number analyzed (Participants) | 931 | 457 | 468
  Not at risk, Week 44 | 7 | 5 | 2
  Not at risk, Week 45: number analyzed (Participants) | 1022 | 482 | 543
  Not at risk, Week 45 | 8 | 6 | 3
  Not at risk, Week 46: number analyzed (Participants) | 1147 | 571 | 576
  Not at risk, Week 46 | 10 | 6 | 3
  Not at risk, Week 47: number analyzed (Participants) | 1220 | 632 | 624
  Not at risk, Week 47 | 11 | 6 | 3
  Not at risk, Week 48: number analyzed (Participants) | 1270 | 656 | 666
  Not at risk, Week 48 | 12 | 7 | 4

105. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis.
Description: as for outcome 101
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1188 | 222 | 214
  At risk, Week 38 | 14 | 0 | 0
  At risk, Week 39: number analyzed (Participants) | 2432 | 138 | 384
  At risk, Week 39 | 19 | 0 | 0
  At risk, Week 40: number analyzed (Participants) | 1980 | 262 | 320
  At risk, Week 40 | 21 | 0 | 0
  At risk, Week 41: number analyzed (Participants) | 2246 | 207 | 304
  At risk, Week 41 | 26 | 0 | 0
  At risk, Week 42: number analyzed (Participants) | 1230 | 172 | 349
  At risk, Week 42 | 13 | 0 | 0
  At risk, Week 43: number analyzed (Participants) | 669 | 106 | 259
  At risk, Week 43 | 6 | 0 | 0
  At risk, Week 44: number analyzed (Participants) | 692 | 134 | 168
  At risk, Week 44 | 5 | 0 | 0
  At risk, Week 45: number analyzed (Participants) | 613 | 88 | 167
  At risk, Week 45 | 8 | 0 | 0
  At risk, Week 46: number analyzed (Participants) | 820 | 183 | 108
  At risk, Week 46 | 2 | 0 | 0
  At risk, Week 47: number analyzed (Participants) | 401 | 71 | 101
  At risk, Week 47 | 0 | 0 | 0
  At risk, Week 48: number analyzed (Participants) | 314 | 56 | 61
  At risk, Week 48 | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 38
  Not at risk, Week 38 | 2 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 194 | 31 | 46
  Not at risk, Week 39 | 1 | 0 | 1
  Not at risk, Week 40: number analyzed (Participants) | 166 | 63 | 37
  Not at risk, Week 40 | 3 | 0 | 3
  Not at risk, Week 41: number analyzed (Participants) | 212 | 127 | 120
  Not at risk, Week 41 | 2 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 132 | 67 | 83
  Not at risk, Week 42 | 2 | 0 | 0
  Not at risk, Week 43: number analyzed (Participants) | 69 | 34 | 97
  Not at risk, Week 43 | 0 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 77 | 45 | 36
  Not at risk, Week 44 | 2 | 0 | 0
  Not at risk, Week 45: number analyzed (Participants) | 91 | 25 | 75
  Not at risk, Week 45 | 0 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 125 | 89 | 33
  Not at risk, Week 46 | 1 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 73 | 61 | 48
  Not at risk, Week 47 | 0 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 50 | 24 | 42
  Not at risk, Week 48 | 0 | 0 | 0

106. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Local Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 101
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1194 | 222 | 291
  At risk, Week 38 | 14 | 0 | 0
  At risk, Week 39: number analyzed (Participants) | 3626 | 360 | 675
  At risk, Week 39 | 33 | 0 | 0
  At risk, Week 40: number analyzed (Participants) | 5606 | 622 | 995
  At risk, Week 40 | 54 | 0 | 0
  At risk, Week 41: number analyzed (Participants) | 7852 | 829 | 1299
  At risk, Week 41 | 80 | 0 | 0
  At risk, Week 42: number analyzed (Participants) | 9082 | 1001 | 1648
  At risk, Week 42 | 93 | 0 | 0
  At risk, Week 43: number analyzed (Participants) | 9751 | 1107 | 1907
  At risk, Week 43 | 99 | 0 | 0
  At risk, Week 44: number analyzed (Participants) | 10443 | 1241 | 2075
  At risk, Week 44 | 104 | 0 | 0
  At risk, Week 45: number analyzed (Participants) | 11056 | 1329 | 2242
  At risk, Week 45 | 112 | 0 | 0
  At risk, Week 46: number analyzed (Participants) | 11876 | 1512 | 2350
  At risk, Week 46 | 114 | 0 | 0
  At risk, Week 47: number analyzed (Participants) | 12277 | 1583 | 2451
  At risk, Week 47 | 114 | 0 | 0
  At risk, Week 48: number analyzed (Participants) | 12591 | 1639 | 2512
  At risk, Week 48 | 114 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 49
  Not at risk, Week 38 | 2 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 275 | 121 | 95
  Not at risk, Week 39 | 3 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 441 | 184 | 132
  Not at risk, Week 40 | 6 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 653 | 311 | 252
  Not at risk, Week 41 | 8 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 785 | 378 | 335
  Not at risk, Week 42 | 10 | 0 | 0
  Not at risk, Week 43: number analyzed (Participants) | 854 | 412 | 432
  Not at risk, Week 43 | 10 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 931 | 457 | 468
  Not at risk, Week 44 | 12 | 0 | 0
  Not at risk, Week 45: number analyzed (Participants) | 1022 | 482 | 543
  Not at risk, Week 45 | 12 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 1147 | 571 | 576
  Not at risk, Week 46 | 13 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 1220 | 632 | 624
  Not at risk, Week 47 | 13 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 1270 | 656 | 666
  Not at risk, Week 48 | 13 | 0 | 0

107. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (General Non-specific Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis.
Description: as for outcome 101
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1188 | 222 | 214
  At risk, Week 38 | 19 | 0 | 0
  At risk, Week 39: number analyzed (Participants) | 2432 | 138 | 384
  At risk, Week 39 | 46 | 1 | 0
  At risk, Week 40: number analyzed (Participants) | 1980 | 262 | 320
  At risk, Week 40 | 46 | 0 | 0
  At risk, Week 41: number analyzed (Participants) | 2246 | 207 | 304
  At risk, Week 41 | 26 | 0 | 0
  At risk, Week 42: number analyzed (Participants) | 1230 | 172 | 349
  At risk, Week 42 | 20 | 0 | 1
  At risk, Week 43: number analyzed (Participants) | 669 | 106 | 259
  At risk, Week 43 | 4 | 0 | 0
  At risk, Week 44: number analyzed (Participants) | 692 | 134 | 168
  At risk, Week 44 | 7 | 0 | 0
  At risk, Week 45: number analyzed (Participants) | 613 | 88 | 167
  At risk, Week 45 | 8 | 0 | 0
  At risk, Week 46: number analyzed (Participants) | 820 | 183 | 108
  At risk, Week 46 | 5 | 0 | 0
  At risk, Week 47: number analyzed (Participants) | 401 | 71 | 101
  At risk, Week 47 | 2 | 0 | 0
  At risk, Week 48: number analyzed (Participants) | 314 | 56 | 61
  At risk, Week 48 | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 38
  Not at risk, Week 38 | 2 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 194 | 31 | 46
  Not at risk, Week 39 | 5 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 166 | 63 | 37
  Not at risk, Week 40 | 2 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 212 | 127 | 120
  Not at risk, Week 41 | 2 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 132 | 67 | 83
  Not at risk, Week 42 | 2 | 0 | 0
  Not at risk, Week 43: number analyzed (Participants) | 69 | 34 | 97
  Not at risk, Week 43 | 1 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 77 | 45 | 36
  Not at risk, Week 44 | 0 | 0 | 0
  Not at risk, Week 45: number analyzed (Participants) | 91 | 25 | 75
  Not at risk, Week 45 | 2 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 125 | 89 | 33
  Not at risk, Week 46 | 2 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 73 | 61 | 48
  Not at risk, Week 47 | 0 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 50 | 24 | 42
  Not at risk, Week 48 | 1 | 0 | 0

108. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (General Non-specific Symptoms) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 101
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Vaccinated_Unknown Group: Volunteered subjects who received influenza vaccination (GSK or Non-GSK not known) in10 volunteer practices.
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1194 | 222 | 291
  At risk, Week 38 | 19 | 0 | 0
  At risk, Week 39: number analyzed (Participants) | 3626 | 360 | 675
  At risk, Week 39 | 65 | 1 | 0
  At risk, Week 40: number analyzed (Participants) | 5606 | 622 | 995
  At risk, Week 40 | 111 | 1 | 0
  At risk, Week 41: number analyzed (Participants) | 7852 | 829 | 1299
  At risk, Week 41 | 137 | 1 | 0
  At risk, Week 42: number analyzed (Participants) | 9082 | 1001 | 1648
  At risk, Week 42 | 157 | 1 | 1
  At risk, Week 43: number analyzed (Participants) | 9751 | 1107 | 1907
  At risk, Week 43 | 161 | 1 | 1
  At risk, Week 44: number analyzed (Participants) | 10443 | 1241 | 2075
  At risk, Week 44 | 168 | 1 | 1
  At risk, Week 45: number analyzed (Participants) | 11056 | 1329 | 2242
  At risk, Week 45 | 176 | 1 | 1
  At risk, Week 46: number analyzed (Participants) | 11876 | 1512 | 2350
  At risk, Week 46 | 181 | 1 | 1
  At risk, Week 47: number analyzed (Participants) | 12277 | 1583 | 2451
  At risk, Week 47 | 183 | 1 | 1
  At risk, Week 48: number analyzed (Participants) | 12591 | 1639 | 2512
  At risk, Week 48 | 183 | 1 | 1
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 49
  Not at risk, Week 38 | 2 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 275 | 121 | 95
  Not at risk, Week 39 | 7 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 441 | 184 | 132
  Not at risk, Week 40 | 9 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 653 | 311 | 252
  Not at risk, Week 41 | 11 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 785 | 378 | 335
  Not at risk, Week 42 | 13 | 0 | 0
  Not at risk, Week 43: number analyzed (Participants) | 854 | 412 | 432
  Not at risk, Week 43 | 14 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 931 | 457 | 468
  Not at risk, Week 44 | 14 | 0 | 0
  Not at risk, Week 45: number analyzed (Participants) | 1022 | 482 | 543
  Not at risk, Week 45 | 16 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 1147 | 571 | 576
  Not at risk, Week 46 | 18 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 1220 | 632 | 624
  Not at risk, Week 47 | 18 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 1270 | 656 | 666
  Not at risk, Week 48 | 19 | 0 | 0

109. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Respiratory/Miscellaneous Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis.
Description: as for outcome 69
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1188 | 222 | 214
  At risk, Week 38 | 32 | 1 | 1
  At risk, Week 39: number analyzed (Participants) | 2432 | 138 | 384
  At risk, Week 39 | 114 | 2 | 0
  At risk, Week 40: number analyzed (Participants) | 1980 | 262 | 320
  At risk, Week 40 | 103 | 2 | 1
  At risk, Week 41: number analyzed (Participants) | 2246 | 207 | 304
  At risk, Week 41 | 77 | 2 | 2
  At risk, Week 42: number analyzed (Participants) | 1230 | 172 | 349
  At risk, Week 42 | 56 | 3 | 3
  At risk, Week 43: number analyzed (Participants) | 669 | 106 | 259
  At risk, Week 43 | 27 | 1 | 4
  At risk, Week 44: number analyzed (Participants) | 692 | 134 | 168
  At risk, Week 44 | 18 | 3 | 1
  At risk, Week 45: number analyzed (Participants) | 613 | 88 | 167
  At risk, Week 45 | 26 | 0 | 0
  At risk, Week 46: number analyzed (Participants) | 820 | 183 | 108
  At risk, Week 46 | 12 | 2 | 0
  At risk, Week 47: number analyzed (Participants) | 401 | 71 | 101
  At risk, Week 47 | 5 | 2 | 0
  At risk, Week 48: number analyzed (Participants) | 314 | 56 | 61
  At risk, Week 48 | 2 | 1 | 0
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 38
  Not at risk, Week 38 | 2 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 194 | 31 | 46
  Not at risk, Week 39 | 6 | 1 | 0
  Not at risk, Week 40: number analyzed (Participants) | 166 | 63 | 37
  Not at risk, Week 40 | 8 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 212 | 127 | 120
  Not at risk, Week 41 | 5 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 132 | 67 | 83
  Not at risk, Week 42 | 9 | 1 | 0
  Not at risk, Week 43: number analyzed (Participants) | 69 | 34 | 97
  Not at risk, Week 43 | 2 | 0 | 1
  Not at risk, Week 44: number analyzed (Participants) | 77 | 45 | 36
  Not at risk, Week 44 | 2 | 1 | 0
  Not at risk, Week 45: number analyzed (Participants) | 91 | 25 | 75
  Not at risk, Week 45 | 3 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 125 | 89 | 33
  Not at risk, Week 46 | 2 | 1 | 0
  Not at risk, Week 47: number analyzed (Participants) | 73 | 61 | 48
  Not at risk, Week 47 | 2 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 50 | 24 | 42
  Not at risk, Week 48 | 0 | 0 | 0

110. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Respiratory/Miscellaneous Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 69
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1194 | 222 | 291
  At risk, Week 38 | 32 | 1 | 1
  At risk, Week 39: number analyzed (Participants) | 3626 | 360 | 675
  At risk, Week 39 | 146 | 3 | 1
  At risk, Week 40: number analyzed (Participants) | 5606 | 622 | 995
  At risk, Week 40 | 249 | 5 | 2
  At risk, Week 41: number analyzed (Participants) | 7852 | 829 | 1299
  At risk, Week 41 | 326 | 7 | 4
  At risk, Week 42: number analyzed (Participants) | 9082 | 1001 | 1648
  At risk, Week 42 | 382 | 10 | 7
  At risk, Week 43: number analyzed (Participants) | 9751 | 1107 | 1907
  At risk, Week 43 | 409 | 11 | 11
  At risk, Week 44: number analyzed (Participants) | 10443 | 1241 | 2075
  At risk, Week 44 | 427 | 14 | 12
  At risk, Week 45: number analyzed (Participants) | 11056 | 1329 | 2242
  At risk, Week 45 | 453 | 14 | 12
  At risk, Week 46: number analyzed (Participants) | 11876 | 1512 | 2350
  At risk, Week 46 | 465 | 16 | 12
  At risk, Week 47: number analyzed (Participants) | 12277 | 1583 | 2451
  At risk, Week 47 | 470 | 18 | 12
  At risk, Week 48: number analyzed (Participants) | 12591 | 1639 | 2512
  At risk, Week 48 | 472 | 19 | 12
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 49
  Not at risk, Week 38 | 2 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 275 | 121 | 95
  Not at risk, Week 39 | 8 | 1 | 0
  Not at risk, Week 40: number analyzed (Participants) | 441 | 184 | 132
  Not at risk, Week 40 | 16 | 1 | 0
  Not at risk, Week 41: number analyzed (Participants) | 653 | 311 | 252
  Not at risk, Week 41 | 21 | 1 | 0
  Not at risk, Week 42: number analyzed (Participants) | 785 | 378 | 335
  Not at risk, Week 42 | 30 | 2 | 0
  Not at risk, Week 43: number analyzed (Participants) | 854 | 412 | 423
  Not at risk, Week 43 | 32 | 2 | 1
  Not at risk, Week 44: number analyzed (Participants) | 931 | 457 | 468
  Not at risk, Week 44 | 34 | 3 | 1
  Not at risk, Week 45: number analyzed (Participants) | 1022 | 482 | 543
  Not at risk, Week 45 | 37 | 3 | 1
  Not at risk, Week 46: number analyzed (Participants) | 1147 | 571 | 576
  Not at risk, Week 46 | 39 | 4 | 1
  Not at risk, Week 47: number analyzed (Participants) | 1220 | 632 | 624
  Not at risk, Week 47 | 41 | 4 | 1
  Not at risk, Week 48: number analyzed (Participants) | 1270 | 656 | 666
  Not at risk, Week 48 | 41 | 4 | 1

111. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Gastrointestinal Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis.
Description: Gastrointestinal AEs include any gastrointestinal AEs, decreased appetite, diarrhoea, nausea and vomiting.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1188 | 222 | 214
  At risk, Week 38 | 16 | 0 | 0
  At risk, Week 39: number analyzed (Participants) | 2432 | 138 | 384
  At risk, Week 39 | 30 | 0 | 0
  At risk, Week 40: number analyzed (Participants) | 1980 | 262 | 320
  At risk, Week 40 | 33 | 0 | 1
  At risk, Week 41: number analyzed (Participants) | 2246 | 207 | 304
  At risk, Week 41 | 22 | 0 | 1
  At risk, Week 42: number analyzed (Participants) | 1230 | 172 | 349
  At risk, Week 42 | 18 | 1 | 0
  At risk, Week 43: number analyzed (Participants) | 669 | 106 | 259
  At risk, Week 43 | 7 | 0 | 0
  At risk, Week 44: number analyzed (Participants) | 692 | 134 | 168
  At risk, Week 44 | 5 | 0 | 0
  At risk, Week 45: number analyzed (Participants) | 613 | 88 | 167
  At risk, Week 45 | 6 | 0 | 0
  At risk, Week 46: number analyzed (Participants) | 820 | 183 | 108
  At risk, Week 46 | 4 | 0 | 1
  At risk, Week 47: number analyzed (Participants) | 401 | 71 | 101
  At risk, Week 47 | 1 | 0 | 0
  At risk, Week 48: number analyzed (Participants) | 314 | 56 | 61
  At risk, Week 48 | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 38
  Not at risk, Week 38 | 2 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 194 | 31 | 46
  Not at risk, Week 39 | 2 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 166 | 63 | 37
  Not at risk, Week 40 | 1 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 212 | 127 | 120
  Not at risk, Week 41 | 3 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 132 | 67 | 83
  Not at risk, Week 42 | 1 | 1 | 0
  Not at risk, Week 43: number analyzed (Participants) | 69 | 34 | 97
  Not at risk, Week 43 | 2 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 77 | 45 | 36
  Not at risk, Week 44 | 0 | 0 | 0
  Not at risk, Week 45: number analyzed (Participants) | 91 | 25 | 75
  Not at risk, Week 45 | 0 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 125 | 89 | 33
  Not at risk, Week 46 | 0 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 73 | 61 | 48
  Not at risk, Week 47 | 0 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 50 | 24 | 42
  Not at risk, Week 48 | 1 | 0 | 0

112. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Gastrointestinal Adverse Events) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: Gastrointestinal AEs include any gastrointestinal AEs, decreased appetite, diarrhoea, nausea and vomiting.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1194 | 222 | 291
  At risk, Week 38 | 16 | 0 | 0
  At risk, Week 39: number analyzed (Participants) | 3626 | 360 | 675
  At risk, Week 39 | 46 | 0 | 0
  At risk, Week 40: number analyzed (Participants) | 5606 | 622 | 995
  At risk, Week 40 | 79 | 0 | 1
  At risk, Week 41: number analyzed (Participants) | 7852 | 829 | 1299
  At risk, Week 41 | 101 | 0 | 2
  At risk, Week 42: number analyzed (Participants) | 9082 | 1001 | 1648
  At risk, Week 42 | 119 | 1 | 2
  At risk, Week 43: number analyzed (Participants) | 9751 | 1107 | 1907
  At risk, Week 43 | 126 | 1 | 2
  At risk, Week 44: number analyzed (Participants) | 10443 | 1241 | 2075
  At risk, Week 44 | 131 | 1 | 2
  At risk, Week 45: number analyzed (Participants) | 11056 | 1329 | 2242
  At risk, Week 45 | 137 | 1 | 2
  At risk, Week 46: number analyzed (Participants) | 11876 | 1512 | 2350
  At risk, Week 46 | 141 | 1 | 3
  At risk, Week 47: number analyzed (Participants) | 12277 | 1583 | 2451
  At risk, Week 47 | 142 | 1 | 3
  At risk, Week 48: number analyzed (Participants) | 12591 | 1639 | 2512
  At risk, Week 48 | 142 | 1 | 3
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 49
  Not at risk, Week 38 | 2 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 275 | 121 | 95
  Not at risk, Week 39 | 4 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 441 | 184 | 132
  Not at risk, Week 40 | 5 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 653 | 311 | 252
  Not at risk, Week 41 | 8 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 785 | 378 | 335
  Not at risk, Week 42 | 9 | 1 | 0
  Not at risk, Week 43: number analyzed (Participants) | 854 | 412 | 432
  Not at risk, Week 43 | 11 | 1 | 0
  Not at risk, Week 44: number analyzed (Participants) | 931 | 457 | 468
  Not at risk, Week 44 | 11 | 1 | 0
  Not at risk, Week 45: number analyzed (Participants) | 1022 | 482 | 543
  Not at risk, Week 45 | 11 | 1 | 0
  Not at risk, Week 46: number analyzed (Participants) | 1147 | 571 | 576
  Not at risk, Week 46 | 11 | 1 | 0
  Not at risk, Week 47: number analyzed (Participants) | 1220 | 632 | 624
  Not at risk, Week 47 | 11 | 1 | 0
  Not at risk, Week 48: number analyzed (Participants) | 1270 | 656 | 666
  Not at risk, Week 48 | 12 | 1 | 0

113. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Sensitivity/Anaphylaxis) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis
Description: as for outcome 73
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1188 | 222 | 214
  At risk, Week 38 | 1 | 1 | 0
  At risk, Week 39: number analyzed (Participants) | 2432 | 138 | 384
  At risk, Week 39 | 2 | 0 | 0
  At risk, Week 40: number analyzed (Participants) | 1980 | 262 | 320
  At risk, Week 40 | 3 | 0 | 0
  At risk, Week 41: number analyzed (Participants) | 2246 | 207 | 304
  At risk, Week 41 | 0 | 0 | 0
  At risk, Week 42: number analyzed (Participants) | 1230 | 172 | 349
  At risk, Week 42 | 1 | 0 | 0
  At risk, Week 43: number analyzed (Participants) | 669 | 106 | 259
  At risk, Week 43 | 2 | 0 | 0
  At risk, Week 44: number analyzed (Participants) | 692 | 134 | 168
  At risk, Week 44 | 1 | 0 | 0
  At risk, Week 45: number analyzed (Participants) | 613 | 88 | 167
  At risk, Week 45 | 1 | 0 | 0
  At risk, Week 46: number analyzed (Participants) | 820 | 183 | 108
  At risk, Week 46 | 0 | 0 | 0
  At risk, Week 47: number analyzed (Participants) | 401 | 71 | 101
  At risk, Week 47 | 0 | 0 | 0
  At risk, Week 48: number analyzed (Participants) | 314 | 56 | 61
  At risk, Week 48 | 1 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 38
  Not at risk, Week 38 | 0 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 194 | 31 | 46
  Not at risk, Week 39 | 0 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 166 | 63 | 37
  Not at risk, Week 40 | 0 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 212 | 127 | 120
  Not at risk, Week 41 | 0 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 132 | 67 | 83
  Not at risk, Week 42 | 2 | 0 | 0
  Not at risk, Week 43: number analyzed (Participants) | 69 | 34 | 97
  Not at risk, Week 43 | 0 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 77 | 45 | 36
  Not at risk, Week 44 | 0 | 0 | 0
  Not at risk, Week 45: number analyzed (Participants) | 91 | 25 | 75
  Not at risk, Week 45 | 0 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 125 | 89 | 33
  Not at risk, Week 46 | 1 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 73 | 61 | 48
  Not at risk, Week 47 | 0 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 50 | 24 | 42
  Not at risk, Week 48 | 0 | 0 | 0

114. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Sensitivity/Anaphylaxis) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 73
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1194 | 222 | 291
  At risk, Week 38 | 1 | 1 | 0
  At risk, Week 39: number analyzed (Participants) | 3626 | 360 | 675
  At risk, Week 39 | 3 | 1 | 0
  At risk, Week 40: number analyzed (Participants) | 5606 | 622 | 995
  At risk, Week 40 | 6 | 1 | 0
  At risk, Week 41: number analyzed (Participants) | 7852 | 829 | 1299
  At risk, Week 41 | 6 | 1 | 0
  At risk, Week 42: number analyzed (Participants) | 9082 | 1001 | 1648
  At risk, Week 42 | 7 | 1 | 0
  At risk, Week 43: number analyzed (Participants) | 9751 | 1107 | 1907
  At risk, Week 43 | 9 | 1 | 0
  At risk, Week 44: number analyzed (Participants) | 10443 | 1241 | 2075
  At risk, Week 44 | 10 | 1 | 0
  At risk, Week 45: number analyzed (Participants) | 11056 | 1329 | 2242
  At risk, Week 45 | 11 | 1 | 0
  At risk, Week 46: number analyzed (Participants) | 11876 | 1512 | 2350
  At risk, Week 46 | 11 | 1 | 0
  At risk, Week 47: number analyzed (Participants) | 12277 | 1583 | 2451
  At risk, Week 47 | 11 | 1 | 0
  At risk, Week 48: number analyzed (Participants) | 12591 | 1639 | 2512
  At risk, Week 48 | 12 | 1 | 0
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 49
  Not at risk, Week 38 | 0 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 275 | 121 | 95
  Not at risk, Week 39 | 0 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 441 | 184 | 132
  Not at risk, Week 40 | 0 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 663 | 311 | 252
  Not at risk, Week 41 | 0 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 785 | 378 | 335
  Not at risk, Week 42 | 2 | 0 | 0
  Not at risk, Week 43: number analyzed (Participants) | 854 | 412 | 432
  Not at risk, Week 43 | 2 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 931 | 457 | 468
  Not at risk, Week 44 | 2 | 0 | 0
  Not at risk, Week 45: number analyzed (Participants) | 1022 | 482 | 543
  Not at risk, Week 45 | 2 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 1147 | 571 | 576
  Not at risk, Week 46 | 3 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 1220 | 632 | 624
  Not at risk, Week 47 | 3 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 1270 | 656 | 666
  Not at risk, Week 48 | 3 | 0 | 0

115. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis
Description: Rash AEs include any rash AEs, generalised rash and rash.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1188 | 222 | 214
  At risk, Week 38 | 2 | 0 | 0
  At risk, Week 39: number analyzed (Participants) | 2432 | 138 | 384
  At risk, Week 39 | 10 | 0 | 0
  At risk, Week 40: number analyzed (Participants) | 1980 | 262 | 320
  At risk, Week 40 | 7 | 2 | 0
  At risk, Week 41: number analyzed (Participants) | 2246 | 207 | 304
  At risk, Week 41 | 7 | 0 | 0
  At risk, Week 42: number analyzed (Participants) | 1230 | 172 | 349
  At risk, Week 42 | 4 | 2 | 0
  At risk, Week 43: number analyzed (Participants) | 669 | 106 | 259
  At risk, Week 43 | 4 | 1 | 0
  At risk, Week 44: number analyzed (Participants) | 692 | 134 | 168
  At risk, Week 44 | 3 | 0 | 0
  At risk, Week 45: number analyzed (Participants) | 613 | 88 | 167
  At risk, Week 45 | 2 | 0 | 0
  At risk, Week 46: number analyzed (Participants) | 820 | 183 | 108
  At risk, Week 46 | 3 | 0 | 1
  At risk, Week 47: number analyzed (Participants) | 401 | 71 | 101
  At risk, Week 47 | 3 | 0 | 1
  At risk, Week 48: number analyzed (Participants) | 314 | 56 | 61
  At risk, Week 48 | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 38
  Not at risk, Week 38 | 0 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 194 | 31 | 46
  Not at risk, Week 39 | 0 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 166 | 63 | 37
  Not at risk, Week 40 | 0 | 1 | 0
  Not at risk, Week 41: number analyzed (Participants) | 212 | 127 | 120
  Not at risk, Week 41 | 0 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 132 | 67 | 83
  Not at risk, Week 42 | 1 | 0 | 0
  Not at risk, Week 43: number analyzed (Participants) | 69 | 34 | 97
  Not at risk, Week 43 | 0 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 77 | 45 | 36
  Not at risk, Week 44 | 0 | 0 | 0
  Not at risk, Week 45: number analyzed (Participants) | 91 | 25 | 75
  Not at risk, Week 45 | 0 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 125 | 89 | 33
  Not at risk, Week 46 | 1 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 73 | 61 | 48
  Not at risk, Week 47 | 0 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 50 | 24 | 42
  Not at risk, Week 48 | 0 | 0 | 0

116. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Rash) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative)
Description: Rash AEs include any rash AEs, generalised rash and rash.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1194 | 222 | 291
  At risk, Week 38 | 2 | 0 | 0
  At risk, Week 39: number analyzed (Participants) | 3626 | 360 | 675
  At risk, Week 39 | 12 | 0 | 0
  At risk, Week 40: number analyzed (Participants) | 5606 | 622 | 995
  At risk, Week 40 | 19 | 2 | 0
  At risk, Week 41: number analyzed (Participants) | 7852 | 829 | 1299
  At risk, Week 41 | 26 | 2 | 0
  At risk, Week 42: number analyzed (Participants) | 9082 | 1001 | 1648
  At risk, Week 42 | 30 | 4 | 0
  At risk, Week 43: number analyzed (Participants) | 9751 | 1107 | 1907
  At risk, Week 43 | 34 | 5 | 0
  At risk, Week 44: number analyzed (Participants) | 10443 | 1241 | 2075
  At risk, Week 44 | 37 | 5 | 0
  At risk, Week 45: number analyzed (Participants) | 11056 | 1329 | 2242
  At risk, Week 45 | 39 | 5 | 0
  At risk, Week 46: number analyzed (Participants) | 11876 | 1512 | 2350
  At risk, Week 46 | 42 | 5 | 1
  At risk, Week 47: number analyzed (Participants) | 12277 | 1583 | 2451
  At risk, Week 47 | 45 | 5 | 2
  At risk, Week 48: number analyzed (Participants) | 12591 | 1639 | 2512
  At risk, Week 48 | 45 | 5 | 2
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 49
  Not at risk, Week 38 | 0 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 275 | 121 | 95
  Not at risk, Week 39 | 0 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 441 | 184 | 132
  Not at risk, Week 40 | 0 | 1 | 0
  Not at risk, Week 41: number analyzed (Participants) | 653 | 311 | 252
  Not at risk, Week 41 | 0 | 1 | 0
  Not at risk, Week 42: number analyzed (Participants) | 785 | 378 | 335
  Not at risk, Week 42 | 1 | 1 | 0
  Not at risk, Week 43: number analyzed (Participants) | 854 | 412 | 432
  Not at risk, Week 43 | 1 | 1 | 0
  Not at risk, Week 44: number analyzed (Participants) | 931 | 457 | 468
  Not at risk, Week 44 | 1 | 1 | 0
  Not at risk, Week 45: number analyzed (Participants) | 1022 | 482 | 543
  Not at risk, Week 45 | 1 | 1 | 0
  Not at risk, Week 46: number analyzed (Participants) | 1147 | 571 | 576
  Not at risk, Week 46 | 2 | 1 | 0
  Not at risk, Week 47: number analyzed (Participants) | 1220 | 632 | 624
  Not at risk, Week 47 | 2 | 1 | 0
  Not at risk, Week 48: number analyzed (Participants) | 1270 | 656 | 666
  Not at risk, Week 48 | 2 | 1 | 0

117. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis
Description: Musculoskeletal AEs include any musculoskeletal AEs, arthropathy and muscle aches/myalgia.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1188 | 222 | 214
  At risk, Week 38 | 29 | 1 | 4
  At risk, Week 39: number analyzed (Participants) | 2432 | 138 | 384
  At risk, Week 39 | 64 | 2 | 2
  At risk, Week 40: number analyzed (Participants) | 1980 | 262 | 320
  At risk, Week 40 | 72 | 1 | 3
  At risk, Week 41: number analyzed (Participants) | 2246 | 207 | 304
  At risk, Week 41 | 43 | 1 | 0
  At risk, Week 42: number analyzed (Participants) | 1230 | 172 | 349
  At risk, Week 42 | 44 | 0 | 2
  At risk, Week 43: number analyzed (Participants) | 669 | 106 | 259
  At risk, Week 43 | 8 | 1 | 0
  At risk, Week 44: number analyzed (Participants) | 692 | 134 | 168
  At risk, Week 44 | 15 | 0 | 0
  At risk, Week 45: number analyzed (Participants) | 613 | 88 | 167
  At risk, Week 45 | 15 | 0 | 2
  At risk, Week 46: number analyzed (Participants) | 820 | 183 | 108
  At risk, Week 46 | 9 | 1 | 0
  At risk, Week 47: number analyzed (Participants) | 401 | 71 | 101
  At risk, Week 47 | 1 | 0 | 1
  At risk, Week 48: number analyzed (Participants) | 314 | 56 | 61
  At risk, Week 48 | 4 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 38
  Not at risk, Week 38 | 3 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 194 | 31 | 46
  Not at risk, Week 39 | 7 | 0 | 1
  Not at risk, Week 40: number analyzed (Participants) | 166 | 63 | 37
  Not at risk, Week 40 | 3 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 212 | 127 | 120
  Not at risk, Week 41 | 5 | 0 | 0
  Not at risk, Week 42: number analyzed (Participants) | 132 | 67 | 83
  Not at risk, Week 42 | 2 | 0 | 0
  Not at risk, Week 43: number analyzed (Participants) | 69 | 34 | 97
  Not at risk, Week 43 | 0 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 77 | 45 | 36
  Not at risk, Week 44 | 0 | 0 | 0
  Not at risk, Week 45: number analyzed (Participants) | 91 | 25 | 75
  Not at risk, Week 45 | 3 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 125 | 89 | 33
  Not at risk, Week 46 | 3 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 73 | 61 | 48
  Not at risk, Week 47 | 1 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 50 | 24 | 42
  Not at risk, Week 48 | 0 | 0 | 0

118. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Musculoskeletal) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative)
Description: Musculoskeletal AEs include any musculoskeletal AEs, arthropathy and muscle aches/myalgia.
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1194 | 222 | 291
  At risk, Week 38 | 29 | 1 | 4
  At risk, Week 39: number analyzed (Participants) | 3626 | 360 | 675
  At risk, Week 39 | 93 | 3 | 6
  At risk, Week 40: number analyzed (Participants) | 5606 | 622 | 995
  At risk, Week 40 | 165 | 4 | 9
  At risk, Week 41: number analyzed (Participants) | 7852 | 829 | 1299
  At risk, Week 41 | 208 | 5 | 9
  At risk, Week 42: number analyzed (Participants) | 9082 | 1001 | 1648
  At risk, Week 42 | 252 | 5 | 11
  At risk, Week 43: number analyzed (Participants) | 9751 | 1107 | 1907
  At risk, Week 43 | 260 | 6 | 11
  At risk, Week 44: number analyzed (Participants) | 10443 | 1241 | 2075
  At risk, Week 44 | 275 | 6 | 11
  At risk, Week 45: number analyzed (Participants) | 11056 | 1329 | 2242
  At risk, Week 45 | 290 | 6 | 13
  At risk, Week 46: number analyzed (Participants) | 11876 | 1512 | 2350
  At risk, Week 46 | 299 | 7 | 13
  At risk, Week 47: number analyzed (Participants) | 12277 | 1583 | 2451
  At risk, Week 47 | 300 | 7 | 14
  At risk, Week 48: number analyzed (Participants) | 12591 | 1639 | 2512
  At risk, Week 48 | 304 | 7 | 14
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 49
  Not at risk, Week 38 | 3 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 275 | 121 | 95
  Not at risk, Week 39 | 10 | 0 | 1
  Not at risk, Week 40: number analyzed (Participants) | 441 | 184 | 132
  Not at risk, Week 40 | 13 | 0 | 1
  Not at risk, Week 41: number analyzed (Participants) | 653 | 311 | 252
  Not at risk, Week 41 | 18 | 0 | 1
  Not at risk, Week 42: number analyzed (Participants) | 785 | 378 | 335
  Not at risk, Week 42 | 20 | 0 | 1
  Not at risk, Week 43: number analyzed (Participants) | 854 | 412 | 432
  Not at risk, Week 43 | 20 | 0 | 1
  Not at risk, Week 44: number analyzed (Participants) | 931 | 457 | 468
  Not at risk, Week 44 | 20 | 0 | 1
  Not at risk, Week 45: number analyzed (Participants) | 1022 | 482 | 543
  Not at risk, Week 45 | 23 | 0 | 1
  Not at risk, Week 46: number analyzed (Participants) | 1147 | 571 | 576
  Not at risk, Week 46 | 26 | 0 | 1
  Not at risk, Week 47: number analyzed (Participants) | 1220 | 632 | 624
  Not at risk, Week 47 | 27 | 0 | 1
  Not at risk, Week 48: number analyzed (Participants) | 1270 | 656 | 666
  Not at risk, Week 48 | 27 | 0 | 1

119. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis
Description: as for outcome 79
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1188 | 222 | 214
  At risk, Week 38 | 19 | 0 | 0
  At risk, Week 39: number analyzed (Participants) | 2432 | 138 | 384
  At risk, Week 39 | 48 | 1 | 0
  At risk, Week 40: number analyzed (Participants) | 1980 | 262 | 320
  At risk, Week 40 | 40 | 1 | 0
  At risk, Week 41: number analyzed (Participants) | 2246 | 207 | 304
  At risk, Week 41 | 30 | 0 | 2
  At risk, Week 42: number analyzed (Participants) | 1230 | 172 | 349
  At risk, Week 42 | 15 | 0 | 0
  At risk, Week 43: number analyzed (Participants) | 669 | 106 | 259
  At risk, Week 43 | 11 | 1 | 2
  At risk, Week 44: number analyzed (Participants) | 692 | 134 | 168
  At risk, Week 44 | 6 | 0 | 0
  At risk, Week 45: number analyzed (Participants) | 613 | 88 | 167
  At risk, Week 45 | 11 | 0 | 0
  At risk, Week 46: number analyzed (Participants) | 820 | 183 | 108
  At risk, Week 46 | 3 | 1 | 0
  At risk, Week 47: number analyzed (Participants) | 401 | 71 | 101
  At risk, Week 47 | 0 | 0 | 0
  At risk, Week 48: number analyzed (Participants) | 314 | 56 | 61
  At risk, Week 48 | 0 | 0 | 0
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 38
  Not at risk, Week 38 | 3 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 194 | 31 | 46
  Not at risk, Week 39 | 4 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 166 | 63 | 37
  Not at risk, Week 40 | 6 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 212 | 127 | 120
  Not at risk, Week 41 | 1 | 0 | 1
  Not at risk, Week 42: number analyzed (Participants) | 132 | 67 | 83
  Not at risk, Week 42 | 2 | 1 | 0
  Not at risk, Week 43: number analyzed (Participants) | 69 | 34 | 97
  Not at risk, Week 43 | 2 | 0 | 0
  Not at risk, Week 44: number analyzed (Participants) | 77 | 45 | 36
  Not at risk, Week 44 | 1 | 1 | 0
  Not at risk, Week 45: number analyzed (Participants) | 91 | 25 | 75
  Not at risk, Week 45 | 2 | 0 | 0
  Not at risk, Week 46: number analyzed (Participants) | 125 | 89 | 33
  Not at risk, Week 46 | 0 | 0 | 0
  Not at risk, Week 47: number analyzed (Participants) | 73 | 61 | 48
  Not at risk, Week 47 | 1 | 0 | 0
  Not at risk, Week 48: number analyzed (Participants) | 50 | 24 | 42
  Not at risk, Week 48 | 1 | 0 | 0

120. Secondary Outcome: Number of Subjects Reporting EMA Defined AEIs (Neurological) and Onset Dates of AEIs Using a Card Based ADR Reporting System by Chief Medical Officer (CMO)-Specified Risk Status, on a Weekly Basis (Cumulative).
Description: as for outcome 79
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Number analyzed (Participants) | 13861 | 2295 | 3178
Participants
  At risk, Week 37: number analyzed (Participants) | 6 | 0 | 77
  At risk, Week 37 | 0 | 0 | 0
  At risk, Week 38: number analyzed (Participants) | 1194 | 222 | 291
  At risk, Week 38 | 19 | 0 | 0
  At risk, Week 39: number analyzed (Participants) | 3626 | 360 | 675
  At risk, Week 39 | 67 | 1 | 0
  At risk, Week 40: number analyzed (Participants) | 5606 | 622 | 995
  At risk, Week 40 | 107 | 2 | 0
  At risk, Week 41: number analyzed (Participants) | 7852 | 829 | 1299
  At risk, Week 41 | 137 | 2 | 2
  At risk, Week 42: number analyzed (Participants) | 9082 | 1001 | 1648
  At risk, Week 42 | 152 | 2 | 2
  At risk, Week 43: number analyzed (Participants) | 9751 | 1107 | 1907
  At risk, Week 43 | 163 | 3 | 4
  At risk, Week 44: number analyzed (Participants) | 10443 | 1241 | 2075
  At risk, Week 44 | 169 | 3 | 4
  At risk, Week 45: number analyzed (Participants) | 11056 | 1329 | 2242
  At risk, Week 45 | 180 | 3 | 4
  At risk, Week 46: number analyzed (Participants) | 11876 | 1512 | 2350
  At risk, Week 46 | 183 | 4 | 4
  At risk, Week 47: number analyzed (Participants) | 12277 | 1583 | 2451
  At risk, Week 47 | 183 | 4 | 4
  At risk, Week 48: number analyzed (Participants) | 12591 | 1639 | 2512
  At risk, Week 48 | 183 | 4 | 4
  Not at risk, Week 37: number analyzed (Participants) | 0 | 0 | 11
  Not at risk, Week 37 | 0 | 0 | 0
  Not at risk, Week 38: number analyzed (Participants) | 81 | 90 | 49
  Not at risk, Week 38 | 3 | 0 | 0
  Not at risk, Week 39: number analyzed (Participants) | 275 | 121 | 95
  Not at risk, Week 39 | 7 | 0 | 0
  Not at risk, Week 40: number analyzed (Participants) | 441 | 184 | 132
  Not at risk, Week 40 | 13 | 0 | 0
  Not at risk, Week 41: number analyzed (Participants) | 653 | 311 | 252
  Not at risk, Week 41 | 14 | 0 | 1
  Not at risk, Week 42: number analyzed (Participants) | 785 | 378 | 335
  Not at risk, Week 42 | 16 | 1 | 1
  Not at risk, Week 43: number analyzed (Participants) | 854 | 412 | 432
  Not at risk, Week 43 | 18 | 1 | 1
  Not at risk, Week 44: number analyzed (Participants) | 931 | 457 | 468
  Not at risk, Week 44 | 19 | 2 | 1
  Not at risk, Week 45: number analyzed (Participants) | 1022 | 482 | 543
  Not at risk, Week 45 | 21 | 2 | 1
  Not at risk, Week 46: number analyzed (Participants) | 1147 | 571 | 576
  Not at risk, Week 46 | 21 | 2 | 1
  Not at risk, Week 47: number analyzed (Participants) | 1220 | 632 | 624
  Not at risk, Week 47 | 22 | 2 | 1
  Not at risk, Week 48: number analyzed (Participants) | 1270 | 656 | 666
  Not at risk, Week 48 | 23 | 2 | 1

ADVERSE EVENTS:
Time Frame: Within 7 days post vaccination (anticipated to be between 01 September 2016 and 30 November 2016)
Description: Subjects who did not report an event were considered as subjects without the event.
Arm/Group | Vaccinated_Fluarix Tetra Group | Vaccinated_Non GSK Group | Vaccinated_Unknown Group
Serious Adverse Events (participants affected / at risk) | 0/13861 | 0/2295 | 0/3178
Other Adverse Events (participants affected / at risk) | 1049/13861 | 62/2295 | 54/3178
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccinated_Fluarix Tetra Group (N=13861) | Vaccinated_Non GSK Group (N=2295) | Vaccinated_Unknown Group (N=3178)
Fever/pyrexia (General disorders) | 133 | 25 | 16
Local erythema (General disorders) | 127 | 0 | 0
Drowsiness (General disorders) | 72 | 0 | 0
Fatigue (General disorders) | 169 | 0 | 1
Irritability (General disorders) | 17 | 0 | 0
Malaise (General disorders) | 4 | 1 | 0
Conjunctivitis (General disorders) | 28 | 2 | 0
Coryza (General disorders) | 96 | 0 | 0
Cough (General disorders) | 210 | 17 | 13
Epistaxis (General disorders) | 12 | 1 | 0
Hoarseness (General disorders) | 71 | 0 | 0
Nasal congestion (General disorders) | 276 | 3 | 0
Oropharyngeal pain (General disorders) | 155 | 2 | 0
Rhinorrhoea (General disorders) | 243 | 2 | 0
Wheezing (General disorders) | 63 | 0 | 1
Decreased appetite (Gastrointestinal disorders) | 50 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 64 | 0 | 2
Nausea (Gastrointestinal disorders) | 71 | 0 | 0
Vomiting (Gastrointestinal disorders) | 19 | 1 | 0
Anaphylactic reactions (General disorders) | 0 | 0 | 0
Facial oedema (General disorders) | 1 | 0 | 0
Hypersensitivity reactions (General disorders) | 14 | 1 | 0
Generalised rash (General disorders) | 31 | 6 | 2
Rash (General disorders) | 16 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 79 | 0 | 0
Muscle aches/myalgia (Musculoskeletal and connective tissue disorders) | 311 | 7 | 15
Bell's palsy (Nervous system disorders) | 0 | 0 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 0 | 0
Headache (General disorders) | 192 | 6 | 5
Peripheral tremor (General disorders) | 24 | 0 | 0
Seizure / Febrile convulsions (General disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.